# The association between mental health conditions and vitiligo: a population-based cohort study in the UK: Statistical Analysis Plan

| SAP version | 1.1 |
|-------------|--------------|
| Date | 05 July 2021 |
| NCT number | NCT04953338 |

## Contents

| List of | abbreviations | 4 |
|----------|-----------------------------------------------------------|----|
| 1. Intro | oduction | 5 |
| 1.1 l | Background | 5 |
| 1.2. | Purposes of analyses | 6 |
| 2. Stud | ly objectives and endpoints | 7 |
| 2.1 5 | Study objectives | 7 |
| 2.2 1 | Primary objectives | 7 |
| 2.3 9 | Secondary objectives: | 7 |
| 2.4 1 | Primary endpoints | 7 |
| 2.5 | Secondary endpoints | 8 |
| 3 Gene | eral Study Design and Plan | 8 |
| 3.1 9 | Study Design | 8 |
| 3.2 1 | Data source and Read codes | 8 |
| 3.3 1 | Data extraction | 8 |
| 3.4 1 | Inclusion-Exclusion Criteria and General Study Population | 9 |
| D | efinition of vitiligo cases | 9 |
| D | efinition of matched controls without vitiligo | 9 |
| D | efinition of mental health outcomes | 9 |
| D | efinition of psychological or work-related complications | 10 |
| 3.5 1 | Baseline characteristics | 10 |
| 4 Sam | ple size calculations | 11 |
| 5 Popı | ılations to be analysed | 11 |
| 5.1 | Inclusion Criteria | 11 |
| 5.2 | Exclusion Criteria | 11 |
| 5.3 | Matching process | 11 |

| 6 Statistical Analysis | 12 |
|-------------------------------------------------|-----|
| 6.1 Statistical principles | 12 |
| 6.2 Primary Endpoint Analysis | 12 |
| Prevalence of mental health conditions | 12 |
| Point prevalence of vitiligo | 13 |
| Incidence of new onset mental health conditions | 13 |
| Healthcare utilisation and management patterns | 14 |
| 6.3 Secondary Objective Analysis | 14 |
| Time off work and unemployment | 14 |
| 6.4 Sensitivity analysis | 15 |
| 6.5 Missing data | 15 |
| 7 Study Limitations | 15 |
| 8 Statistical software | 16 |
| 9 Ethics | 16 |
| References | 17 |
| Appendix 1 | 19 |
| Appendix 2 | 32 |
| Appendix 3 | 33 |
| Appendix 4 | 168 |

# List of abbreviations

| Abbreviation | Full Form |
|---|---|
| AD | Anxiety disorder |
| ADEPT | Anonymised Data Ethics Protocols and Transparency |
| BMI | Body mass index |
| CI | Confidence Interval |
| DE | Depressive episode |
| GEP | Good Epidemiological Practice |
| GP | General Practitioner |
| GPP | Guidelines for Good Pharmacoepidemiology Practices |
| HR | Hazard Ratio |
| IEA | International Epidemiological Association |
| IMD | Index of multiple deprivation |
| IQR | Interquartile range |
| ISPE | International Society for Pharmacoepidemiology |
| MDD | Major depressive disorder |
| OPC | Optimum Patient Care |
| OPCRD | Optimum Patient Care Research Database |
| QoL | Quality of life |
| RECORD | Reporting of studies conducted using observational routinely collected data |
| SD | Standard deviation |
| SES | Socio-economic status |
| THIN | The Health Improvement Network |
| UK | United Kingdom |

#### 1. Introduction

#### 1.1 Background

Vitiligo is an acquired skin disorder characterised by depigmented patches of skin that may appear in a localised or generalised distribution. Vitiligo is estimated to affect 0.5-2% of the global population with an equal incidence between genders, age or racial/ethnic groups (1). The exact cause of the loss of functioning melanocytes in vitiligo remains unknown but is likely to be resulted from the complex interplay of genetics, oxidative stress, and autoimmunity (2).

Although vitiligo is typically asymptomatic, it may substantially affect the psychological wellbeing of people living with the condition (3-5). This could be due to the unpredictable prognosis, the current lack of cure or the perception and emotional burden associated with the visibility of vitiligo. A recent systematic review has shown that people with vitiligo are significantly more likely to suffer from depression and anxiety compared to the healthy controls (6). However, there is a lack of knowledge of the other types of psychological symptoms/disorders that people with vitiligo experience (7).

Human society places a profound significance on appearance, aesthetics and pigmentation (8). Vitiligo is visible on all skin types, and is particularly noticeable on dark skin tones because of the strong contrast. Given the visible difference in appearance of affected and unaffected areas of the skin the condition has been construed as being disfiguring. Some studies have suggested in those with darker skin vitiligo is correlated with a worse quality of life (QoL) (9, 10). However, these studies have small sample sizes and psychiatric comorbidities and psychological wellbeing were not evaluated in the analyses. Further, there are other studies that indicate that people with lighter skin tones may also experience distress (11).

In addition to skin colour, the location of vitiligo lesions may also influence the overall well-being and stigmatisation experience of patients. However, inconsistent findings have been reported. A few studies showed that patients had a more significant QoL impairment

when lesions were located on visible sites (e.g. face, neck and hand) (12, 13) whilst other studies did not find any relationship (14, 15). By contrast, some studies report vitiligo lesions on more central body parts (e.g. chest, arms and trunks) are more likely to have an adverse impact on emotional wellbeing of people with the condition, perhaps because there remains anxiety as to how they might be judged by others if the condition were to be revealed (9, 16). Indeed, the nature of reactions received from others is also likely to play an integral role in adjustment and the extent to which stigmatisation is experienced (17, 18). Additional data from mixed method studies is needed to further understand this topic and how this may affect the possible comorbid burden of mental health conditions.

There is currently a lack of large population-based studies providing reliable estimates of the risks of psychological comorbidities associated with vitiligo in the UK. A recent observational study using the UK-THIN database (19) highlighted the burden of depression in vitiligo patients and found a bidirectional relationship between the two conditions. However, the study did not explore the associations with other forms of psychological distress and did not use a validated definition for depression. An analysis of the depression risk on the populations of different ethnicity and location of the vitiligo lesions, which can be potential sources of heterogeneity, were also not conducted.

## 1.2. Purposes of analyses

To the best of our knowledge, there has only been one large population-based study assessing psychosocial comorbidities in vitiligo compared to those without the condition (19). This study was limited only to exploring major depressive disorder (MDD, also termed recurrent depressive disorder) and used an unvalidated case definition for MDD. There have been no large-scale population studies looking at the association between vitiligo and depressive episodes (not meeting the criteria for MDD), anxiety, social phobias and other potential psychological complications of vitiligo. No current study explores the relationship with ethnicity and psychological outcomes or the associations between vitiligo location and a broader range of psychological outcomes beyond MDD. The purpose of this study is therefore to fill this evidence gap.

## 2. Study objectives and endpoints

## 2.1 Study objectives

The objective of this study is to determine the risks of comorbid mental health conditions (including depression, anxiety and other potential psychological complications of vitiligo) in people with vitiligo compared to a control population and to evaluate whether the relative risks may vary by different ethnicities.

## 2.2 Primary objectives

- Briefly describe the epidemiology of vitiligo in the dataset: vitiligo incidence of vitiligo over time and by age, sex, ethnicity and sociodemographic factors and lifetime prevalence by age and sex.
- Describe the prevalence of common mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorder), overall and stratified by sociodemographic factors and location of lesion.
- Describe the incidence of common mental health conditions (depressive episodes, recurrent depressive disorder and anxiety disorders), overall and stratified by sociodemographic factors and lesion location.
- Describe current primary care service utilisation in those vitiligo cases and matched controls having a prevalent depressive illness of anxiety disorder at their index date.
- Describe management patterns in those vitiligo cases and matched controls having a prevalent depressive illness of anxiety disorder at their index date.

## 2.3 Secondary objectives:

 Describe the baseline prevalence and post diagnosis incidence of other potential psychological or work-related complications of vitiligo.

## 2.4 Primary endpoints

- Vitiligo prevalence: A diagnosis of vitiligo at any time prior to 31 December 2020.
- Mental health condition prevalence: A diagnosis of the relevant common mental health condition prior to the index date in vitiligo cases and matched controls

- Incidence: Time to first diagnosis of the relevant mental health condition in the two years following the index date in vitiligo cases and matched controls
- Primary care service utilisation: Number of primary care visits in the one year following the index date in vitiligo cases and matched controls
- Management patterns: Secondary care dermatology referrals in the one year following the index date in vitiligo cases.

## 2.5 Secondary endpoints

- Psychological or work-related complications consist of time of work for illness, unemployment, social phobia, adjustment disorder, substance abuse, self-harm, overdose, and parasuicide or suicide attempts
- Prevalence: A diagnosis or recording of the relevant psychological or work-related complication prior to the index date in vitiligo cases and matched controls
- Incidence: Time to first diagnosis or recording of the relevant psychological or work-related complication in the year following the index date in vitiligo cases and matched controls

## 3 General Study Design and Plan

## 3.1 Study Design

Matched-cohort design

#### 3.2 Data source and Read codes

This study will use routinely collected and collated data from the Optimum Patient Care Research Database (OPCRD) (20). This database incorporates pseudonymised primary care records from up to 700 GP practices distributed across England, Wales, Scotland and Northern Ireland. The current OPCRD cohort size is over 5 million actively registered people, and historic records available for 10.1 million people.

#### 3.3 Data extraction

Individual patient data is anonymised at the point of data extraction. Queries will be executed to extract relevant data from the OPCRD using the codes listed in Appendix 1.

All data will remain in anonymised form and will be held on a secure server. The data will not be used for any purposes other than for the research which is described in the respective protocols and which has been approved by OPC. The sponsor, Pfizer Ltd, will not have access to the individual anonymised patient data.

#### 3.4 Inclusion-Exclusion Criteria and General Study Population

### Definition of vitiligo cases

We will identify all people diagnosed with vitiligo using diagnostic Read and SNOMED CT codes which are specific to vitiligo (Appendix 1). A diagnostic algorithm will be used to facilitate robust case identification of vitiligo. This algorithm will identify anyone with a vitiligo specific diagnosis code followed by exclusion of anyone with a diagnosis code for an alternative depigmenting disorder coded within a one-year period (six months before or after their first vitiligo diagnosis code). The list of alternative depigmenting disorders is shown in Appendix 2.

The study index date for people diagnosed with vitiligo will be the latest of; the start date of follow-up (1st Jan 2010), date of registration with GP plus six months, or the date of diagnosis of vitiligo.

#### Definition of matched controls without vitiligo

Eligible controls at each index date will comprise people actively registered with the GP practice at that date without a history of vitiligo and a minimum one-year registration with their GP practice (to minimise the risk they had a non-recorded existing vitiligo diagnosis). After matching (refer to section 5.3), the index date for each control will be set at the index date of their matched counterpart. People diagnosed with vitiligo during the study period will be included in the pool of eligible unexposed people for matching, but if matched, will be censored on the date of their vitiligo diagnosis. Such people are thus eligible to contribute to the study as matched controls until the date of their vitiligo diagnosis.

#### Definition of mental health outcomes

We will identify three common mental health outcomes which will be examined separately; depressive episodes (DE), MDD, and non-phobia related anxiety disorder (AD),

chosen as they represent the most common mental health conditions presenting to primary care (21). Each condition will be identified using algorithms validated in UK primary care (22). The codes used to identify these conditions are provided in Appendix 3. We will use a concurrent diagnosis and treatment code to identify acute episodes (DE and AD) and for MDD either a historical code for any depression and current treatment or a depressive disorder specific diagnosis code (22). We will also identified less common mental health conditions; social phobia, adjustment disorder, substance abuse, self-harm, overdose and suicide attempt or parasuicide, using specific diagnostic codes.

#### Definition of psychological or work-related complications

Time-off work will be defined by the issue of Med 3 certificates of fitness for work (23), which are issued to patients to provide to their employers as evidence of being medically unable to perform usual work activities, and thus indicate absenteeism. Unemployment will be defined by the presence of a Read code relating to unemployment or issue of either an IB113 or ESA113 form to indicate incapacity from work (24). We will not evaluate whether time-off work and incapacity from work related specifically to vitiligo or mental health as this information is not available in the clinical record.

#### 3.5 Baseline characteristics

Sociodemographic groups will be defined by 10-year age category, sex, socio-economic status (SES), and ethnicity. SES will be defined using the official national deprivation measure; index of multiple deprivation (IMD) (25). This will be calculated at the point using patient postcode, with the resultant scores stratified by deprivation quintile according to the national distribution. Ethnicity will be grouped into major ethnic groups to be consistent with the UK official census categories: White, Black African/Caribbean, Asian, Mixed, and Other (26, 27). Other clinical covariates comprised BMI category, smoking status, alcohol use, and common comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, stroke, heart failure, chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease, and dementia). These will be identified using clinical codes and test results recorded in the patient record.

## 4 Sample size calculations

No previous studies have examined mental health risk in people with vitiligo to provide an estimation of effect size to inform our sample size calculation. Assuming 80% power, a 1:1 ratio of vitiligo cases to controls, and an overall probability of 15% for anxiety and 10% for depression (conservative estimates based on a previous analysis of DSM\_IV disorders) in the general population (21) a sample size of between 3,350 and 5,023 will be required to detect a minimum clinically relevant effect size of a 27% increased risk of a mental health condition in the vitiligo cohort compared to population controls. We anticipate c.22,500 people in our study cohort will be defined as vitiligo cases, these will be 1:1 matched to population controls providing a study cohort well in excess of this required sample size.

## 5 Populations to be analysed

#### 5.1 Inclusion Criteria

All eligible adults (≥18) (as at date of index date) registered with GP practices contributing data to OPCRD between January 1, 2004 and December 31, 2020, are eligible for inclusion in the study. Eligible vitiligo cases will comprise all incident cases of vitiligo over the last 15 years (2004-2020).

#### 5.2 Exclusion Criteria

People with less than 1 year of follow up available.

## 5.3 Matching process

Each adult with vitiligo will be 1:1 matched at their index date using, nearest neighbour matching (30) with an unaffected control (people without vitiligo prior to or during the study period). Matching variables will comprise age, sex, duration of practice registration and within primary care practice where numbers allow. After matching, the index date for each control will be set at the index date of their matched counterpart. Refer also to section 3.4 -Definition of matched controls without vitiligo.

## 6 Statistical Analysis

#### 6.1 Statistical principles

The mean, standard deviation (sd) and any other statistical measures, will be reported to one decimal place. Continuous data will be summarised in the form of means, sd, median, interquartile range (IQR) and range as appropriate. Categorical data will be summarised using frequencies and proportions. Chi-squared and t-tests will be performed to compare the frequency of dichotomous variables and the values of continuous variables where relevant. 95% CIs will be reported for main effect sizes. Statistical significance will be assessed using p<0.05. Actual p-values will be reported except for p-values less than 3 decimal places which will be reported as "<0.001". P-values >0.1 will be reported to one decimal place, p-values between 0.01 and 0.1 will be reported to three decimal places.

The assessment of any associations with baseline characteristics and the primary endpoint will be assessed using Cox proportional hazards models. A standard set of features will be used in all multivariable models as listed in section 6.2.

Assumptions of statistical approaches will be assessed, and transformations used if necessary (although it is not anticipated that the data will violate model assumptions).

## **6.2 Primary Endpoint Analysis**

#### Prevalence of mental health conditions

Prevalence of mental health conditions will be estimated at the index date for both cases and matched controls.

Prevalence of the three common mental health conditions (MDD, DE, and AD) in vitiligo cases will be compared to matched controls without vitiligo, overall, and by sociodemographic subgroups defined by age, sex, SES, and ethnicity. For cases and controls, prevalence will be calculated by dividing the total number of people in each cohort fulfilling the diagnostic inclusion criteria for the indicated mental health condition,

by the total number of people in each cohort. The concomitant prevalence of MDD and AD, and DE and AD, will be estimated using the same approach.

Prevalence of social phobia, adjustment disorder, substance abuse, self-harm, and suicide attempt or parasuicide will also be examined in cases and controls.

#### Point prevalence of vitiligo

Point prevalence of vitiligo will be used as an estimate for lifetime prevalence. We will estimate point prevalence overall and by age and sex, on 31 December, 2020, the last date of follow-up. Point prevalence will be calculated by dividing the total number of actively registered people with a vitiligo diagnostic code (at any prior time point) by the total number of actively registered people in OPCRD. New episodes or recurrent episodes of vitiligo in those already coded as vitiligo will be excluded. All people will be included regardless of the date of vitiligo diagnosis in relation to the date of registration with a practice. People with <365 days of follow up from date of registration will be excluded from the analysis.

#### Incidence of new onset mental health conditions

Incidence of new onset mental health conditions will be assessed prospectively in vitiligo cases and matched controls from the index date. Only case and control pairs who both are without the relevant mental health condition at the index date will be included, We will then estimate incidence rates for each common mental health conditions within two years of the index date for both vitiligo cases and controls, overall by sociodemographic subgroups defined by age, sex, SES and ethnicity.

The end of follow-up will be defined as the earliest of the study end-date (December 31, 2020), the date of patient transfer from an included general practice, date of death, or the date an individual first developed a mental health condition of interest, or two years after the index date.

Incidence will be calculated by dividing the number of incident people by the sum of person-years of follow-up. Risk of developing each mental health condition will then be examined using time to failure analysis. Initially, unadjusted Cox proportional hazards models, stratified by matched set (vitiligo cases versus matched controls), will be used to provide overall hazard ratios (HRs) as summary estimates for the association of the presence of vitiligo with the time to each mental health condition category. Models will be subsequently adjusted for sociodemographic features (age, sex, SES, and ethnicity) and common comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, stroke, heart failure, chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease, and dementia) in multivariable analysis.

#### Healthcare utilisation and management patterns

We will prospectively examine primary care visit frequency and secondary care dermatology referral rates within one year of index date in the subset of vitiligo cases and matched controls, comprising of those individuals with a prevalent depressive illness of anxiety disorder at their index date using Cox proportional hazards models adjusted for sociodemographic factors (age, sex, SES, and ethnicity) and common comorbidities (hypertension, hyperlipidaemia, type 2 diabetes, atrial fibrillation, angina, myocardial infarction, stroke, heart failure, chronic kidney disease stages 3-5, chronic obstructive pulmonary disease, asthma, chronic liver disease, and dementia).

We will also report the overall primary care visit frequency and secondary care referral rate for comparison.

## 6.3 Secondary Objective Analysis

## Time off work and unemployment

Risk of either being issued a time-off work certificate or having a record of unemployment in the one year following the index date will be examined in people of normal working age (18-65) using time to failure analysis. For each outcome, proportions will be

estimated as the cumulative one-year incidence using the Kaplan-Meier method, which will allow for differential follow-up time as not all people had a full year of follow-up available. Adjusted Cox models (same covariate set as for mental health outcomes) will be used to estimate the relative association of the presence of vitiligo with issue of Med3 certificate and unemployment.

#### 6.4 Sensitivity analysis

To evaluate the magnitude of potential bias from including, as matched controls, people who are registered with GP practices but who do not attend their practice, we will repeat the primary analysis including only controls with a least one primary care consultation in the year preceding their index date.

#### 6.5 Missing data

This study will use the missing indicator variable method as missing data are considered likely not to be missing at random, meaning multiple imputation approaches will lack validity.

Patient will need to be excluded from analyses based on a matched design if they have incomplete data in the fields (age, sex) required to run the matching process. In similar studies, the exclusion rate due to incomplete data has been low (28, 29).

## 7 Study Limitations

Although the data is derived from a validated and nationally representative sample of the UK, results should not be extrapolated to dissimilar populations. Important limitations of the study include the reliance on comprehensive code lists to identify any given baseline or outcome variable. This limitation is common to all studies using routinely recorded data and will be mitigated through the use of a validated approach for defining baseline and outcome parameters. (30)

Limitations exist in the amount of clinical detail presently recorded in routine primary care electronic health records. Routine primary care databases offer the benefit of large cohorts at the expense of granularity; a limitation that is universal in epidemiological studies of this type. Some analyses will be restricted to people in whom complete information is available which may introduce selection bias as a result. Finally, the data presented will be observational in nature and although attempts will be made to reduce confounding by statistical adjustment where relevant, it is not possible to exclude the possibility of residual confounding as part of the explanation for any findings.

#### 8 Statistical software

All statistical analyses will be performed using R software version 3.4.1.

#### 9 Ethics

This study requires approval by the Anonymised Data Ethics Protocols and Transparency (ADEPT) Committee. It has been uploaded to ClinicalTrials.gov.

This study will be conducted in accordance with legal and regulatory requirements, as well as with scientific purpose, value, and rigor and follow generally accepted research practices described in Guidelines for Good Pharmacoepidemiology Practices (GPP) issued by the International Society for Pharmacoepidemiology (ISPE), and Good Epidemiological Practice (GEP) guidelines issued by the International Epidemiological Association (IEA). Study reporting will be conducted in accordance with the RECORD (Reporting of studies conducted using observational routinely collected data) guidelines.(31)

#### References

- 1. Steiner D, Bedin V, Moraes MB, Villas RT, Steiner T. Vitiligo. Anais Brasileiros de Dermatologia. 2004;79:335-51.
- 2. Grimes PE, Miller MM. Vitiligo: Patient stories, self-esteem, and the psychological burden of disease. Int J Womens Dermatol. 2018;4(1):32-7.
- 3. Vernwal D. A study of anxiety and depression in Vitiligo patients: New challenges to treat. European Psychiatry. 2017;41:S321.
- 4. Sangma LN, Nath J, Bhagabati D. Quality of life and psychological morbidity in vitiligo patients: a study in a teaching hospital from north-East India. Indian J Dermatol. 2015;60(2):142-6.
- 5. Papadopoulos L, Bor R, Legg C. Coping with the disfiguring effects of vitiligo: a preliminary investigation into the effects of cognitive-behavioural therapy. Br J Med Psychol. 1999;72 ( Pt 3):385-96.
- 6. Lai YC, Yew YW, Kennedy C, Schwartz RA. Vitiligo and depression: a systematic review and meta-analysis of observational studies. Br J Dermatol. 2017;177(3):708-18.
- 7. Osinubi O, Grainge MJ, Hong L, Ahmed A, Batchelor JM, Grindlay D, et al. The prevalence of psychological comorbidity in people with vitiligo: a systematic review and meta-analysis. Br J Dermatol. 2018;178(4):863-78.
- 8. Thompson AR. Research directions in appearance research: models for the future. In Rumsey, N., & Harcourt, D. (Eds.), Oxford handbook of appearance. Oxford: Oxford University Press 2012.
- 9. Homan M, Spuls P, Korte J, Bos J, Sprangers M, Veen J. The burden of vitiligo: Patient characteristics associated with quality of life. Journal of the American Academy of Dermatology. 2009;61:411-20.
- 10. Dolatshahi M, Ghazi P, Feizy V, Hemami MR. Life quality assessment among patients with vitiligo: comparison of married and single patients in Iran. Indian J Dermatol Venereol Leprol. 2008;74(6):700.
- 11. Thompson AR, Kent G, Smith JA. Living with vitiligo: dealing with difference. Br J Health Psychol. 2002;7(Pt 2):213-25.
- 12. Bae JM, Lee SC, Kim TH, Yeom SD, Shin JH, Lee WJ, et al. Factors affecting quality of life in patients with vitiligo: a nationwide study. British Journal of Dermatology. 2018;178(1):238-44.
- 13. Patvekar M, Deo K, Verma S, Kothari P, Gupta A. Quality of life in vitiligo: Relationship to clinical severity and demographic data. Pigment International. 2017;4:104-8.
- 14. Chen D, Tuan H, Zhou EY, Liu D, Zhao Y. Quality of life of adult vitiligo patients using camouflage: A survey in a Chinese vitiligo community. PLOS ONE. 2019;14(1):e0210581.
- 15. Ongenae K, Van Geel N, De Schepper S, Naeyaert JM. Effect of vitiligo on self-reported health-related quality of life. Br J Dermatol. 2005;152(6):1165-72.
- 16. Kruger C, Schallreuter KU. Stigmatisation, Avoidance Behaviour and Difficulties in Coping are Common Among Adult Patients with Vitiligo. Acta Derm Venereol. 2015;95(5):553-8.
- 17. Thompson AR, Clarke SA, Newell RJ, Gawkrodger DJ. Vitiligo linked to stigmatization in British South Asian women: a qualitative study of the experiences of living with vitiligo. Br J Dermatol. 2010;163(3):481-6.
- 18. Kent G, Al'Abadie M. Psychologic effects of vitiligo: A critical incident analysis. Journal of the American Academy of Dermatology. 1996;35(6):895-8.
- 19. Vallerand IA, Lewinson RT, Parsons LM, Hardin J, Haber RM, Lowerison MW, et al. Vitiligo and major depressive disorder: A bidirectional population-based cohort study. Journal of the American Academy of Dermatology. 2019;80(5):1371-9.

- 20. OPCRD. OPCRD The Optimum Patient Care Research Database 2016 [Available from: <a href="http://optimumpatientcare.org/opcrd/">http://optimumpatientcare.org/opcrd/</a>.
- 21. Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005;62(6):617-27.
- 22. John A, McGregor J, Fone D, Dunstan F, Cornish R, Lyons RA, et al. Case-finding for common mental disorders of anxiety and depression in primary care: an external validation of routinely collected data. BMC Medical Informatics and Decision Making. 2016;16(1):35.
- 23. Chan T, Cohen A, de Lusignan S. Using routine data to conduct small area health needs assessment through observing trends in demographics, recording of common mental health problems (CMHPs) and sickness certificates: longitudinal analysis of a northern and London locality. Informatics in primary care. 2010;18(4):273-82.
- 24. Trost LB, Bergfeld WF, Calogeras E. The diagnosis and treatment of iron deficiency and its potential relationship to hair loss. Journal of the American Academy of Dermatology. 2006;54(5):824-44.
- 25. Department for Communities and Local Government. The English Indices of Deprivation. 2015.2015. Available from: <a href="https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015">https://www.gov.uk/government/statistics/english-indices-of-deprivation-2015</a>.
- 26. Office for National Statistics. Ethnicity2018 2nd January 2020. Available from: <a href="https://www.ons.gov.uk/peoplepopulationandcommunity/culturalidentity/ethnicity">https://www.ons.gov.uk/peoplepopulationandcommunity/culturalidentity/ethnicity</a>.
- 27. Tippu Z, Correa A, Liyanage H, Burleigh D, McGovern A, Van Vlymen J, et al. Ethnicity Recording in Primary Care Computerised Medical Record Systems: An Ontological Approach. J Innov Health Inform. 2017;23(4):920.
- 28. Kumar S, de Lusignan S, McGovern A, Correa A, Hriskova M, Gatenby P, et al. Ischaemic stroke, haemorrhage, and mortality in older patients with chronic kidney disease newly started on anticoagulation for atrial fibrillation: a population based study from UK primary care. Bmj. 2018;360:k342.
- 29. Rayner LH, Mcgovern A, Sherlock J, Gatenby P, Correa A, Creagh-Brown B, et al. The impact of therapy on the risk of asthma in type 2 diabetes. Clin Respir J. 2019;13(5):299-305.
- 30. de Lusignan S, Liaw ST, Michalakidis G, Jones S. Defining datasets and creating data dictionaries for quality improvement and research in chronic disease using routinely collected data: an ontology-driven approach. Informatics in primary care. 2011;19(3):127-34.
- 31. Benchimol EI, Smeeth L, Guttmann A, Harron K, Moher D, Petersen I, et al. The REporting of studies Conducted using Observational Routinely-collected health Data (RECORD) statement. PLoS Med. 2015;12(10):e1001885.

# Appendix 1

Codes to be used to identify cases of vitiligo and important exclusion conditions.

Read and SNOMED codes to be used to identify cases of vitiligo

| Read V2 Code | Term ID | Description |
|---|---|---|
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Leucoderma |
| M295z | All | Leucoderma NOS |
| Read CTV3 Code | Term ID | Description |
| M2951 | All | Vitiligo |
| M293. | All | Hypopigmentation disorder |
| F4E53 | All | Vitiligo of eyelid |
| M295. | All | Acquired hypomelanosis |
| M295z | All | Leucoderma NOS |
| SNOMED Code | Term ID | Description |
| 56727007 | | Vitiligo (disorder) |
| 87666009 | | Vitiligo of eyelid (disorder) |
| 721539008 | | Vitiligo of eyelid and periocular area (disorder) |
| 403271008 | | Kobner vitiligo (disorder) |
| 403270009 | | Trichrome vitiligo (disorder) |
| 403267005 | | Localised vitiligo (disorder) |
| 403268000 | | Segmental vitiligo (disorder) |
| 402621008 | | Idiopathic vitiligo (disorder) |
| 403269008 | | Generalised vitiligo (disorder) |
| 330931000119106 | | Vitiligo of skin of left eyelid and periocular area (disorder) |
| 330931000119104 | | Vitiligo of skin of right eyelid and periocular area (disorder) |
| 330911000119101 | | Vitiligo of skin of left upper eyelid and periocular area (disorder) |
| 330881000119101 | | Vitiligo of skin of right upper eyelid and periocular area (disorder) |
| 726608002 | | Spastic paraparesis, vitiligo, premature greying, characteristic facies syndrome |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 89031001 | | Hypopigmentation (morphological abnormality) |
| 68210006 | | Hypopigmentation of eyelid |
| 18655006 | | Dipigmentation |
| 23267004 | | Achromia of skin (disorder) |
| 402807009 | | Circumscribed hypomelanosis (disorder) |

Read codes and SNOMED codes to be used to identify alternative depigmenting disorders for exclusion

| Congenital and Genetic | Hypomela | noses |
|---|---|---|
| Read V2 Code | Term ID | Description |
| C302A | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| PKy54 | All | Waardenburg's syndrome |
| C3029 | All | Hermansky-Pudlak |
| PKy92 | All | Menke's syndrome |
| Read CTV3 Code | Term ID | Description |
| X78Ve | All | Hypomelanosis of Ito |
| XaZqX | All | Piebaldism |
| PK5 | All | Tuberous sclerosis |
| X78E7 | All | Ash leaf spot, tuberous sclerosis |
| X78E8 | All | Shargreen patch |
| X78E9 | All | Adenoma sebaceum |
| X20Ex | All | Hermansky-Pudlak syndrome |
| X20ij | All | Griscelli syndrome with immunodeficiency |
| PKy92 | All | Menkes syndrome |
| SNOMED Code | Term ID | Description |
| 218358001 | | Incontinentia pigmenti achromians syndrome (disorder) |
| 718122005 | | Piebaldism (disorder) |
| 7199000 | | Tuberous sclerosus syndrome (disorder) |
| 254243001 | | Ash leaf spot, tuberous sclerosis (disorder) |
| 36025004 | | Fibrous skin tumor of tuberous sclerosis (disorder) |
| 254244007 | | Shagreen patch (disorder) |
| 9311003 | | Hermansky-Pudlak syndrome (disorder) |
| 37548006 | | Hypopigmentation-immunodeficiency disease (disorder) |
| 59178007 | | Menkes kinky-hair syndrome (disorder) |
| 47434006 | | Waardenburg's syndrome (disorder) |
| 715952000 | | Waardenburg syndrome co-occurrent with Hirschsprung disease (disorder) |
| 773575001 | | Ocular albinism with congenital sensorineural deafness (disorder) |
| 765325002 | | Peripheral demyelinating neuropathy, central dysmyelinating leukodystrophy, Waardenburg syndrome, Hirschsprung disease (disorder) |
| Post-inflammatory Hyp | omelanose | S |
| Read V2 Code | Term ID | Description |
| M2920 | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |
| M1700 | All | Lichen planus actinicus |
| M1701 | All | Lichen planus annularis |
| M1702 | All | Lichen planus atrophicus |
| M1703 | All | Lichen planus bullosus |
| M1704 | All | Lichen planus hypertrophicus |
| M1705 | All | Lichen planus linearis |
| M1707 | All | Lichen planus obtusus |
| M1708 | All | Subacute active lichen planus |

| M1709 | All | Follicular lichen planus |
|---|---|---|
| M170z | All | Lichen planus NOS |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus and atrophicus |
| K276. | All | Balanitis xerotica obliterans |
| Read CTV3 Code | Term ID | Description |
| Xa0WM | All | Post inflammatory hypopigmentation |
| M170. | All | Lichen planus |
| X507Y | All | Confluent lichen planus |
| X507Z | All | Micropaplular lichen planus |
| X507a | All | Guttate lichen planus |
| X507b | All | Follicular lichen planus |
| M1703 | All | Bullous lichen planus |
| M1701 | All | Annular lichen planus |
| M1704 | All | Hypertrophic lichen planus |
| M1702 | All | Atrophic lichen planus |
| M1705 | All | Linear lichen planus |
| X507c | All | Zosteriform lichen planus |
| M1700 | All | Acintic lichen planus |
| X507d | All | Post inflammatory hyperpigmentation in lichen planus |
| X507e | All | Wickham's striae in lichen planus |
| X507f | All | Lichen planus - lupus erythematosus overlap |
| X507g | All | Lichen planus pemphigoides |
| X507h | All | Site-specific lichen planus |
| X507i | All | Lichen planus of scalp |
| X507j | All | Lichen planus of palms and soles |
| X507k | All | Ulcerative lichen planus of palms and soles |
| X507n | All | Mutilating lichen planus of fingers and toes |
| X507I | All | Lichen planus of nail |
| X507w | All | Genital lichen planus |
| X408F | All | Lichen planus of vuvla |
| X507y | All | Erosive lichen planus of vulva |
| X507z | All | Lichen planus of penis |
| X5080 | All | Lichen planus of glans penis |
| M1707 | All | Lichen planus obtusus |
| M1708 | All | Subacute active lichen planus |
| M170z | All | Lichen planus NOS |
| Myu32 | All | [X]Other lichen planus |
| M17y0 | All | Lichen ruber moniliforme |
| M1650 | All | Pityriasis alba |
| M2102 | All | Lichen sclerosus |
| X50FC | All | Genital lichen sclerosus |
| K276. | All | Balanitis xerotica obliterans |

| X50FE | All | Lichen sclerosus of vulva |
|---|---|---|
| X50FF | All | Extra genital lichen sclerosus |
| X50FG | All | Guttate lichen sclerosus |
| SNOMED Code | Term ID | Description |
| 277787003 | | Post-inflammatory hypopigmentation (disorder) |
| 403272001 | | Post-infective hypomelanosis (disorder) |
| 403276003 | | Acquired hypomelanosis of uncertain etiology (disorder) |
| 4776004 | | Lichen planus (disorder) |
| 263797007 | | Lichen planus-like (qualifier value) |
| 4459000 | | Linear lichen planus (disorder) |
| 6111009 | | Bullous lichen planus (disorder) |
| 238666005 | | Lichen planus of lips (disorder) |
| 201001005 | | Lichen planus obtusus (disorder) |
| 200999007 | | Actinic lichen planus (disorder) |
| 238658001 | | Lichen planus of nail (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 201000006 | | Annular lichen planus (disorder) |
| 238647005 | | Guttate lichen planus (disorder) |
| 237112004 | | Lichen planus of vulva (disorder) |
| 400108007 | | Flexural lichen planus (disorder) |
| 238655003 | | Lichen planus of scalp (disorder) |
| 44509000 | | Linear lichen planus (disorder) |
| 25858008 | | Atrophic lichen planus (disorder) |
| 238670002 | | Lichen planus of penis (disorder) |
| 238645002 | | Confluent lichen planus (disorder) |
| 717061002 | | Lichen planus pigmentosus (disorder) |
| 238648000 | | Zosteriform lichen planus (disorder) |
| 238653005 | | Lichen planus pemphigoides (disorder) |
| 68266006 | | Hypertrophic lichen planus (disorder) |
| 238646001 | | Micropapular lichen planus (disorder) |
| 64540004 | | Lichen planopilaris (disorder) |
| 238654004 | | Site-specific lichen planus (disorder) |
| 238652000 | | Lichen planus-lupus erythematosus overlap (disorder) |
| 403198004 | | Lichenoid actinic keratosis (disorder) |
| 723003004 | | Acute eruptive lichen planus (disorder) |
| 238671003 | | Lichen planus of glans penis (disorder) |
| 68266006 | | Hypertrophic lichen planus (disorder) |
| 201002003 | | Subacute active lichen planus (disorder) |
| 720493003 | | Annular atrophic lichen planus (disorder) |
| 238651007 | | Wickham's striae in lichen planus (disorder) |
| 201001005 | | Lichen planus obtusus (disorder) |
| 402349005 | | Chronic lichen planus (disorder) |
| 238668006 | | Genital lichen planus (disorder) |
| 238656002 | | Lichen planus of palms and soles (disorder) |
| 402352002 | | Poikiloderma due to lichen planus (disorder) |

| 721171007 | | Hypertrophic lichen planus of vulva (disorder) |
|---|---|---|
| 402348002 | | Köbner reaction from lichen planus (disorder) |
| 238657006 | | Ulcerative lichen planus of palms and soles (disorder) |
| 238660004 | | Mutilating lichen planus of fingers and toes (disorder) |
| 726476005 | | Lichen planus co-occurrent with onycholysis (disorder) |
| 238649008 | | Post-inflammatory hyperpigmentation in lichen planus (disorder) |
| 402296004 | | Pityriasis alba (disorder) |
| 402298003 | | Diffuse pityriasis alba (disorder) |
| 402297008 | | Localised pityriasis alba (disorder) |
| 25674000 | | Lichen sclerosus et atrophicus (disorder) |
| 402423004 | | Adult lichen sclerosus (disorder) |
| 782666006 | | Lichen sclerosus of anus (disorder) |
| 238934003 | | Guttate lichen sclerosus (disorder) |
| 238932004 | | Genital lichen sclerosus (disorder) |
| 700082001 | | Lichen sclerosus of penis (disorder) |
| 26348009 | | Lichen sclerosus et atrophicus of the vulva (disorder) |
| 402424005 | | Childhood lichen sclerosus (disorder) |
| 403566002 | | Anogenital lichen sclerosus (disorder) |
| 238933009 | | Extragenital lichen sclerosus (disorder) |
| 402714001 | | Lichen sclerosus of male genitalia (disorder) |
| 402715000 | | Lichen sclerosus of female genitalia (disorder) |
| 402422009 | | Bullous extragenital lichen sclerosus (disorder) |
| 721199003 | | Prepubertal lichen sclerosus of vulva (disorder) |
| 403568001 | | Localized extragenital lichen sclerosus (disorder) |
| 402421002 | | Generalized extragenital lichen sclerosus (disorder) |
| 403564004 | | Lichen sclerosus of penis, childhood form (disorder) |
| 111023000 | | Lichen sclerosus et atrophicus, bullous type (disorder) |
| 403565003 | | Vulval lichen sclerosus, childhood form (disorder) |
| 198033005 | | Balanitis xerotica obliterans (disorder) |
| Post Traumatic Leukode | erma | |
| SNOMED Code | Term ID | Description |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 18655006 | | Depigmentation (morphologic abnormality) |
| 23006000 | | Hypopigmentation of skin (disorder) |
| 398656003 | | Acquired hypomelanotic disorder (disorder) |
| Para-Malignant Hypome | elanoses | |
| Read V2 Code | Term ID | Description |
| B621. | All | Mycosis fungoides |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6211 | All | Mycosis fungoides of lymph nodes of head, face and neck |
| B6212 | All | Mycosis fungoides of intrathoracic lymph nodes |
| B6213 | All | Mycosis fungoides of intra-abdominal lymph nodes |
| B6214 | All | Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6215 | All | Mycosis fungoides of lymph nodes of inguinal region and leg |
| <u> </u> | • | • |

| B6216 | All | Mycosis fungoides of intrapelvic lymph nodes |
|---|---|---|
| B6217 | All | Mycosis fungoides of spleen |
| B6218 | All | Mycosis fungoides of lymph nodes of multiple sites |
| B621z | All | Mycosis fungoides NOS |
| BBI | All | [M]Mycosis fungoides |
| BBIO. | All | [M]Mycosis fungoides |
| BBI1. | All | [M]Sezary's disease |
| BBIz. | All | [M]Mycosis fungoides NOS |
| B62xX | All | Oth and unspecif peripheral & cutaneous T-cell lymphomas |
| | All | Subcutaneous panniculitis like T-cell lymphoma |
| BBmD. | All | [M]Cutaneous lymphoma |
| B622. | All | Sezary's disease |
| B6220 | All | Sezary's disease of unspecified site |
| | All | Sezary's disease of lymph nodes of head, face and neck |
| B6222 | All | Sezary's disease of intrathoracic lymph nodes |
| B6223 | All | Sezary's disease of intra-abdominal lymph nodes |
| B6224 | All | Sezary's disease of lymph nodes of axilla and upper limb |
| B6225 | All | Sezary's disease of lymph nodes of inguinal region and leg |
| B6226 | All | Sezary's disease of intrapelvic lymph nodes |
| B6227 | All | Sezary's disease of spleen |
| | All | Sezary's disease of lymph nodes of multiple sites |
| B622z | All | Sezary's disease NOS |
| BBEA. | All | Amelanotic melanoma |
| Read CTV3 Code | Term ID | Description |
| B621. | All | Mycosis fungoides |
| XaQbT | All | Poikiloderma vasculare atrophicans |
| X78hm | All | Mycosis fungoides of skin |
| | /AII | |
| B6210 | All | Mycosis fungoides of unspecified site |
| B6210<br>B6211 | | |
| | All | Mycosis fungoides of unspecified site |
| B6211<br>B6212 | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck |
| B6211<br>B6212<br>B6213 | All<br>All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes |
| B6211<br>B6212<br>B6213<br>B6214 | All<br>All<br>All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes |
| B6211<br>B6212<br>B6213<br>B6214<br>B6215 | All All All All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb |
| B6211<br>B6212<br>B6213<br>B6214<br>B6215 | All All All All All All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 | AII AII AII AII AII AII | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 | AII | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 B621z B622. | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites Mycosis fungoides NOS |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 B621z B622. | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites Mycosis fungoides NOS Sezary's disease |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 B621z B622. B6220 | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites Mycosis fungoides NOS Sezary's disease Sezary's disease of unspecified site |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 B621z B6220 B6221 | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites Mycosis fungoides NOS Sezary's disease Sezary's disease of unspecified site Sezary's disease of lymph nodes of head, face and neck |
| B6211 B6212 B6213 B6214 B6215 B6216 B6217 B6218 B621z B6222 B6222 B6223 | All | Mycosis fungoides of unspecified site Mycosis fungoides of lymph nodes of head, face and neck Mycosis fungoides of intrathoracic lymph nodes Mycosis fungoides of intra-abdominal lymph nodes Mycosis fungoides of lymph nodes of axilla and upper limb Mycosis fungoides of lymph nodes of inguinal region and leg Mycosis fungoides of intrapelvic lymph nodes Mycosis fungoides of spleen Mycosis fungoides of lymph nodes of multiple sites Mycosis fungoides NOS Sezary's disease Sezary's disease of unspecified site Sezary's disease of lymph nodes of head, face and neck Sezary's disease of intrathoracic lymph nodes |

| B6226 | All | Sezary's disease of intrapelvic lymph nodes |
|---|---|---|
| B6227 | All | Sezary's disease of spleen |
| B6228 | All | Sezary's disease of lymph nodes of multiple sites |
| B622z | All | Sezary's disease NOS |
| X78hn | All | Sezary's disease of skin |
| X78hl | All | Cutaneous lymphoma |
| XaYin | All | Cutaneous follicle centre lymphoma |
| Xa0Sz | All | Cutaneous/peripheral T-cell lymphoma |
| XaYjf | All | Subcutaneous panniculitis like T-cell lymphoma |
| ByuDD | All | [X]0th and unspecif peripheral & cutaneous T-cell lymphomas |
| XaYjl | All | Primary cutaneous CD30 antigen positive large T-cell lymphoma |
| XaOCE | All | Amelanotic malignant melanoma of skin |
| SNOMED Code | Term ID | Description |
| 90120004 | | Mycosis fungoides (morphologic abnormality) |
| 118618005 | | Mycosis fungoides (disorder) |
| 765328000 | | Classic mycosis fungoides (disorder) |
| 404115006 | | Bullous mycosis fungoides (disorder) |
| 94714002 | | Mycosis fungoides of spleen (disorder) |
| 404117003 | | Spongiotic mycosis fungoides (disorder) |
| 681291000119105 | | History of mycosis fungoides (situation) |
| 418628003 | | Follicular mycosis fungoides (morphologic abnormality) |
| 404113004 | | Tumour stage mycosis fungoides (disorder) |
| 404118008 | | Syrngotropic mycosis fungoides (disorder) |
| 404112009 | | Granulomatous mycosis fungoides (disorder) |
| 404114005 | | Erythrodermic mycosis fungoides (disorder) |
| 404110001 | | Hypomelanocytic mycosis fungoides (disorder) |
| 404109006 | | Folliculotropic mycosis fungoides (disorder) |
| 404108003 | | Pokilodermatous mycosis fungoides (disorder) |
| 404107008 | | Patch/plaque stage mycosis fungoides (disorder) |
| 404116007 | | Mycosis fungoides with systemic infiltration (disorder) |
| 94708009 | | Mycosis fungoides of intrapelvic lymph nodes (disorder) |
| 94707004 | | Mycosis fungoides of intra-abdominal lymph nodes (disorder) |
| 188627002 | | Mycosis fungoides of lymph nodes of multiple sites (disorder) |
| 404111002 | | Lymphomatoid papulosis-associated mycosis fungoides (disorder) |
| 404104001 | | Lymphomatoid papulosis type B mycosis fungoides-like (disorder) |
| 94715001 | | Mycosis fungoides of extranodal AND/OR solid organ site (disorder) |
| 94709001 | | Mycosis fungoides of intrathoracic lymph nodes (disorder) |
| 94711005 | | Mycosis fungoides of lymph nodes of head, face AND/OR neck (disorder) |
| 94710006 | | Mycosis fungoides of lymph nodes of axilla AND/OR upper limb (disorder) |
| 188627002 | | Mycosis fungoides of lymph nodes of multiple sites (disorder) |
| 94712003 | | Mycosis fungoides of lymph nodes of inguinal region AND/OR lower limb (disorder) |
| 28054005 | | Cutaneous T-cell lymphoma, no International Classification of Diseases for oncology subtype (morphologic abnormality) |

| 40012207 | Primary cutaneous T-cell lymphoma (disorder) |
|---|---|
| 277613000 | Cutaneous/peripheral T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutanoeus T-cell lymphoma (disorder) |
| 419283005 | Primary cutaneous T-cell lymphoma - category (morphologic abnormality) |
| 128804002 | Primary cutaneous CD30 antigen positive T-cell lymphoproliferative disorder (morphologic abnormality) |
| 450908002 | Primary cutaneous gamma-delta T-cell lymphoma (morphologic abnormality) |
| 122571000119106 | History of primary cutaneous T-cell lymphoma (situation) |
| 419018000 | Primary cutaneous large T-cell lymphoma - category (morphologic abnormality) |
| 402880009 | Primary cutaneous large T-cell lymphoma (disorder) |
| 404133000 | Subcutaneous panniculitic cutaneous T-cell lymphoma (disorder) |
| 404128004 | CD-30 negative cutaneous T-cell lymphoma (disorder) |
| 787198005 | Primary cutaneous acral CD8 positive T-cell lymphoma (morphologic abnormality) |
| 397352006 | Primary cutaneous anaplastic large T-cell lymphoma, CD30-positive (morphologic abnormality) |
| 733627006 | Primary cutaneous gamma-delta-positive T-cell lymphoma (disorder) |
| 404129007 | CD-30 negative anaplastic large T-cell cutaneous lymphoma (disorder) |
| 122571000119106 | History of malignant cutaneous T-cell lymphoma (situation) |
| 404130002 | CD-30 negative pleomorphic large T-cell cutaneous lymphoma (disorder) |
| 404126000 | CD-30 positive pleomorphic large T-cell cutaneous lymphoma (disorder) |
| 419283005 | Primary cutaneous T-cell lymphoma - category (morphologic abnormality) |
| 450908002 | Primary cutaneous gamma-delta T-cell lymphoma - category (morphologic abnormality) |
| 765136002 | Primary cutaneous CD8 positive aggressicve epidermotropic cytotoxic T-cell lymphoma (disorder) |
| 128875000 | Primary cutaneous CD30 antigen positive large T-cell lymphoma (disorder) |
| 733895005 | Primary cutaneous CD8 positive aggressicve epidermotropic cytotoxic T-cell lymphoma (morphologic abnormality) |
| 419586003 | Primary cutaneous T-cell lymphoma, large cell, CD30-negative (morphological abnormality) |
| 118611004 | Sezary's disease (disorder) |
| 4950009 | Sezary's disease (morphologic abnormality) |
| 255101006 | Sezary disease of skin (disorder) |
| 95263006 | Sezary's disase of spleen (disorder) |
| 188632001 | Sezary's disase of intra-abdominal lymph nodes (disorder) |
| 188635004 | Sezary's disase of intrapelvic lymph nodes (disorder) |
| 188631008 | Sezary's disase of intrathoracic lymph nodes (disorder) |
| 188637007 | Sezary disease of lymph nodes of multiple sites (disorder) |
| 95264000 | Sézary's disease of extranodal AND/OR solid organ site (disorder) |
| 188633006 | Sézary's disease of lymph nodes of axilla and upper limb (disorder) |
| 95260009 | Sézary's disease of lymph nodes of head, face AND/OR neck (disorder) |
| 188634000 | Sézary's disease of lymph nodes of inguinal region and lower limb (disorder) |

| | | Sézary's disease of lymph nodes of inguinal region AND/OR lower limb |
|---|---|---|
| 95261008 | | (disorder) |
| 419392005 | | Primary cutaneous lymphoma (morphologic abnormality) |
| | | Tumour and germline whole genome sequencing for anaplastic |
| 8232100000106 | | lymphoma kinase negative anaplastic large cell lymphoma including primary cutaneous subtypes (procedure) |
| 403274000 | | Hypomelanosis surrounding malignant melanoma (disorder) |
| 402563000 | | Metastatic malignant melanoma with diffuse hypermelanosis (disorder) |
| 276751004 | | Amelanotic malignant melanoma of skin (disorder) |
| 70594002 | | Amelanotic melanoma (morphologic abnormality) |
| 404110001 | | Hypomelanotic mycosis fungoides (disorder) |
| 402623006 | | Hypomelanosis surrounding melanocytic neoplasm (disorder) |
| Occupational/drug indu | uced hypon | |
| Read V2 Code | Term ID | Description |
| M293. | All | Hypopigmentation |
| Read CTV3 Code | Term ID | Description |
| X508z | All | Occupational vitiligo |
| X78VE | All | Chemically-induced hypomelanosis |
| X50Gx | All | Drug-induced hypomelanosis |
| Xa1aV | All | Chemically-induced hypomelanosis |
| M2950 | All | Leucoderma aestivale |
| M295. | All | Acquired hypomelanosis |
| SNOMED Code | Term ID | Description |
| 238713002 | | Occupational vitiligo (disorder) |
| 280962005 | | Chemically-induced hypomelanosis (disorder) |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 403807001 | | Phylloid hypomelanosis (disorder) |
| 398656003 | | Acquired hypomelanotic disorder (disorder) |
| 238999005 | | Drug-induced hypomelanosis (disorder) |
| 403698000 | | Laser-induced hypopigmentation (disorder) |
| 402622001 | | Hypomelanosis due to scarring (disorder) |
| 280962005 | | Chemically-induced hypomelanosis (disorder) |
| 403692004 | | Hypomelanosis due to cryotherapy (disorder) |
| 403744007 | | Arsenic-induced "rain-drop" hypomelanosis (disorder) |
| 403698000 | | Laser-induced hypopigmentation (disorder) |
| 201290009 | | Leukoderma estivale (disorder) |
| Para-infectious hypopig | | |
| Read V2 Code | Term ID | Description |
| | All | Pityriasis versicolor |
| AB10. | All | |
| AB10. Read CTV3 Code | Term ID | Description |
| | | <b>Description</b> Pityriasis versicolor |
| Read CTV3 Code | Term ID | |
| Read CTV3 Code AB10. | Term ID | Pityriasis versicolor |

| 721794002 | | Infection caused by Malassezia (disorder) |
|---|---|---|
| 402133004 | | Malassezia infection of the skin (disorder) |
| 29619007 | | Malassezia furfur (organism) |
| - | - | oea, Idiopathic guttate hypomelanosis, Xeroderma pigmentosum, |
| Read V2 Code | Term ID | Description Cutaneous sarcoidosis) |
| M290. | All | Melasma |
| M2900 | All | Chloasma bronzinum |
| M2901 | All | Chloasma cachecticorum |
| M2902 | All | Chloasma caloricum |
| M2903 | All | Chloasma gravidarum |
| M2903 | All | Chloasma gravidarum |
| M2903 | All | Chloasma gravidarum |
| M290z | All | Chloasma NOS |
| M2103 | All | Morphoea |
| M2104 | All | Linear Morphoea |
| M210. | All | Circumscribed scleroderma |
| M2100 | All | Unspecified circumscribed scleroderma |
| M2101 | All | Localised dermatosclerosis |
| M210z | All | Circumscribed scleroderma NOS |
| PH322 | All | Xeroderma pigmentosum |
| BBE9. | All | [M]Nonpigmented naevus |
| AD530 | All | Lupus Pernio |
| AD53. | All | Sarcoidosis of skin |
| Read CTV3 Code | Term ID | Description |
| M290. | All | Melasma |
| Xa1aM | All | Drug-induced melasma |
| M2900 | All | Chloasma bronzinum |
| M2901 | All | Chloasma cachecticorum |
| M2902 | All | Chloasma caloricum |
| M2904 | All | Chloasma hepaticum |
| M2905 | All | Chloasma toxicum |
| M2906 | All | Chloasma traumaticum |
| M290z | All | Chloasma NOS |
| M2903 | All | Melasma of pregnancy |
| Xa1aM | All | Drug-induced melasma |
| M2103 | All | Morphoea |
| X7053 | All | Generalised morphoea |
| M2101 | All | Localised morphoea |
| M2100 | All | Unspecified circumscribed scleroderma |
| M210z | All | Circumscribed scleroderma NOS |
| X7055 | All | Linear morphoea |
| PH322 | All | Xeroderma pigmentosum |
| X78Cz | All | Xeroderma pigmentosum group A |
| X78D0 | All | Xeroderma pigmentosum group B |

| X78D1 | All | Xeroderma pigmentosum group C |
|-------------|---------|-----------------------------------------|
| X78D2 | All | Xeroderma pigmentosum group D |
| X78D3 | All | Xeroderma pigmentosum group E |
| X78D4 | All | Xeroderma pigmentosum group F |
| X78D5 | All | Xeroderma pigmentosum group G |
| X78D6 | All | Xeroderma pigmentosum XP variant |
| X78D7 | All | De Sanctis-Cacchione syndrome |
| X78D8 | All | Xerodermoid, pigmented |
| X50lw | All | Symmetrical progressive leucopathy |
| X20GW | All | Cutaneous sarcoid |
| X20GX | All | Orofacial sarcoid |
| X20GY | All | Lupus pernio |
| X5089 | All | Acute skin sarcoidosis |
| X508A | All | Sarcoidosis-induced erythema nodosum |
| X508B | All | Lofgrens syndrome |
| X508C | All | Maculopapular sarcoidosis |
| X508D | All | Chronic skin sarcoidosis |
| X508E | All | Sarcoidosis in scar |
| X508F | All | Papular sarcoidosis |
| X508G | All | Lichenoid sarcoidosis |
| X508H | All | Nodular sarcoidosis |
| X508I | All | Angiolupoid sarcoidosis |
| X00YQ | All | Sarcoid skin of eyelid |
| X20G5 | All | Sarcoid dactylitis |
| X50Dy | All | Subacute nodular migratory panniculitis |
| X50Dz | All | Subcutaneous lipogranulomatosis |
| SNOMED Code | Term ID | Description |
| 36209000 | | Melasma |
| 201274009 | | Chloasma bronzinum (disorder) |
| 201275005 | | Chloasma cachecticorum (disorder) |
| 201276006 | | Chloasma caloricum (disorder) |
| 201277002 | | Chloasma hepaticum (disorder) |
| 201278007 | | Chloasma toxicum (disorder) |
| 280955001 | | Drug-induced melasma (disorder) |
| 79840007 | | Idiopathic chloasma (disorder) |
| 111208003 | | Melasma gravidarum (disorder) |
| 54397000 | | Symptomatic chloasma (disorder) |
| 201279004 | | Chloasma traumaticum (disorder) |
| 201049004 | | Morphea (disorder) |
| 128458002 | | Plaque morphea (disorder) |
| 22784002 | | Linear scleroderma (disorder) |
| 403521006 | | Guttate morphea (disorder) |
| 201048007 | | Localised morphea (disorder) |
| 7513007 | | Generalized morphea (disorder) |

| 403522004 | Subcutaneous morphea (disorder) |
|---|---|
| 51156002 | Coup de sabre scleroderma (disorder) |
| 403523009 | Disabling pansclerotic morphea of children (disorder) |
| 128460000 | Diffuse cutaneous scleroderma (disorder) |
| 403524003 | Scleroderma-like secondary cutaneous sclerosis (disorder) |
| 1717003 | Idiopathic guttate hypomelanosis (disorder) |
| 711154007 | Guttate hypopigmentation and punctate palmoplantar keratoderma with or without ectopic calcification (disorder) |
| 44600005 | Xeroderma pigmentosum (disorder) |
| 56048001 | Xeroderma pigmentosum, group E (disorder) |
| 25784009 | Xeroderma pigmentosum, group C (disorder) |
| 36454001 | Xeroderma pigmentosum, group G (disorder) |
| 1073003 | Xeroderma pigmentosum, group B (disorder) |
| 68637004 | Xeroderma pigmentosum, group D (disorder) |
| 42530008 | Xeroderma pigmentosum, group F (disorder) |
| 43477006 | Xeroderma pigmentosum, group A (disorder) |
| 73663008 | Neurologic xeroderma pigmentosum (disorder) |
| 88877002 | Xeroderma pigmentosum, variant form (disorder) |
| 7806002 | Non-neurologic xeroderma pigmentosum (disorder) |
| 719819004 | Xeroderma pigmentosum and Cockayne syndrome complex (disorder) |
| 239083007 | Symmetrical progressive leucopathy (disorder) |
| 763368004 | Familial progressive hyper and hypopigmentation of skin (disorder) |
| 403541001 | Nevus depigmentosus |
| 112680001 | Naevus depigmentosus |
| 55941000 | Cutaneous sarcoidosis (disorder) |
| 238680003 | Papular sarcoidosis (disorder) |
| 238679001 | Sarcoidosis in scar (disorder) |
| 402369000 | Atrophic sarcoidosis (disorder) |
| 402371000 | Verrucous sarcoidosis (disorder) |
| 238681004 | Lichenoid sarcoidosis (disorder) |
| 238674006 | Acute skin sarcoidosis (disorder) |
| 402370004 | Ulcerative sarcoidosis (disorder) |
| 58870009 | Sarcoidosis, anular type (disorder) |
| 54515008 | Sarcoidosis, plaque type (disorder) |
| 80941006 | Subcutaneous sarcoidosis (disorder) |
| 870334009 | Palmoplantar sarcoidosis (disorder) |
| 238678009 | Chronic skin sarcoidosis (disorder) |
| 238677004 | Maculopapular sarcoidosis (disorder) |
| 402368008 | Ichthyosiform sarcoidosis (disorder) |
| 402373002 | Hypomelanotic sarcoidosis (disorder) |
| 9529007 | Sarcoidosis, erythrodermic type (disorder) |
| 72470008 | Sarcoidosis, lupus pernio type (disorder) |
| 402372007 | Subcutaneous nodular sarcoidosis (disorder) |
| 238675007 | Sarcoidosis-induced erythema nodosum (disorder) |
| 238676008 | Lofgrens syndrome (disorder) |

| 31541009 | Lupus pernio of Besnier |
|-----------|-----------------------------------|
| 231799005 | Sarcoid skin of eyelid (disorder) |

## **Appendix 2**

Potential differential diagnoses for vitiligo which will be used as exclusion criteria if they appear as diagnoses in the medical record within six months of the initial diagnosis of vitiligo (six months before or after the vitiligo diagnosis). \*As these conditions are extremely uncommon in the UK they will not be used in the exclusion process. Codes for these conditions are listed in Appendix 1.

| Condition group | Conditions/causes included |
|---|---|
| Congenital and genetic hypomelanoses | Piebaldism |
| | Tuberous sclerosis |
| | Hypomelanosis of Ito |
| | Waardenburg syndrome |
| | Hermanski-Pudlak syndrome |
| | Griscelli syndrome |
| | Menkes syndrome |
| Post-inflammatory hypomelanoses | Post-inflammatory leukoderma including after |
| | Atopic eczema or Psoriasis |
| | Lichen planus |
| | Pityriasis alba |
| | Lichen sclerosus |
| Post traumatic leukoderma | Post traumatic leukoderma |
| Para-malignant hypomelanoses | Cutaneous T-cell lymphoma (mycosis fungoides) |
| | Melanoma associated depigmentation |
| Occupational/drug induced | Occupational vitiligo |
| hypomelanoses | Other induced hypomelanoses |
| Para-infectious hypopigmentation | Pityriasis versicolor (or tinea versicolor) |
| | Leprosy* |
| | Leishmaniasis* |
| Others | Melasma |
| | Morphoea |
| | Idiopathic guttate hypomelanosis |
| | Xeroderma pigmentosum |
| | Progressive macular hypomelanosis |
| | Nevus depigmentosus |
| | Cutaneous sarcoidosis |

# Appendix 3

Read and SNOMED codes to be used to identify mental health conditions and related clinical entities (mental health symptoms and treatments) used to correctly identify people with mental health conditions. The full algorithms used to identify these conditions are described elsewhere (22).

| Depressive Episode | Depressive Episode | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| E0013 | All | Presenile dementia with depression |
| E0021 | All | Senile dementia with depression |
| E112. | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E118. | All | Seasonal affective disorder |
| E11y2 | All | Atypical depressive disorder |
| E11z2 | All | Masked depression |
| E130. | All | Reactive depressive psychosis |
| E135. | All | Agitated depression |
| E2003 | All | Anxiety with depression |
| E291. | All | Prolonged depressive reaction |
| E2B | All | Depressive disorder NEC |
| E2B1. | All | Chronic depression |
| E2B0. | All | Postviral depression |
| Eu204 | All | [X]Post-schizophrenic depression |
| Eu251 | All | [X]Schizoaffective disorder, depressive type |
| Eu32. | All | [X]Depressive episode |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu322 | All | [X]Severe depressive episode without psychotic symptoms |
| Eu323 | All | [X]Severe depressive episode with psychotic symptoms |
| Eu324 | All | [X]Mild depression |
| Eu325 | All | [X]Major depression, mild |
| Eu326 | All | [X]Major depression, moderately severe |

| Eu327 | All | [X]Major depression, severe without psychotic symptoms |
|---|---|---|
| Eu328 | All | [X]Major depression, severe with psychotic symptoms |
| Eu32y | All | [X]Other depressive episodes |
| Eu32z | All | [X]Depressive episode, unspecified |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| Eu332 | All | [X]Recurrent depressive disorder, current episode severe without |
| Eu333 | All | psychotic symptoms [X]Recurrent depressive disorder, current episode severe with psychotic symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Eu412 | All | [X]Mixed anxiety and depressive disorder |
| Read CTV3 Code | Term ID | Description |
| X00Sb | All | Mixed anxiety and depressive disorder |
| X00SO | All | Depressive disorder |
| X761L | All | Seasonal affective disorder |
| Xa0wV | All | Recurrent brief depressive disorder |
| X00SQ | All | Agitated depression |
| XE1YC | All | Reactive depression |
| XOOSR | All | Endogenous depression |
| XOOSS | All | Endogenous depression first episode |
| XE1Y0 | All | Single major depressive episode |
| E1120 | All | Single major depressive episode, unspecified |
| E1121 | All | Single major depressive episode, mild |
| E1122 | All | Single major depressive episode, moderate |
| E1123 | All | Single major depressive episode, severe, without mention of psychosis |
| E1124 | All | Single major depressive episode, severe, with psychosis |
| XaX53 | All | Single major depressive episode, severe, with psychosis, psychosis in remission |
| E1125 | All | Single major depressive episode, in partial or unspecified remission |
| E1126 | All | Single major depressive episode, in full remission |
| E112z | All | Single major depressive episode NOS |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| X00SU | All | Masked depression |
| E11y2 | All | Atypical depressive disorder |
| X00S8 | All | Post-schizophrenic depression |
| XSEGJ | All | Major depressive disorder |
| XSKr7 | All | Cotard syndrome |
| XSGol | All | Moderate major depression |
| 73001 | 711 | moderate major depression |

| XSGok | All | Mild major depression |
|---|---|---|
| XSGom | All | Severe major depression without psychotic features |
| XSGon | All | Severe major depression without psychotic features |
| E1137 | All | Recurrent depression |
| E130. | All | Reactive depressive psychosis |
| E2B | All | Depressive disorder NEC |
| E2B0. | All | Postviral depression |
| E2B1. | All | Chronic depression |
| Eu320 | All | [X]Mild depressive episode |
| Eu321 | All | [X]Moderate depressive episode |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |
| | All | |
| XE1ZY | | [X]Severe depressive episode without psychotic symptoms |
| XE1ZZ | All | [X]Severe depressive episode with psychotic symptoms |
| XE1Za | All | [X]Other depressive episodes |
| XE1Zb | All | [X]Depressive episode, unspecified [X]Recurrent depressive disorder, current episode severe without |
| XE1Zd | All | psychotic symptoms |
| VE47- | A.II | [X]Recurrent depressive disorder, current episode severe with psychotic |
| XE1Ze | All | symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |
| XaB9J | All | Depression NOS |
| XaCHr | All | [X] Single episode agitated depression without psychotic symptoms |
| XaCHs | All | [X] Single episode major depression without psychotic symptoms |
| XaCls | All | Mild depression |
| XaClt | All | Moderate depression |
| XaClu | All | Severe depression |
| E0013 | All | Presenile dementia with depression |
| E0021 | All | Senile dementia with depression |
| SNOMED Code | Term ID | Description |
| 832007 | | Moderate major depression (disorder) |
| 2618002 | | Chronic recurrent major depressive disorder (disorder) |
| 14070001 | | Multi-infarct dementia with depression (disorder) |
| 14183003 | | Chronic major depressive disorder, single episode (disorder) |
| 15193003 | | Severe recurrent major depression with psychotic features, mood- |
| | | incongruent (disorder) |
| 15639000 | | Moderate major depression, single episode (disorder) |
| 18818009 | | Moderate recurrent major depression (disorder) |
| 19527009 | | Single episode of major depression in full remission (disorder) |
| 20250007 | | Severe major depression, single episode, with psychotic features, mood-incongruent (disorder) |
| 25922000 | | Major depressive disorder, single episode with postpartum onset (disorder) |
| 26852004 | | Primary degenerative dementia of the Alzheimer type, senile onset, with depression (disorder) |
| 28475009 | | Severe recurrent major depression with psychotic features (disorder) |
| 30605009 | | Major depression in partial remission (disorder) |
| 33078009 | | Severe recurrent major depression with psychotic features, mood-congruent (disorder) |
| 33135002 | | Recurrent major depression in partial remission (disorder) |
| 33736005 | | Severe major depression with psychotic features, mood-congruent (disorder) |

| 35489007 | Depressive disorder (disorder) |
|---|---|
| 36474008 | Severe recurrent major depression without psychotic features (disorder) |
| 36923009 | Major depression, single episode (disorder) |
| 38694004 | Recurrent major depressive disorder with atypical features (disorder) |
| 39809009 | Recurrent major depressive disorder with catatonic features (disorder) |
| 40379007 | Mild recurrent major depression (disorder) |
| 40568001 | Recurrent brief depressive disorder (disorder) |
| | Major depressive disorder, single episode with atypical features |
| 42925002 | (disorder) |
| 48589009 | Minor depressive disorder (disorder) |
| 58703003 | Postpartum depression (disorder) |
| 60099002 | Severe major depression with psychotic features, mood-incongruent (disorder) |
| 66344007 | Recurrent major depression (disorder) |
| 69392006 | Major depressive disorder, single episode with catatonic features (disorder) |
| 70747007 | Major depression single episode, in partial remission (disorder) |
| 71336009 | Recurrent major depressive disorder with postpartum onset (disorder) |
| 73867007 | Severe major depression with psychotic features (disorder) |
| 75084000 | Severe major depression without psychotic features (disorder) |
| 76441001 | Severe major depression, single episode, without psychotic features (disorder) |
| 77911002 | Severe major depression, single episode, with psychotic features, mood-congruent (disorder) |
| 79298009 | Mild major depression, single episode (disorder) |
| 79842004 | Stuporous depression (disorder) |
| 82218004 | Postoperative depression (disorder) |
| 83458005 | Agitated depression (disorder) |
| 84788008 | Menopausal depression (disorder) |
| 87414006 | Reactive depression (situational) (disorder) |
| 87512008 | Mild major depression (disorder) |
| 161469008 | History of depression (situation) |
| 191457008 | Senile dementia with depressive or paranoid features (disorder) |
| 191459006 | Senile dementia with depression (disorder) |
| 191466007 | Arteriosclerotic dementia with depression (disorder) |
| 191495003 | Drug-induced depressive state (disorder) |
| 191604000 | Single major depressive episode, severe, with psychosis (disorder) |
| 191610000 | Recurrent major depressive episodes, mild (disorder) |
| 191611001 | Recurrent major depressive episodes, moderate (disorder) |
| 191613003 | Recurrent major depressive episodes, severe, with psychosis (disorder) |
| 191616006 | Recurrent depression (disorder) |
| 191659001 | Atypical depressive disorder (disorder) |
| 191676002 | Reactive depressive psychosis (disorder) |
| 192046006 | Brief depressive adjustment reaction (disorder) |
| 192049004 | Prolonged depressive adjustment reaction (disorder) |
| 192079006 | Postviral depression (disorder) |
| 192080009 | Chronic depression (disorder) |
| 231485007 | Post-schizophrenic depression (disorder) |
| 231499006 | Endogenous depression first episode (disorder) |
| 231500002 | Masked depression (disorder) |
| 231504006 | Mixed anxiety and depressive disorder (disorder) |
| 237349002 | Mild postnatal depression (disorder) |
|---|---|
| 237350002 | Severe postnatal depression (disorder) |
| 237739002 | Pseudo-Cushings syndrome of depression (disorder) |
| 247803002 | Seasonal affective disorder (disorder) |
| 268621008 | Recurrent major depressive episodes (disorder) |
| 272022009 | Complaining of feeling depressed (finding) |
| 274948002 | Endogenous depression - recurrent (disorder) |
| 300706003 | Endogenous depression (disorder) |
| 310495003 | Mild depression (disorder) |
| 310496002 | Moderate depression (disorder) |
| 310497006 | Severe depression (disorder) |
| 319768000 | Recurrent major depressive disorder with melancholic features (disorder) |
| 320751009 | Major depression, melancholic type (disorder) |
| 321717001 | Involutional depression (disorder) |
| 366979004 | Depressed mood (finding) |
| 370143000 | Major depressive disorder (disorder) |
| 394924000 | Symptoms of depression (finding) |
| 395072006 | Counseling for postnatal depression (procedure) |
| 430852001 | Severe major depression, single episode, with psychotic features (disorder) |
| 450714000 | Severe major depression (disorder) |
| 704678007 | Depressed mood with postpartum onset (finding) |
| 712823008 | Acute depression (disorder) |
| 718636001 | Minimal depression (disorder) |
| 719592004 | Moderately severe major depression (disorder) |
| 719593009 | Moderately severe depression (disorder) |
| 720451004 | Minimal recurrent major depression (disorder) |
| 720452006 | Moderately severe recurrent major depression (disorder) |
| 720453001 | Moderately severe major depression single episode (disorder) |
| 720454007 | Minimal major depression single episode (disorder) |
| 720455008 | Minimal major depression (disorder) |
| 723928009 | Mood disorder with depressive symptoms caused by alcohol (disorder) |
| 723930006 | Mood disorder with mixed manic and depressive symptoms caused by alcohol (disorder) |
| 724676000 | Mood disorder with depressive symptoms caused by sedative (disorder) |
| 724677009 | Mood disorder with depressive symptoms caused by hypnotic (disorder) |
| 724678004 | Mood disorder with depressive symptoms caused by anxiolytic (disorder) |
| 724690002 | Mood disorder with depressive symptoms caused by cocaine (disorder) |
| 724757005 | Depressive symptoms due to primary psychotic disorder (disorder) |
| 726772006 | Major depression with psychotic features (disorder) |
| 762321000 | Mood disorder with depressive symptoms caused by opioid (disorder) |
| 762329003 | Mood disorder with depressive symptoms caused by stimulant (disorder) |
| 762336002 | Mood disorder with depressive symptoms caused by hallucinogen (disorder) |
| 762339009 | Mood disorder with depressive symptoms caused by volatile inhalant (disorder) |
| 762512002 | Mood disorder with depressive symptoms caused by synthetic cathinone (disorder) |
| 768835002 | Depression care management (procedure) |

| 788120007 | Antenatal depression (disorder) |
|---|---|
| 838529004 | Mood disorder with mixed depressive and manic symptoms caused by |
| 838529004 | amfetamine and amfetamine derivative (disorder) |
| 871840004 | Episode of depression (finding) |
| 251000119105 | Severe major depression, single episode (disorder) |
| 281000119103 | Severe recurrent major depression (disorder) |
| 10211000132109 | Perinatal depression (disorder) |
| 94631000119100 | Depressive disorder in mother complicating pregnancy (disorder) |
| 133121000119109 | Severe seasonal affective disorder (disorder) |
| 142001000119106 | Depressed mood in Alzheimers disease (disorder) |
| 199111000000100 | Referral for guided self-help for depression (procedure) |
| 286711000000107 | Counseling for depression (procedure) |
| 288751000119101 | Reactive depressive psychosis, single episode (disorder) |
| 361761000000106 | On full dose long term treatment for depression (finding) |
| 755321000000106 | Single major depressive episode, severe, with psychosis, psychosis in remission (disorder) |
| 755331000000108 | Recurrent major depressive episodes, severe, with psychosis, psychosis in remission (disorder) |
| 764611000000100 | Recurrent major depressive episodes, severe (disorder) |
| 764691000000109 | Recurrent major depressive episodes, in partial remission (disorder) |
| 764701000000109 | Recurrent major depressive episodes, in remission (disorder) |
| 764711000000106 | Single major depressive episode, in remission (disorder) |
| 923921000000104 | Referral for depression self-help video (procedure) |
| 1086471000000100 | Recurrent reactive depressive episodes, severe, with psychosis (disorder) |
| 1086661000000100 | Reactive depression, prolonged single episode (disorder) |
| 1086671000000100 | Reactive depression, single episode (disorder) |
| 1086681000000100 | Reactive depression, recurrent (disorder) |
| 1086691000000100 | Reactive depression, first episode (disorder) |
| 1089511000000100 | Recurrent depression with current severe episode and psychotic features (disorder) |
| 1089631000000100 | Recurrent depression with current severe episode without psychotic features (disorder) |
| 1089641000000100 | Recurrent depression with current moderate episode (disorder) |
| 10811121000119100 | Major depressive disorder in mother complicating childbirth (disorder) |
| 10811161000119100 | Major depressive disorder in mother complicating pregnancy (disorder) |
| 10835871000119100 | Depressive disorder in mother complicating childbirth (disorder) |
| 16238181000119100 | Depressive disorder caused by amphetamine (disorder) |
| 16238221000119100 | Depressive disorder caused by methamphetamine (disorder) |
| 16264621000119100 | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100 | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |
| 16264901000119100 | Recurrent moderate major depressive disorder co-occurrent with anxiety (disorder) |
| 16265301000119100 | Recurrent major depressive disorder in partial remission co-occurrent with anxiety (disorder) |
| 16265951000119100 | Mild major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266831000119100 | Moderate major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266991000119100 | Severe major depressive disorder co-occurrent with anxiety single episode (disorder) |
| <b>Recurrent Depressive Disorder</b> | |

| Read V2 Code | Term ID | Description |
|---|---|---|
| E113. | All | Recurrent major depressive episode |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E1137 | All | Recurrent depression |
| E113z | All | Recurrent major depressive episode NOS |
| E2B1. | All | Chronic depression |
| Eu32A | All | [X]Recurrent major depressive episodes, severe, with psychosis, psychosis in remission |
| Eu33. | All | [X]Recurrent depressive disorder |
| Eu330 | All | [X]Recurrent depressive disorder, current episode mild |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| Eu332 | All | [X]Recurrent depressive disorder, current episode severe without psychotic symptoms |
| Eu333 | All | [X]Recurrent depressive disorder, current episode severe with psychotic symptoms |
| Eu334 | All | [X]Recurrent depressive disorder, currently in remission |
| Eu33y | All | [X]Other recurrent depressive disorders |
| Eu33z | All | [X]Recurrent depressive disorder, unspecified |
| Read CTV3 Code | Term ID | Description |
| Xa0wV | All | Recurrent brief depressive disorder |
| XM1GC | All | Endogenous depression - recurrent |
| E1130 | All | Recurrent major depressive episodes, unspecified |
| E1131 | All | Recurrent major depressive episodes, mild |
| E1132 | All | Recurrent major depressive episodes, moderate |
| E1133 | All | Recurrent major depressive episodes, severe, without mention of psychosis |
| E1134 | All | Recurrent major depressive episodes, severe, with psychosis |
| XaX54 | All | Recurrent major depressive episodes, severe, with psychosis, psychosis in remission |
| E1135 | All | Recurrent major depressive episodes, in partial or unspecified remission |
| E1136 | All | Recurrent major depressive episodes, in full remission |
| E113z | All | Recurrent major depressive episode NOS |
| E1137 | All | Recurrent depression |
| E2B1. | All | Chronic depression |
| Eu331 | All | [X]Recurrent depressive disorder, current episode moderate |
| XE1Y1 | All | Recurrent major depressive episodes |
| XE1Zd | All | [X]Recurrent depressive disorder, current episode severe without psychotic symptoms |
| XE1Ze | All | [X]Recurrent depressive disorder, current episode severe with psychotic symptoms |
| XE1Zf | All | [X]Recurrent depressive disorder, unspecified |
| SNOMED Code | Term ID | Description |
| | | Severe recurrent major depression with psychotic features, mood- |
| 15193003 | | incongruent (disorder) Recurrent mild major depressive disorder co-occurrent with anxiety |

| 16264821000119100 | | Recurrent severe major depressive disorder co-occurrent with anxiety |
|---|---|---|
| | | (disorder) Recurrent moderate major depressive disorder co-occurrent with |
| 16264901000119100 | | anxiety (disorder) |
| 16265061000119100 | | Recurrent major depressive disorder co-occurrent with anxiety in full remission (disorder) |
| 16265301000119100 | | Recurrent major depressive disorder in partial remission co-occurrent with anxiety (disorder) |
| 18818009 | | Moderate recurrent major depression (disorder) |
| 191610000 | | Recurrent major depressive episodes, mild (disorder) |
| 191611001 | | Recurrent major depressive episodes, moderate (disorder) |
| 191613003 | | Recurrent major depressive episodes, severe, with psychosis (disorder) |
| 2618002 | | Chronic recurrent major depressive disorder (disorder) |
| 268621008 | | Recurrent major depressive episodes (disorder) |
| 274948002 | | Endogenous depression - recurrent (disorder) |
| 281000119103 | | Severe recurrent major depression (disorder) |
| 28475009 | | Severe recurrent major depression with psychotic features (disorder) |
| 319768000 | | Recurrent major depressive disorder with melancholic features (disorder) |
| 33078009 | | Severe recurrent major depression with psychotic features, mood-congruent (disorder) |
| 33135002 | | Recurrent major depression in partial remission (disorder) |
| 36474008 | | Severe recurrent major depression without psychotic features (disorder) |
| 38694004 | | Recurrent major depressive disorder with atypical features (disorder) |
| 39809009 | | Recurrent major depressive disorder with catatonic features (disorder) |
| 40379007 | | Mild recurrent major depression (disorder) |
| 66344007 | | Recurrent major depression (disorder) |
| 68019004 | | Recurrent major depression in remission (disorder) |
| 71336009 | | Recurrent major depressive disorder with postpartum onset (disorder) |
| 720451004 | | Minimal recurrent major depression (disorder) |
| 720452006 | | Moderately severe recurrent major depression (disorder) |
| 755331000000108 | | Recurrent major depressive episodes, severe, with psychosis, psychosis in remission (disorder) |
| 764611000000100 | | Recurrent major depressive episodes, severe (disorder) |
| 764691000000109 | | Recurrent major depressive episodes, in partial remission (disorder) |
| 764701000000109 | | Recurrent major depressive episodes, in remission (disorder) |
| Depressive Symptoms | | |
| Read V2 Code | Term ID | Description |
| 1B17. | All | Depressed |
| 1B1U. | All | Symptoms of depression |
| 1BQ | All | Loss of capacity for enjoyment |
| 1BT | All | Depressed mood |
| 1BU | All | Loss of hope for the future |
| 2257 | All | O/E - depressed |
| Read CTV3 Code | Term ID | Description |
| XE0re | All | Depressed mood |
| XalmU | All | Symptoms of depression |
| X761E | All | Loss of capacity for enjoyment |
| X761G | All | Loss of hope for the future |
| | , | |
| Xa3Xh | All | Feeling of hopelessness |
| Xa3Xh<br>2257. | | Feeling of hopelessness O/E - depressed |

| Eu413 | All | [X]Other mixed anxiety disorders |
|---|---|---|
| Eu41z | All | [X]Anxiety disorder, unspecified |
| XE1Zj | All | [X]Other specified anxiety disorders |
| SNOMED Code | Term ID | Description |
| 1037451000000100 | | Referral for psychological management of anxiety (procedure) |
| 1053831000000100 | | Signposting to Anxiety UK (procedure) |
| 10586006 | | Occupation-related stress disorder (disorder) |
| 10743001000119100 | | Anxiety disorder in mother complicating childbirth (disorder) |
| 109006 | | Anxiety disorder of childhood OR adolescence (disorder) |
| 111487009 | | Dream anxiety disorder (disorder) |
| 11458009 | | Anticipatory anxiety, mild (finding) |
| 11806006 | | Separation anxiety disorder of childhood (disorder) |
| 12398201000119100 | | Anxiety disorder caused by methamphetamine (disorder) |
| 126943008 | | Separation anxiety (disorder) |
| 13438001 | | Overanxious disorder of childhood (disorder) |
| 15277004 | | Hallucinogen-induced anxiety disorder (disorder) |
| 161470009 | | History of anxiety state (situation) |
| 16264621000119100 | | Recurrent mild major depressive disorder co-occurrent with anxiety (disorder) |
| 16264821000119100 | | Recurrent severe major depressive disorder co-occurrent with anxiety (disorder) |
| 16264901000119100 | | Recurrent moderate major depressive disorder co-occurrent with anxiety (disorder) |
| 16265301000119100 | | Recurrent major depressive disorder in partial remission co-occurrent with anxiety (disorder) |
| 16265701000119100 | | Illness anxiety disorder (disorder) |
| 16265951000119100 | | Mild major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266831000119100 | | Moderate major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 16266991000119100 | | Severe major depressive disorder co-occurrent with anxiety single episode (disorder) |
| 162723006 | | On examination - anxious (finding) |
| 1686006 | | Sedative, hypnotic AND/OR anxiolytic-induced anxiety disorder (disorder) |
| 17496003 | | Organic anxiety disorder (disorder) |
| 191708009 | | Chronic anxiety (finding) |
| 191709001 | | Recurrent anxiety (finding) |
| 192108001 | | Disturbance of anxiety and fearfulness in childhood and adolescence (disorder) |
| 192611004 | | Childhood phobic anxiety disorder (disorder) |
| 197480006 | | Anxiety disorder (disorder) |
| 198288003 | | Anxiety state (finding) |
| 207363009 | | Anxiety neurosis (finding) |
| 21897009 | | Generalized anxiety disorder (disorder) |
| 225216003 | | Acknowledging anxiety (procedure) |
| 225624000 | | Panic attack (finding) |
| 22621000119103 | | Anxiety disorder caused by drug (disorder) |
| 228560001 | | Anxiety management training (procedure) |
| 231502005 | | Situational panic attack (finding) |
| 231503000 | | Non-situational panic attack (finding) |
| 231504006 | | Mixed anxiety and depressive disorder (disorder) |
| 231506008 | | Anxiety hysteria (finding) |

| 231528008 | Anxious personality disorder (disorder) |
|---|---|
| 247805009 | Anxiety and fear (finding) |
| 286644009 | Level of anxiety (finding) |
| 286710008 | Anxious character (finding) |
| 286711007 | Over-anxious character (finding) |
| 286712000 | Fearful character (finding) |
| 300895004 | Anxiety attack (finding) |
| 313087008 | Counseling for anxiety (procedure) |
| 34938008 | Alcohol-induced anxiety disorder (disorder) |
| 351861000000106 | Stranger anxiety (disorder) |
| 35429005 | Anticipatory anxiety (finding) |
| 35607004 | Panic disorder with agoraphobia (disorder) |
| 36646009 | Anticipatory anxiety, moderate (finding) |
| 371631005 | Panic disorder (disorder) |
| 37868008 | Anxiety disorder of adolescence (disorder) |
| 37872007 | Avoidant disorder of childhood OR adolescence (disorder) |
| 386808001 | Phobia (finding) |
| 386810004 | Phobic anxiety disorder (disorder) |
| 395017009 | Complaining of panic attack (finding) |
| 405051006 | Level of anxiety (observable entity) |
| 417676004 | On examination - panic attack (finding) |
| 43150009 | Panic disorder without agoraphobia with severe panic attacks (disorder) |
| 47372000 | Adjustment disorder with anxious mood (disorder) |
| 48694002 | Anxiety (finding) |
| 50026000 | Psychoactive substance-induced organic anxiety disorder (disorder) |
| 51493001 | Cocaine-induced anxiety disorder (disorder) |
| 51916003 | Biofeedback training by electroencephalogram application in anxiety (regime/therapy) |
| 52910006 | Anxiety disorder due to a general medical condition (disorder) |
| 53467004 | Anxiety disorder of childhood (disorder) |
| 53956006 | Panic disorder without agoraphobia with panic attacks in partial remission (disorder) |
| 5509004 | Panic disorder with agoraphobia AND severe panic attacks (disorder) |
| 55967005 | Phencyclidine-induced anxiety disorder (disorder) |
| 56576003 | Panic disorder without agoraphobia (disorder) |
| 5874002 | Anticipatory anxiety, severe (finding) |
| 61387006 | Moderate anxiety (finding) |
| 63909006 | Panic disorder with agoraphobia AND panic attacks in partial remission (disorder) |
| 64165008 | Avoidant disorder of childhood (disorder) |
| 65064003 | Panic disorder without agoraphobia with moderate panic attacks (disorder) |
| 69479009 | Anxiety hyperventilation (disorder) |
| 70997004 | Mild anxiety (finding) |
| 710060004 | Management of anxiety (procedure) |
| 710841007 | Assessment of anxiety (procedure) |
| 724708007 | Anxiety disorder caused by methylenedioxymethamphetamine (disorder) |
| 724722007 | Anxiety disorder caused by dissociative drug (disorder) |
| 724723002 | Anxiety disorder caused by ketamine (disorder) |
| 72861004 | Panic disorder without agoraphobia with mild panic attacks (disorder) |

| 737341006 | | Anxiety disorder caused by synthetic cannabinoid (disorder) |
|---|---|---|
| 762331007 | | Anxiety disorder caused by stimulant (disorder) |
| 788866004 | | Anxiety due to dementia (finding) |
| 80583007 | | Severe anxiety (panic) (finding) |
| 81350009 | | Free-floating anxiety (finding) |
| 8185002 | | Panic disorder with agoraphobia AND moderate panic attacks (disorder) |
| 82339009 | | Amphetamine-induced anxiety disorder (disorder) |
| 85061001 | | Separation anxiety disorder of childhood, early onset (disorder) |
| | | Provision of written information about generalised anxiety disorder |
| 858991000000101 | | (procedure) |
| 859891000000103 | | Able to manage anxiety (finding) |
| 861611000000100 | | Education about anxiety (procedure) |
| 89948007 | | Panic disorder with agoraphobia AND mild panic attacks (disorder) |
| 90790003 | | Avoidant disorder of adolescence (disorder) |
| 94641000119109 | | Anxiety in pregnancy (disorder) |
| Anxiety Symptoms | | |
| Read V2 Code | Term ID | Description |
| 1B13. | All | Anxiousness |
| 2258. | All | O/E - anxious |
| 1B12. | All | Nerves - nervousness |
| R2y2. | All | [D]Nervousness |
| 2259. | All | O/E - nervous |
| Read CTV3 Code | Term ID | Description |
| XE0rb | All | Anxiety |
| XE0ra | All | Nervousness |
| 1B1 | All | General nervous symptoms |
| 1B1Z. | All | General nervous symptom NOS |
| Xa7kB | All | Anxiety attack |
| 2258. | All | O/E - anxious |
| 2259. | All | O/E - nervous |
| R2y2. | All | [D]Nervousness |
| SNOMED Code | Term ID | Description |
| 79015004 | | Worried (finding) |
| 424196004 | | Feeling nervous (finding) |
| 162189001 | | General nervous symptoms (finding) |
| 162724000 | | On examination - nervous (finding) |
| 425131000 | | Nervous tension (finding) |
| 48694002 | | Anxiety (finding) |
| 35429005 | | Anticipatory anxiety (finding) |
| 11458009 | | Anticipatory anxiety, mild (finding) |
| 36646009 | | Anticipatory anxiety, moderate (finding) |
| 5874002 | | Anticipatory anxiety, severe (finding) |
| 247825008 | | Anxiety about behavior or performance (finding) |
| 277838008 | | Anxiety about appearing ridiculous (finding) |
| 225643000 | | Anxiety about making mistakes (finding) |
| 277839000 | | Anxiety about saying the wrong thing (finding) |
| 247808006 | | Anxiety about body function or health (finding) |
| 225644006 | | Anxiety about altered body image (finding) |
| 277831002 | | Anxiety about becoming fat (finding) |
| 277031002 | | Trixiety about becoming fat (mains) |

| 323351000000104 | Anxiety about mood (finding) |
|-----------------|--------------------------------------------------|
| 225636006 | Anxiety about forced dependence (finding) |
| 225637002 | Anxiety about loss of control (finding) |
| 277829006 | Anxiety about losing emotional control (finding) |
| 300895004 | Anxiety attack (finding) |
| 286710008 | Anxious character (finding) |
| 286712000 | Fearful character (finding) |
| 286711007 | Over-anxious character (finding) |
| 69479009 | Anxiety hyperventilation (disorder) |
| 198288003 | Anxiety state (finding) |
| 231506008 | Anxiety hysteria (finding) |
| 207363009 | Anxiety neurosis (finding) |
| 191708009 | Chronic anxiety (finding) |
| 386808001 | Phobia (finding) |
| 191709001 | Recurrent anxiety (finding) |
| 81350009 | Free-floating anxiety (finding) |
| 70997004 | Mild anxiety (finding) |
| 61387006 | Moderate anxiety (finding) |
| 162723006 | On examination - anxious (finding) |
| 417676004 | On examination - panic attack (finding) |
| 225624000 | Panic attack (finding) |
| 395017009 | Complaining of panic attack (finding) |
| 231503000 | Non-situational panic attack (finding) |
| 231502005 | Situational panic attack (finding) |
| 405051006 | Level of anxiety (observable entity) |
| 286644009 | Level of anxiety (finding) |
| 247805009 | Anxiety and fear (finding) |

| Counselling | | |
|----------------|---------|--------------------------------------------|
| Read V2 Code | Term ID | Description |
| 67 | 11 | Counselling/health education |
| 671 | All | Counselling - general |
| 6712 | All | Counselling offered |
| 6714 | All | Counselling carried out |
| 6715 | All | Counselling by other agency |
| 6716 | All | Counselling of benefit |
| 6717 | All | Counselling of no benefit |
| 671Z. | All | Counselling - general NOS |
| 6735 | All | Counselled by a social worker |
| 6736 | All | Counselled by a counsellor |
| 6737 | All | Counselled by a vol. worker |
| 673Z. | All | Counselled by person NOS |
| 8M8 | All | Counselling requested |
| 9NJ1. | All | In-house counselling |
| 9NJR. | All | In-house counselling first appointment |
| 9NJT. | All | In-house counselling follow-up appointment |
| Read CTV3 Code | Term ID | Description |
| X71Ec | All | Counselling |
| X71Ep | All | Coping strategy counselling |
| XaEC1 | All | Phobia counselling |
| XaD27 | All | Family counselling |
| 6779. | All | Psychological counselling |
| XaECG | All | Anxiety counselling |
| XaECF | All | Self-esteem counselling |
| Xal8j | All | Stress counselling |
| 6715. | All | Counselling by other agency |
| 6735. | All | Counselled by a social worker |
| 6736. | All | Counselled by a counsellor |
| 6737. | All | Counselled by voluntary worker |
| 673Z. | All | Counselled by person NOS |
| 9N2B. | All | Seen by counsellor |
| XaAS4 | All | Seen by mental health counsellor |
| XaBT1 | All | Refer to counsellor |
| XaAfJ | All | Referral to mental health counsellor |
| 9NJ1. | All | In-house counselling |
| XaLnp | All | In-house counselling first appointment |
| XaLnr | All | In-house counselling follow-up appointment |
| 671 | All | Counselling - general |
| 6712. | All | Counselling offered |
| 6714. | All | Counselling carried out |
| 6716. | All | Counselling of benefit |
| 6717. | All | Counselling of no benefit |
| 671Z. | All | Counselling - general NOS |
| XaAOd | All | Under care of counsellor |
| XaAOh | All | Under care of mental health counsellor |
| XaAen | All | Referral for mental health counselling |
| SNOMED Code | Term ID | Description |

| 409063005 | Counseling (procedure) |
|---|---|
| 413473000 | Counseling about alcohol consumption (procedure) |
| 243068007 | Counseling about bullying (procedure) |
| 243067002 | Counseling about coping strategies (procedure) |
| 247871000000103 | Anger management counselling (procedure) |
| 313075001 | Counseling for phobia (procedure) |
| 445142003 | Counseling about disease (procedure) |
| 24165007 | Alcoholism counseling (procedure) |
| 784055004 | Counseling for acquired polycystic kidney disease (procedure) |
| 784054000 | Counseling for acquired polycystic kidney disease (procedure) Counseling for congenital polycystic kidney disease (procedure) |
| 286711000000107 | |
| 395072006 | Counseling for depression (procedure) Counseling for postnatal depression (procedure) |
| 313076000 | Counseling for eating disorder (procedure) |
| 428997004 | Psychosocial counseling about cancer (procedure) |
| 710199005 | Counseling about fear (procedure) |
| 711030000 | Counseling about level of hope (procedure) |
| 441331000124108 | Counseling about nutrition using cognitive restructuring strategy (procedure) |
| 441201000124108 | Counseling about nutrition using cognitive-behavioral theoretical |
| | approach (procedure) |
| 441271000124102 | Counseling about nutrition using goal setting strategy (procedure) |
| 441231000124100 | Counseling about nutrition using health belief model (procedure) |
| 441261000124109 | Counseling about nutrition using motivational interviewing strategy (procedure) |
| 441291000124101 | Counseling about nutrition using problem solving strategy (procedure) |
| 441341000124103 | Counseling about nutrition using relapse prevention strategy (procedure) |
| 441351000124101 | Counseling about nutrition using rewards and contingency management strategy (procedure) |
| 441281000124104 | Counseling about nutrition using self-monitoring strategy (procedure) |
| 441241000124105 | Counseling about nutrition using social learning theory approach (procedure) |
| 441301000124100 | Counseling about nutrition using social support strategy (procedure) |
| 441321000124105 | Counseling about nutrition using stimulus control strategy (procedure) |
| | Counseling about nutrition using stimulus control strategy (procedure) |
| 441311000124102 | (procedure) |
| 441251000124107 | Counseling about nutrition using transtheoretical model and stages of |
| | change approach (procedure) |
| 310358004 | Counseling about serious diagnosis (procedure) |
| 710198002 | Counseling about spiritual distress (procedure) |
| 711028002 | Counseling about tobacco use (procedure) |
| 105393000 | Counseling by chaplain (regime/therapy) |
| 105394006 | Inpatient counseling by chaplain (regime/therapy) |
| 105395007 | Outpatient counseling by chaplain (regime/therapy) |
| 243069004 | Counseling for abuse (procedure) |
| 313070006 | Counseling for domestic abuse (procedure) |
| 243071004 | Counseling for physical abuse (procedure) |
| 313072003 | Counseling for racial abuse (procedure) |
| 243070003 | Counseling for sexual abuse (procedure) |
| 313071005 | Counseling for substance abuse (procedure) |
| 60112009 | Drug addiction counseling (procedure) |
| 299941000000103 | Substance misuse structured counselling (procedure) |

| 313069005 | Counseling for verbal abuse (procedure) |
|---|---|
| 737598000 | Counseling for end of life issues (procedure) |
| 313078004 | Counseling for loss (procedure) |
| 395184006 | Counseling following miscarriage (procedure) |
| 171007003 | Counseling for bereavement (procedure) |
| 171006007 | Counseling for grieving (procedure) |
| 514171000000100 | Counselling about diagnosis (procedure) |
| 33697008 | Geriatric counseling (procedure) |
| 310359007 | Prognosis counseling (procedure) |
| 171001002 | Counseling about benefits (procedure) |
| 313084001 | Redundancy counseling (procedure) |
| 171004005 | Retirement counseling (procedure) |
| 313083007 | Unemployment counseling (procedure) |
| 171002009 | Vocational counseling (procedure) |
| 1103851000000109 | Counselling offered (situation) |
| 185490001 | In-house counseling (procedure) |
| 247181000000106 | In-house counselling discharge (procedure) |
| 247171000000109 | In-house counselling first appointment (procedure) |
| 247191000000108 | In-house counselling follow-up appointment (procedure) |
| 129441002 | Counseling - action (qualifier value) |
| 439495000 | Counseling declined (situation) |
| 19260001000004109 | Abuse counseling for non-offending parent (situation) |
| 19270001000004103 | Abuse counseling for offending parent (situation) |
| 170986003 | Patient counseled (situation) |
| 268532004 | Person counseled by (situation) |
| 170997003 | Counseled by counselor (situation) |
| 170992009 | Counseled by doctor (situation) |
| 276497001 | Counseled by member of primary health care team (situation) |
| 170995006 | Counseled by midwife (situation) |
| 170993004 | Counseled by nurse (situation) |
| 170996007 | Counseled by social worker (situation) |
| 170998008 | Counseled by voluntary worker (situation) |
| 1052641000000102 | Counselled by health visitor (situation) |
| 306225008 | Referral to counseling service (procedure) |
| 385720006 | Patient counseling management (procedure) |
| 306227000 | Referral for mental health counseling (procedure) |
| 1239851000000103 | Referral to debt counselling service (procedure) |
| 306226009 | Referral to mental health counseling service (procedure) |
| 385719000 | Patient counseling education (procedure) |
| 439853000 | Consent given for counseling (finding) |
| 440611006 | Home visit for marriage counseling (procedure) |
| 166871000000108 | Date children offered counselling (observable entity) |
| 527961000000108 | Counselling about alcohol by other agency (procedure) |
| 1037431000000105 | Recommendation to self-refer for counselling (procedure) |
| 1104491000000102 | Signposting to family support counselling (procedure) |
| 1104501000000108 | Signposting to counselling (procedure) |
| 1109931000000108 | Signposting to general practice based counselling (procedure) |
| 171022008 | Psychological counseling (procedure) |

| 225421002 | Counseling for change in body image (procedure) |
|---|---|
| 313086004 | Counseling for self-esteem (procedure) |
| 698505007 | Counseling for trauma (procedure) |
| 445428001 | Person centered counseling (procedure) |
| 171023003 | Psychosexual counseling (procedure) |
| 737365009 | Counseling about sexual attitude (procedure) |
| 313079007 | Counseling for homosexuality (procedure) |
| 243066006 | Counseling for sexual dysfunction (procedure) |
| 737302009 | Counseling related to sexuality (procedure) |
| 66800001 | Counseling by physiotherapist (procedure) |
| 315600006 | Counseling for stress (procedure) |
| 10383002 | Counseling for termination of pregnancy (procedure) |
| 225326008 | Counseling following termination of pregnancy (procedure) |
| 225327004 | Counseling prior to the termination of pregnancy (procedure) |
| 440215007 | Counseling for unwanted pregnancy (procedure) |
| 313073008 | Counseling of crime victim (procedure) |
| 410273004 | Behavior modification education, guidance, and counseling (procedure) |
| 762449006 | Behavioral counseling (procedure) |
| 423640000 | Community outreach worker services education, guidance, and |
| 422649009 | counseling (procedure) |
| 410282005 | Coping skills education, guidance, and counseling (procedure) |
| 410304007 | Relaxation/breathing techniques education, guidance, and counseling (procedure) |
| 171014001 | Medical counseling (procedure) |
| 171000001 | Social counseling (procedure) |
| 313085000 | Relationship counseling (procedure) |
| 68168001 | Marital counseling (procedure) |
| 86515003 | Premarital counseling (procedure) |
| 313080005 | Work-related counseling (procedure) |
| 108226001 | Specific patient counseling session (procedure) |
| 698506008 | Supportive counseling (procedure) |
| 737375007 | Group counseling (procedure) |
| 311764000 | Family counseling (procedure) |
| 719111000000107 | School counselling (qualifier value) |
| 443913008 | Counseling procedure with explicit context (situation) |
| 19260001000004100 | Abuse counseling for non-offending parent (situation) |
| 19270001000004100 | Abuse counseling for offending parent (situation) |
| 359101000000103 | Active listening offered (situation) |
| 170978003 | Counseling not wanted (situation) |
| 170982001 | Counseling of benefit (situation) |
| 394890004 | Counseling requested (situation) |
| 170983006 | Counseling of no benefit (situation) |
| 1103851000000100 | Counselling offered (situation) |
| 170985004 | Person counseled (situation) |
| 170987007 | Family counseled (situation) |
| 170988002 | Relative counseled (situation) |
| 1104501000000100 | Signposting to counselling (procedure) |
| | Signiposting to counselling (procedure) |
| 1104491000000100 | Signposting to family support counselling (procedure) |
| 1104491000000100<br>1109931000000100 | |

| 810891000000103 | | Referral to counselling assessment referral advice and throughcare drug |
|---|---|---|
| | | service (procedure) |
| 185288004 | | Seen by counselor (finding) |
| 305622007 | | Seen by bereavement counselor (finding) |
| 372501000000100 | | Seen by counsellor for alcohol misuse (finding) |
| 305624008 | | Seen by marriage guidance counselor (finding) |
| 305625009 | | Seen by mental health counselor (finding) |
| 305918000 | | Referral by counselor (procedure) |
| 305919008 | | Referral by bereavement counselor (procedure) |
| 305922005 | | Referral by mental health counselor (procedure) |
| 824191000000109 | | Liaison with counsellor (procedure) |
| 305439002 | | Under care of counselor (finding) |
| 305440000 | | Under care of bereavement counselor (finding) |
| 305442008 | | Under care of marriage guidance counselor (finding) |
| 305443003 | | Under care of mental health counselor (finding) |
| 306383002 | | Discharge by counselor (procedure) |
| 306385009 | | Discharge by bereavement counselor (procedure) |
| 306387001 | | Discharge by marriage guidance counselor (procedure) |
| 306388006 | | Discharge by mental health counselor (procedure) |
| Cognitive Behavioural Tl | nerapy | |
| Read V2 Code | Term ID | Description |
| 8G13. | All | Cognitive-behaviour therapy |
| 8G130 | All | Cognitive behavioural therapy parenting programme |
| 8G131 | All | CBTp - cognitive behavioural therapy for psychosis |
| 7L1a. | All | Cognitive behavioural therapy |
| 7L1a0 | All | Cognitive behavioural therapy by unidisciplinary team |
| 7L1a1 | All | Cognitive behavioural therapy by multidisciplinary team |
| 7L1ay | All | Other specified cognitive behavioural therapy |
| 7L1az | All | Cognitive behavioural therapy NOS |
| 8G510 | All | Group cognitive behavioural therapy |
| 8G15. | All | Computerised cognitive behavioural therapy |
| 8HIK. | All | Referral for cognitive behavioural therapy |
| Read CTV3 Code | Term ID | Description |
| Ub0qp | All | Cognitive and behavioural therapy |
| XaABO | All | Cognitive - behaviour therapy |
| Xad6J | All | Cognitive behavioural therapy for psychosis |
| Xaaa6 | All | Cognitive behavioural therapy parenting programme |
| XaQC0 | All | Guided self help cognitive behavioural therapy |
| XaKzQ | All | Computerised cognitive behavioural therapy |
| Xa8I9 | All | Generic cognitive behavioural therapy |
| XaM2I | All | Cognitive behavioural therapy by unidisciplinary team |
| XaM2J | All | Cognitive behavioural therapy by multidisciplinary team |
| XaM2K | All | Other specified cognitive behavioural therapy |
| XaM2L | All | Cognitive behavioural therapy NOS |
| XaR2j | All | Referral to cognitive behavioural therapist |
| XaR5D | All | Referral for cognitive behavioural therapy |
| XaYgB | All | Referral for high intensity cognitive behavioural therapy |
| XaZsD | All | Group cognitive behavioural therapy |
| SNOMED Code | Term ID | Description |
| 228557008 | | Cognitive and behavioral therapy (regime/therapy) |
| | | O |

| 405500000 | | |
|---|---|---|
| 425680009 | | Cognitive behavioral therapy by multidisciplinary team (regime/therapy) |
| 868185009 | | Cognitive behavioral therapy for insomnia (regime/therapy) |
| 718026005 | | Cognitive behavioral therapy for psychosis (regime/therapy) |
| 231621000000108 | | Cognitive behavioural therapy by unidisciplinary team (regime/therapy) |
| 1111811000000100 | | Cognitive behavioural therapy for eating disorders (regime/therapy) |
| 88384100000104 | | Cognitive behavioural therapy parenting programme (regime/therapy) |
| 228553007 | | Cognitive therapy (regime/therapy) |
| 302234000 | | Becks cognitive therapy (regime/therapy) |
| 702474001 | | Cognitive rehabilitation therapy (regime/therapy) |
| 304637004 | | Cognitive restructuring (regime/therapy) |
| 386241007 | | Cognitive stimulation (regime/therapy) |
| 1024851000000100 | | Cognitive-linguistic therapy (regime/therapy) |
| 975281000000106 | | Rapid instructional pacing (regime/therapy) |
| 228555000 | | Rational emotive therapy (regime/therapy) |
| 429329005 | | Computerized cognitive behavioral therapy (regime/therapy) |
| 1109721000000100 | | Digital cognitive behavioural therapy for insomnia (regime/therapy) |
| 302230009 | | Generic cognitive behavioral therapy (regime/therapy) |
| 444175001 | | Guided self-help cognitive behavioral therapy (regime/therapy) |
| 439916005 | | Paradoxical intention behavior therapy (regime/therapy) |
| 859501000000107 | | Group cognitive behavioural therapy (regime/therapy) |
| 519101000000109 | | Referral for cognitive behavioural therapy (procedure) |
| 1097161000000100 | | Referral for cognitive behavioural therapy for psychosis (procedure) |
| 110719100000100 | | Referral for digital cognitive behavioural therapy for insomnia (procedure) |
| 814131000000101 | | Referral for high intensity cognitive behavioural therapy (procedure) |
| 110718100000100 | | Signposting for digital cognitive behavioural therapy for insomnia (procedure) |
| 110720100000100 | | Self referral for digital cognitive behavioural therapy for insomnia (procedure) |
| Psychotherapy | | , |
| Read V2 Code | Term ID | Description |
| 8G | All | Psychotherapy |
| 8G1 | All | General psychotherapy |
| 8G10. | All | Psychotherapy - behavioural |
| 8G100 | | · |
| | All | Behavioural activation therapy |
| 8G101 | All | Behavioural activation therapy Dialectical behaviour therapy |
| 8G101<br>8G102 | All | Dialectical behaviour therapy |
| 8G101<br>8G102<br>8G11. | | Dialectical behaviour therapy Behavioural parent training |
| 8G102 | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive |
| 8G102<br>8G11.<br>8G12. | All<br>All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic |
| 8G102<br>8G11.<br>8G12.<br>8G120 | All All All All All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121 | All All All All All All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122 | All All All All All All All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15.<br>8G16. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy Interpersonal psychotherapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15.<br>8G16.<br>8G18. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy Interpersonal psychotherapy Cognitive stimulation therapy |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15.<br>8G16.<br>8G18.<br>9NIK. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy Interpersonal psychotherapy Cognitive stimulation therapy Seen by psychotherapist |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15.<br>8G16.<br>8G18.<br>9NIK. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy Interpersonal psychotherapy Cognitive stimulation therapy Seen by psychotherapist Seen by trainee psychotherapist |
| 8G102<br>8G11.<br>8G12.<br>8G120<br>8G121<br>8G122<br>8G14.<br>8G15.<br>8G16.<br>8G18.<br>9NIK. | All | Dialectical behaviour therapy Behavioural parent training Psychotherapy - cognitive Psychotherapy - psychodynamic Short-term psychodynamic therapy Dynamic interpersonal therapy Focal psychodynamic therapy Cognitive analytic therapy Computerised cognitive behavioural therapy Interpersonal psychotherapy Cognitive stimulation therapy Seen by psychotherapist |

| ZV673 | All | [V]Psychotherapy or other treatment for mental disorder follow-up |
|---|---|---|
| 8G9Z. | All | Other psychotherapy NOS |
| 8G9 | All | Other psychotherapy |
| 8GZ | All | Psycho./socio therapy NOS |
| Read CTV3 Code | Term ID | Description |
| X71bp | All | Psychotherapy |
| XaaUO | All | Cognitive rehabilitation therapy |
| Xaltc | All | Brief solution focused psychotherapy |
| Xa8IG | All | Psychoanalytic and psychodynamic therapy |
| Xa8IJ | All | Long-term exploratory psychotherapy |
| 3841. | All | Psychoanalysis |
| XaA8V | All | Generic psychoanalysis |
| XaA8W | All | Independent psychoanalysis |
| XaA8T | All | Kleinian psychoanalysis |
| XaA8U | All | Bion-based group psychoanalysis |
| XaA8X | All | Classical psychoanalysis |
| XaA8Y | All | Lacanian psychoanalysis |
| XaA8g | All | Group psychoanalysis |
| 384Z. | All | Psychological analysis NOS |
| Xa8IM | All | Jungian-based therapy |
| Xa8IN | All | Generic Jungian-based therapy |
| Xa8IP | All | Analytical psychology |
| Xa8IR | All | Long-term psychodynamic psychotherapy |
| XaA8Z | All | Developmental psychodynamic psychotherapy |
| XaA8c | All | Supportive expressive psychodynamic psychotherapy |
| XaA8d | All | Psychodynamic-interpersonal psychotherapy |
| XaEVq | All | Psychodynamic psychotherapy |
| Xad7C | All | Focal psychodynamic therapy |
| Xa8II | All | Short-term psychodynamic therapy |
| XaXuc | All | Dynamic interpersonal therapy |
| XaA9g | All | Specific task orientated psychotherapy |
| XE0iL | All | Psychotherapy/sociotherapy |
| 8G9Z. | All | Other psychotherapy NOS |
| 8G9 | All | Other psychotherapy |
| 8G1 | All | General psychotherapy |
| 8G10. | All | Psychotherapy - behavioural |
| 8G11. | All | Psychotherapy - cognitive |
| 8G12. | All | Psychotherapy - psychodynamic |
| XaAUN | All | Seen by psychotherapist |
| Xaa4f | All | Seen by trainee psychotherapist |
| SNOMED Code | Term ID | Description |
| 75516001 | | Psychotherapy (regime/therapy) |
| 183405004 | | Anti-criminal psychotherapy (regime/therapy) |
| 183401008 | | Anti-suicide psychotherapy (regime/therapy) |
| 700445002 | | Attachment-based therapy (regime/therapy) |
| 166001 | | Behavioral therapy (regime/therapy) |
| 3518004 | | Aversive psychotherapy (regime/therapy) |
| 228557008 | | Cognitive and behavioral therapy (regime/therapy) |
| 401157001 | | Brief solution focused psychotherapy (regime/therapy) |

| 429159005 | Child psychotherapy (regime/therapy) |
|---|---|
| 427954006 | Child psychoanalytic psychotherapy (regime/therapy) |
| 38678006 | Client-centered psychotherapy (regime/therapy) |
| 41035007 | Conjoint psychotherapy (regime/therapy) |
| 440274001 | Couple psychotherapy (regime/therapy) |
| 723619005 | Behavioral couple psychotherapy (regime/therapy) |
| 183398005 | Daily life psychotherapy (regime/therapy) |
| 405793004 | Eclectic psychotherapy (regime/therapy) |
| 15558000 | Expressive psychotherapy (regime/therapy) |
| 736861004 | Systemic psychotherapy (regime/therapy) |
| 302245002 | Family, systemic, couple and sex therapy (regime/therapy) |
| 405792009 | Formal psychological therapy (regime/therapy) |
| 183385001 | Functional psychotherapy (regime/therapy) |
| 183381005 | General psychotherapy (regime/therapy) |
| 183382003 | Psychotherapy - behavioral (regime/therapy) |
| 183383008 | Psychotherapy - cognitive (regime/therapy) |
| 76168009 | Group psychotherapy (regime/therapy) |
| 1555005 | Brief group psychotherapy (regime/therapy) |
| 108313002 | Family psychotherapy procedure (regime/therapy) |
| 302247005 | Narrative family psychotherapy (regime/therapy) |
| 361229007 | Structural family psychotherapy (regime/therapy) |
| 27591006 | Group analytical psychotherapy (regime/therapy) |
| 28868002 | Interactive group medical psychotherapy (regime/therapy) |
| 1106951000000100 | Interpersonal psychotherapy for group (regime/therapy) |
| 106681100000100 | High intensity psychological intervention in combination with |
| 1066811000000100 | medication (regime/therapy) |
| 302243009 | Humanistic and integrative therapy (regime/therapy) |
| 313105004 | Action therapy (regime/therapy) |
| 304825004 | Humanistic psychotherapy (regime/therapy) |
| 304826003 | Integrative psychotherapy (regime/therapy) |
| 390773006 | Cognitive analytic therapy (regime/therapy) |
| 440582002 | Psychosynthesis (regime/therapy) |
| 18512000 | Individual psychotherapy (regime/therapy) |
| 8411005 | Interactive individual medical psychotherapy (regime/therapy) |
| 443730003 | Interpersonal psychotherapy (regime/therapy) |
| 1108261000000100 | Interpersonal and social rhythm therapy (regime/therapy) |
| 700446001 | Parent-infant psychotherapy (regime/therapy) |
| 302235004 | Psychoanalytic and psychodynamic therapy (regime/therapy) |
| 440646003 | Educational psychotherapy (regime/therapy) |
| 302236003 | Long-term exploratory psychotherapy (regime/therapy) |
| 302238002 | Jungian-based therapy (regime/therapy) |
| 302240007 | Analytical psychology (regime/therapy) |
| 302239005 | Generic Jungian-based therapy (regime/therapy) |
| 302242004 | Long-term psychodynamic psychotherapy (regime/therapy) |
| 304820009 | Developmental psychodynamic psychotherapy (regime/therapy) |
| 304020003 | Developmental psychodynamic psychotherapy (regime/therapy) |
| 304822001 | Psychodynamic-interpersonal psychotherapy (regime/therapy) |
| | Psychodynamic-interpersonal psychotherapy (regime/therapy) |
| 304822001 | Psychodynamic-interpersonal psychotherapy (regime/therapy) Supportive expressive psychodynamic psychotherapy (regime/therapy) |
| 304822001<br>304821008 | Psychodynamic-interpersonal psychotherapy (regime/therapy) |

| 1323681000000100 | Eating-disorder-focused focal psychodynamic therapy (regime/therapy) |
|---|---|
| 429048003 | Short-term psychodynamic therapy (regime/therapy) |
| 786721000000109 | Dynamic interpersonal therapy (regime/therapy) |
| 1111671000000100 | Transference focused psychotherapy (regime/therapy) |
| 397074006 | Psychologic desensitization therapy (regime/therapy) |
| 302248000 | Psychotherapeutic approaches using specific settings (regime/therapy) |
| 266744007 | Psychotherapy/sociotherapy (regime/therapy) |
| 6227009 | Relationship psychotherapy (regime/therapy) |
| 345181000000108 | Marital psychotherapy (regime/therapy) |
| 63386006 | Sexual psychotherapy (regime/therapy) |
| 15142007 | Sexual psychotherapy, female therapist - female patient (regime/therapy) |
| 113144009 | Sexual psychotherapy, female therapist - male patient (regime/therapy) |
| 26693005 | Sexual psychotherapy, group (regime/therapy) |
| 33661004 | Sexual psychotherapy, group, all female (regime/therapy) |
| 41653002 | Sexual psychotherapy, group, all male (regime/therapy) |
| 31408009 | Sexual psychotherapy, group, male and female (regime/therapy) |
| 305111000000109 | Relationship psychosexual therapy (regime/therapy) |
| 66060003 | Sexual psychotherapy, male therapist - female patient (regime/therapy) |
| 73139001 | Sexual psychotherapy, male therapist - male patient (regime/therapy) |
| 90102008 | Social psychotherapy (regime/therapy) |
| 304851002 | Specific task orientated psychotherapy (regime/therapy) |
| 183391004 | Stimulative psychotherapy (regime/therapy) |
| 361230002 | Structural psychotherapy (regime/therapy) |
| 85925008 | Supportive verbal psychotherapy (regime/therapy) |
| 84892007 | Suppressive psychotherapy (regime/therapy) |
| 183411001 | Therapeutic psychology (regime/therapy) |
| 394913002 | Psychotherapy (specialty) (qualifier value) |
| 1323761000000100 | Medical psychotherapy (qualifier value) |
| 773451003 | Psychotherapy care plan (record artifact) |
| 305878005 | Seen by psychotherapy service (finding) |
| 299695005 | Competitive games psychotherapy (regime/therapy) |
| 81294000 | Patient referral for psychotherapy (procedure) |
| 183374003 | Convalescence after psychotherapy (finding) |
| 763151000000107 | Did not attend psychotherapy appointment (finding) |
| 1079251000000100 | Emergency hospital admission to psychotherapy service (procedure) |
| 305761008 | Seen by psychotherapist (finding) |
| 865241000000103 | Seen by trainee psychotherapist (finding) |
| 306055009 | Referral by psychotherapist (procedure) |
| 824211000000108 | Liaison with psychotherapist (procedure) |
| 306526008 | Discharge by psychotherapist (procedure) |
| 305589008 | Under care of psychotherapist (finding) |
| 305744005 | Seen by nurse psychotherapist (finding) |
| 306038005 | Referral by nurse psychotherapist (procedure) |
| 306503001 | Discharge by nurse psychotherapist (procedure) |
| 305567009 | Under care of nurse psychotherapist (finding) |

| SSRIs | | |
|--------------|---------|-------------------------------------------|
| Read V2 Code | Term ID | Description |
| da9 | All | CITALOPRAM |
| da91. | All | CITALOPRAM 20mg tablets |
| da92. | All | CIPRAMIL 20mg tablets |
| da93. | All | CITALOPRAM 10mg tablets |
| da94. | All | *CIPRAMIL 10mg tablets |
| da95. | All | CITALOPRAM 40mg tablets |
| da96. | All | *CIPRAMIL 40mg tablets |
| da97. | All | CIPRAMIL 40mg/mL oral drops 15mL |
| da98. | All | *PAXORAN 10mg tablets |
| da99. | All | *PAXORAN 20mg tablets |
| da9A. | All | *PAXORAN 40mg tablets |
| da9z. | All | CITALOPRAM 40mg/mL oral drops |
| gde | All | DULOXETINE |
| gde1. | All | YENTREVE 20mg gastro-resistant capsules |
| gde2. | All | YENTREVE 40mg gastro-resistant capsules |
| gde3. | All | CYMBALTA 30mg gastro-resistant capsules |
| gde4. | All | CYMBALTA 60mg gastro-resistant capsules |
| gdew. | All | DULOXETINE 60mg gastro-resistant capsules |
| gdex. | All | DULOXETINE 30mg gastro-resistant capsules |
| gdey. | All | DULOXETINE 20mg gastro-resistant capsules |
| gdez. | All | DULOXETINE 40mg gastro-resistant capsules |
| daC | All | ESCITALOPRAM |
| daC1. | All | ESCITALOPRAM 10mg tablets |
| daC2. | All | CIPRALEX 10mg tablets |
| daC3. | All | ESCITALOPRAM 20mg tablets |
| daC4. | All | CIPRALEX 20mg tablets |
| daC5. | All | ESCITALOPRAM 5mg tablets |
| daC6. | All | CIPRALEX 5mg tablets |
| daC7. | All | ESCITALOPRAM 10mg/mL oral drops |
| daC8. | All | *CIPRALEX 10mg/mL oral drops |
| daC9. | All | CIPRALEX 20mg/mL oral drops |
| daC9. | All | CIPRALEX 20mg/mL oral drops |
| da4 | All | FLUOXETINE HYDROCHLORIDE |
| da41. | All | FLUOXETINE 20mg capsules |
| da42. | All | *PROZAC 20mg capsules x30 |
| da43. | All | FLUOXETINE 20mg/5mL oral liquid |
| da44. | All | PROZAC 20mg/5mL oral liquid |
| da45. | All | PROZAC 20mg capsules |
| da46. | All | FLUOXETINE 60mg capsules |
| da47. | All | *PROZAC 60mg capsules |
| da48. | All | *FELICIUM 20mg capsules |
| da49. | All | OXACTIN 20mg capsules |
| da4A. | All | RANFLUTIN 20mg capsules |
| da4B. | All | PROZIT 20mg/5mL oral solution |
| da4C. | All | PROZEP 20mg/5mL oral solution |
| da4D. | All | OLENA 20mg dispersible tablets |
| da4E. | All | FLUOXETINE 20mg dispersible tablets |

| da3 | All | FLUVOXAMINE MALEATE |
|---|---|---|
| da31. | All | FAVERIN 50mg tablets |
| da32. | All | FLUVOXAMINE MALEATE 50mg tablets |
| da32. | All | FLUVOXAMINE MALEATE 50mg tablets |
| da32. | All | FLUVOXAMINE MALEATE 50mg tablets |
| da6 | All | PAROXETINE HYDROCHLORIDE |
| da61. | All | PAROXETINE 20mg tablets |
| da62. | All | SEROXAT 20mg tablets x30 |
| da63. | All | PAROXETINE 30mg tablets |
| da64. | All | SEROXAT 30mg tablets x30 |
| da65. | All | PAROXETINE 10mg/5mL sugar free liquid |
| da66. | All | SEROXAT 10mg/5mL sugar free liquid |
| da67. | All | PAROXETINE 10mg tablets |
| da68. | All | SEROXAT 10mg tablets |
| da5 | All | SERTRALINE HYDROCHLORIDE |
| da51. | All | SERTRALINE 50mg tablets |
| da52. | All | SERTRALINE 100mg tablets |
| da53. | All | LUSTRAL 50mg tablets |
| da54. | All | LUSTRAL 100mg tablets |
| da7 | All | VENLAFAXINE |
| da71. | All | VENLAFAXINE 37.5mg tablets |
| da72. | All | VENLAFAXINE 75mg tablets |
| da73. | All | *EFEXOR 37.5mg tablets |
| da74. | All | *EFEXOR 75mg tablets |
| da75. | All | *VENLAFAXINE 50mg tablets |
| da76. | All | *EFEXOR 50mg tablets |
| da77. | All | VENLAFAXINE 75mg m/r capsules |
| da78. | All | EFEXOR XL 75mg m/r capsules |
| da79. | All | VENLAFAXINE 150mg m/r capsules |
| da7A. | All | EFEXOR XL 150mg m/r capsules |
| da7B. | All | RODOMEL XL 75mg m/r capsules |
| da7C. | All | RODOMEL XL 150mg m/r capsules |
| da7D. | All | WINFEX XL 75mg m/r capsules |
| da7E. | All | WINFEX XL 150mg m/r capsules |
| da7F. | All | TRIXAT XL 75mg m/r capsules |
| da7G. | All | TRIXAT XL 150mg m/r capsules |
| da7H. | All | VIEPAX XL 75mg m/r tablets |
| da7I. | All | VENLAFAXINE 75mg m/r tablets |
| da7J. | All | VIEPAX XL 150mg m/r tablets |
| da7K. | All | VENLAFAXINE 150mg m/r tablets |
| da7L. | All | *TARDCAPS XL 75mg m/r capsules |
| da7M. | All | *TARDCAPS XL 150mg m/r capsule |
| da7N. | All | VIEPAX 37.5mg tablets |
| da7O. | All | VIEPAX 75mg tablets |
| da7P. | All | VENSIR XL 75mg m/r capsules |
| | | <u> </u> |
| aa/Q. | All | VENSIR XL 150mg m/r capsules |
| da7Q. | All All | VENSIR XL 150mg m/r capsules TIFAXIN XL 75mg m/r capsules |
| da7Q.<br>da7R.<br>da7S. | | VENSIR XL 150mg m/r capsules TIFAXIN XL 75mg m/r capsules TIFAXIN XL 150mg m/r capsules |

| da7U. | All | VEXARIN XL 150mg m/r capsules |
|---|---|---|
| da7V. | All | VENLALIC XL 75mg m/r tablets |
| da7W. | All | VENLALIC XL 150mg m/r tablets |
| da7X. | All | VENLALIC XL 225mg m/r tablets |
| da7Y. | All | VENLAFAXINE 225mg m/r tablets |
| da71. | All | VENAXX XL 75mg m/r capsules |
| da7a. | All | VENAXX XL 150mg m/r capsules |
| da7b. | All | VAXALIN XL 75mg m/r capsules |
| da7c. | All | VAXALIN XL 150mg m/r capsules |
| da7d. | All | ALVENTA XL 75mg m/r capsules |
| da7e. | All | ALVENTA XL 150mg m/r capsules |
| da7f. | All | RANFAXINE XL 150mg m/r capsules |
| da7g. | All | RANFAXINE XL 75mg m/r capsules |
| da7h. | All | BONILUX XL 75mg m/r capsules |
| da7i. | All | BONILUX XL 150mg m/r capsules |
| da7i. | All | TONPULAR XL 75mg m/r capsules |
| da7k. | All | TONPULAR XL 75Hig Hi/T capsules TONPULAR XL 150mg m/r capsules |
| da7k. | All | FORAVEN XL 75mg m/r capsules |
| da7n. | All | |
| da7m. | All | FORAVEN XL 150mg m/r capsules DEPEFEX XL 75mg m/r capsules |
| da7n. | All | DEPEFEX XL 150mg m/r capsules |
| da7p. | All | VENLALIC XL 37.5mg m/r tablets |
| da7p. | All | VENLAFAXINE 37.5mg m/r tablets |
| da7q. | All | SUNVENIZ XL 75mg m/r tablets |
| da7s. | All | SUNVENIZ XL 75mg m/r tablets SUNVENIZ XL 150mg m/r tablets |
| da7s. | All | VENLADEX XL 75mg m/r tablets |
| da7u. | All | VENLADEX XL 75mg m/r tablets VENLADEX XL 150mg m/r tablets |
| daA | All | REBOXETINE |
| daA1. | All | REBOXETINE 4mg tablets |
| | All | |
| daA2. | All | EDRONAX 4mg tablets MIRTAZAPINE |
| daB1. | All | MIRTAZAPINE MIRTAZAPINE 30mg tablets |
| daB1. | All | *ZISPIN 30mg tablets |
| daB3. | All | MIRTAZAPINE 30mg oro-dispersible tablets |
| daB4. | All | ZISPIN SOLTAB 30mg oro-dispersible tablets |
| daB5. | All | MIRTAZAPINE 15mg oro-dispersible tablets |
| | | ZISPIN SOLTAB 15mg oro-dispersible tablets |
| daB6.<br>daB7. | All | MIRTAZAPINE 45mg oro-dispersible tablets |
| daB8. | All | ZISPIN SOLTAB 45mg oro-dispersible tablets |
| | All | MIRTAZAPINE 45mg tablets |
| daBy. | All | MIRTAZAPINE 45mg tablets MIRTAZAPINE 15mg tablets |
| daBz. | All | AGOMELATINE AGOMELATINE |
| daD | All | VALDOXAN 25mg tablets |
| daD1. | All | AGOMELATINE 25mg tablets |
| Read CTV3 Code | Term ID | Description |
| da9 | All | Citalopram |
| da93. | All | Citalopram 10mg tablet |
| da94.<br>da98. | All | Cipramil 10mg tablet Paxoran 10mg tablet |
| uajo. | All | Layoran Tollik ranier |

| da91. | All | Citalopram 20mg tablet |
|-------|-----|-------------------------------------|
| da92. | All | Cipramil 20mg tablet |
| da99. | All | Paxoran 20mg tablet |
| da95. | All | Citalopram 40mg tablet |
| da96. | All | Cipramil 40mg tablet |
| da9A. | All | Paxoran 40mg tablet |
| da9z. | All | Citalopram 40mg/mL oral drops |
| x054r | All | Cipramil 40mg/mL oral drops |
| da97. | All | Cipramil 40mg/mL oral drops 15mL |
| gm1 | All | DAPOXETINE |
| gm11. | All | PRILIGY 30mg tablets |
| gm12. | All | DAPOXETINE 30mg tablets |
| gm13. | All | PRILIGY 60mg tablets |
| gm14. | All | DAPOXETINE 60mg tablets |
| daC | All | Escitalopram |
| daC5. | All | Escitalopram 5mg tablet |
| daC6. | All | Cipralex 5mg tablet |
| daC7. | All | ESCITALOPRAM 10mg/mL oral drops |
| daC8. | All | CIPRALEX 10mg/mL oral drops |
| daC1. | All | Escitalopram 10mg tablet |
| daC2. | All | Cipralex 10mg tablet |
| daC3. | All | Escitalopram 20mg tablet |
| daC4. | All | Cipralex 20mg tablet |
| daC9. | All | CIPRALEX 20mg/mL oral drops |
| daCA. | All | ESCITALOPRAM 20mg/mL oral drops |
| x01Ar | All | Fluoxetine |
| da41. | All | Fluoxetine 20mg capsule |
| da48. | All | Felicium 20mg capsule |
| da49. | All | Oxactin 20mg capsule |
| da45. | All | Prozac 20mg capsule |
| da42. | All | Prozac 20mg capsules x30 |
| da4A. | All | Ranflutin 20mg capsule |
| da46. | All | Fluoxetine 60mg capsule |
| da47. | All | Prozac 60mg capsule |
| da43. | All | Fluoxetine 20mg/5mL oral liquid |
| da44. | All | Prozac 20mg/5mL liquid |
| da4C. | All | PROZEP 20mg/5mL oral solution |
| da4B. | All | Prozit 20mg/5mL oral solution |
| da4 | All | Fluoxetine hydrochloride |
| da4D. | All | OLENA 20mg dispersible tablets |
| da4E. | All | FLUOXETINE 20mg dispersible tablets |
| x01As | All | Fluvoxamine |
| da32. | All | Fluvoxamine maleate 50mg tablet |
| da31. | All | Faverin 50mg tablet |
| da34. | All | Fluvoxamine maleate 100mg tablet |
| da33. | All | Faverin 100mg tablet |
| da3 | T | |
| | All | Fluvoxamine maleate |
| da6 | All | Paroxetine |

| da68. | All | SEROXAT 10mg tablets |
|---|---|---|
| da61. | All | Paroxetine 20mg tablet |
| x00fz | All | Seroxat 20mg tablet |
| da62. | All | Seroxat 20mg tablets x30 |
| da63. | All | Paroxetine 30mg tablet |
| | All | Seroxat 30mg tablet |
| x00g0<br>da64. | All | |
| | | Seroxat 30mg tablets x30 |
| da65. | All | Paroxetine 10mg/5mL s/f liquid |
| da66. | All | Seroxat 10mg/5mL s/f liquid |
| da5 | All | Sertraline Controlling 50 or a table to |
| da51. | All | Sertraline 50mg tablet |
| da53. | All | Lustral 50mg tablet |
| da52. | All | Sertraline 100mg tablet |
| da54. | All | Lustral 100mg tablet |
| daE | All | VORTIOXETINE |
| daE1. | All | BRINTELLIX 5mg tablets |
| daE2. | All | VORTIOXETINE 5mg tablets |
| daE3. | All | BRINTELLIX 10mg tablets |
| daE4. | All | VORTIOXETINE 10mg tablets |
| daE5. | All | BRINTELLIX 20mg tablets |
| daE6. | All | VORTIOXETINE 20mg tablets |
| SNOMED Code | Term ID | Description |
| 37431011000001109 | | Brintellix 10mg tablets - CST Pharma Ltd |
| 38122011000001109 | | Brintellix 10mg tablets - DE Pharmaceuticals |
| 37622111000001101 | | Brintellix 10mg tablets - Ethigen Ltd |
| 30248111000001105 | | Brintellix 10mg tablets - Lundbeck Ltd |
| 37352011000001105 | | Brintellix 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 37431111000001105 | | Brintellix 10mg tablets 28 tablet - CST Pharma Ltd |
| 38122111000001105 | | Brintellix 10mg tablets 28 tablet - DE Pharmaceuticals |
| 37622211000001107 | | Brintellix 10mg tablets 28 tablet - Ethigen Ltd |
| 30248211000001104 | | Brintellix 10mg tablets 28 tablet - Lundbeck Ltd |
| 37352211000001100 | | Brintellix 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 30247811000001102 | | Brintellix 20mg tablets - Lundbeck Ltd |
| 30247911000001107 | | Brintellix 20mg tablets 28 tablet - Lundbeck Ltd |
| 37431211000001104 | | Brintellix 5mg tablets - CST Pharma Ltd |
| 38121811000001107 | | Brintellix 5mg tablets - DE Pharmaceuticals |
| 37622311000001104 | | Brintellix 5mg tablets - Ethigen Ltd |
| 30247511000001100 | | Brintellix 5mg tablets - Lundbeck Ltd |
| 37351811000001108 | | Brintellix 5mg tablets - Mawdsley-Brooks & Company Ltd |
| 37431311000001107 | | Brintellix 5mg tablets 28 tablet - CST Pharma Ltd |
| 38121911000001102 | | Brintellix 5mg tablets 28 tablet - DE Pharmaceuticals |
| 37622411000001106 | | Brintellix 5mg tablets 28 tablet - Ethigen Ltd |
| 30247611000001101 | | Brintellix 5mg tablets 28 tablet - Lundbeck Ltd |
| 37351911000001103 | | Brintellix 5mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 37376411000001102 | | Cipralex 10mg tablets - CST Pharma Ltd |
| 13849211000001102 | | Cipralex 10mg tablets - DE Pharmaceuticals |
| 13106711000001102 | | Cipralex 10mg tablets - Dowelhurst Ltd |
| 16148211000001109 | | Cipralex 10mg tablets - Lexon (UK) Ltd |
| 3388511000001100 | | Cipralex 10mg tablets - Lundbeck Ltd |

| 16501911000001108 | Cipralex 10mg tablets - Mawdsley-Brooks & Company Ltd |
|---|---|
| 18220311000001108 | Cipralex 10mg tablets - Necessity Supplies Ltd |
| 17534811000001109 | Cipralex 10mg tablets - Sigma Pharmaceuticals Plc |
| 10505911000001102 | Cipralex 10mg tablets - Waymade Healthcare Plc |
| 37376511000001103 | Cipralex 10mg tablets 28 tablet - CST Pharma Ltd |
| 13849311000001105 | Cipralex 10mg tablets 28 tablet - DE Pharmaceuticals |
| 13106811000001105 | Cipralex 10mg tablets 28 tablet - Dowelhurst Ltd |
| 16148411000001108 | Cipralex 10mg tablets 28 tablet - Lexon (UK) Ltd |
| 3388811000001102 | Cipralex 10mg tablets 28 tablet - Lundbeck Ltd |
| 16502011000001101 | Cipralex 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 18220411000001101 | Cipralex 10mg tablets 28 tablet - Necessity Supplies Ltd |
| 17534911000001104 | Cipralex 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 10506211000001100 | Cipralex 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 10364011000001102 | Cipralex 10mg/ml oral drops - Lundbeck Ltd |
| 10364111000001101 | Cipralex 10mg/ml oral drops 28 ml - Lundbeck Ltd |
| 19540411000001109 | Cipralex 5mg tablets - DE Pharmaceuticals |
| 7331811000001105 | Cipralex 5mg tablets - Lundbeck Ltd |
| 16501611000001102 | Cipralex 5mg tablets - Mawdsley-Brooks & Company Ltd |
| 13364711000001104 | Cipralex 5mg tablets - Waymade Healthcare Plc |
| 19540511000001108 | Cipralex 5mg tablets 28 tablet - DE Pharmaceuticals |
| 7331911000001100 | Cipralex 5mg tablets 28 tablet - Lundbeck Ltd |
| 16501711000001106 | Cipralex 5mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 13364811000001107 | Cipralex 5mg tablets 28 tablet - Waymade Healthcare Plc |
| 62511000001109 | Cipramil 10mg tablets - Lundbeck Ltd |
| 5347911000001108 | Cipramil 10mg tablets - Waymade Healthcare Plc |
| 1421111000001108 | Cipramil 10mg tablets 28 tablet - Lundbeck Ltd |
| 5348011000001105 | Cipramil 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 13849411000001103 | Cipramil 20mg tablets - DE Pharmaceuticals |
| 5532311000001109 | Cipramil 20mg tablets - Dowelhurst Ltd |
| 16148511000001107 | Cipramil 20mg tablets - Lexon (UK) Ltd |
| 847211000001102 | Cipramil 20mg tablets - Lundbeck Ltd |
| 16502511000001109 | Cipramil 20mg tablets - Mawdsley-Brooks & Company Ltd |
| 14496111000001103 | Cipramil 20mg tablets - Sigma Pharmaceuticals Plc |
| 5348211000001100 | Cipramil 20mg tablets - Waymade Healthcare Plc |
| 13849511000001104 | Cipramil 20mg tablets 28 tablet - DE Pharmaceuticals |
| 5532411000001102 | Cipramil 20mg tablets 28 tablet - Dowelhurst Ltd |
| 5580611000001109 | Cipramil 20mg tablets 28 tablet - Dowelhurst Ltd |
| 16148611000001106 | Cipramil 20mg tablets 28 tablet - Lexon (UK) Ltd |
| 1421511000001104 | Cipramil 20mg tablets 28 tablet - Lundbeck Ltd |
| 16502611000001108 | Cipramil 20mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 14496211000001109 | Cipramil 20mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 5348311000001108 | Cipramil 20mg tablets 28 tablet - Waymade Healthcare Plc |
| 18522611000001107 | Cipramil 20mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 13849611000001100 | Cipramil 40mg tablets - DE Pharmaceuticals |
| 13107111000001100 | Cipramil 40mg tablets - Dowelhurst Ltd |
| 16148811000001105 | Cipramil 40mg tablets - Lexon (UK) Ltd |
| 695611000001105 | Cipramil 40mg tablets - Lundbeck Ltd |
| 19736911000001101 | Cipramil 40mg tablets - Mawdsley-Brooks & Company Ltd |
| 14496311000001101 | Cipramil 40mg tablets - Sigma Pharmaceuticals Plc |
| 14430311000001101 | Cipidinii Honig tablets - Sigina Filanniaceutitais Fit |

| 10850111000001102 | Cipramil 40mg tablets - Waymade Healthcare Plc |
|---|---|
| 13849711000001109 | Cipramil 40mg tablets 28 tablet - DE Pharmaceuticals |
| 13107311000001103 | Cipramil 40mg tablets 28 tablet - Dowelhurst Ltd |
| 16148911000001100 | Cipramil 40mg tablets 28 tablet - Lexon (UK) Ltd |
| 1422011000001104 | Cipramil 40mg tablets 28 tablet - Lundbeck Ltd |
| 19737011000001102 | Cipramil 40mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 14496411000001108 | Cipramil 40mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 10850211000001108 | Cipramil 40mg tablets 28 tablet - Waymade Healthcare Plc |
| 18629411000001109 | Cipramil 40mg/ml drops - DE Pharmaceuticals |
| 16149011000001109 | Cipramil 40mg/ml drops - Lexon (UK) Ltd |
| 1211000001102 | Cipramil 40mg/ml drops - Lundbeck Ltd |
| 16502311000001103 | Cipramil 40mg/ml drops - Mawdsley-Brooks & Company Ltd |
| 18221011000001101 | Cipramil 40mg/ml drops - Necessity Supplies Ltd |
| 14495911000001107 | Cipramil 40mg/ml drops - Sigma Pharmaceuticals Plc |
| 15883911000001109 | Cipramil 40mg/ml drops - Waymade Healthcare Plc |
| 18629511000001108 | Cipramil 40mg/ml drops 15 ml - DE Pharmaceuticals |
| 16149111000001105 | Cipramil 40mg/ml drops 15 ml - Lexon (UK) Ltd |
| 2730011000001105 | Cipramil 40mg/ml drops 15 ml - Lundbeck Ltd |
| 16502411000001105 | Cipramil 40mg/ml drops 15 ml - Mawdsley-Brooks & Company Ltd |
| 18221111000001100 | Cipramil 40mg/ml drops 15 ml - Necessity Supplies Ltd |
| 14496011000001104 | Cipramil 40mg/ml drops 15 ml - Sigma Pharmaceuticals Plc |
| 15884011000001107 | Cipramil 40mg/ml drops 15 ml - Waymade Healthcare Plc |
| 321989000 | Citalopram 10mg tablets |
| 4011011000001101 | Citalopram 10mg tablets - A A H Pharmaceuticals Ltd |
| 18460711000001104 | Citalopram 10mg tablets - Accord Healthcare Ltd |
| 7394711000001106 | Citalopram 10mg tablets - Actavis UK Ltd |
| 4247611000001101 | Citalopram 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9785611000001105 | Citalopram 10mg tablets - Almus Pharmaceuticals Ltd |
| 10394011000001100 | Citalopram 10mg tablets - Arrow Generics Ltd |
| 15989511000001105 | Citalopram 10mg tablets - Bristol Laboratories Ltd |
| 19714411000001107 | Citalopram 10mg tablets - DE Pharmaceuticals |
| 13224311000001101 | Citalopram 10mg tablets - Dowelhurst Ltd |
| 9448211000001104 | Citalopram 10mg tablets - IVAX Pharmaceuticals UK Ltd |
| 4011411000001105 | Citalopram 10mg tablets - Kent Pharmaceuticals Ltd |
| 37052811000001100 | Citalopram 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 38836011000001102 | Citalopram 10mg tablets - Medihealth (Northern) Ltd |
| 36107611000001101 | Citalopram 10mg tablets - Medinealth (Northern) Eta |
| 19188711000001104 | Citalopram 10mg tablets - Medietch Fit Citalopram 10mg tablets - Milpharm Ltd |
| 4817511000001102 | Citalopram 10mg tablets - Milpharm Etu Citalopram 10mg tablets - Mylan |
| 10443011000001102 | Citalopram 10mg tablets - Mylan Citalopram 10mg tablets - Niche Generics Ltd |
| 37505611000001103 | Citalogram 10mg tablets - Noumed Life Sciences Ltd |
| 17859011000001102 | Citalogram 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 9411011000001105 | Citalogram 10mg tablets - PLIVA Pharma Ltd |
| 7457811000001107 | Citalogram 10mg tablets - Ranbaxy (UK) Ltd |
| 28690311000001101 | Citalogram 10mg tablets - Rivopharm (UK) Ltd |
| 4011711000001104 | Citalopram 10mg tablets - Sandoz Ltd |
| 15079211000001109 | Citalopram 10mg tablets - Sigma Pharmaceuticals Plc |
| 36513711000001107 | Citalopram 10mg tablets - Sovereign Medical Ltd |
| 7396211000001109 | Citalopram 10mg tablets - Teva UK Ltd |

| 13745011000001108 | Citalopram 10mg tablets - Tillomed Laboratories Ltd |
|---|---|
| 21853711000001104 | Citalopram 10mg tablets - Waymade Healthcare Plc |
| 4468311000001101 | Citalopram 10mg tablets - Zentiva Pharma UK Ltd |
| 38194711000001106 | Citalopram 10mg tablets 250 tablet |
| 38194811000001103 | Citalopram 10mg tablets 250 tablet - Mylan |
| 1201711000001104 | Citalopram 10mg tablets 28 tablet Citalopram 10mg tablets 28 tablet |
| 4011211000001106 | Citalopram 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 18461011000001105 | Citalopram 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 7394811000001103 | Citalopram 10mg tablets 28 tablet - Actavis UK Ltd |
| 4247711000001105 | Citalopram 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 9785711000001101 | Citalopram 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 10394211000001105 | Citalopram 10mg tablets 28 tablet - Arrow Generics Ltd |
| 15989611000001109 | Citalopram 10mg tablets 28 tablet - Bristol Laboratories Ltd |
| 19714511000001106 | Citalopram 10mg tablets 28 tablet - DE Pharmaceuticals |
| 13224611000001106 | Citalopram 10mg tablets 28 tablet - Dowelhurst Ltd |
| 9448311000001107 | Citalopram 10mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 4011611000001108 | Citalopram 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 37052911000001105 | Citalopram 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38836111000001101 | Citalopram 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 36107711000001105 | Citalopram 10mg tablets 28 tablet - Medreich Plc |
| 19188811000001107 | Citalopram 10mg tablets 28 tablet - Milpharm Ltd |
| 4817611000001103 | Citalopram 10mg tablets 28 tablet - Mylan |
| 10443111000001104 | Citalopram 10mg tablets 28 tablet - Niche Generics Ltd |
| 37505711000001107 | Citalopram 10mg tablets 28 tablet - Noumed Life Sciences Ltd |
| 17859111000001101 | Citalopram 10mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 9411111000001106 | Citalopram 10mg tablets 28 tablet - PLIVA Pharma Ltd |
| 7457911000001102 | Citalopram 10mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 28690511000001107 | Citalopram 10mg tablets 28 tablet - Rivopharm (UK) Ltd |
| 4011811000001107 | Citalopram 10mg tablets 28 tablet - Sandoz Ltd |
| 15079311000001101 | Citalopram 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 36513811000001104 | Citalopram 10mg tablets 28 tablet - Sovereign Medical Ltd |
| 7396411000001108 | Citalopram 10mg tablets 28 tablet - Teva UK Ltd |
| 13745111000001109 | Citalopram 10mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 21853811000001107 | Citalopram 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 4468511000001107 | Citalopram 10mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 12021011000001104 | Citalopram 10mg/5ml oral suspension |
| 11970211000001108 | Citalopram 10mg/5ml oral suspension - Special Order |
| 11970011000001103 | Citalopram 10mg/5ml oral suspension 1 ml |
| 11970411000001107 | Citalopram 10mg/5ml oral suspension 1 ml - Special Order |
| 321987003 | Citalopram 20mg tablets |
| 4011911000001102 | Citalopram 20mg tablets - A A H Pharmaceuticals Ltd |
| 18460911000001102 | Citalopram 20mg tablets - Accord Healthcare Ltd |
| 7394911000001108 | Citalopram 20mg tablets - Actavis UK Ltd |
| 4247811000001102 | Citalopram 20mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9785811000001109 | Citalopram 20mg tablets - Almus Pharmaceuticals Ltd |
| 13764611000001109 | Citalopram 20mg tablets - Apotex UK Ltd |
| 10394411000001109 | Citalopram 20mg tablets - Arrow Generics Ltd |
| 15989711000001100 | Citalopram 20mg tablets - Bristol Laboratories Ltd |
| 19714611000001105 | Citalopram 20mg tablets - DE Pharmaceuticals |
| | The property of the second sec |

| 5455511000001101 | Citalopram 20mg tablets - Dowelhurst Ltd |
|---|---|
| 9180011000001104 | Citalopram 20mg tablets - IVAX Pharmaceuticals UK Ltd |
| 4012111000001105 | Citalopram 20mg tablets - Kent Pharmaceuticals Ltd |
| 37053111000001101 | Citalopram 20mg tablets - Mawdsley-Brooks & Company Ltd |
| 38836211000001107 | Citalopram 20mg tablets - Medihealth (Northern) Ltd |
| 9180111000001103 | Citalopram 20mg tablets - Medreich Plc |
| 4817711000001107 | Citalopram 20mg tablets - Mylan |
| 10443511000001108 | Citalopram 20mg tablets - Niche Generics Ltd |
| 37505811000001104 | Citalopram 20mg tablets - Noumed Life Sciences Ltd |
| 17859211000001107 | Citalopram 20mg tablets - Phoenix Healthcare Distribution Ltd |
| 9410811000001107 | Citalopram 20mg tablets - PLIVA Pharma Ltd |
| 7458011000001100 | Citalopram 20mg tablets - Ranbaxy (UK) Ltd |
| 28690711000001102 | Citalopram 20mg tablets - Rivopharm (UK) Ltd |
| 4012311000001107 | Citalopram 20mg tablets - Sandoz Ltd |
| 15079511000001107 | Citalopram 20mg tablets - Sigma Pharmaceuticals Plc |
| 36755911000001104 | Citalopram 20mg tablets - Sovereign Medical Ltd |
| 7396511000001107 | Citalopram 20mg tablets - Teva UK Ltd |
| 13745211000001103 | Citalopram 20mg tablets - Tillomed Laboratories Ltd |
| 10508411000001100 | Citalopram 20mg tablets - Waymade Healthcare Plc |
| 21853911000001102 | Citalopram 20mg tablets - Waymade Healthcare Plc |
| 4468611000001106 | Citalopram 20mg tablets - Zentiva Pharma UK Ltd |
| 38195111000001109 | Citalopram 20mg tablets 250 tablet |
| 38195211000001103 | Citalopram 20mg tablets 250 tablet - Mylan |
| 1112911000001109 | Citalopram 20mg tablets 28 tablet |
| 4012011000001109 | Citalopram 20mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 18470011000001107 | Citalopram 20mg tablets 28 tablet - Accord Healthcare Ltd |
| 7395011000001108 | Citalopram 20mg tablets 28 tablet - Actavis UK Ltd |
| 4247911000001107 | Citalopram 20mg tablets 28 tablet - Alliance Healthcare (Distribution)<br>Ltd |
| 9786011000001107 | Citalopram 20mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 13764711000001100 | Citalopram 20mg tablets 28 tablet - Apotex UK Ltd |
| 10394611000001107 | Citalopram 20mg tablets 28 tablet - Arrow Generics Ltd |
| 15989811000001108 | Citalopram 20mg tablets 28 tablet - Bristol Laboratories Ltd |
| 19714711000001101 | Citalopram 20mg tablets 28 tablet - DE Pharmaceuticals |
| 5455611000001102 | Citalopram 20mg tablets 28 tablet - Dowelhurst Ltd |
| 4012211000001104 | Citalopram 20mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 37053211000001107 | Citalopram 20mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38836311000001104 | Citalopram 20mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 4817811000001104 | Citalopram 20mg tablets 28 tablet - Mylan |
| 10443711000001103 | Citalopram 20mg tablets 28 tablet - Niche Generics Ltd |
| 37505911000001109 | Citalopram 20mg tablets 28 tablet - Noumed Life Sciences Ltd |
| 17859311000001104 | Citalopram 20mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 9410911000001102 | Citalopram 20mg tablets 28 tablet - PLIVA Pharma Ltd |
| 7458111000001104 | Citalopram 20mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 28690811000001105 | Citalopram 20mg tablets 28 tablet - Rivopharm (UK) Ltd |
| 4012411000001100 | Citalopram 20mg tablets 28 tablet - Sandoz Ltd |
| 15079711000001102 | Citalopram 20mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 36756011000001107 | Citalopram 20mg tablets 28 tablet - Sovereign Medical Ltd |
| 7396611000001106 | Citalopram 20mg tablets 28 tablet - Teva UK Ltd |
| 13745311000001106 | Citalopram 20mg tablets 28 tablet - Tillomed Laboratories Ltd |
| | 1 . • |

| 10500711000001106 | Citalanuara 20ma tablata 20 tablata Waynaada Haalkhaara Dla |
|---|---|
| 10508711000001106 | Citalogram 20mg tablets 28 tablet - Waymade Healthcare Plc |
| 21854011000001104 | Citalopram 20mg tablets 28 tablet - Waymade Healthcare Plc |
| 4468811000001105 | Citalogram 20mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 18522511000001108 | Citalopram 20mg tablets 30 tablet |
| 11970711000001101 | Citalopram 20mg/5ml oral suspension - Special Order |
| 11970911000001104 | Citalogram 20mg/5ml oral suspension 1 ml - Special Order |
| 321991008 | Citalopram 40mg tablets |
| 4012511000001101 | Citalopram 40mg tablets - A A H Pharmaceuticals Ltd |
| 18470111000001108 | Citalopram 40mg tablets - Accord Healthcare Ltd |
| 7395111000001109 | Citalopram 40mg tablets - Actavis UK Ltd |
| 4248011000001109 | Citalopram 40mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9786311000001105 | Citalopram 40mg tablets - Almus Pharmaceuticals Ltd |
| 13764811000001108 | Citalopram 40mg tablets - Apotex UK Ltd |
| 10394811000001106 | Citalopram 40mg tablets - Arrow Generics Ltd |
| 15989911000001103 | Citalopram 40mg tablets - Bristol Laboratories Ltd |
| 19714811000001109 | Citalopram 40mg tablets - DE Pharmaceuticals |
| 13224811000001105 | Citalopram 40mg tablets - Dowelhurst Ltd |
| 9180211000001109 | Citalopram 40mg tablets - IVAX Pharmaceuticals UK Ltd |
| 4012711000001106 | Citalopram 40mg tablets - Kent Pharmaceuticals Ltd |
| 38836411000001106 | Citalopram 40mg tablets - Medihealth (Northern) Ltd |
| 36438811000001108 | Citalopram 40mg tablets - Medreich Plc |
| 19189311000001109 | Citalopram 40mg tablets - Milpharm Ltd |
| 4817911000001109 | Citalopram 40mg tablets - Mylan |
| 10444011000001103 | Citalopram 40mg tablets - Niche Generics Ltd |
| 37506011000001101 | Citalopram 40mg tablets - Noumed Life Sciences Ltd |
| 17859411000001106 | Citalopram 40mg tablets - Phoenix Healthcare Distribution Ltd |
| 9411411000001101 | Citalopram 40mg tablets - PLIVA Pharma Ltd |
| 7458311000001102 | Citalopram 40mg tablets - Ranbaxy (UK) Ltd |
| 28692211000001105 | Citalopram 40mg tablets - Rivopharm (UK) Ltd |
| 4012911000001108 | Citalopram 40mg tablets - Sandoz Ltd |
| 15079911000001100 | Citalopram 40mg tablets - Sigma Pharmaceuticals Plc |
| 36756111000001108 | Citalopram 40mg tablets - Sovereign Medical Ltd |
| 7396711000001102 | Citalopram 40mg tablets - Teva UK Ltd |
| 13745411000001104 | Citalopram 40mg tablets - Tillomed Laboratories Ltd |
| 21854111000001103 | Citalopram 40mg tablets - Waymade Healthcare Plc |
| 4469011000001109 | Citalopram 40mg tablets - Zentiva Pharma UK Ltd |
| 38195411000001104 | Citalopram 40mg tablets 100 tablet |
| 38195511000001100 | Citalopram 40mg tablets 100 tablet - Mylan |
| 944011000001105 | Citalopram 40mg tablets 28 tablet |
| 4012611000001102 | Citalopram 40mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 18470211000001102 | Citalopram 40mg tablets 28 tablet - Accord Healthcare Ltd |
| 7395211000001103 | Citalopram 40mg tablets 28 tablet - Actavis UK Ltd |
| 4248111000001105 | Citalopram 40mg tablets 28 tablet - Alliance Healthcare (Distribution)<br>Ltd |
| 9786411000001103 | Citalopram 40mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 13764911000001103 | Citalopram 40mg tablets 28 tablet - Apotex UK Ltd |
| 10394911000001101 | Citalopram 40mg tablets 28 tablet - Arrow Generics Ltd |
| 15000011000001100 | Citalopiani 40mg tablets 28 tablet - Arrow Generics Etu |
| 15990011000001106 | Citalopram 40mg tablets 28 tablet - Bristol Laboratories Ltd |
| 15990011000001106<br>19714911000001104 | |

| 9180311000001101<br>4012811000001103 | Citalopram 40mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
|---|---|
| 4012811000001103 | |
| 4012811000001103 | Citalopram 40mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 38836511000001105 | Citalopram 40mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 36438911000001103 | Citalopram 40mg tablets 28 tablet - Medreich Plc |
| 19189411000001102 | Citalopram 40mg tablets 28 tablet - Milpharm Ltd |
| 4818011000001106 | Citalopram 40mg tablets 28 tablet - Mylan |
| 10444111000001102 | Citalopram 40mg tablets 28 tablet - Niche Generics Ltd |
| 37506111000001100 | Citalopram 40mg tablets 28 tablet - Noumed Life Sciences Ltd |
| 17859511000001105 | Citalopram 40mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 9411511000001102 | Citalopram 40mg tablets 28 tablet - PLIVA Pharma Ltd |
| 7458411000001109 | Citalopram 40mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 28692411000001109 | Citalopram 40mg tablets 28 tablet - Rivopharm (UK) Ltd |
| 4013111000001104 | Citalopram 40mg tablets 28 tablet - Sandoz Ltd |
| 15080011000001104 | Citalopram 40mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 36756211000001102 | Citalopram 40mg tablets 28 tablet - Sovereign Medical Ltd |
| 7396811000001105 | Citalopram 40mg tablets 28 tablet - Teva UK Ltd |
| 13745511000001100 | Citalopram 40mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 21854211000001109 | Citalopram 40mg tablets 28 tablet - Waymade Healthcare Plc |
| 4469111000001105 | Citalopram 40mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 321994000 | Citalopram 40mg/ml oral drops sugar free |
| 15262111000001107 | Citalopram 40mg/ml oral drops sugar free - A A H Pharmaceuticals Ltd |
| 16741611000001107 | Citalopram 40mg/ml oral drops sugar free - Actavis UK Ltd |
| 17664211000001107 | Citalopram 40mg/ml oral drops sugar free - Advanz Pharma |
| 17004211000001100 | Citalopram 40mg/ml oral drops sugar free - Advanz Frianna Citalopram 40mg/ml oral drops sugar free - Alliance Healthcare |
| 15247311000001101 | (Distribution) Ltd |
| 17964911000001101 | Citalopram 40mg/ml oral drops sugar free - Almus Pharmaceuticals Ltd |
| 30137211000001101 | Citalopram 40mg/ml oral drops sugar free - DE Pharmaceuticals |
| 38836611000001109 | Citalopram 40mg/ml oral drops sugar free - Medihealth (Northern) Ltd |
| 18100511000001109 | Citalopram 40mg/ml oral drops sugar free - Phoenix Healthcare Distribution Ltd |
| 16421711000001105 | Citalopram 40mg/ml oral drops sugar free - Rosemont Pharmaceuticals Ltd |
| 29788911000001108 | Citalopram 40mg/ml oral drops sugar free - Sigma Pharmaceuticals Plc |
| 15067911000001101 | Citalopram 40mg/ml oral drops sugar free - Teva UK Ltd |
| 37591611000001104 | Citalopram 40mg/ml oral drops sugar free - Thame Laboratories Ltd |
| 21853511000001109 | Citalopram 40mg/ml oral drops sugar free - Waymade Healthcare Plc |
| 1104311000001103 | Citalopram 40mg/ml oral drops sugar free 15 ml |
| 15262311000001109 | Citalopram 40mg/ml oral drops sugar free 15 ml - A A H Pharmaceuticals Ltd |
| 16741711000001103 | Citalopram 40mg/ml oral drops sugar free 15 ml - Actavis UK Ltd |
| 17664311000001103 | Citalopram 40mg/ml oral drops sugar free 15 ml - Advanz Pharma |
| 15247411000001108 | Citalopram 40mg/ml oral drops sugar free 15 ml - Alliance Healthcare (Distribution) Ltd |
| 17965111000001100 | Citalopram 40mg/ml oral drops sugar free 15 ml - Almus<br>Pharmaceuticals Ltd |
| 30137311000001109 | Citalopram 40mg/ml oral drops sugar free 15 ml - DE Pharmaceuticals |
| 38836711000001100 | Citalopram 40mg/ml oral drops sugar free 15 ml - Medihealth (Northern) Ltd |
| 18100611000001108 | Citalopram 40mg/ml oral drops sugar free 15 ml - Phoenix Healthcare Distribution Ltd |

| | Citalopram 40mg/ml oral drops sugar free 15 ml - Sigma |
|---|---|
| 29789011000001104 | Pharmaceuticals Plc |
| 15068111000001103 | Citalopram 40mg/ml oral drops sugar free 15 ml - Teva UK Ltd |
| 37591711000001108 | Citalopram 40mg/ml oral drops sugar free 15 ml - Thame Laboratories Ltd |
| 21853611000001108 | Citalopram 40mg/ml oral drops sugar free 15 ml - Waymade Healthcare Plc |
| 17013011000001106 | Dapoxetine 30mg tablets |
| 21559511000001107 | Dapoxetine 30mg tablets - Special Order |
| 21559411000001108 | Dapoxetine 30mg tablets 1 tablet |
| 21559611000001106 | Dapoxetine 30mg tablets 1 tablet - Special Order |
| 16989211000001105 | Dapoxetine 30mg tablets 3 tablet |
| 16989311000001102 | Dapoxetine 30mg tablets 6 tablet |
| 17013111000001107 | Dapoxetine 60mg tablets |
| 16989711000001103 | Dapoxetine 60mg tablets 3 tablet |
| 16989811000001106 | Dapoxetine 60mg tablets 6 tablet |
| 407915000 | Escitalopram 10mg tablets |
| 3404611000001102 | Escitalopram 10mg tablets |
| 24620411000001102 | Escitalopram 10mg tablets - A A H Pharmaceuticals Ltd |
| 34934011000001102 | Escitalopram 10mg tablets - Accord Healthcare Ltd |
| 24604411000001103 | Escitalopram 10mg tablets - Actavis UK Ltd |
| 24600211000001105 | Escitalopram 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 32496611000001100 | Escitalopram 10mg tablets - Brown & Burk UK Ltd |
| 35923211000001101 | Escitalopram 10mg tablets - Consilient Health Ltd |
| 30054011000001109 | Escitalopram 10mg tablets - DE Pharmaceuticals |
| 32406211000001100 | Escitalopram 10mg tablets - Kent Pharmaceuticals Ltd |
| 29671611000001109 | Escitalopram 10mg tablets - Macleods Pharma UK Ltd |
| 30126011000001105 | Escitalopram 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 38890611000001104 | Escitalopram 10mg tablets - Medihealth (Northern) Ltd |
| 35160211000001103 | Escitalopram 10mg tablets - Milpharm Ltd |
| 33594411000001108 | Escitalopram 10mg tablets - Mylan |
| 14223811000001105 | Escitalopram 10mg tablets - Sigma Pharmaceuticals Plc |
| 29856811000001106 | Escitalopram 10mg tablets - Sigma Pharmaceuticals Plc |
| 24599011000001102 | Escitalopram 10mg tablets - Teva UK Ltd |
| 36829911000001101 | Escitalopram 10mg tablets - Torrent Pharma (UK) Ltd |
| 3388211000001103 | Escitalopram 10mg tablets 28 tablet |
| 24620511000001103 | Escitalopram 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 34934111000001101 | Escitalopram 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 24604511000001104 | Escitalopram 10mg tablets 28 tablet - Actavis UK Ltd |
| 24600311000001102 | Escitalopram 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 32496711000001109 | Escitalopram 10mg tablets 28 tablet - Brown & Burk UK Ltd |
| 35923311000001109 | Escitalopram 10mg tablets 28 tablet - Consilient Health Ltd |
| 30054111000001105 | Escitalopram 10mg tablets 28 tablet - DE Pharmaceuticals |
| 32406311000001108 | Escitalopram 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 29671711000001100 | Escitalopram 10mg tablets 28 tablet - Macleods Pharma UK Ltd |
| 30126111000001106 | Escitalopram 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38890711000001108 | Escitalopram 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 35160311000001106 | Escitalopram 10mg tablets 28 tablet - Milpharm Ltd |
| 33594711000001102 | Escitalopram 10mg tablets 28 tablet - Mylan |
| 14223911000001100 | Escitalopram 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1.223311000001100 | 2501tatoprant 20116 tableto 20 tablet Signia i natifiaceuticais i it |

| 29856911000001101 | Escitalopram 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
|---|---|
| 24599111000001101 | Escitalopram 10mg tablets 28 tablet - Teva UK Ltd |
| 36830011000001106 | Escitalopram 10mg tablets 28 tablet - Torrent Pharma (UK) Ltd |
| 10364811000001108 | Escitalopram 10mg/ml oral drops sugar free |
| 10363911000001100 | Escitalopram 10mg/ml oral drops sugar free 28 ml |
| 409150001 | Escitalopram 5mg tablets |
| 7335411000001106 | Escitalopram 5mg tablets |
| 24620211000001101 | Escitalopram 5mg tablets - A A H Pharmaceuticals Ltd |
| 34934411000001106 | Escitalopram 5mg tablets - Accord Healthcare Ltd |
| 24604211000001102 | Escitalopram 5mg tablets - Actavis UK Ltd |
| 24600011000001100 | Escitalopram 5mg tablets - Alliance Healthcare (Distribution) Ltd |
| 35923011000001106 | Escitalopram 5mg tablets - Consilient Health Ltd |
| 30053811000001101 | Escitalopram 5mg tablets - DE Pharmaceuticals |
| 29671411000001106 | Escitalopram 5mg tablets - Macleods Pharma UK Ltd |
| 30122211000001101 | Escitalopram 5mg tablets - Mawdsley-Brooks & Company Ltd |
| 38891011000001102 | Escitalopram 5mg tablets - Medihealth (Northern) Ltd |
| 33595111000001104 | Escitalopram 5mg tablets - Mylan |
| 29857211000001107 | Escitalopram 5mg tablets - Sigma Pharmaceuticals Plc |
| 24598811000001101 | Escitalopram 5mg tablets - Teva UK Ltd |
| 36829711000001103 | Escitalopram 5mg tablets - Torrent Pharma (UK) Ltd |
| 25557111000001108 | Escitalopram 5mg tablets - Zentiva Pharma UK Ltd |
| 7331711000001102 | Escitalopram 5mg tablets 28 tablet |
| 24620311000001109 | Escitalopram 5mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 34934511000001105 | Escitalopram 5mg tablets 28 tablet - Accord Healthcare Ltd |
| 24604311000001105 | Escitalopram 5mg tablets 28 tablet - Actavis UK Ltd |
| 24600111000001104 | Escitalopram 5mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 35923111000001107 | Escitalopram 5mg tablets 28 tablet - Consilient Health Ltd |
| 30053911000001106 | Escitalopram 5mg tablets 28 tablet - DE Pharmaceuticals |
| 29671511000001105 | Escitalopram 5mg tablets 28 tablet - Macleods Pharma UK Ltd |
| 30122311000001109 | Escitalopram 5mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38891111000001101 | Escitalopram 5mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 33595211000001105 | Escitalopram 5mg tablets 28 tablet - Mylan |
| 29857311000001104 | Escitalopram 5mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 24598911000001106 | Escitalopram 5mg tablets 28 tablet - Teva UK Ltd |
| 36829811000001106 | Escitalopram 5mg tablets 28 tablet - Torrent Pharma (UK) Ltd |
| 25557311000001105 | Escitalopram 5mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 24604611000001100 | Escitalopram 20mg tablets - Actavis UK Ltd |
| 24604711000001109 | Escitalopram 20mg tablets 28 tablet - Actavis UK Ltd |
| 408067001 | Escitalopram 20mg tablets |
| 4942411000001101 | Escitalopram 20mg tablets 28 tablet |
| 30126211000001100 | Escitalopram 20mg tablets - Mawdsley-Brooks & Company Ltd |
| 30126311000001108 | Escitalopram 20mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 32489411000001109 | Escitalopram 20mg tablets - Brown & Burk UK Ltd |
| 32489511000001108 | Escitalopram 20mg tablets 28 tablet - Brown & Burk UK Ltd |
| 29671811000001108 | Escitalopram 20mg tablets - Macleods Pharma UK Ltd |
| 29671911000001103 | Escitalopram 20mg tablets 28 tablet - Macleods Pharma UK Ltd |
| 35160411000001104 | Escitalopram 20mg tablets - Milpharm Ltd |
| 35160511000001100 | Escitalopram 20mg tablets 28 tablet - Milpharm Ltd |
| 34933811000001105 | Escitalopram 20mg tablets - Accord Healthcare Ltd |

| 34933911000001100 | Escitalopram 20mg tablets 28 tablet - Accord Healthcare Ltd |
|---|---|
| 24601911000001108 | Escitalopram 20mg tablets - Alliance Healthcare (Distribution) Ltd |
| 24602011000001101 | Escitalopram 20mg tablets 28 tablet - Alliance Healthcare (Distribution) |
| 33594211000001109 | Ltd Escitalopram 20mg tablets - Mylan |
| 33594311000001101 | Escitalopram 20mg tablets - Mylan Escitalopram 20mg tablets 28 tablet - Mylan |
| 36830111000001107 | Escitalopram 20mg tablets - Torrent Pharma (UK) Ltd |
| 36830211000001107 | Escitalopram 20mg tablets - Torrent Pharma (UK) Ltd Escitalopram 20mg tablets 28 tablet - Torrent Pharma (UK) Ltd |
| 35923411000001102 | Escitalopram 20mg tablets - Consilient Health Ltd |
| 35923511000001103 | Escitalopram 20mg tablets 28 tablet - Consilient Health Ltd |
| 30054211000001104 | Escitalogram 20mg tablets - DE Pharmaceuticals |
| 30054311000001107 | Escitalogram 20mg tablets 28 tablet - DE Pharmaceuticals |
| 38890811000001100 | Escitalopram 20mg tablets - Medihealth (Northern) Ltd |
| 38890911000001105 | Escitalopram 20mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 29857011000001102 | Escitalopram 20mg tablets - Sigma Pharmaceuticals Plc |
| 29857111000001101 | Escitalopram 20mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 24620611000001104 | Escitalopram 20mg tablets - A A H Pharmaceuticals Ltd |
| 24620711000001108 | Escitalopram 20mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 24599211000001107 | Escitalopram 20mg tablets - Teva UK Ltd |
| 24599311000001104 | Escitalopram 20mg tablets 28 tablet - Teva UK Ltd |
| 595611000001101 | Faverin 100mg tablets - Mylan |
| 2614511000001107 | Faverin 100mg tablets 30 tablet - Mylan |
| 542511000001103 | Faverin 50mg tablets - Mylan |
| 2611511000001105 | Faverin 50mg tablets 60 tablet - Mylan |
| 456311000001103 | Felicium 20mg capsules - Opus Pharmaceuticals Ltd |
| 1402111000001109 | Felicium 20mg capsules 30 capsule - Opus Pharmaceuticals Ltd |
| 373959000 | Fluoxetine 10mg capsules |
| 33424811000001109 | Fluoxetine 10mg capsules - A A H Pharmaceuticals Ltd |
| 35850211000001104 | Fluoxetine 10mg capsules - Accord Healthcare Ltd |
| 32907711000001107 | Fluoxetine 10mg capsules - Alliance Healthcare (Distribution) Ltd |
| 37381911000001108 | Fluoxetine 10mg capsules - DE Pharmaceuticals |
| 37069211000001101 | Fluoxetine 10mg capsules - Mawdsley-Brooks & Company Ltd |
| 38916811000001106 | Fluoxetine 10mg capsules - Medihealth (Northern) Ltd |
| 32745811000001106 | Fluoxetine 10mg capsules - Medreich Plc |
| 35989211000001105 | Fluoxetine 10mg capsules - Morningside Healthcare Ltd |
| 32745711000001103 | Fluoxetine 10mg capsules 30 capsule |
| 33424911000001104 | Fluoxetine 10mg capsules 30 capsule - A A H Pharmaceuticals Ltd |
| 35850311000001107 | Fluoxetine 10mg capsules 30 capsule - Accord Healthcare Ltd |
| 32907811000001104 | Fluoxetine 10mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd |
| 37382111000001100 | Fluoxetine 10mg capsules 30 capsule - DE Pharmaceuticals |
| 37069311000001109 | Fluoxetine 10mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| 38916911000001101 | Fluoxetine 10mg capsules 30 capsule - Medihealth (Northern) Ltd |
| 32745911000001101 | Fluoxetine 10mg capsules 30 capsule - Medreich Plc |
| 35989311000001102 | Fluoxetine 10mg capsules 30 capsule - Morningside Healthcare Ltd |
| 373965000 | Fluoxetine 10mg tablets |
| 34894211000001108 | Fluoxetine 10mg tablets - A A H Pharmaceuticals Ltd |
| 34905711000001108 | Fluoxetine 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37384811000001101 | Fluoxetine 10mg tablets - DE Pharmaceuticals |
| 34732311000001100 | Fluoxetine 10mg tablets - Endo Ventures Ltd |
| 3-73231100001100 | Transcribe Tonig tablets - Lilao ventales eta |

| 38962111000001102 | Fluoxetine 10mg tablets - Imported |
|---|---|
| 38917011000001102 | Fluoxetine 10mg tablets - Medihealth (Northern) Ltd |
| 16676011000001103 | Fluoxetine 10mg tablets - Special Order |
| 16675911000001106 | Fluoxetine 10mg tablets 1 tablet |
| 16676111000001102 | Fluoxetine 10mg tablets 1 tablet - Special Order |
| 34732211000001108 | Fluoxetine 10mg tablets 30 tablet |
| 34894311000001100 | Fluoxetine 10mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 34905811000001100 | Fluoxetine 10mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 37384911000001106 | Fluoxetine 10mg tablets 30 tablet - DE Pharmaceuticals |
| 34732411000001107 | Fluoxetine 10mg tablets 30 tablet - Endo Ventures Ltd |
| 38962211000001108 | Fluoxetine 10mg tablets 30 tablet - Imported |
| 38917111000001101 | Fluoxetine 10mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 36002911000001103 | Fluoxetine 10mg/5ml oral suspension |
| 35989511000001108 | Fluoxetine 10mg/5ml oral suspension - Special Order |
| 35989411000001109 | Fluoxetine 10mg/5ml oral suspension 1 ml |
| 35989611000001107 | Fluoxetine 10mg/5ml oral suspension 1 ml - Special Order |
| 8516511000001104 | Fluoxetine 2.5mg/5ml oral solution |
| 8483611000001103 | Fluoxetine 2.5mg/5ml oral solution - Special Order |
| 8483111000001106 | Fluoxetine 2.5mg/5ml oral solution 1 ml |
| 8483811000001104 | Fluoxetine 2.5mg/5ml oral solution 1 ml - Special Order |
| 8516611000001100 | Fluoxetine 2.5mg/5ml oral suspension |
| 8484111000001108 | Fluoxetine 2.5mg/5ml oral suspension - Special Order |
| 8484011000001107 | Fluoxetine 2.5mg/5ml oral suspension 1 ml |
| 8484411000001103 | Fluoxetine 2.5mg/5ml oral suspension 1 ml - Special Order |
| 321949006 | Fluoxetine 20mg capsules |
| 723711000001104 | Fluoxetine 20mg capsules - A A H Pharmaceuticals Ltd |
| 18461711000001107 | Fluoxetine 20mg capsules - Accord Healthcare Ltd |
| 335911000001100 | Fluoxetine 20mg capsules - Actavis UK Ltd |
| 453911000001108 | Fluoxetine 20mg capsules - Alliance Healthcare (Distribution) Ltd |
| 9799811000001108 | Fluoxetine 20mg capsules - Almus Pharmaceuticals Ltd |
| 10408211000001105 | Fluoxetine 20mg capsules - Arrow Generics Ltd |
| 23587411000001103 | Fluoxetine 20mg capsules - Bristol Laboratories Ltd |
| 32489611000001107 | Fluoxetine 20mg capsules - Brown & Burk UK Ltd |
| 23909011000001106 | Fluoxetine 20mg capsules - DE Pharmaceuticals |
| 5505911000001108 | Fluoxetine 20mg capsules - Dowelhurst Ltd |
| 11018011000001101 | Fluoxetine 20mg capsules - Dr Reddys Laboratories (UK) Ltd |
| 18074311000001105 | Fluoxetine 20mg capsules - Fannin (UK) Ltd |
| 37593011000001107 | Fluoxetine 20mg capsules - Flamingo Pharma (UK) Ltd |
| 33555411000001101 | Fluoxetine 20mg capsules - Genesis Pharmaceuticals Ltd |
| 848111000001109 | Fluoxetine 20mg capsules - Genus Pharmaceuticals Ltd |
| 258111000001102 | Fluoxetine 20mg capsules - IVAX Pharmaceuticals UK Ltd |
| 614811000001109 | Fluoxetine 20mg capsules - Kent Pharmaceuticals Ltd |
| 30131811000001107 | Fluoxetine 20mg capsules - Mawdsley-Brooks & Company Ltd |
| 38917611000001109 | Fluoxetine 20mg capsules - Medihealth (Northern) Ltd |
| 32938411000001107 | Fluoxetine 20mg capsules - Medreich Plc |
| 19193611000001100 | Fluoxetine 20mg capsules - Medielch Fluoxetine 20mg capsules - Milpharm Ltd |
| 24132411000001103 | Fluoxetine 20mg capsules - Minmarin Ltu Fluoxetine 20mg capsules - Morningside Healthcare Ltd |
| 252411000001105 | Fluoxetine 20mg capsules - Morningside Healthcare Ltd Fluoxetine 20mg capsules - Mylan |
| 10444811000001109 | Fluoxetine 20mg capsules - Nylan Fluoxetine 20mg capsules - Niche Generics Ltd |
| 10444011000001103 | Fluoxetine Zonig capsules - Niche Generics Lta |

| 17909511000001108 | Fluoxetine 20mg capsules - Phoenix Healthcare Distribution Ltd |
|---|---|
| 166911000001109 | Fluoxetine 20mg capsules - Ranbaxy (UK) Ltd |
| 37091511000001101 | Fluoxetine 20mg capsules - Relonchem Ltd |
| 527811000001100 | Fluoxetine 20mg capsules - Sandoz Ltd |
| 15209011000001100 | Fluoxetine 20mg capsules - Sigma Pharmaceuticals Plc |
| 18282511000001107 | Fluoxetine 20mg capsules - Strides Pharma UK Ltd |
| 756611000001101 | Fluoxetine 20mg capsules - Teva UK Ltd |
| 13751411000001100 | Fluoxetine 20mg capsules - Tillomed Laboratories Ltd |
| 22014311000001108 | Fluoxetine 20mg capsules - Waymade Healthcare Plc |
| 12909311000001100 | Fluoxetine 20mg capsules - Wockhardt UK Ltd |
| 560111000001104 | Fluoxetine 20mg capsules - Zentiva Pharma UK Ltd |
| 37765011000001107 | Fluoxetine 20mg capsules 100 capsule |
| 37765111000001107 | |
| | Fluoretine 20mg capsules 100 capsule - Mylan |
| 5404511000001109 | Fluoxetine 20mg capsules 28 capsule |
| 5506111000001104 | Fluoxetine 20mg capsules 28 capsule - Dowelhurst Ltd |
| 15209111000001104 | Fluoxetine 20mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 1214811000001107 | Fluoxetine 20mg capsules 30 capsule |
| 1400511000001101 | Fluoxetine 20mg capsules 30 capsule - A A H Pharmaceuticals Ltd |
| 18461811000001104 | Fluoxetine 20mg capsules 30 capsule - Accord Healthcare Ltd |
| 1400711000001106 | Fluoxetine 20mg capsules 30 capsule - Actavis UK Ltd |
| 1402811000001102 | Fluoxetine 20mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd |
| 9799911000001103 | Fluoxetine 20mg capsules 30 capsule - Almus Pharmaceuticals Ltd |
| 10408311000001102 | Fluoxetine 20mg capsules 30 capsule - Arrow Generics Ltd |
| 23587511000001104 | Fluoxetine 20mg capsules 30 capsule - Bristol Laboratories Ltd |
| 32489711000001103 | Fluoxetine 20mg capsules 30 capsule - Brown & Burk UK Ltd |
| 23909111000001107 | Fluoxetine 20mg capsules 30 capsule - DE Pharmaceuticals |
| 11018211000001106 | Fluoxetine 20mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd |
| 18074611000001100 | Fluoxetine 20mg capsules 30 capsule - Fannin (UK) Ltd |
| 37593211000001102 | Fluoxetine 20mg capsules 30 capsule - Flamingo Pharma (UK) Ltd |
| 33555511000001102 | Fluoxetine 20mg capsules 30 capsule - Genesis Pharmaceuticals Ltd |
| 1401111000001104 | Fluoxetine 20mg capsules 30 capsule - Genus Pharmaceuticals Ltd |
| 1401311000001102 | Fluoxetine 20mg capsules 30 capsule - IVAX Pharmaceuticals UK Ltd |
| 1401611000001107 | Fluoxetine 20mg capsules 30 capsule - Kent Pharmaceuticals Ltd |
| 30131911000001102 | Fluoxetine 20mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| 38917711000001100 | Fluoxetine 20mg capsules 30 capsule - Medihealth (Northern) Ltd |
| 32938511000001106 | Fluoxetine 20mg capsules 30 capsule - Medreich Plc |
| 19193711000001109 | Fluoxetine 20mg capsules 30 capsule - Milpharm Ltd |
| 24132611000001100 | Fluoxetine 20mg capsules 30 capsule - Morningside Healthcare Ltd |
| 1400911000001108 | Fluoxetine 20mg capsules 30 capsule - Mylan |
| 10445011000001104 | Fluoxetine 20mg capsules 30 capsule - Niche Generics Ltd |
| 17909611000001107 | Fluoxetine 20mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd |
| 1402511000001100 | Fluoxetine 20mg capsules 30 capsule - Ranbaxy (UK) Ltd |
| 37091811000001103 | Fluoxetine 20mg capsules 30 capsule - Relonchem Ltd |
| 1401711000001103 | Fluoxetine 20mg capsules 30 capsule - Sandoz Ltd |
| 15209411000001109 | Fluoxetine 20mg capsules 30 capsule - Samuoz Etu Fluoxetine 20mg capsules 30 capsule - Sigma Pharmaceuticals Plc |
| 18282611000001106 | Fluoxetine 20mg capsules 30 capsule - Strides Pharma UK Ltd |
| 1400811000001103 | Fluoretine 20mg capsules 30 capsule - Teva UK Ltd |
| 13751511000001101 | Fluoxetine 20mg capsules 30 capsule - Tillomed Laboratories Ltd |

| 22014411000001101 | Fluoxetine 20mg capsules 30 capsule - Waymade Healthcare Plc |
|---|---|
| 12909511000001101 | Fluoxetine 20mg capsules 30 capsule - Waymade Healthcare Fit |
| 1402711000001105<br>321951005 | Fluoxetine 20mg capsules 30 capsule - Zentiva Pharma UK Ltd Fluoxetine 20mg/5ml oral solution |
| 437511000001107 | Fluoxetine 20mg/5ml oral solution - A A H Pharmaceuticals Ltd Fluoxetine 20mg/5ml oral solution - Alliance Healthcare (Distribution) |
| 476511000001107 | Ltd |
| 17970711000001104 | Fluoxetine 20mg/5ml oral solution - Almus Pharmaceuticals Ltd |
| 23980211000001107 | Fluoxetine 20mg/5ml oral solution - DE Pharmaceuticals |
| 5504511000001102 | Fluoxetine 20mg/5ml oral solution - Dowelhurst Ltd |
| 18073311000001108 | Fluoxetine 20mg/5ml oral solution - Fannin (UK) Ltd |
| 10307911000001105 | Fluoxetine 20mg/5ml oral solution - Focus Pharmaceuticals Ltd |
| 4576111000001104 | Fluoxetine 20mg/5ml oral solution - IVAX Pharmaceuticals UK Ltd |
| 321711000001101 | Fluoxetine 20mg/5ml oral solution - Kent Pharmaceuticals Ltd |
| 30810711000001106 | Fluoxetine 20mg/5ml oral solution - Mawdsley-Brooks & Company Ltd |
| 38918211000001106 | Fluoxetine 20mg/5ml oral solution - Medihealth (Northern) Ltd |
| 9480011000001103 | Fluoxetine 20mg/5ml oral solution - Mylan |
| 18108111000001103 | Fluoxetine 20mg/5ml oral solution - Phoenix Healthcare Distribution Ltd |
| 13621511000001108 | Fluoxetine 20mg/5ml oral solution - Pinewood Healthcare |
| 4331011000001108 | Fluoxetine 20mg/5ml oral solution - Sandoz Ltd |
| 29866111000001106 | Fluoxetine 20mg/5ml oral solution - Sigma Pharmaceuticals Plc |
| 263811000001105 | Fluoxetine 20mg/5ml oral solution - Teva UK Ltd |
| 22014711000001107 | Fluoxetine 20mg/5ml oral solution - Waymade Healthcare Plc |
| 1074111000001101 | Fluoxetine 20mg/5ml oral solution 70 ml |
| 2182611000001102 | Fluoxetine 20mg/5ml oral solution 70 ml - A A H Pharmaceuticals Ltd |
| 2183011000001100 | Fluoxetine 20mg/5ml oral solution 70 ml - Alliance Healthcare (Distribution) Ltd |
| 17970911000001102 | Fluoxetine 20mg/5ml oral solution 70 ml - Almus Pharmaceuticals Ltd |
| 23980311000001104 | Fluoxetine 20mg/5ml oral solution 70 ml - DE Pharmaceuticals |
| 5504711000001107 | Fluoxetine 20mg/5ml oral solution 70 ml - Dowelhurst Ltd |
| 18073411000001101 | Fluoxetine 20mg/5ml oral solution 70 ml - Fannin (UK) Ltd |
| 10308111000001108 | Fluoxetine 20mg/5ml oral solution 70 ml - Focus Pharmaceuticals Ltd |
| 4576211000001105 | Fluoxetine 20mg/5ml oral solution 70 ml - IVAX Pharmaceuticals UK Ltd |
| 2257911000001101 | Fluoxetine 20mg/5ml oral solution 70 ml - Kent Pharmaceuticals Ltd |
| 30810811000001103 | Fluoxetine 20mg/5ml oral solution 70 ml - Mawdsley-Brooks & Company Ltd |
| 38918311000001103 | Fluoxetine 20mg/5ml oral solution 70 ml - Medihealth (Northern) Ltd |
| 9480111000001102 | Fluoxetine 20mg/5ml oral solution 70 ml - Mylan |
| 18108211000001109 | Fluoxetine 20mg/5ml oral solution 70 ml - Phoenix Healthcare Distribution Ltd |
| 13621611000001107 | Fluoxetine 20mg/5ml oral solution 70 ml - Pinewood Healthcare |
| 4331111000001109 | Fluoxetine 20mg/5ml oral solution 70 ml - Sandoz Ltd |
| 29866211000001100 | Fluoxetine 20mg/5ml oral solution 70 ml - Sigma Pharmaceuticals Plc |
| 2182411000001100 | Fluoxetine 20mg/5ml oral solution 70 ml - Teva UK Ltd |
| 22014811000001104 | Fluoxetine 20mg/5ml oral solution 70 ml - Waymade Healthcare Plc |
| 11590211000001106 | Fluoxetine 20mg/5ml oral solution sugar free |
| 34036311000001104 | Fluoxetine 20mg/5ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 18802911000001109 | Fluoxetine 20mg/5ml oral solution sugar free - Accord Healthcare Ltd |
| 32332211000001102 | Fluoxetine 20mg/5ml oral solution sugar free - Colorama Pharmaceuticals Ltd |
| 37384511000001104 | Fluoxetine 20mg/5ml oral solution sugar free - DE Pharmaceuticals |
| | - |

| 26055211000001106 | Fluoxetine 20mg/5ml oral solution sugar free - Ennogen Healthcare Ltd |
|---|---|
| 31406111000001105 | Fluoxetine 20mg/5ml oral solution sugar free - J M McGill Ltd |
| 38918411000001105 | Fluoxetine 20mg/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 24227311000001107 | Fluoxetine 20mg/5ml oral solution sugar free - Morningside Healthcare Ltd |
| 11581111000001107 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml |
| 34036411000001106 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - A A H Pharmaceuticals Ltd |
| 18803011000001101 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - Accord Healthcare Ltd |
| 32332511000001104 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - Colorama<br>Pharmaceuticals Ltd |
| 37384711000001109 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - DE Pharmaceuticals |
| 26055411000001105 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - Ennogen Healthcare Ltd |
| 31406211000001104 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - J M McGill Ltd |
| 38918511000001109 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - Medihealth (Northern) Ltd |
| 24227411000001100 | Fluoxetine 20mg/5ml oral solution sugar free 70 ml - Morningside<br>Healthcare Ltd |
| 15880011000001100 | Fluoxetine 2mg/5ml oral solution |
| 15862311000001100 | Fluoxetine 2mg/5ml oral solution - Special Order |
| 15862211000001108 | Fluoxetine 2mg/5ml oral solution 1 ml |
| 15862411000001107 | Fluoxetine 2mg/5ml oral solution 1 ml - Special Order |
| 15880111000001104 | Fluoxetine 2mg/5ml oral suspension |
| 15863111000001108 | Fluoxetine 2mg/5ml oral suspension - Special Order |
| 15862811000001109 | Fluoxetine 2mg/5ml oral suspension 1 ml |
| 15863311000001105 | Fluoxetine 2mg/5ml oral suspension 1 ml - Special Order |
| 32960811000001102 | Fluoxetine 30mg capsules |
| 33425011000001104 | Fluoxetine 30mg capsules - A A H Pharmaceuticals Ltd |
| 33427811000001100 | Fluoxetine 30mg capsules - Alliance Healthcare (Distribution) Ltd |
| 37384011000001107 | Fluoxetine 30mg capsules - DE Pharmaceuticals |
| 38962311000001100 | Fluoxetine 30mg capsules - Imported |
| 37077011000001105 | Fluoxetine 30mg capsules - Mawdsley-Brooks & Company Ltd |
| 38917811000001108 | Fluoxetine 30mg capsules - Medihealth (Northern) Ltd |
| 32938711000001101 | Fluoxetine 30mg capsules - Medreich Plc |
| 32938611000001105 | Fluoxetine 30mg capsules 30 capsule |
| 33425111000001103 | Fluoxetine 30mg capsules 30 capsule - A A H Pharmaceuticals Ltd |
| 33427911000001105 | Fluoxetine 30mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd |
| 37384111000001108 | Fluoxetine 30mg capsules 30 capsule - DE Pharmaceuticals |
| 38962511000001106 | Fluoxetine 30mg capsules 30 capsule - Imported |
| 37077411000001101 | Fluoxetine 30mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| 38917911000001103 | Fluoxetine 30mg capsules 30 capsule - Medihealth (Northern) Ltd |
| 32938811000001109 | Fluoxetine 30mg capsules 30 capsule - Medreich Plc |
| 376803002 | Fluoxetine 40mg capsules |
| 33425211000001109 | Fluoxetine 40mg capsules - A A H Pharmaceuticals Ltd |
| 33428011000001107 | Fluoxetine 40mg capsules - Alliance Healthcare (Distribution) Ltd |
| 37384211000001102 | Fluoxetine 40mg capsules - DE Pharmaceuticals |
| 38962811000001109 | Fluoxetine 40mg capsules - Imported |
| 37077611000001103 | Fluoxetine 40mg capsules - Mawdsley-Brooks & Company Ltd |
| Fluoxetine 40mg capsules - Special Order | 32939011000001108 | Fluoxetine 40mg capsules - Medreich Plc |
|---|---|---|
| Sepsein Fluoxetine Fluoxe | | |
| Fluoxetine 40mg capsules 1 capsule - Special Order | | |
| Pluoxetine 40mg capsules 30 capsule - A A H Pharmaceuticals Ltd | | |
| Fluoxetine 40mg capsules 30 capsule - A A H Pharmaceuticals Ltd | | |
| Fluoxetine 40mg capsules 30 capsule - Alliance Healthcare (Distribution) It | | |
| Ital | | |
| Fluoxetine 40mg capsules 30 capsule - Imported | 33428111000001108 | |
| Fluoxetine 40mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd | 37384311000001105 | Fluoxetine 40mg capsules 30 capsule - DE Pharmaceuticals |
| Fluoxetine 40mg capsules 30 capsule - Medreich Plc | 38962911000001104 | Fluoxetine 40mg capsules 30 capsule - Imported |
| Fluoxetine 60mg capsules Fluoxetine 60mg cap | 37077711000001107 | Fluoxetine 40mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| Fluoxetine 60mg capsules - A A H Pharmaceuticals Ltd | 32939111000001109 | Fluoxetine 40mg capsules 30 capsule - Medreich Plc |
| 17219811000001108 | 321954002 | Fluoxetine 60mg capsules |
| Fluoxetine 60mg capsules - Advanz Pharma | 9530611000001107 | Fluoxetine 60mg capsules - A A H Pharmaceuticals Ltd |
| 4572511000001107 Fluoxetine 60mg capsules - Alliance Healthcare (Distribution) Ltd 19818411000001100 Fluoxetine 60mg capsules - Almus Pharmaceuticals Ltd 23980011000001102 Fluoxetine 60mg capsules - Bristol Laboratories Ltd 23980011000001102 Fluoxetine 60mg capsules - DE Pharmaceuticals 18475711000001104 Fluoxetine 60mg capsules - DE Pharmaceuticals 18475711000001102 Fluoxetine 60mg capsules - DE Pharmaceuticals Ltd 30132011000001109 Fluoxetine 60mg capsules - Kent Pharmaceuticals Ltd 30132011000001101 Fluoxetine 60mg capsules - Medihealth (Northern) Ltd 32938211000001108 Fluoxetine 60mg capsules - Medihealth (Northern) Ltd 32938211000001107 Fluoxetine 60mg capsules - Medihealth (Northern) Ltd 32938211000001107 Fluoxetine 60mg capsules - Milpharm Ltd 33162011000001107 Fluoxetine 60mg capsules - Milpharm Ltd 33162011000001101 Fluoxetine 60mg capsules - Mylan 33162011000001101 Fluoxetine 60mg capsules - Phoenix Healthcare Distribution Ltd 34956411000001101 Fluoxetine 60mg capsules - Sigma Pharmaceuticals Ptc 34956411000001102 Fluoxetine 60mg capsules - Waymade Healthcare Ptc 328011000001103 Fluoxetine 60mg capsules - Waymade Healthcare Ptc 328011000001103 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 37219911000001103 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 37219911000001103 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 3721911000001107 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 3721911000001106 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 3726611000001106 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 37267711000001107 Fluoxetine 60mg capsules 30 capsule - A Harmaceuticals Ltd 372687711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 372687711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 372687711000001109 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Ltd 372687711000001109 Fluoxetine 60mg capsules 30 caps | 17219811000001108 | Fluoxetine 60mg capsules - Actavis UK Ltd |
| 19818411000001100 | 29922611000001103 | Fluoxetine 60mg capsules - Advanz Pharma |
| Fluoxetine 60mg capsules - Bristol Laboratories Ltd | 4572511000001107 | Fluoxetine 60mg capsules - Alliance Healthcare (Distribution) Ltd |
| Fluoxetine 60mg capsules - DE Pharmaceuticals | 19818411000001100 | Fluoxetine 60mg capsules - Almus Pharmaceuticals Ltd |
| Fluoxetine 60mg capsules - Dr Reddys Laboratories (UK) Ltd | 23587611000001100 | Fluoxetine 60mg capsules - Bristol Laboratories Ltd |
| Fluoxetine 60mg capsules - Kent Pharmaceuticals Ltd 30132011000001109 Fluoxetine 60mg capsules - Mawdsley-Brooks & Company Ltd 38918011000001101 Fluoxetine 60mg capsules - Medihealth (Northern) Ltd 32938211000001107 Fluoxetine 60mg capsules - Medireich Plc 35162011000001107 Fluoxetine 60mg capsules - Milipharm Ltd 3962111000001101 Fluoxetine 60mg capsules - Mylan 17909711000001103 Fluoxetine 60mg capsules - Mylan 17909711000001101 Fluoxetine 60mg capsules - Phoenix Healthcare Distribution Ltd 15088111000001101 Fluoxetine 60mg capsules - Sigma Pharmaceuticals Plc 14956411000001101 Fluoxetine 60mg capsules - Teva UK Ltd 22014511000001102 Fluoxetine 60mg capsules - Waymade Healthcare Plc 1288011000001108 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001103 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001106 Fluoxetine 60mg capsules 30 capsule - Advanz Pharma 4572611000001106 Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd 23587711000001101 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23587711000001109 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Ltd 36132111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Ltd 764711000001108 Fluoxetine 60mg capsules 30 capsule - De Pharmaceuticals Ltd 3898111000001107 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38981811000001100 Fluoxetine 60mg capsules 30 capsule - Medriech Plc 3182111000001100 Fluoxetine 60mg capsules 30 capsule - Medriech Plc 31938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 319081100001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 319081100001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 319081100001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 319081100001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 319081100001100 Fluoxetine 60mg capsules | 23980011000001102 | Fluoxetine 60mg capsules - DE Pharmaceuticals |
| Silvantine 60mg capsules - Mawdsley-Brooks & Company Ltd | 18475711000001104 | Fluoxetine 60mg capsules - Dr Reddys Laboratories (UK) Ltd |
| 38918011000001101 Fluoxetine 60mg capsules - Medihealth (Northern) Ltd 32938211000001107 Fluoxetine 60mg capsules - Medreich Plc 35162011000001107 Fluoxetine 60mg capsules - Milpharm Ltd 3962111000001101 Fluoxetine 60mg capsules - Mylan 17909711000001103 Fluoxetine 60mg capsules - Phoenix Healthcare Distribution Ltd 15088111000001101 Fluoxetine 60mg capsules - Sigma Pharmaceuticals Plc 14956411000001101 Fluoxetine 60mg capsules - Teva UK Ltd 22014511000001102 Fluoxetine 60mg capsules - Waymade Healthcare Plc 1288011000001103 Fluoxetine 60mg capsules 30 capsule 953071100001103 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001103 Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd 29922711000001107 Fluoxetine 60mg capsules 30 capsule - Advanz Pharma 4572611000001106 Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23587711000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Ltd 17764711000001103 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001101 Fluoxetine 60mg capsules 30 capsule - DR Reddys Laboratories (UK) Ltd 17764711000001108 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 33938111000001105 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 31032111000001106 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 31032111000001106 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 31032111000001106 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 31032111000001106 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 3103211000001106 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 3103211000001106 Fluoxeti | 7764411000001102 | Fluoxetine 60mg capsules - Kent Pharmaceuticals Ltd |
| Fluoxetine 60mg capsules - Medreich Plc | 30132011000001109 | Fluoxetine 60mg capsules - Mawdsley-Brooks & Company Ltd |
| Fluoxetine 60mg capsules - Milpharm Ltd | 38918011000001101 | Fluoxetine 60mg capsules - Medihealth (Northern) Ltd |
| Fluoxetine 60mg capsules - Mylan | 32938211000001108 | Fluoxetine 60mg capsules - Medreich Plc |
| Fluoxetine 60mg capsules - Phoenix Healthcare Distribution Ltd | 35162011000001107 | Fluoxetine 60mg capsules - Milpharm Ltd |
| Fluoxetine 60mg capsules - Sigma Pharmaceuticals Plc | 3962111000001101 | Fluoxetine 60mg capsules - Mylan |
| 1495641100001101Fluoxetine 60mg capsules - Teva UK Ltd22014511000001102Fluoxetine 60mg capsules - Waymade Healthcare Plc1288011000001108Fluoxetine 60mg capsules 30 capsule9530711000001103Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd17219911000001103Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd29922711000001107Fluoxetine 60mg capsules 30 capsule - Advanz Pharma4572611000001106Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution)<br>Ltd19818511000001101Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd23587711000001109Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals18475811000001101Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals18475811000001107Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd7764711000001108Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd30132111000001105Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd32938311000001100Fluoxetine 60mg capsules 30 capsule - Medreich Plc35162111000001108Fluoxetine 60mg capsules 30 capsule - Medreich Plc35162111000001106Fluoxetine 60mg capsules 30 capsule - Mylan17909811000001106Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution<br>Ltd | 17909711000001103 | Fluoxetine 60mg capsules - Phoenix Healthcare Distribution Ltd |
| Fluoxetine 60mg capsules - Waymade Healthcare Plc 1288011000001108 Fluoxetine 60mg capsules 30 capsule 9530711000001103 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001103 Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd 29922711000001107 Fluoxetine 60mg capsules 30 capsule - Advanz Pharma 4572611000001106 Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd 23587711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23980111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001107 Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 3293831100001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 15088111000001101 | Fluoxetine 60mg capsules - Sigma Pharmaceuticals Plc |
| Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001103 Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd 17219911000001107 Fluoxetine 60mg capsules 30 capsule - Advanz Pharma 4572611000001106 Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd 23587711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23980111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001107 Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 14956411000001101 | Fluoxetine 60mg capsules - Teva UK Ltd |
| Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - A Ctavis UK Ltd Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd Fluoxetine 60mg capsules 30 capsule - Advanz Pharma Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - DF Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 22014511000001102 | Fluoxetine 60mg capsules - Waymade Healthcare Plc |
| Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd 29922711000001107 Fluoxetine 60mg capsules 30 capsule - Advanz Pharma 4572611000001106 Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd 23587711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23980111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001107 Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 1288011000001108 | Fluoxetine 60mg capsules 30 capsule |
| Fluoxetine 60mg capsules 30 capsule - Advanz Pharma Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 9530711000001103 | Fluoxetine 60mg capsules 30 capsule - A A H Pharmaceuticals Ltd |
| Fluoxetine 60mg capsules 30 capsule - Alliance Healthcare (Distribution) Ltd Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - DF Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - DF Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 17219911000001103 | Fluoxetine 60mg capsules 30 capsule - Actavis UK Ltd |
| 19818511000001101 Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd 23587711000001109 Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd 23980111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001107 Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 29922711000001107 | Fluoxetine 60mg capsules 30 capsule - Advanz Pharma |
| Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 4572611000001106 | |
| 23980111000001101 Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals 18475811000001107 Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 19818511000001101 | Fluoxetine 60mg capsules 30 capsule - Almus Pharmaceuticals Ltd |
| Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd Fluoxetine 60mg capsules 30 capsule - Medreich Plc Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd Fluoxetine 60mg capsules 30 capsule - Mylan Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution | 23587711000001109 | Fluoxetine 60mg capsules 30 capsule - Bristol Laboratories Ltd |
| 7764711000001108 Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 23980111000001101 | Fluoxetine 60mg capsules 30 capsule - DE Pharmaceuticals |
| 30132111000001105 Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 18475811000001107 | Fluoxetine 60mg capsules 30 capsule - Dr Reddys Laboratories (UK) Ltd |
| 38918111000001100 Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 7764711000001108 | Fluoxetine 60mg capsules 30 capsule - Kent Pharmaceuticals Ltd |
| 32938311000001100 Fluoxetine 60mg capsules 30 capsule - Medreich Plc 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 30132111000001105 | Fluoxetine 60mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| 35162111000001108 Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 38918111000001100 | Fluoxetine 60mg capsules 30 capsule - Medihealth (Northern) Ltd |
| 3962411000001106 Fluoxetine 60mg capsules 30 capsule - Mylan 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 32938311000001100 | Fluoxetine 60mg capsules 30 capsule - Medreich Plc |
| 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 35162111000001108 | Fluoxetine 60mg capsules 30 capsule - Milpharm Ltd |
| 17909811000001106 Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution Ltd | 3962411000001106 | Fluoxetine 60mg capsules 30 capsule - Mylan |
| | 17909811000001106 | Fluoxetine 60mg capsules 30 capsule - Phoenix Healthcare Distribution |
| 15088211000001107 Huoxetine 60mg capsules 30 capsule - Sigma Pharmaceuticals Plc | 15088211000001107 | Fluoxetine 60mg capsules 30 capsule - Sigma Pharmaceuticals Plc |

| 14956511000001102 | Fluoxetine 60mg capsules 30 capsule - Teva UK Ltd |
|---|---|
| 22014611000001103 | Fluoxetine 60mg capsules 30 capsule - Waymade Healthcare Plc |
| 36613911000001100 | Fluoxetine 60mg capsules 60 capsule |
| 36614011000001102 | Fluoxetine 60mg capsules 60 capsule - Bristol Laboratories Ltd |
| 321947008 | Fluvoxamine 100mg tablets |
| 544211000001105 | Fluvoxamine 100mg tablets - A A H Pharmaceuticals Ltd |
| 767511000001108 | Fluvoxamine 100mg tablets - Actavis UK Ltd |
| 658411000001109 | Fluvoxamine 100mg tablets - Alliance Healthcare (Distribution) Ltd |
| 10408911000001101 | Fluvoxamine 100mg tablets - Arrow Generics Ltd |
| 23981011000001106 | Fluvoxamine 100mg tablets - DE Pharmaceuticals |
| 630711000001101 | Fluvoxamine 100mg tablets - IVAX Pharmaceuticals UK Ltd |
| 813511000001102 | Fluvoxamine 100mg tablets - Kent Pharmaceuticals Ltd |
| 30133311000001102 | Fluvoxamine 100mg tablets - Mawdsley-Brooks & Company Ltd |
| 38923611000001109 | Fluvoxamine 100mg tablets - Medihealth (Northern) Ltd |
| 15054811000001109 | Fluvoxamine 100mg tablets - Sigma Pharmaceuticals Plc |
| 387511000001107 | Fluvoxamine 100mg tablets - Teva UK Ltd |
| 26778111000001105 | Fluvoxamine 100mg tablets - Tillomed Laboratories Ltd |
| 22015911000001108 | Fluvoxamine 100mg tablets - Waymade Healthcare Plc |
| 529111000001101 | Fluvoxamine 100mg tablets - Wockhardt UK Ltd |
| 1297111000001109 | Fluvoxamine 100mg tablets 30 tablet |
| 2613111000001100 | Fluvoxamine 100mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 2613311000001103 | Fluvoxamine 100mg tablets 30 tablet - Actavis UK Ltd |
| 2614911000001100 | Fluvoxamine 100mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 10409111000001106 | Fluvoxamine 100mg tablets 30 tablet - Arrow Generics Ltd |
| 23981111000001107 | Fluvoxamine 100mg tablets 30 tablet - DE Pharmaceuticals |
| 2613611000001108 | Fluvoxamine 100mg tablets 30 tablet - IVAX Pharmaceuticals UK Ltd |
| 2613911000001102 | Fluvoxamine 100mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 30133411000001109 | Fluvoxamine 100mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 38923711000001100 | Fluvoxamine 100mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 15054911000001104 | Fluvoxamine 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 2613411000001105 | Fluvoxamine 100mg tablets 30 tablet - Teva UK Ltd |
| 26778311000001107 | Fluvoxamine 100mg tablets 30 tablet - Tillomed Laboratories Ltd |
| 22016011000001100 | Fluvoxamine 100mg tablets 30 tablet - Waymade Healthcare Plc |
| 2613511000001109 | Fluvoxamine 100mg tablets 30 tablet - Wockhardt UK Ltd |
| 321945000 | Fluvoxamine 50mg tablets |
| 895911000001106 | Fluvoxamine 50mg tablets - A A H Pharmaceuticals Ltd |
| 530911000001107 | Fluvoxamine 50mg tablets - Actavis UK Ltd |
| 634411000001101 | Fluvoxamine 50mg tablets - Alliance Healthcare (Distribution) Ltd |
| 10408611000001107 | Fluvoxamine 50mg tablets - Arrow Generics Ltd |
| 23981211000001101 | Fluvoxamine 50mg tablets - DE Pharmaceuticals |
| 156311000001102 | Fluvoxamine 50mg tablets - IVAX Pharmaceuticals UK Ltd |
| 410311000001105 | Fluvoxamine 50mg tablets - Kent Pharmaceuticals Ltd |
| 30133111000001104 | Fluvoxamine 50mg tablets - Mawdsley-Brooks & Company Ltd |
| 38923811000001108 | Fluvoxamine 50mg tablets - Medihealth (Northern) Ltd |
| 15055011000001104 | Fluvoxamine 50mg tablets - Sigma Pharmaceuticals Plc |
| 242611000001105 | Fluvoxamine 50mg tablets - Teva UK Ltd |
| 13751611000001102 | Fluvoxamine 50mg tablets - Tillomed Laboratories Ltd |
| 22015711000001106 | Fluvoxamine 50mg tablets - Waymade Healthcare Plc |
| 154211000001100 | Fluvoxamine 50mg tablets - Wockhardt UK Ltd |
| | <u> </u> |

| 1004811000001103 | Fluvoxamine 50mg tablets 60 tablet |
|---|---|
| | Fluvoxamine 50mg tablets 60 tablet - A A H Pharmaceuticals Ltd |
| 2610211000001101<br>2610311000001109 | Fluvoxamine 50mg tablets 60 tablet - A A II Fliatiliaceuticals Etu |
| 2010311000001109 | Fluvoxamine 50mg tablets 60 tablet - Actavis OK Etu Fluvoxamine 50mg tablets 60 tablet - Alliance Healthcare (Distribution) |
| 2611911000001103 | Ltd |
| 10408711000001103 | Fluvoxamine 50mg tablets 60 tablet - Arrow Generics Ltd |
| 23981311000001109 | Fluvoxamine 50mg tablets 60 tablet - DE Pharmaceuticals |
| 2611111000001101 | Fluvoxamine 50mg tablets 60 tablet - IVAX Pharmaceuticals UK Ltd |
| 2611311000001104 | Fluvoxamine 50mg tablets 60 tablet - Kent Pharmaceuticals Ltd |
| 30133211000001105 | Fluvoxamine 50mg tablets 60 tablet - Mawdsley-Brooks & Company Ltd |
| 38923911000001103 | Fluvoxamine 50mg tablets 60 tablet - Medihealth (Northern) Ltd |
| 15055211000001109 | Fluvoxamine 50mg tablets 60 tablet - Sigma Pharmaceuticals Plc |
| 2610411000001102 | Fluvoxamine 50mg tablets 60 tablet - Teva UK Ltd |
| 13751711000001106 | Fluvoxamine 50mg tablets 60 tablet - Tillomed Laboratories Ltd |
| 22015811000001103 | Fluvoxamine 50mg tablets 60 tablet - Waymade Healthcare Plc |
| 2610811000001100 | Fluvoxamine 50mg tablets 60 tablet - Wockhardt UK Ltd |
| 8517111000001106 | Fluvoxamine 50mg/5ml oral suspension |
| 8483011000001105 | Fluvoxamine 50mg/5ml oral suspension - Special Order |
| 8482911000001102 | Fluvoxamine 50mg/5ml oral suspension 1 ml |
| 8483211000001100 | Fluvoxamine 50mg/5ml oral suspension 1 ml - Special Order |
| 13927411000001102 | Lustral 100mg tablets - DE Pharmaceuticals |
| 5523011000001104 | Lustral 100mg tablets - Dowelhurst Ltd |
| 19968211000001105 | Lustral 100mg tablets - Lexon (UK) Ltd |
| 16514711000001106 | Lustral 100mg tablets - Mawdsley-Brooks & Company Ltd |
| 14375011000001106 | Lustral 100mg tablets - Sigma Pharmaceuticals Plc |
| 16582411000001109 | Lustral 100mg tablets - Stephar (U.K.) Ltd |
| 687611000001102 | Lustral 100mg tablets - Upjohn UK Ltd |
| 10920611000001104 | Lustral 100mg tablets - Waymade Healthcare Plc |
| 16582611000001107 | Lustral 100mg tablets 14 tablet - Stephar (U.K.) Ltd |
| 13927511000001103 | Lustral 100mg tablets 28 tablet - DE Pharmaceuticals |
| 16514911000001108 | Lustral 100mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 14375211000001101 | Lustral 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1422311000001101 | Lustral 100mg tablets 28 tablet - Upjohn UK Ltd |
| 10920711000001101 | Lustral 100mg tablets 28 tablet - Waymade Healthcare Plc |
| 13927711000001108 | Lustral 100mg tablets 30 tablet - DE Pharmaceuticals |
| 5523111000001103 | Lustral 100mg tablets 30 tablet - Dc Frialmaceuticals Lustral 100mg tablets 30 tablet - Dowelhurst Ltd |
| | Lustral 100mg tablets 30 tablet - Dowelliust Ltd Lustral 100mg tablets 30 tablet - Lexon (UK) Ltd |
| 19968311000001102<br>18666711000001103 | Lustral 100mg tablets 30 tablet - Lexon (OK) Ltd Lustral 100mg tablets 30 tablet - Waymade Healthcare Plc |
| 13927211000001101 | Lustral 50mg tablets - DE Pharmaceuticals |
| 5523311000001101 | Lustral 50mg tablets - Dowelhurst Ltd |
| 16203811000001107 | Lustral 50mg tablets - Lexon (UK) Ltd |
| 37540711000001109 | Lustral 50mg tablets - Mawdsley-Brooks & Company Ltd |
| 936411000001108 | Lustral 50mg tablets - Upjohn UK Ltd |
| 10767811000001100 | Lustral 50mg tablets - Waymade Healthcare Plc |
| 13927311000001109 | Lustral 50mg tablets 28 tablet - DE Pharmaceuticals |
| 5616411000001103 | Lustral 50mg tablets 28 tablet - Dowelhurst Ltd |
| 16203911000001102 | Lustral 50mg tablets 28 tablet - Lexon (UK) Ltd |
| 37540811000001101 | Lustral 50mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 1422211000001109 | Lustral 50mg tablets 28 tablet - Upjohn UK Ltd |
| 25400511000001103 | Lustral 50mg tablets 28 tablet - Waymade Healthcare Plc |

| 5523511000001107 | Lustral 50mg tablets 30 tablet - Dowelhurst Ltd |
|---|---|
| 10767911000001105 | Lustral 50mg tablets 30 tablet - Waymade Healthcare Plc |
| 24397511000001101 | Olena 20mg dispersible tablets - Advanz Pharma |
| 24397611000001102 | Olena 20mg dispersible tablets 28 tablet - Advanz Pharma |
| 689411000001109 | Oxactin 20mg capsules - Discovery Pharmaceuticals |
| 1616411000001104 | Oxactin 20mg capsules 30 capsule - Discovery Pharmaceuticals |
| 39701911000001102 | Paroxetine 10mg tablets |
| 421041006 | Paroxetine 10mg tablets |
| 21548411000001103 | Paroxetine 10mg tablets - A A H Pharmaceuticals Ltd |
| 21541611000001108 | Paroxetine 10mg tablets - Accord Healthcare Ltd |
| 22247311000001102 | Paroxetine 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 35429511000001104 | Paroxetine 10mg tablets - Crescent Pharma Ltd |
| 30074111000001108 | Paroxetine 10mg tablets - DE Pharmaceuticals |
| 30855811000001101 | Paroxetine 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 39176211000001102 | Paroxetine 10mg tablets - Medihealth (Northern) Ltd |
| 35851411000001109 | Paroxetine 10mg tablets - Medreich Plc |
| 33471411000001106 | Paroxetine 10mg tablets - Morningside Healthcare Ltd |
| 29982911000001101 | Paroxetine 10mg tablets - Sigma Pharmaceuticals Plc |
| 33387311000001107 | Paroxetine 10mg tablets - Teva UK Ltd |
| 34581311000001101 | Paroxetine 10mg tablets - Zentiva Pharma UK Ltd |
| 11270511000001105 | Paroxetine 10mg tablets 28 tablet |
| 21548511000001104 | Paroxetine 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 21541711000001104 | Paroxetine 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 22247411000001109 | Paroxetine 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 35429611000001100 | Paroxetine 10mg tablets 28 tablet - Crescent Pharma Ltd |
| 30074211000001102 | Paroxetine 10mg tablets 28 tablet - DE Pharmaceuticals |
| 30855911000001106 | Paroxetine 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 39176311000001105 | Paroxetine 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 35851511000001108 | Paroxetine 10mg tablets 28 tablet - Medreich Plc |
| 33471511000001105 | Paroxetine 10mg tablets 28 tablet - Morningside Healthcare Ltd |
| 29983011000001109 | Paroxetine 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 33387411000001100 | Paroxetine 10mg tablets 28 tablet - Teva UK Ltd |
| 34581411000001108 | Paroxetine 10mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 13004411000001105 | Paroxetine 10mg/5ml oral solution |
| 12983011000001102 | Paroxetine 10mg/5ml oral solution - Special Order |
| 12982611000001104 | Paroxetine 10mg/5ml oral solution 1 ml |
| 12983111000001101 | Paroxetine 10mg/5ml oral solution 1 ml - Special Order |
| 13004511000001109 | Paroxetine 10mg/5ml oral suspension |
| 12982111000001107 | Paroxetine 10mg/5ml oral suspension - Special Order |
| 12981811000001109 | Paroxetine 10mg/5ml oral suspension 1 ml |
| 12982411000001102 | Paroxetine 10mg/5ml oral suspension 1 ml - Special Order |
| 36565911000001109 | Paroxetine 10mg/5ml oral suspension sugar free |
| 321968009 | Paroxetine 10mg/5ml oral suspension sugar free |
| 5307311000001101 | Paroxetine 10mg/5ml oral suspension sugar free - Dowelhurst Ltd |
| | Paroxetine 10mg/5ml oral suspension sugar free - Sigma |
| 14708411000001101 | Pharmaceuticals Plc |
| 1240411000001106 | Paroxetine 10mg/5ml oral suspension sugar free 150 ml |
| 5307511000001107 | Paroxetine 10mg/5ml oral suspension sugar free 150 ml - Dowelhurst Ltd |
| 14708511000001102 | Paroxetine 10mg/5ml oral suspension sugar free 150 ml - Sigma<br>Pharmaceuticals Plc |

| 321964006 | Paroxetine 20mg tablets |
|---|---|
| 570611000001104 | Paroxetine 20mg tablets - A A H Pharmaceuticals Ltd |
| 4116911000001101 | Paroxetine 20mg tablets - Accord Healthcare Ltd |
| 115611000001107 | Paroxetine 20mg tablets - Alliance Healthcare (Distribution) Ltd |
| 11427211000001106 | Paroxetine 20mg tablets - Almus Pharmaceuticals Ltd |
| 13767011000001105 | Paroxetine 20mg tablets - Apotex UK Ltd |
| 34346311000001101 | Paroxetine 20mg tablets - Crescent Pharma Ltd |
| 30074311000001105 | Paroxetine 20mg tablets - DE Pharmaceuticals |
| 13234911000001103 | Paroxetine 20mg tablets - Dowelhurst Ltd |
| 9034711000001106 | Paroxetine 20mg tablets - Genus Pharmaceuticals Ltd |
| 31211000001109 | Paroxetine 20mg tablets - IVAX Pharmaceuticals UK Ltd |
| 485211000001109 | Paroxetine 20mg tablets - Kent Pharmaceuticals Ltd |
| 39176411000001103 | Paroxetine 20mg tablets - Medihealth (Northern) Ltd |
| 21410111000001106 | Paroxetine 20mg tablets - Medreich Plc |
| 19195811000001102 | Paroxetine 20mg tablets - Milpharm Ltd |
| 21811000001107 | Paroxetine 20mg tablets - Mylan |
| 16696911000001107 | Paroxetine 20mg tablets - Pfizer Ltd |
| 17953511000001100 | Paroxetine 20mg tablets - Phoenix Healthcare Distribution Ltd |
| 9729511000001102 | Paroxetine 20mg tablets - PLIVA Pharma Ltd |
| 13722411000001109 | Paroxetine 20mg tablets - Ranbaxy (UK) Ltd |
| 7489711000001103 | Paroxetine 20mg tablets - Sandoz Ltd |
| 15154911000001107 | Paroxetine 20mg tablets - Sigma Pharmaceuticals Plc |
| 7836711000001105 | Paroxetine 20mg tablets - Sterwin Medicines |
| 7941011000001105 | Paroxetine 20mg tablets - Teva UK Ltd |
| 35861411000001100 | Paroxetine 20mg tablets - Tillomed Laboratories Ltd |
| 21841411000001109 | Paroxetine 20mg tablets - Waymade Healthcare Plc |
| 5533611000001109 | Paroxetine 20mg tablets 14 tablet |
| 5408911000001109 | Paroxetine 20mg tablets 28 tablet |
| 1083911000001105 | Paroxetine 20mg tablets 30 tablet |
| 1930611000001109 | Paroxetine 20mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 4117011000001102 | Paroxetine 20mg tablets 30 tablet - Accord Healthcare Ltd |
| 1931011000001106 | Paroxetine 20mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 11427311000001103 | Paroxetine 20mg tablets 30 tablet - Almus Pharmaceuticals Ltd |
| 13767111000001106 | Paroxetine 20mg tablets 30 tablet - Apotex UK Ltd |
| 34346411000001108 | Paroxetine 20mg tablets 30 tablet - Crescent Pharma Ltd |
| 30074411000001103 | Paroxetine 20mg tablets 30 tablet - DE Pharmaceuticals |
| 13235011000001103 | Paroxetine 20mg tablets 30 tablet - Dowelhurst Ltd |
| 9034811000001103 | Paroxetine 20mg tablets 30 tablet - Genus Pharmaceuticals Ltd |
| 1930811000001108 | Paroxetine 20mg tablets 30 tablet - IVAX Pharmaceuticals UK Ltd |
| 1930911000001103 | Paroxetine 20mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 39176511000001104 | Paroxetine 20mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 21410211000001100 | Paroxetine 20mg tablets 30 tablet - Medreich Plc |
| 19195911000001107 | Paroxetine 20mg tablets 30 tablet - Milpharm Ltd |
| 1930711000001100 | Paroxetine 20mg tablets 30 tablet - Mylan |
| 16697011000001106 | Paroxetine 20mg tablets 30 tablet - Pfizer Ltd |
| 17953611000001101 | Paroxetine 20mg tablets 30 tablet - Phoenix Healthcare Distribution Ltd |
| 9729611000001103 | Paroxetine 20mg tablets 30 tablet - PLIVA Pharma Ltd |
| 13722611000001107 | Paroxetine 20mg tablets 30 tablet - Ranbaxy (UK) Ltd |
| 7489911000001101 | Paroxetine 20mg tablets 30 tablet - Sandoz Ltd |

| 15155011000001107 | Paroxetine 20mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
|---|---|
| 7836811000001102 | Paroxetine 20mg tablets 30 tablet - Sterwin Medicines |
| 7941211000001100 | Paroxetine 20mg tablets 30 tablet - Teva UK Ltd |
| 35861511000001101 | Paroxetine 20mg tablets 30 tablet - Tillomed Laboratories Ltd |
| 21841511000001108 | Paroxetine 20mg tablets 30 tablet - Waymade Healthcare Plc |
| 13004611000001108 | Paroxetine 20mg/5ml oral solution |
| 12983911000001103 | Paroxetine 20mg/5ml oral solution - Special Order |
| 12983811000001108 | Paroxetine 20mg/5ml oral solution 1 ml |
| 12984011000001100 | Paroxetine 20mg/5ml oral solution 1 ml - Special Order |
| 13004711000001104 | Paroxetine 20mg/5ml oral suspension |
| 12983611000001109 | |
| | Paroxetine 20mg/5ml oral suspension - Special Order |
| 12983411000001106<br>12983711000001100 | Paroxetine 20mg/5ml oral suspension 1 ml |
| | Paroxetine 20mg/5ml oral suspension 1 ml - Special Order |
| 321966008 | Paroxetine 30mg tablets |
| 7384811000001104 | Paroxetine 30mg tablets - A A H Pharmaceuticals Ltd |
| 6330111000001108 | Paroxetine 30mg tablets - Accord Healthcare Ltd |
| 7332211000001102 | Paroxetine 30mg tablets - Alliance Healthcare (Distribution) Ltd |
| 11427011000001101 | Paroxetine 30mg tablets - Almus Pharmaceuticals Ltd |
| 13767211000001100 | Paroxetine 30mg tablets - Apotex UK Ltd |
| 36005511000001104 | Paroxetine 30mg tablets - Crescent Pharma Ltd |
| 30074511000001104 | Paroxetine 30mg tablets - DE Pharmaceuticals |
| 13235111000001102 | Paroxetine 30mg tablets - Dowelhurst Ltd |
| 7476911000001103 | Paroxetine 30mg tablets - Kent Pharmaceuticals Ltd |
| 39176611000001100 | Paroxetine 30mg tablets - Medihealth (Northern) Ltd |
| 21410311000001108 | Paroxetine 30mg tablets - Medreich Plc |
| 19196111000001103 | Paroxetine 30mg tablets - Milpharm Ltd |
| 8112711000001103 | Paroxetine 30mg tablets - Mylan |
| 16696711000001105 | Paroxetine 30mg tablets - Pfizer Ltd |
| 17953711000001105 | Paroxetine 30mg tablets - Phoenix Healthcare Distribution Ltd |
| 9729711000001107 | Paroxetine 30mg tablets - PLIVA Pharma Ltd |
| 11533011000001102 | Paroxetine 30mg tablets - Sandoz Ltd |
| 15154711000001105 | Paroxetine 30mg tablets - Sigma Pharmaceuticals Plc |
| 9526211000001105 | Paroxetine 30mg tablets - Teva UK Ltd |
| 21842211000001103 | Paroxetine 30mg tablets - Waymade Healthcare Plc |
| 7837611000001104 | Paroxetine 30mg tablets - Zentiva Pharma UK Ltd |
| 1249611000001103 | Paroxetine 30mg tablets 30 tablet |
| 7384911000001109 | Paroxetine 30mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 6331011000001103 | Paroxetine 30mg tablets 30 tablet - Accord Healthcare Ltd |
| 7332311000001105 | Paroxetine 30mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 11427111000001100 | Paroxetine 30mg tablets 30 tablet - Almus Pharmaceuticals Ltd |
| 13767311000001108 | Paroxetine 30mg tablets 30 tablet - Apotex UK Ltd |
| 36005611000001100 | Paroxetine 30mg tablets 30 tablet - Crescent Pharma Ltd |
| 30074611000001100 | Paroxetine 30mg tablets 30 tablet - DE Pharmaceuticals |
| 13235311000001100 | Paroxetine 30mg tablets 30 tablet - Dowelhurst Ltd |
| 7477311000001101 | Paroxetine 30mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 39176711000001109 | Paroxetine 30mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 21410511000001102 | Taroxetine soring tablets so tablet. Weatheatti (Northern) Eta |
| 21-1100111000001102 | Paroxetine 30mg tablets 30 tablet - Medreich Plc |
| 19196211000001109 | |

| 16606811000001103 | Developed 20mg tablets 20 tablet Distant Ltd |
|---|---|
| 16696811000001102<br>17953811000001102 | Paroxetine 30mg tablets 30 tablet - Pfizer Ltd |
| | Paroxetine 30mg tablets 30 tablet - Phoenix Healthcare Distribution Ltd |
| 9729811000001104<br>11533111000001101 | Paroxetine 30mg tablets 30 tablet - PLIVA Pharma Ltd Paroxetine 30mg tablets 30 tablet - Sandoz Ltd |
| | - |
| 15154811000001102 | Paroxetine 30mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 9526311000001102 | Paroxetine 30mg tablets 30 tablet - Teva UK Ltd |
| 21842311000001106 | Paroxetine 30mg tablets 30 tablet - Waymade Healthcare Plc |
| 7837711000001108 | Paroxetine 30mg tablets 30 tablet - Zentiva Pharma UK Ltd |
| 13004811000001107 | Paroxetine 30mg/5ml oral solution |
| 12985011000001101 | Paroxetine 30mg/5ml oral solution - Special Order |
| 12984811000001106 | Paroxetine 30mg/5ml oral solution 1 ml |
| 12985211000001106 | Paroxetine 30mg/5ml oral solution 1 ml - Special Order |
| 13004911000001102 | Paroxetine 30mg/5ml oral suspension |
| 12984411000001109 | Paroxetine 30mg/5ml oral suspension - Special Order |
| 12984211000001105 | Paroxetine 30mg/5ml oral suspension 1 ml |
| 12984611000001107 | Paroxetine 30mg/5ml oral suspension 1 ml - Special Order |
| 422084009 | Paroxetine 40mg tablets |
| 35031511000001106 | Paroxetine 40mg tablets - A A H Pharmaceuticals Ltd |
| 34575911000001105 | Paroxetine 40mg tablets - Alliance Healthcare (Distribution) Ltd |
| 33181811000001102 | Paroxetine 40mg tablets - Crescent Pharma Ltd |
| 37772211000001101 | Paroxetine 40mg tablets - DE Pharmaceuticals |
| 37125911000001107 | Paroxetine 40mg tablets - Mawdsley-Brooks & Company Ltd |
| 39325411000001100 | Paroxetine 40mg tablets - Medihealth (Northern) Ltd |
| 33470811000001100 | Paroxetine 40mg tablets - Morningside Healthcare Ltd |
| 33563711000001101 | Paroxetine 40mg tablets - Teva UK Ltd |
| 33470711000001108 | Paroxetine 40mg tablets 28 tablet |
| 35031611000001105 | Paroxetine 40mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 37772311000001109 | Paroxetine 40mg tablets 28 tablet - DE Pharmaceuticals |
| 37126011000001104 | Paroxetine 40mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 39325511000001101 | Paroxetine 40mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 33471211000001107 | Paroxetine 40mg tablets 28 tablet - Morningside Healthcare Ltd |
| 33563811000001109 | Paroxetine 40mg tablets 28 tablet - Teva UK Ltd |
| 33181711000001105 | Paroxetine 40mg tablets 30 tablet |
| 37191811000001107 | Paroxetine 40mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 34576011000001102 | Paroxetine 40mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 33181911000001107 | Paroxetine 40mg tablets 30 tablet - Crescent Pharma Ltd |
| 23362111000001107 | Priligy 30mg tablets - A. Menarini Farmaceutica Internazionale SRL |
| 16989411000001109 | Priligy 30mg tablets - Imported (Germany) |
| 23362211000001101 | Priligy 30mg tablets 3 tablet - A. Menarini Farmaceutica Internazionale SRL |
| 16989511000001108 | Priligy 30mg tablets 3 tablet - Imported (Germany) |
| 23362311000001109 | Priligy 30mg tablets 6 tablet - A. Menarini Farmaceutica Internazionale SRL |
| 16989611000001107 | Priligy 30mg tablets 6 tablet - Imported (Germany) |
| 23361611000001105 | Priligy 60mg tablets - A. Menarini Farmaceutica Internazionale SRL |
| 16989911000001101 | Priligy 60mg tablets - Imported (Germany) |
| | Priligy 60mg tablets 3 tablet - A. Menarini Farmaceutica Internazionale |
| 23361711000001101 | SRL |
| 16990011000001109 | Priligy 60mg tablets 3 tablet - Imported (Germany) |
| 23361811000001109 | Priligy 60mg tablets 6 tablet - A. Menarini Farmaceutica Internazionale SRL |

| 16000111000001105 | Drillian COma tableta C tablet Imported (Cormonn) |
|---|---|
| 16990111000001105 | Priligy 60mg tablets 6 tablet - Imported (Germany) |
| 13949811000001105 | Prozac 20mg capsules - DE Pharmaceuticals |
| 5577211000001101 | Prozac 20mg capsules - Dowelhurst Ltd |
| 573011000001101 | Prozac 20mg capsules - Eli Lilly and Company Ltd |
| 16229811000001102 | Prozac 20mg capsules - Lexon (UK) Ltd |
| 17424311000001105 | Prozac 20mg capsules - Mawdsley-Brooks & Company Ltd |
| 18174111000001100 | Prozac 20mg capsules - Necessity Supplies Ltd |
| 5405011000001102 | Prozac 20mg capsules - Waymade Healthcare Plc |
| 13949911000001100 | Prozac 20mg capsules 28 capsule - DE Pharmaceuticals |
| 5577411000001102 | Prozac 20mg capsules 28 capsule - Dowelhurst Ltd |
| 5577311000001109 | Prozac 20mg capsules 28 capsule - Dowelhurst Ltd |
| 16229911000001107 | Prozac 20mg capsules 28 capsule - Lexon (UK) Ltd |
| 17424511000001104 | Prozac 20mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 18174211000001106 | Prozac 20mg capsules 28 capsule - Necessity Supplies Ltd |
| 5405111000001101 | Prozac 20mg capsules 28 capsule - Waymade Healthcare Plc |
| 1616811000001102 | Prozac 20mg capsules 30 capsule - Eli Lilly and Company Ltd |
| 17424611000001100 | Prozac 20mg capsules 30 capsule - Mawdsley-Brooks & Company Ltd |
| 13952011000001108 | Prozac 20mg/5ml liquid - DE Pharmaceuticals |
| 5309711000001105 | Prozac 20mg/5ml liquid - Dowelhurst Ltd |
| 695811000001109 | Prozac 20mg/5ml liquid - Eli Lilly and Company Ltd |
| 16229611000001101 | Prozac 20mg/5ml liquid - Lexon (UK) Ltd |
| 17424711000001109 | Prozac 20mg/5ml liquid - Mawdsley-Brooks & Company Ltd |
| 18174311000001103 | Prozac 20mg/5ml liquid - Necessity Supplies Ltd |
| 14380011000001108 | Prozac 20mg/5ml liquid - Sigma Pharmaceuticals Plc |
| 5405411000001106 | Prozac 20mg/5ml liquid - Waymade Healthcare Plc |
| 13952111000001109 | Prozac 20mg/5ml liquid 70 ml - DE Pharmaceuticals |
| 5309811000001102 | Prozac 20mg/5ml liquid 70 ml - Dowelhurst Ltd |
| 2182211000001104 | Prozac 20mg/5ml liquid 70 ml - Eli Lilly and Company Ltd |
| 16229711000001105 | Prozac 20mg/5ml liquid 70 ml - Lexon (UK) Ltd |
| 17424811000001101 | Prozac 20mg/5ml liquid 70 ml - Mawdsley-Brooks & Company Ltd |
| 18174411000001105 | Prozac 20mg/5ml liquid 70 ml - Necessity Supplies Ltd |
| 14380411000001104 | Prozac 20mg/5ml liquid 70 ml - Sigma Pharmaceuticals Plc |
| 5405511000001105 | Prozac 20mg/5ml liquid 70 ml - Waymade Healthcare Plc |
| 142311000001103 | Prozac 60mg capsules - Eli Lilly and Company Ltd |
| 2180911000001109 | Prozac 60mg capsules 30 capsule - Eli Lilly and Company Ltd |
| 11581211000001101 | Prozep 20mg/5ml oral solution - Chemidex Pharma Ltd |
| 11581311000001109 | Prozep 20mg/5ml oral solution 70 ml - Chemidex Pharma Ltd |
| 10065611000001109 | Prozit 20mg/5ml oral solution - Pinewood Healthcare |
| 10065711000001100 | Prozit 20mg/5ml oral solution 70 ml - Pinewood Healthcare |
| 683911000001104 | Ranflutin 20mg capsules - Ranbaxy (UK) Ltd |
| 1402211000001103 | Ranflutin 20mg capsules 30 capsule - Ranbaxy (UK) Ltd |
| 11270611000001109 | Seroxat 10mg tablets - GlaxoSmithKline UK Ltd |
| 27991411000001109 | Seroxat 10mg tablets - Waymade Healthcare Plc |
| 11270711000001100 | Seroxat 10mg tablets 28 tablet - GlaxoSmithKline UK Ltd |
| 27991511000001108 | Seroxat 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 18612611000001107 | Seroxat 20mg tablets - DE Pharmaceuticals |
| 5533411000001106 | Seroxat 20mg tablets - Dowelhurst Ltd |
| 477511000001109 | Seroxat 20mg tablets - Boweringst Etd Seroxat 20mg tablets - GlaxoSmithKline UK Ltd |
| 16243511000001100 | Seroxat 20mg tablets - Glaxosmithtime on Eta |
| 10273311000001100 | Scronat Zoriig tableto Lenori (Ori) Lta |

| 17449311000001109 | Carayat 20mg tablets Maudelay Procks & Company Ltd |
|---|---|
| 5408211000001109 | Seroxat 20mg tablets - Mawdsley-Brooks & Company Ltd |
| | Seroxat 20mg tablets - Waymade Healthcare Plc |
| 5533811000001108 | Seroxat 20mg tablets 14 tablet - Dowelhurst Ltd |
| 5534011000001100 | Seroxat 20mg tablets 28 tablet - Dowelhurst Ltd |
| 5409411000001109 | Seroxat 20mg tablets 28 tablet - Waymade Healthcare Plc |
| 18612711000001103 | Seroxat 20mg tablets 30 tablet - DE Pharmaceuticals |
| 13204011000001107 | Seroxat 20mg tablets 30 tablet - Dowelhurst Ltd |
| 1931111000001107 | Seroxat 20mg tablets 30 tablet - GlaxoSmithKline UK Ltd |
| 16243611000001101 | Seroxat 20mg tablets 30 tablet - Lexon (UK) Ltd |
| 17449411000001102 | Seroxat 20mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 11056811000001103 | Seroxat 20mg tablets 30 tablet - Waymade Healthcare Plc |
| 37596511000001107 | Seroxat 20mg/10ml liquid - CST Pharma Ltd |
| 14001011000001102 | Seroxat 20mg/10ml liquid - DE Pharmaceuticals |
| 5319311000001108 | Seroxat 20mg/10ml liquid - Dowelhurst Ltd |
| 16811000001109 | Seroxat 20mg/10ml liquid - GlaxoSmithKline UK Ltd |
| 16243311000001106 | Seroxat 20mg/10ml liquid - Lexon (UK) Ltd |
| 18187711000001102 | Seroxat 20mg/10ml liquid - Necessity Supplies Ltd |
| 17595111000001106 | Seroxat 20mg/10ml liquid - Sigma Pharmaceuticals Plc |
| 5411611000001109 | Seroxat 20mg/10ml liquid - Waymade Healthcare Plc |
| 37596611000001106 | Seroxat 20mg/10ml liquid 150 ml - CST Pharma Ltd |
| 14001111000001101 | Seroxat 20mg/10ml liquid 150 ml - DE Pharmaceuticals |
| 5319411000001101 | Seroxat 20mg/10ml liquid 150 ml - Dowelhurst Ltd |
| 2157911000001104 | Seroxat 20mg/10ml liquid 150 ml - GlaxoSmithKline UK Ltd |
| 16243411000001104 | Seroxat 20mg/10ml liquid 150 ml - Lexon (UK) Ltd |
| 18188011000001103 | Seroxat 20mg/10ml liquid 150 ml - Necessity Supplies Ltd |
| 17595411000001101 | Seroxat 20mg/10ml liquid 150 ml - Sigma Pharmaceuticals Plc |
| 5411811000001108 | Seroxat 20mg/10ml liquid 150 ml - Waymade Healthcare Plc |
| 13204111000001108 | Seroxat 30mg tablets - Dowelhurst Ltd |
| 738111000001107 | Seroxat 30mg tablets - GlaxoSmithKline UK Ltd |
| 16243711000001105 | Seroxat 30mg tablets - Lexon (UK) Ltd |
| 17449511000001103 | Seroxat 30mg tablets - Mawdsley-Brooks & Company Ltd |
| 12561311000001107 | Seroxat 30mg tablets - Waymade Healthcare Plc |
| 13204211000001102 | Seroxat 30mg tablets 30 tablet - Dowelhurst Ltd |
| 1931211000001101 | Seroxat 30mg tablets 30 tablet - GlaxoSmithKline UK Ltd |
| 16243811000001102 | Seroxat 30mg tablets 30 tablet - Lexon (UK) Ltd |
| 17449611000001104 | Seroxat 30mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 12561411000001100 | Seroxat 30mg tablets 30 tablet - Waymade Healthcare Plc |
| 39704011000001103 | Sertraline 100mg tablets |
| 321960002 | Sertraline 100mg tablets |
| 9751511000001104 | Sertraline 100mg tablets - A A H Pharmaceuticals Ltd |
| 20169911000001105 | Sertraline 100mg tablets - Accord Healthcare Ltd |
| 9745111000001107 | Sertraline 100mg tablets - Actors UK Ltd |
| 9840311000001107 | Sertraline 100mg tablets - Actavis OK Ltu Sertraline 100mg tablets - Alliance Healthcare (Distribution) Ltd |
| 11409011000001100 | Sertraline 100mg tablets - Almarce Heattricare (Distribution) Ltd Sertraline 100mg tablets - Almus Pharmaceuticals Ltd |
| 13770311000001100 | Sertraline 100mg tablets - Apotex UK Ltd |
| 10438111000001109 | Sertraline 100mg tablets - Arrow Generics Ltd |
| 16066511000001109 | Sertraline 100mg tablets - Bristol Laboratories Ltd |
| 14130511000001101 | Sertraline 100mg tablets - Consilient Health Ltd |
| 28988311000001101 | Sertraline 100mg tablets - Crescent Pharma Ltd |

| 20006011000001107 | Cortrolino 100mg tablets DE Pharmacouticals |
|---|---|
| 30096011000001107 | Sertraline 100mg tablets - DE Pharmaceuticals |
| 5509011000001106 | Sertraline 100mg tablets - Dowelhurst Ltd |
| 11011511000001104 | Sertraline 100mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 10296111000001100 | Sertraline 100mg tablets - Focus Pharmaceuticals Ltd |
| 33654511000001107 | Sertraline 100mg tablets - Genesis Pharmaceuticals Ltd |
| 9841611000001104 | Sertraline 100mg tablets - IVAX Pharmaceuticals UK Ltd |
| 9764911000001101 | Sertraline 100mg tablets - Kent Pharmaceuticals Ltd |
| 27701711000001107 | Sertraline 100mg tablets - Lupin Healthcare (UK) Ltd |
| 37139711000001109 | Sertraline 100mg tablets - Mawdsley-Brooks & Company Ltd |
| 39242711000001109 | Sertraline 100mg tablets - Medihealth (Northern) Ltd |
| 19734911000001109 | Sertraline 100mg tablets - Medreich Plc |
| 19197211000001106 | Sertraline 100mg tablets - Milpharm Ltd |
| 9842911000001104 | Sertraline 100mg tablets - Mylan |
| 10442611000001102 | Sertraline 100mg tablets - Niche Generics Ltd |
| 39623411000001108 | Sertraline 100mg tablets - NorthStar Healthcare Unlimited Company |
| 36699811000001106 | Sertraline 100mg tablets - Noumed Life Sciences Ltd |
| 17928211000001105 | Sertraline 100mg tablets - Phoenix Healthcare Distribution Ltd |
| 9738611000001109 | Sertraline 100mg tablets - PLIVA Pharma Ltd |
| 10567411000001103 | Sertraline 100mg tablets - Ranbaxy (UK) Ltd |
| 10294911000001105 | Sertraline 100mg tablets - Relonchem Ltd |
| 36619111000001100 | Sertraline 100mg tablets - Ria Generics Ltd |
| 9775011000001107 | Sertraline 100mg tablets - Sandoz Ltd |
| 15211411000001106 | Sertraline 100mg tablets - Sigma Pharmaceuticals Plc |
| 9746211000001107 | Sertraline 100mg tablets - Teva UK Ltd |
| 13762711000001105 | Sertraline 100mg tablets - Tillomed Laboratories Ltd |
| 21896311000001103 | Sertraline 100mg tablets - Waymade Healthcare Plc |
| 5413411000001105 | Sertraline 100mg tablets - Waymade Healthcare Plc |
| 9781211000001105 | Sertraline 100mg tablets - Wockhardt UK Ltd |
| 9751911000001106 | Sertraline 100mg tablets - Zentiva Pharma UK Ltd |
| 16582511000001108 | Sertraline 100mg tablets 14 tablet |
| 1209011000001102 | Sertraline 100mg tablets 28 tablet |
| 9751611000001100 | Sertraline 100mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 20170011000001109 | Sertraline 100mg tablets 28 tablet - Accord Healthcare Ltd |
| 9745211000001101 | Sertraline 100mg tablets 28 tablet - Actavis UK Ltd |
| 9840511000001105 | Sertraline 100mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 11409211000001105 | Sertraline 100mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 13770411000001107 | Sertraline 100mg tablets 28 tablet - Apotex UK Ltd |
| 10438311000001106 | Sertraline 100mg tablets 28 tablet - Arrow Generics Ltd |
| 16382911000001103 | Sertraline 100mg tablets 28 tablet - Bristol Laboratories Ltd |
| 14130611000001102 | Sertraline 100mg tablets 28 tablet - Consilient Health Ltd |
| 28988411000001108 | Sertraline 100mg tablets 28 tablet - Crescent Pharma Ltd |
| 30096111000001108 | Sertraline 100mg tablets 28 tablet - DE Pharmaceuticals |
| 11011611000001100 | Sertraline 100mg tablets 28 tablet - Dr Reddys Laboratories (UK) Ltd |
| 10296211000001106 | Sertraline 100mg tablets 28 tablet - Focus Pharmaceuticals Ltd |
| 33654611000001106 | Sertraline 100mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 9841711000001108 | Sertraline 100mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 9765011000001101 | Sertraline 100mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 27702111000001101 | Sertraline 100mg tablets 28 tablet - Lupin Healthcare (UK) Ltd |
| 37140011000001100 | Sertraline 100mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 571.0011000001100 | 1 33. 3. |

| 19735111000001105 Sertraline 100mg tablets 28 tablet - Medreich Plc 19197311000001103 Sertraline 100mg tablets 28 tablet - Milpharm Ltd 1943111000001106 Sertraline 100mg tablets 28 tablet - Milpharm Ltd 39623511000001107 Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Unlimited Company Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Unlimited Company Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Unlimited Company Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Distribution Ltd 17928311000001100 Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd 1873711000001100 Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd 10295211000001100 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 10295211000001106 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 10295211000001106 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 10295211000001108 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 13762811000001105 Sertraline 100mg tablets 28 tablet - Signa Pharmaceuticals Plc 9746311000001104 Sertraline 100mg tablets 28 tablet - Teva UK Ltd 13762811000001104 Sertraline 100mg tablets 28 tablet - Teva UK Ltd 13762811000001102 Sertraline 100mg tablets 28 tablet - Teva UK Ltd 13762811000001102 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 97831311000001103 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 97831311000001103 Sertraline 100mg tablets 30 tablet Sertraline Ltd 1509611000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 1509611000001101 Sertraline 100mg tablets 500 tablet - A H Pharmaceuticals Plc 15413611000001102 Sertraline 100mg tablets 500 tablet - A H Pharmaceuticals Plc 15413611000001103 Sertraline 100mg/5ml oral suspension 1 ml - Drug T | 39242811000001101 | Sertraline 100mg tablets 28 tablet - Medihealth (Northern) Ltd |
|---|---|---|
| 19197311000001103 Sertraline 100mg tablets 28 tablet - Milpharm Ltd | | |
| 9843111000001108 Sertraline 100mg tablets 28 tablet - Mylan 10442711000001106 Sertraline 100mg tablets 28 tablet - Niche Generics Ltd 39623511000001107 Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Unlimited Company 36699911000001101 Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Distribution Ltd 9738711000001102 Sertraline 100mg tablets 28 tablet - PluVA Pharma Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - PluVA Pharma Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 36619211000001106 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 3677511000001108 Sertraline 100mg tablets 28 tablet - Sandoz Ltd 3775111000001108 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc 3746311000001104 Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd 21896511000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 3782811000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 378311000001100 Sertraline 100mg tablets 30 tablet 38131000001101 Sertraline 100mg tablets 30 tablet 38131000001103 Sertraline 100mg tablets 30 tablet 38131000001100 Sertraline | | - |
| 1044271100001106 | | |
| Sertraline 100mg tablets 28 tablet - NorthStar Healthcare Unlimited Company 36699911000001101 Sertraline 100mg tablets 28 tablet - Noumed Life Sciences Ltd 17928311000001102 Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 36619211000001106 Sertraline 100mg tablets 28 tablet - Relonchem Ltd 36619211000001105 Sertraline 100mg tablets 28 tablet - Sandoz Ltd 15211511000001105 Sertraline 100mg tablets 28 tablet - Samoz Ltd 15211511000001104 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc 9746311000001104 Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd 21896511000001109 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001103 Sertraline 100mg tablets 28 tablet - Vaymade Healthcare Plc 9781311000001103 Sertraline 100mg tablets 30 tablet 16066611000001108 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37720411000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37720411000001108 Sertraline 100mg tablets 500 tablet - AA H Pharmaceuticals Plc 4313611000001108 Sertraline 100mg tablets 500 tablet - AA H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - AN J Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 8696011000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 869611000001108 Sertraline 100mg/5ml oral suspension 1 ml - Special Order 869611000001100 Sertraline 100mg/5ml oral suspension 1 ml - Special Order 8696311000001100 Sertraline 100mg/5ml oral suspension | | |
| 39925311000001107 Company | | |
| 17928311000001102 | 39623511000001107 | |
| 9738711000001100 Sertraline 100mg tablets 28 tablet - PLIVA Pharma Ltd 10567511000001100 Sertraline 100mg tablets 28 tablet - Ranbaxy (UK) Ltd 36619211000001106 Sertraline 100mg tablets 28 tablet - Ria Generics Ltd 3775111000001108 Sertraline 100mg tablets 28 tablet - Ria Generics Ltd 9775111000001108 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc 9746311000001104 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc 9746311000001104 Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd 13762811000001109 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 9752011000001103 Sertraline 100mg tablets 30 tablet - Zentiva Pharma UK Ltd 9431311000001104 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 9509211000001107 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 978111000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 978111000001109 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 978111000001100 Sertraline 100mg tablets 500 tablet - Waymade Healthcare Plc | 36699911000001101 | Sertraline 100mg tablets 28 tablet - Noumed Life Sciences Ltd |
| 10567511000001104 | 17928311000001102 | Sertraline 100mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 10295211000001100 | 9738711000001100 | Sertraline 100mg tablets 28 tablet - PLIVA Pharma Ltd |
| Sertraline 100mg tablets 28 tablet - Ria Generics Ltd | 10567511000001104 | Sertraline 100mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 9775111000001108 Sertraline 100mg tablets 28 tablet - Sandoz Ltd 15211511000001104 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc 9746311000001102 Sertraline 100mg tablets 28 tablet - Teva UK Ltd 13762811000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001103 Sertraline 100mg tablets 30 tablet - Zentiva Pharma UK Ltd 5433311000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37220511000001107 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696111000001105 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001100 Sertraline 100mg/5ml oral suspension 1 ml Drug Tariff Special Order < | 10295211000001100 | Sertraline 100mg tablets 28 tablet - Relonchem Ltd |
| 15211511000001105 Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc | 36619211000001106 | Sertraline 100mg tablets 28 tablet - Ria Generics Ltd |
| 9746311000001104 Sertraline 100mg tablets 28 tablet - Teva UK Ltd 13762811000001102 Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd 21896511000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 5413311000001103 Sertraline 100mg tablets 30 tablet 5509211000001101 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001100 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet - Waymade Healthcare Plc 37220411000001102 Sertraline 100mg tablets 500 tablet - Maylan 37220411000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg/5ml oral suspension 8696111000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001103 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 82439411000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 829651100000 | 9775111000001108 | Sertraline 100mg tablets 28 tablet - Sandoz Ltd |
| 13762811000001102 Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd 21896511000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 5413311000001103 Sertraline 100mg tablets 30 tablet 16066611000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 3722041100001108 Sertraline 100mg tablets 500 tablet 3722041100001108 Sertraline 100mg tablets 500 tablet 37220511000001107 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 3721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696211000001103 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439511000001108 Sertraline 100mg/5ml oral suspension 1 0ml - Drug Tariff Special Order 8696311000001107 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001107 | 15211511000001105 | Sertraline 100mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 21896511000001109 Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 5413311000001103 Sertraline 100mg tablets 30 tablet 16066611000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet - Waymade Healthcare Plc 37220511000001107 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 869611000001105 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696111000001102 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 869611000001107 Sertraline 100mg/5ml oral suspension 1 ml 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml | 9746311000001104 | Sertraline 100mg tablets 28 tablet - Teva UK Ltd |
| 9781311000001102 Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 5413311000001103 Sertraline 100mg tablets 30 tablet 16066611000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 1521171100001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001107 Sertraline 100mg/5ml oral suspension 8696111000001103 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696211000001103 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8696311000001107 Sertraline 10mg/5ml oral suspension 1 ml - Drug Tariff Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001101 <td>13762811000001102</td> <td>Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd</td> | 13762811000001102 | Sertraline 100mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 9752011000001104 Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd 5413311000001103 Sertraline 100mg tablets 30 tablet 16066611000001101 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696211000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439411000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8696311000001107 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001100 Sertra | 21896511000001109 | Sertraline 100mg tablets 28 tablet - Waymade Healthcare Plc |
| 5413311000001103 Sertraline 100mg tablets 30 tablet 16066611000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 869611100001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 869601100001103 Sertraline 100mg/5ml oral suspension 1 ml 869621100001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension - Special Order 869641100001107 Sertraline 10mg/5ml oral suspension 1 ml - Drug Tariff Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696511000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 3 | 9781311000001102 | Sertraline 100mg tablets 28 tablet - Wockhardt UK Ltd |
| 16066611000001108 Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg/5ml oral suspension 8696111000001105 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8696311000001107 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 3697311000001101 Sertraline 12.5mg tablets - Special Order 3687481100000110 | 9752011000001104 | Sertraline 100mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 5509211000001101 Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd 15211711000001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001101 Sertraline 12.5mg tablets 36874811000001103 Sertraline 12.5mg tablets - Special Order 36875011000001104 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg/5ml oral suspension | 5413311000001103 | Sertraline 100mg tablets 30 tablet |
| 15211711000001100 Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 8696511000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension <td>16066611000001108</td> <td>Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd</td> | 16066611000001108 | Sertraline 100mg tablets 30 tablet - Bristol Laboratories Ltd |
| 5413611000001108 Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 869611100001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets 36874811000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order | 5509211000001101 | Sertraline 100mg tablets 30 tablet - Dowelhurst Ltd |
| 37220411000001108 Sertraline 100mg tablets 500 tablet 37768711000001107 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension 8696411000001100 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36875011000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg/5ml oral suspension | 15211711000001100 | Sertraline 100mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 37768711000001102 Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001107 Sertraline 10mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8696411000001100 Sertraline 10mg/5ml oral suspension - Special Order 8696511000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36875011000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 5413611000001108 | Sertraline 100mg tablets 30 tablet - Waymade Healthcare Plc |
| 37220511000001107 Sertraline 100mg tablets 500 tablet - Mylan 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 10mg/5ml oral suspension 8696411000001102 Sertraline 10mg/5ml oral suspension 8696311000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 37220411000001108 | Sertraline 100mg tablets 500 tablet |
| 8721711000001105 Sertraline 100mg/5ml oral suspension 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001107 Sertraline 100mg/5ml oral suspension 100 ml 8721811000001107 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 37768711000001102 | Sertraline 100mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 8696111000001102 Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001102 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001101 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg/5ml oral suspension | 37220511000001107 | Sertraline 100mg tablets 500 tablet - Mylan |
| 8696011000001103 Sertraline 100mg/5ml oral suspension 1 ml 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001102 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36875011000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg/5ml oral suspension | 8721711000001105 | Sertraline 100mg/5ml oral suspension |
| 8696211000001108 Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001102 Sertraline 10mg/5ml oral suspension - Special Order 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36875011000001103 Sertraline 12.5mg tablets 1 tablet 36875011000001104 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696111000001102 | Sertraline 100mg/5ml oral suspension - Drug Tariff Special Order |
| 24439411000001108 Sertraline 100mg/5ml oral suspension 100 ml 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001102 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696011000001103 | Sertraline 100mg/5ml oral suspension 1 ml |
| 24439511000001107 Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order 8721811000001102 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696211000001108 | Sertraline 100mg/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 8721811000001102 Sertraline 10mg/5ml oral suspension 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 24439411000001108 | Sertraline 100mg/5ml oral suspension 100 ml |
| 8696411000001107 Sertraline 10mg/5ml oral suspension - Special Order 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 24439511000001107 | Sertraline 100mg/5ml oral suspension 100 ml - Drug Tariff Special Order |
| 8696311000001100 Sertraline 10mg/5ml oral suspension 1 ml 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8721811000001102 | Sertraline 10mg/5ml oral suspension |
| 8696511000001106 Sertraline 10mg/5ml oral suspension 1 ml - Special Order 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696411000001107 | Sertraline 10mg/5ml oral suspension - Special Order |
| 36905311000001101 Sertraline 12.5mg tablets 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696311000001100 | Sertraline 10mg/5ml oral suspension 1 ml |
| 36874911000001103 Sertraline 12.5mg tablets - Special Order 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 8696511000001106 | Sertraline 10mg/5ml oral suspension 1 ml - Special Order |
| 36874811000001108 Sertraline 12.5mg tablets 1 tablet 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 36905311000001101 | Sertraline 12.5mg tablets |
| 36875011000001103 Sertraline 12.5mg tablets 1 tablet - Special Order 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 36874911000001103 | Sertraline 12.5mg tablets - Special Order |
| 13045611000001104 Sertraline 12.5mg/5ml oral suspension | 36874811000001108 | Sertraline 12.5mg tablets 1 tablet |
| | 36875011000001103 | Sertraline 12.5mg tablets 1 tablet - Special Order |
| 13030011000001104 | 13045611000001104 | Sertraline 12.5mg/5ml oral suspension |
| Sertraline 12.5mg/5ml oral suspension - Special Order | 13030011000001104 | Sertraline 12.5mg/5ml oral suspension - Special Order |
| 13029811000001104 Sertraline 12.5mg/5ml oral suspension 1 ml | 13029811000001104 | Sertraline 12.5mg/5ml oral suspension 1 ml |
| 13030111000001103 Sertraline 12.5mg/5ml oral suspension 1 ml - Special Order | 13030111000001103 | Sertraline 12.5mg/5ml oral suspension 1 ml - Special Order |
| 13045711000001108 Sertraline 150mg/5ml oral suspension | 13045711000001108 | Sertraline 150mg/5ml oral suspension |
| 13030411000001108 Sertraline 150mg/5ml oral suspension - Special Order | 13030411000001108 | Sertraline 150mg/5ml oral suspension - Special Order |
| 13030311000001101 Sertraline 150mg/5ml oral suspension 1 ml | 13030311000001101 | Sertraline 150mg/5ml oral suspension 1 ml |
| 13030511000001107 Sertraline 150mg/5ml oral suspension 1 ml - Special Order | 13030511000001107 | Sertraline 150mg/5ml oral suspension 1 ml - Special Order |

| 22750711000001105 | Cortroline 15mg/5ml arel suspension |
|---|---|
| 32750711000001105 | Sertraline 15mg/5ml oral suspension |
| 32727211000001100 | Sertraline 15mg/5ml oral suspension - Special Order |
| 32727111000001106 | Sertraline 15mg/5ml oral suspension 1 ml |
| 32727311000001108 | Sertraline 15mg/5ml oral suspension 1 ml - Special Order |
| 13045811000001100 | Sertraline 20mg/5ml oral suspension |
| 13030711000001102 | Sertraline 20mg/5ml oral suspension - Special Order |
| 13030611000001106 | Sertraline 20mg/5ml oral suspension 1 ml |
| 13030811000001105 | Sertraline 20mg/5ml oral suspension 1 ml - Special Order |
| 36003511000001103 | Sertraline 25mg/5ml oral solution |
| 35993811000001105 | Sertraline 25mg/5ml oral solution - Special Order |
| 35993711000001102 | Sertraline 25mg/5ml oral solution 1 ml |
| 35994011000001102 | Sertraline 25mg/5ml oral solution 1 ml - Special Order |
| 13045911000001105 | Sertraline 25mg/5ml oral suspension |
| 13031011000001108 | Sertraline 25mg/5ml oral suspension - Drug Tariff Special Order |
| 13030911000001100 | Sertraline 25mg/5ml oral suspension 1 ml |
| 13031111000001109 | Sertraline 25mg/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 36533111000001101 | Sertraline 25mg/5ml oral suspension 150 ml |
| 36533211000001107 | Sertraline 25mg/5ml oral suspension 150 ml - Drug Tariff Special Order |
| 39704111000001102 | Sertraline 50mg tablets |
| 321959007 | Sertraline 50mg tablets |
| 9751311000001105 | Sertraline 50mg tablets - A A H Pharmaceuticals Ltd |
| 20169711000001108 | Sertraline 50mg tablets - Accord Healthcare Ltd |
| 9744911000001106 | Sertraline 50mg tablets - Actavis UK Ltd |
| 9840111000001101 | Sertraline 50mg tablets - Alliance Healthcare (Distribution) Ltd |
| 11408711000001107 | Sertraline 50mg tablets - Almus Pharmaceuticals Ltd |
| 13770511000001106 | Sertraline 50mg tablets - Apotex UK Ltd |
| 10437511000001104 | Sertraline 50mg tablets - Arrow Generics Ltd |
| 16066211000001106 | Sertraline 50mg tablets - Bristol Laboratories Ltd |
| 14130111000001105 | Sertraline 50mg tablets - Consilient Health Ltd |
| 28988111000001103 | Sertraline 50mg tablets - Crescent Pharma Ltd |
| 30095811000001109 | Sertraline 50mg tablets - DE Pharmaceuticals |
| 5452311000001101 | Sertraline 50mg tablets - Dowelhurst Ltd |
| 11011711000001109 | Sertraline 50mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 10296311000001103 | Sertraline 50mg tablets - Focus Pharmaceuticals Ltd |
| 33654711000001102 | Sertraline 50mg tablets - Genesis Pharmaceuticals Ltd |
| 9841411000001102 | Sertraline 50mg tablets - IVAX Pharmaceuticals UK Ltd |
| 9764711000001103 | Sertraline 50mg tablets - Kent Pharmaceuticals Ltd |
| 27700611000001108 | Sertraline 50mg tablets - Lupin Healthcare (UK) Ltd |
| 37139311000001105 | Sertraline 50mg tablets - Mawdsley-Brooks & Company Ltd |
| 39242911000001106 | Sertraline 50mg tablets - Medihealth (Northern) Ltd |
| 19734711000001107 | Sertraline 50mg tablets - Medreich Plc |
| 19197011000001101 | Sertraline 50mg tablets - Milpharm Ltd |
| 9842711000001101 | Sertraline 50mg tablets - Mylan |
| 10442311000001107 | Sertraline 50mg tablets - Niche Generics Ltd |
| 39623611000001106 | Sertraline 50mg tablets - NorthStar Healthcare Unlimited Company |
| 36699611000001107 | Sertraline 50mg tablets - Noumed Life Sciences Ltd |
| 17928011000001100 | Sertraline 50mg tablets - Phoenix Healthcare Distribution Ltd |
| 9738411000001106 | Sertraline 50mg tablets - PLIVA Pharma Ltd |
| 10567211000001102 | Sertraline 50mg tablets - Ranbaxy (UK) Ltd |
| 1030721100001102 | Jertranne Jonig tablets - Natibaxy (OK) Ltu |

| 10295311000001108 | Sertraline 50mg tablets - Relonchem Ltd |
|---|---|
| 36619311000001103 | Sertraline 50mg tablets - Ria Generics Ltd |
| 9774711000001105 | Sertraline 50mg tablets - Sandoz Ltd |
| 15187911000001107 | Sertraline 50mg tablets - Sigma Pharmaceuticals Plc |
| 9746011000001102 | Sertraline 50mg tablets - Teva UK Ltd |
| 13762511000001100 | Sertraline 50mg tablets - Tillomed Laboratories Ltd |
| 21896011000001101 | Sertraline 50mg tablets - Waymade Healthcare Plc |
| 5413111000001100 | Sertraline 50mg tablets - Waymade Healthcare Plc |
| 9779311000001107 | Sertraline 50mg tablets - Wockhardt UK Ltd |
| 9751711000001109 | Sertraline 50mg tablets - Zentiva Pharma UK Ltd |
| 1040511000001102 | Sertraline 50mg tablets 28 tablet |
| 9751411000001103 | Sertraline 50mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 20169811000001100 | Sertraline 50mg tablets 28 tablet - Accord Healthcare Ltd |
| 9745011000001106 | Sertraline 50mg tablets 28 tablet - Actavis UK Ltd |
| 9840211000001107 | Sertraline 50mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 11408811000001104 | Sertraline 50mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 13770611000001105 | Sertraline 50mg tablets 28 tablet - Apotex UK Ltd |
| 10437711000001109 | Sertraline 50mg tablets 28 tablet - Arrow Generics Ltd |
| 16066311000001103 | Sertraline 50mg tablets 28 tablet - Bristol Laboratories Ltd |
| 14130211000001104 | Sertraline 50mg tablets 28 tablet - Consilient Health Ltd |
| 28988211000001109 | Sertraline 50mg tablets 28 tablet - Crescent Pharma Ltd |
| 30095911000001104 | Sertraline 50mg tablets 28 tablet - DE Pharmaceuticals |
| 11011811000001101 | Sertraline 50mg tablets 28 tablet - Dr Reddys Laboratories (UK) Ltd |
| 10296411000001105 | Sertraline 50mg tablets 28 tablet - Focus Pharmaceuticals Ltd |
| 33654811000001105 | Sertraline 50mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 9841511000001103 | Sertraline 50mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 9764811000001106 | Sertraline 50mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 27700711000001104 | Sertraline 50mg tablets 28 tablet - Lupin Healthcare (UK) Ltd |
| 37139411000001103 | Sertraline 50mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 39243011000001103 | Sertraline 50mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 19734811000001104 | Sertraline 50mg tablets 28 tablet - Medreich Plc |
| 19197111000001100 | Sertraline 50mg tablets 28 tablet - Milpharm Ltd |
| 9842811000001109 | Sertraline 50mg tablets 28 tablet - Mylan |
| 10442411000001100 | Sertraline 50mg tablets 28 tablet - Niche Generics Ltd |
| 39623711000001102 | Sertraline 50mg tablets 28 tablet - NorthStar Healthcare Unlimited |
| 39623711000001102 | Company |
| 36699711000001103 | Sertraline 50mg tablets 28 tablet - Noumed Life Sciences Ltd |
| 17928111000001104 | Sertraline 50mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 9738511000001105 | Sertraline 50mg tablets 28 tablet - PLIVA Pharma Ltd |
| 10567311000001105 | Sertraline 50mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 10295511000001102 | Sertraline 50mg tablets 28 tablet - Relonchem Ltd |
| 36619411000001105 | Sertraline 50mg tablets 28 tablet - Ria Generics Ltd |
| 9774811000001102 | Sertraline 50mg tablets 28 tablet - Sandoz Ltd |
| 15188111000001105 | Sertraline 50mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 9746111000001101 | Sertraline 50mg tablets 28 tablet - Teva UK Ltd |
| 13762611000001101 | Sertraline 50mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 21896211000001106 | Sertraline 50mg tablets 28 tablet - Waymade Healthcare Plc |
| 9779511000001101 | Sertraline 50mg tablets 28 tablet - Wockhardt UK Ltd |
| 9751811000001101 | Sertraline 50mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 5412911000001109 | Sertraline 50mg tablets 30 tablet |

| 5452511000001107 | Sertraline 50mg tablets 30 tablet - Dowelhurst Ltd |
|---|---|
| 5413211000001106 | Sertraline 50mg tablets 30 tablet - Waymade Healthcare Plc |
| 37220211000001109 | Sertraline 50mg tablets 500 tablet |
| 37768811000001105 | Sertraline 50mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 37220311000001101 | Sertraline 50mg tablets 500 tablet - Mylan |
| 35993411000001108 | Sertraline 50mg/5ml oral solution - Special Order |
| 35993611000001106 | Sertraline 50mg/5ml oral solution 1 ml - Special Order |
| 8721911000001107 | Sertraline 50mg/5ml oral suspension |
| 8696711000001101 | Sertraline 50mg/5ml oral suspension - Drug Tariff Special Order |
| 8696611000001105 | Sertraline 50mg/5ml oral suspension 1 ml |
| 8696811000001109 | Sertraline 50mg/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 19605211000001101 | Sertraline 50mg/5ml oral suspension 150 ml |
| 19605311000001109 | Sertraline 50mg/5ml oral suspension 150 ml - Drug Tariff Special Order |
| 34684211000001100 | Sertraline 5mg/5ml oral suspension |
| 34673611000001108 | Sertraline 5mg/5ml oral suspension - Special Order |
| 34673411000001105 | Sertraline 5mg/5ml oral suspension 1 ml |
| 34673711000001104 | Sertraline 5mg/5ml oral suspension 1 ml - Special Order |
| 35575611000001108 | Sertraline 75mg/5ml oral suspension |
| 35547611000001102 | Sertraline 75mg/5ml oral suspension - Special Order |
| 35547411000001100 | Sertraline 75mg/5ml oral suspension 1 ml |
| 35547811000001103 | Sertraline 75mg/5ml oral suspension 1 ml - Special Order |
| 30738611000001105 | Vortioxetine 10mg tablets |
| 30248011000001109 | Vortioxetine 10mg tablets 28 tablet |
| 30738711000001101 | Vortioxetine 20mg tablets |
| 30247711000001105 | Vortioxetine 20mg tablets 28 tablet |
| 30738811000001109 | Vortioxetine 5mg tablets |
| 30247411000001104 | Vortioxetine 5mg tablets 28 tablet |

| Tricyclic Antidepressants | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| d71 | All | AMITRIPTYLINE HYDROCHLORIDE [ANTIDEPRESSANT] |
| d711. | All | AMITRIPTYLINE 10mg tablets |
| d712. | All | AMITRIPTYLINE 25mg tablets |
| d713. | All | AMITRIPTYLINE 50mg tablets |
| d714. | All | *DOMICAL 10mg tablets |
| d715. | All | *DOMICAL 25mg tablets |
| d716. | All | *DOMICAL 50mg tablets |
| d717. | All | ELAVIL 10mg tablets |
| d718. | All | ELAVIL 25mg tablets |
| d719. | All | *LENTIZOL 25mg m/r capsules |
| d71a. | All | *LENTIZOL 50mg m/r capsules |
| d71b. | All | *TRYPTIZOL 75mg m/r capsules |
| d71c. | All | *TRYPTIZOL 10mg tablets |
| d71d. | All | *TRYPTIZOL 25mg tablets |
| d71e. | All | *TRYPTIZOL 50mg tablets |
| d71f. | All | *TRYPTIZOL 10mg/5mL syrup |
| d71g. | All | TRYPTIZOL 100mg/10mL injection |
| d71h. | All | AMITRIPTYLINE 25mg/5mL sugar free solution |
| d71i. | All | AMITRIPTYLINE 50mg/5mL sugar free solution |
| d71u. | All | AMITRIPTYLINE 25mg m/r capsules |
| d71v. | All | AMITRIPTYLINE 50mg m/r capsules |
| d71w. | All | AMITRIPTYLINE 75mg m/r capsules |
| d71y. | All | *AMITRIPTYLINE 10mg/5mL syrup |
| d71z. | All | AMITRIPTYLINE HYDROCHLORIDE 100mg/10mL injection |
| d73 | All | CLOMIPRAMINE HYDROCHLORIDE |
| d731. | All | *ANAFRANIL 10mg capsules |
| d732. | All | *ANAFRANIL 25mg capsules |
| d733. | All | *ANAFRANIL 50mg capsules |
| d734. | All | *ANAFRANIL 25mg/5mL syrup |
| d735. | All | *ANAFRANIL 25mg/2mL injection |
| d736. | All | ANAFRANIL SR 75mg m/r tablets |
| d737. | All | *TRANQUAX 10mg capsules |
| d738. | All | *TRANQUAX 25mg capsules |
| d739. | All | TRANQUAX 50mg capsules |
| d73r. | All | *CLOMIPRAMINE HCL 50mg tablets |
| d73s. | All | *CLOMIPRAMINE HCL 10mg tablets |
| d73t. | All | *CLOMIPRAMINE HCL 25mg tablets |
| d73u. | All | CLOMIPRAMINE HCL 10mg capsules |
| d73v. | All | CLOMIPRAMINE HCL 25mg capsules |
| d73w. | All | CLOMIPRAMINE HCL 50mg capsules |
| d73x. | All | CLOMIPRAMINE HYDROCHLORIDE 25mg/5mL syrup |
| d73y. | All | CLOMIPRAMINE HCL 25mg/2mL injection |
| d73z. | All | CLOMIPRAMINE HCL 75mg m/r tabs |
| d75 | All | DOSULEPIN HYDROCHLORIDE |
| d751. | All | PROTHIADEN 25mg capsules |
| d752. | All | PROTHIADEN 75mg tablets |

| d754. | All | *PREPADINE 75mg tablets |
|-------|-----|-------------------------------------------------|
| d755. | All | *DOTHAPAX 25mg capsules |
| d756. | All | *DOTHAPAX 75mg tablets |
| d759. | All | *THADEN 25mg capsules |
| d75A. | All | *THADEN 75mg tablets |
| d75y. | All | DOSULEPIN HYDROCHLORIDE 25mg capsules |
| d75z. | All | DOSULEPIN HYDROCHLORIDE 75mg tablets |
| d76 | All | DOXEPIN |
| d761. | All | *SINEQUAN 10mg capsules x56CP |
| d762. | All | *SINEQUAN 25mg capsules x28CP |
| d763. | All | *SINEQUAN 50mg capsules x28CP |
| d764. | All | *SINEQUAN 75mg capsules x28CP |
| d765. | All | *SINEPIN 25mg capsules |
| d766. | All | *SINEPIN 50mg capsules |
| d76w. | All | *DOXEPIN 10mg capsules |
| d76x. | All | DOXEPIN 25mg capsules |
| d76y. | All | DOXEPIN 50mg capsules |
| d76z. | All | *DOXEPIN 75mg capsules |
| d77 | All | IMIPRAMINE HYDROCHLORIDE [ANTIDEPRESSANT] |
| d771. | All | IMIPRAMINE 10mg tabs |
| d772. | All | IMIPRAMINE 25mg tablets |
| d773. | All | *PRAMINIL 10mg tablets |
| d774. | All | *PRAMINIL 25mg tablets |
| d775. | All | *TOFRANIL 10mg tablets |
| d776. | All | *TOFRANIL 25mg tablets |
| d777. | All | *TOFRANIL 25mg/5mL syrup |
| d77w. | All | IMIPRAMINE HYDROCHLORIDE 25mg/5mL oral solution |
| d77x. | All | IMIPRAMINE HYDROCHLORIDE 10mg tablets |
| d77y. | All | IMIPRAMINE HYDROCHLORIDE 25mg tablets |
| d77z. | All | IMIPRAMINE HYDROCHLORIDE 25mg/5mL syrup |
| d79 | All | LOFEPRAMINE |
| d791. | All | *GAMANIL 70mg tablets x56CP |
| d792. | All | LOMONT 70mg/5mL sugar free suspension |
| d793. | All | *FEPRAPAX 70mg tablets |
| d794. | All | *GAMANIL 70mg tablets |
| d79y. | All | LOFEPRAMINE 70mg/5mL sugar free suspension |
| d79z. | All | LOFEPRAMINE 70mg tablets |
| d7b | All | MIANSERIN HYDROCHLORIDE |
| d7b1. | All | MIANSERIN 10mg tablets |
| d7b2. | All | MIANSERIN 20mg tablets |
| d7b3. | All | MIANSERIN 30mg tablets |
| d7b4. | All | *BOLVIDON 10mg tablets |
| d7b5. | All | *BOLVIDON 20mg tablets |
| d7b6. | All | *BOLVIDON 30mg tablets |
| d7b7. | All | *NORVAL 10mg tablets |
| d7b8. | All | *NORVAL 20mg tablets |
| d7b9. | All | *NORVAL 30mg tablets |
| d7c | All | NORTRIPTYLINE |
| d7c1. | All | *ALLEGRON 10mg tablets |
| 4/61. | | ALLEGION TOTAL MOTEUS |

| d7c2. | All | *ALLEGRON 25mg tablets |
|---|---|---|
| d7c3. | All | *AVENTYL 10mg capsules |
| d7c4. | All | *AVENTYL 25mg capsules |
| d7c5. | All | *AVENTYL 10mg/5mL liquid |
| d7c6. | All | NORTRIPTYLINE 10mg tablets |
| d7c7. | All | *NORTRIPTYLINE 10mg/5mL liquid |
| d7c8. | All | NORTRIPTYLINE 25mg tablets |
| d7c9. | All | *NORTRIPTYLINE 10mg capsules |
| d7cy. | All | *NORTRIPTYLINE 25mg capsules |
| d7e | All | TRAZODONE HYDROCHLORIDE |
| d7e1. | All | MOLIPAXIN 50mg capsules x84CP |
| d7e2. | All | MOLIPAXIN 100mg capsules x56CP |
| d7e3. | All | *MOLIPAXIN 50mg/5mL liquid |
| d7e4. | All | MOLIPAXIN 150mg tablets x28CP |
| d7e5. | All | TRAZODONE HYDROCHLORIDE 150mg tablets |
| d7e6. | All | MOLIPAXIN CR 150mg m/r tablets x28 |
| d7e7. | All | TRAZODONE HYDROCHLORIDE 150mg m/r tablets |
| d7ew. | All | TRAZODONE HYDROCHLORIDE 190mg myr tablets TRAZODONE HYDROCHLORIDE 100mg capsules |
| d7ex. | All | TRAZODONE HYDROCHLORIDE 50mg capsules |
| d7ez. | All | TRAZODONE HYDROCHLORIDE 50mg capsules TRAZODONE HYDROCHLORIDE 50mg/5mL liquid |
| d7f | All | TRIMIPRAMINE |
| d7f1. | All | *SURMONTIL 50mg capsules x28CP |
| d7f2. | All | *SURMONTIL 10mg tablets |
| d7f3. | All | *SURMONTIL 25mg tablets |
| d7fx. | All | TRIMIPRAMINE 50mg capsules |
| d7fy. | All | TRIMIPRAMINE 10mg tablets |
| d7fz. | All | TRIMIPRAMINE 25mg tablets |
| Read CTV3 Code | Term ID | Description Description |
| x01Aw | All | Amitriptyline |
| d711. | All | Amitriptyline hydrochloride 10mg tablet |
| d714. | All | Domical 10mg tablet |
| d717. | All | Elavil 10mg tablet |
| d71c. | All | Tryptizol 10mg tablet |
| d712. | All | Amitriptyline hydrochloride 25mg tablet |
| d715. | All | Domical 25mg tablet |
| d718. | All | Elavil 25mg tablet |
| d71d. | All | Tryptizol 25mg tablet |
| d713. | All | Amitriptyline hydrochloride 50mg tablet |
| d716. | All | Domical 50mg tablet |
| d71e. | All | Tryptizol 50mg tablet |
| d71u. | All | Amitriptyline hydrochloride 25mg m/r capsule |
| d719. | All | Lentizol 25mg m/r capsule |
| d71v. | All | Amitriptyline hydrochloride 50mg m/r capsule |
| d71a. | All | Lentizol 50mg m/r capsule |
| d71w. | All | Amitriptyline hydrochloride 75mg m/r capsule |
| d71b. | All | Tryptizol 75mg m/r capsule |
| d71y. | All | Amitriptyline 10mg/5mL oral suspension |
| · · | | |
| d71f. | All | Tryptizol 10mg/5mL mixture |
| d71f.<br>d71h. | | |

| d71i. | All | Amitriptyline 50mg/5mL s/f oral solution |
|-------|-----|--------------------------------------------------------|
| d71z. | All | Amitriptyline hydrochloride 100mg/10mL injection |
| d71g. | All | Tryptizol 100mg/10mL injection |
| d71 | All | Amitriptyline hydrochloride [antidepressant] |
| d71j. | All | AMITRIPTYLINE 10mg/5mL sugar free oral solution |
| gd1 | All | Amitriptyline hydrochloride [enuresis - no drugs here] |
| x01Ax | All | Clomipramine |
| d73s. | All | Clomipramine hydrochloride 10mg tablet |
| d73t. | All | Clomipramine hydrochloride 25mg tablet |
| d73r. | All | Clomipramine hydrochloride 50mg tablet |
| d73u. | All | Clomipramine hydrochloride 10mg capsule |
| d731. | All | Anafranil 10mg capsule |
| d737. | All | Tranquax 10mg capsule |
| d73v. | All | Clomipramine hydrochloride 25mg capsule |
| d732. | | Anafranil 25mg capsule |
| | All | |
| d738. | All | Tranquax 25mg capsule |
| d73w. | All | Clomipramine hydrochloride 50mg capsule |
| d733. | All | Anafranil 50mg capsule |
| d739. | All | Tranquax 50mg capsule |
| d73z. | All | Clomipramine hydrochloride 75mg m/r tablet |
| d736. | All | Anafranil SR 75mg tablet |
| d73x. | All | Clomipramine hydrochloride 25mg/5mL syrup |
| d734. | All | Anafranil 25mg/5mL syrup |
| d73y. | All | Clomipramine hydrochloride 25mg/2mL injection |
| d735. | All | Anafranil 25mg/2mL injection |
| d73 | All | Clomipramine hydrochloride |
| d76 | All | Doxepin |
| d76w. | All | Doxepin 10mg capsule |
| x00E9 | All | Sinequan 10mg capsule |
| d761. | All | Sinequan 10mg capsules x56CP |
| d76x. | All | Doxepin 25mg capsule |
| d765. | All | SINEPIN 25mg capsules |
| x00EA | All | Sinequan 25mg capsule |
| d762. | All | Sinequan 25mg capsules x28CP |
| d76y. | All | Doxepin 50mg capsule |
| d766. | All | SINEPIN 50mg capsules |
| x00EB | All | Sinequan 50mg capsule |
| d763. | All | Sinequan 50mg capsules x28CP |
| d76z. | All | Doxepin 75mg capsule |
| x00EC | All | Sinequan 75mg capsule |
| d764. | All | Sinequan 75mg capsules x28CP |
| x01B0 | All | Imipramine |
| d771. | All | Imipramine hydrochloride 10mg tablet |
| d773. | All | Praminil 10mg tablet |
| d775. | All | Tofranil 10mg tablet |
| d772. | All | Imipramine hydrochloride 25mg tablet |
| d774. | All | Praminil 25mg tablet |
| d776. | All | Tofranil 25mg tablet |
| d77z. | All | Imipramine hydrochloride 25mg/5mL syrup |

| d777. | All | Tofranil 25mg/5mL syrup |
|-------|-----|--------------------------------------------------------|
| d77 | All | Imipramine hydrochloride [antidepressant] |
| d77w. | All | IMIPRAMINE HYDROCHLORIDE 25mg/5mL oral solution |
| gd5 | All | Imipramine hydrochloride [enuresis - no drugs here] |
| x01Ay | All | Desipramine |
| d74z. | All | Desipramine hydrochloride 25mg tablet |
| d741. | All | Pertofran 25mg tablet |
| d74 | All | Desipramine hydrochloride |
| d7c | All | Nortriptyline |
| d7c6. | All | Nortriptyline 10mg tablet |
| d7c1. | All | Allegron 10mg tablet |
| d7c8. | All | Nortriptyline 25mg tablet |
| d7c2. | All | Allegron 25mg tablet |
| d7c9. | All | Nortriptyline 10mg capsule |
| d7c3. | All | Aventyl 10mg capsule |
| d7cy. | All | Nortriptyline 25mg capsule |
| d7c4. | All | Aventyl 25mg capsule |
| d7c7. | All | Nortriptyline 10mg/5mL liquid |
| d7c5. | All | Aventyl 10mg/5mL liquid |
| gd6 | All | Nortriptyline hydrochloride [enuresis - no drugs here] |
| x01B2 | All | Trazodone |
| d7ex. | All | Trazodone hydrochloride 50mg capsule |
| x00E4 | All | Molipaxin 50mg capsule |
| d7e1. | All | Molipaxin 50mg capsules x84CP |
| d7ew. | All | Trazodone hydrochloride 100mg capsule |
| x00E5 | All | Molipaxin 100mg capsule |
| d7e2. | All | Molipaxin 100mg capsules x56CP |
| d7e5. | All | Trazodone hydrochloride 150mg tablet |
| x00fa | All | Molipaxin 150mg tablet |
| d7e4. | All | Molipaxin 150mg tablets x28CP |
| d7e7. | All | Trazodone hydrochloride 150mg m/r tablet |
| x00fb | All | Molipaxin CR 150mg tablet |
| d7e6. | All | Molipaxin CR 150mg m/r tablets x28 |
| d7ez. | All | Trazodone hydrochloride 50mg/5mL liquid |
| d7e3. | All | Molipaxin 50mg/5mL liquid |
| d7e | All | Trazodone hydrochloride |
| x01Az | All | Dosulepin |
| d75y. | All | Dosulepin hydrochloride 25mg capsule |
| d755. | All | Dothapax 25mg capsule |
| d753. | All | Prepadine 25mg capsule |
| d751. | All | Prothiaden 25mg capsule |
| d759. | All | Thaden 25mg capsule |
| d75z. | All | Dosulepin hydrochloride 75mg tablet |
| d756. | All | Dothapax 75mg tablet |
| d754. | All | Prepadine 75mg tablet |
| d752. | All | Prothiaden 75mg tablet |
| d75A. | All | Thaden 75mg tablet |
| d757. | All | Dosulepin hydrochloride 25mg/5mL s/f elixir |
| d758. | All | Dosulepin hydrochloride 75mg/5mL s/f elixir |

| d75 | All | Dothiepin hydrochloride |
|---|---|---|
| d79 | All | Lofepramine |
| d79z. | All | Lofepramine 70mg tablet |
| d793. | All | Feprapax 70mg tablet |
| d794. | All | Gamanil 70mg tablet |
| d791. | All | Gamanil 70mg tablets x56CP |
| d79y. | All | Lofepramine 70mg/5mL s/f suspension |
| d792. | All | Lomont 70mg/5mL s/f suspension |
| d7c | All | Nortriptyline |
| d7c6. | All | Nortriptyline 10mg tablet |
| d7c1. | All | Allegron 10mg tablet |
| d7c8. | All | Nortriptyline 25mg tablet |
| d7c2. | All | Allegron 25mg tablet |
| d7c9. | All | Nortriptyline 10mg capsule |
| d7c3. | All | Aventyl 10mg capsule |
| d7cy. | All | Nortriptyline 25mg capsule |
| d7c4. | All | Aventyl 25mg capsule |
| d7c4. | All | Nortriptyline 10mg/5mL liquid |
| d7c5. | All | |
| | All | Aventyl 10mg/5mL liquid Nortriptyline hydrochloride [enuresis - no drugs here] |
| gd6<br>d7f | All | Trimipramine |
| d7fy. | All | Trimipramine 10mg tablet |
| d7f2. | All | Surmontil 10mg tablet |
| d7fz. | All | Trimipramine 25mg tablet |
| d7f3. | All | <del> </del> |
| d7fx. | All | Surmontil 25mg tablet Trimipramine 50mg capsule |
| x00ED | All | Surmontil 50mg capsule |
| d7f1. | All | Surmontil 50mg capsules x28CP |
| SNOMED Code | Term ID | Description |
| 893811000001100 | Termin | Allegron 10mg tablets - King Pharmaceuticals Ltd |
| 16136611000001100 | | Allegron 10mg tablets - King Pharmaceuticals Ltu Allegron 10mg tablets - Lexon (UK) Ltd |
| 16259011000001109 | | Allegron 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 17532311000001107 | | Allegron 10mg tablets - Sigma Pharmaceuticals Plc |
| 2391711000001107 | | Allegron 10mg tablets 100 tablet - King Pharmaceuticals Ltd |
| 16136711000001100 | | Allegron 10mg tablets 100 tablet - King Frial maceuticals Eta |
| 16259111000001105 | | Allegron 10mg tablets 100 tablet - Lexon (OK) Eta Allegron 10mg tablets 100 tablet - Mawdsley-Brooks & Company Ltd |
| 17532411000001100 | | Allegron 10mg tablets 100 tablet - Mawdsley-Brooks & Company Ltd Allegron 10mg tablets 100 tablet - Sigma Pharmaceuticals Plc |
| 18544911000001108 | | Allegron 25mg tablets - DE Pharmaceuticals |
| 629711000001106 | | Allegron 25mg tablets - Be Pharmaceuticals Allegron 25mg tablets - King Pharmaceuticals Ltd |
| 16136811000001108 | | Allegron 25mg tablets - King Pharmaceuticals Ltu Allegron 25mg tablets - Lexon (UK) Ltd |
| 16259211000001104 | | Allegron 25mg tablets - Lexon (OK) Ltd Allegron 25mg tablets - Mawdsley-Brooks & Company Ltd |
| 17579111000001104 | | Allegron 25mg tablets - Necessity Supplies Ltd |
| 14053811000001100 | | Allegron 25mg tablets - Necessity Supplies Ltu Allegron 25mg tablets - Sigma Pharmaceuticals Plc |
| 18545011000001108 | | Allegron 25mg tablets 100 tablet - DE Pharmaceuticals |
| 2392811000001107 | | Allegron 25mg tablets 100 tablet - BE Frialmaceuticals Allegron 25mg tablets 100 tablet - King Pharmaceuticals Ltd |
| 16136911000001107 | | Allegron 25mg tablets 100 tablet - King Pharmaceuticals Ltd Allegron 25mg tablets 100 tablet - Lexon (UK) Ltd |
| 16259311000001107 | | Allegron 25mg tablets 100 tablet - Lexon (Ox) Ltd Allegron 25mg tablets 100 tablet - Mawdsley-Brooks & Company Ltd |
| 17579611000001107 | | Allegron 25mg tablets 100 tablet - Mawasiey-Brooks & Company Ltd Allegron 25mg tablets 100 tablet - Necessity Supplies Ltd |
| | | Allegron 25mg tablets 100 tablet - Necessity Supplies Ltd Allegron 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc |
| 17532511000001101 | | Allegion zoing tablets for tablet - Sigma Marmaceuticals Mc |

| 14053911000001105 | Allegron 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc |
|---|---|
| 11711211000001100 | Amitriptyline 1.25mg/5ml oral solution |
| 11682311000001109 | Amitriptyline 1.25mg/5ml oral solution - Special Order |
| 11682211000001101 | Amitriptyline 1.25mg/5ml oral solution 1 ml |
| 11682411000001102 | Amitriptyline 1.25mg/5ml oral solution 1 ml - Special Order |
| 11711311000001108 | Amitriptyline 100mg/5ml oral solution |
| 11682611000001104 | Amitriptyline 100mg/5ml oral solution - Special Order |
| 11682511000001103 | Amitriptyline 100mg/5ml oral solution 1 ml |
| 11682711000001108 | Amitriptyline 100mg/5ml oral solution 1 ml - Special Order |
| 310911000001104 | Amitriptyline 10mg tablets - A A H Pharmaceuticals Ltd |
| 18457211000001101 | Amitriptyline 10mg tablets - Accord Healthcare Ltd |
| 179011000001109 | Amitriptyline 10mg tablets - Actord Healthcare (Distribution) Ltd |
| 9784511000001105 | Amitriptyline 10mg tablets - Almus Pharmaceuticals Ltd |
| 20438711000001109 | Amitriptyline 10mg tablets - Arrow Generics Ltd |
| 36612511000001100 | Amitriptyline 10mg tablets - Arrow deficits Ltd Amitriptyline 10mg tablets - Bristol Laboratories Ltd |
| 22589711000001107 | Amitriptyline 10mg tablets - DE Pharmaceuticals |
| 13109811000001104 | Amitriptyline 10mg tablets - Develhurst Ltd |
| 34103511000001104 | Amitriptyline 10mg tablets - Dowelliurst Ltd Amitriptyline 10mg tablets - Genesis Pharmaceuticals Ltd |
| 105411000001106 | Amitriptyline 10mg tablets - Genesis Friannaceuticals Ltd Amitriptyline 10mg tablets - IVAX Pharmaceuticals UK Ltd |
| 47511000001100 | |
| | Amitriptyline 10mg tablets - Kent Pharmaceuticals Ltd |
| 29991511000001104 | Amitriptyline 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 38784611000001108 | Amitriptyline 10mg tablets - Medihealth (Northern) Ltd |
| 34966211000001108 | Amitriptyline 10mg tablets - NorthStar Healthcare Unlimited Company |
| 17778011000001106 | Amitriptyline 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 29763811000001106 | Amitriptyline 10mg tablets - Sigma Pharmaceuticals Plc |
| 865611000001103 | Amitriptyline 10mg tablets - Teva UK Ltd |
| 21762711000001103 | Amitriptyline 10mg tablets - Waymade Healthcare Plc |
| 13059111000001107 | Amitriptyline 10mg tablets - Wockhardt UK Ltd |
| 1420111000001102 | Amitriptyline 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 18457311000001109 | Amitriptyline 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 1420411000001107 | Amitriptyline 10mg tablets 28 tablet - Actavis UK Ltd |
| 1421611000001100 | Amitriptyline 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 9784611000001109 | Amitriptyline 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 20438811000001101 | Amitriptyline 10mg tablets 28 tablet - Arrow Generics Ltd |
| 36612611000001101 | Amitriptyline 10mg tablets 28 tablet - Bristol Laboratories Ltd |
| 22589811000001104 | Amitriptyline 10mg tablets 28 tablet - DE Pharmaceuticals |
| 13109911000001109 | Amitriptyline 10mg tablets 28 tablet - Dowelhurst Ltd |
| 34103611000001101 | Amitriptyline 10mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 1421911000001106 | Amitriptyline 10mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1421211000001102 | Amitriptyline 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 29991611000001100 | Amitriptyline 10mg tablets 28 tablet - Mawdsley-Brooks & Company<br>Ltd |
| 38784711000001104 | Amitriptyline 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 34966311000001100 | Amitriptyline 10mg tablets 28 tablet - NorthStar Healthcare Unlimited Company |
| 17778311000001109 | Amitriptyline 10mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 29763911000001101 | Amitriptyline 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1420711000001101 | Amitriptyline 10mg tablets 28 tablet - Teva UK Ltd |
| 21762911000001101 | Amitriptyline 10mg tablets 28 tablet - Waymade Healthcare Plc |

| 13059211000001101 | Amitriptyline 10mg tablets 28 tablet - Wockhardt UK Ltd |
|---|---|
| 13892411000001104 | Amitriptyline 10mg/5ml oral solution |
| 13879011000001108 | Amitriptyline 10mg/5ml oral solution - Special Order |
| 13878911000001104 | Amitriptyline 10mg/5ml oral solution 1 ml |
| 13879911000001107 | Amitriptyline 10mg/5ml oral solution 1 ml - Special Order |
| 19593711000001107 | Amitriptyline 10mg/5ml oral solution 150 ml |
| 19593811000001106 | Amitriptyline 10mg/5ml oral solution 150 ml - Special Order |
| 29686711000001103 | Amitriptyline 10mg/5ml oral solution sugar free |
| | Amitriptyline 10mg/5ml oral solution sugar free - A A H |
| 30125611000001108 | Pharmaceuticals Ltd |
| 30800511000001103 | Amitriptyline 10mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 37105611000001109 | Amitriptyline 10mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 38783611000001105 | Amitriptyline 10mg/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 32871411000001108 | Amitriptyline 10mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc |
| 29496211000001107 | Amitriptyline 10mg/5ml oral solution sugar free - Thame Laboratories Ltd |
| 29681411000001103 | Amitriptyline 10mg/5ml oral solution sugar free - Wockhardt UK Ltd |
| 29495711000001108 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml |
| 30125711000001104 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 268711000001108 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 30800611000001104 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 37105711000001100 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals |
| 38783911000001104 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - Medihealth (Northern) Ltd |
| 32871611000001106 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - Sigma Pharmaceuticals Plc |
| 29497511000001107 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - Thame Laboratories Ltd |
| 29681811000001101 | Amitriptyline 10mg/5ml oral solution sugar free 150 ml - Wockhardt UK Ltd |
| 8277811000001102 | Amitriptyline 10mg/5ml oral suspension |
| 8242611000001100 | Amitriptyline 10mg/5ml oral suspension - Special Order |
| 8242311000001105 | Amitriptyline 10mg/5ml oral suspension 1 ml |
| 8242811000001101 | Amitriptyline 10mg/5ml oral suspension 1 ml - Special Order |
| 19593911000001101 | Amitriptyline 10mg/5ml oral suspension 100 ml |
| 19594011000001103 | Amitriptyline 10mg/5ml oral suspension 100 ml - Special Order |
| 11711411000001101 | Amitriptyline 150mg/5ml oral solution |
| 11682911000001105 | Amitriptyline 150mg/5ml oral solution - Special Order |
| 11682811000001100 | Amitriptyline 150mg/5ml oral solution 1 ml |
| 11683011000001102 | Amitriptyline 150mg/5ml oral solution 1 ml - Special Order |
| 11711511000001102 | Amitriptyline 15mg/5ml oral solution |
| 11683211000001107 | Amitriptyline 15mg/5ml oral solution - Special Order |
| 11683111000001101 | Amitriptyline 15mg/5ml oral solution 1 ml |
| 11683311000001104 | Amitriptyline 15mg/5ml oral solution 1 ml - Special Order |
| 11711611000001103 | Amitriptyline 2.5mg/5ml oral solution |
| 11683511000001105 | Amitriptyline 2.5mg/5ml oral solution - Special Order |
| 11683411000001106 | Amitriptyline 2.5mg/5ml oral solution 1 ml |
| | 1 / 0/1 11 11 11 |

| 11683611000001109 | Amitriptyline 2.5mg/5ml oral solution 1 ml - Special Order |
|---|---|
| 190511000001102 | Amitriptyline 25mg tablets - A A H Pharmaceuticals Ltd |
| 18457411000001102 | Amitriptyline 25mg tablets - Accord Healthcare Ltd |
| 78811000001102 | Amitriptyline 25mg tablets - Actavis UK Ltd |
| 735211000001108 | Amitriptyline 25mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9784711000001100 | Amitriptyline 25mg tablets - Almus Pharmaceuticals Ltd |
| 20438911000001106 | Amitriptyline 25mg tablets - Arrow Generics Ltd |
| 36613511000001107 | Amitriptyline 25mg tablets - Bristol Laboratories Ltd |
| 28978311000001109 | Amitriptyline 25mg tablets - Crescent Pharma Ltd |
| 22589911000001109 | Amitriptyline 25mg tablets - DE Pharmaceuticals |
| 13110011000001104 | Amitriptyline 25mg tablets - Dowelhurst Ltd |
| 34103711000001105 | Amitriptyline 25mg tablets - Genesis Pharmaceuticals Ltd |
| 788611000001109 | Amitriptyline 25mg tablets - IVAX Pharmaceuticals UK Ltd |
| 440811000001107 | Amitriptyline 25mg tablets - Kent Pharmaceuticals Ltd |
| 29991711000001109 | Amitriptyline 25mg tablets - Mawdsley-Brooks & Company Ltd |
| 38784011000001101 | Amitriptyline 25mg tablets - Medihealth (Northern) Ltd |
| 34966411000001107 | Amitriptyline 25mg tablets - NorthStar Healthcare Unlimited Company |
| 17778711000001108 | Amitriptyline 25mg tablets - Phoenix Healthcare Distribution Ltd |
| 666511000001101 | Amitriptyline 25mg tablets - Ranbaxy (UK) Ltd |
| 5162711000001107 | Amitriptyline 25mg tablets - Sandoz Ltd |
| 15051511000001109 | Amitriptyline 25mg tablets - Sigma Pharmaceuticals Plc |
| 40611000001100 | Amitriptyline 25mg tablets - Teva UK Ltd |
| 21763111000001105 | Amitriptyline 25mg tablets - Waymade Healthcare Plc |
| 11176611000001109 | Amitriptyline 25mg tablets - Wockhardt UK Ltd |
| 1422511000001107 | Amitriptyline 25mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 18457511000001103 | Amitriptyline 25mg tablets 28 tablet - Accord Healthcare Ltd |
| 1422811000001105 | Amitriptyline 25mg tablets 28 tablet - Actavis UK Ltd |
| | Amitriptyline 25mg tablets 28 tablet - Alliance Healthcare |
| 1423111000001109 | (Distribution) Ltd |
| 9784811000001108 | Amitriptyline 25mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 20439011000001102 | Amitriptyline 25mg tablets 28 tablet - Arrow Generics Ltd |
| 36613611000001106 | Amitriptyline 25mg tablets 28 tablet - Bristol Laboratories Ltd |
| 28978411000001102 | Amitriptyline 25mg tablets 28 tablet - Crescent Pharma Ltd |
| 22590011000001101 | Amitriptyline 25mg tablets 28 tablet - DE Pharmaceuticals |
| 13110111000001103 | Amitriptyline 25mg tablets 28 tablet - Dowelhurst Ltd |
| 34103811000001102 | Amitriptyline 25mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 1423311000001106 | Amitriptyline 25mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1423011000001108 | Amitriptyline 25mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 29991811000001101 | Amitriptyline 25mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38784111000001100 | Amitriptyline 25mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 34966511000001106 | Amitriptyline 25mg tablets 28 tablet - NorthStar Healthcare Unlimited Company |
| 17778811000001100 | Amitriptyline 25mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 5162811000001104 | Amitriptyline 25mg tablets 28 tablet - Sandoz Ltd |
| 15051711000001104 | Amitriptyline 25mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1422911000001100 | Amitriptyline 25mg tablets 28 tablet - Teva UK Ltd |
| 21768011000001102 | Amitriptyline 25mg tablets 28 tablet - Waymade Healthcare Plc |
| 11176711000001100 | Amitriptyline 25mg tablets 28 tablet - Wockhardt UK Ltd |
| 1422411000001108 | Amitriptyline 25mg tablets 500 tablet - A A H Pharmaceuticals Ltd |

| 1423211000001103 | Amitriptyline 25mg tablets 500 tablet - Ranbaxy (UK) Ltd |
|---|---|
| 35901411000001107 | Amitriptyline 25mg/5ml oral solution sugar free |
| 321761009 | Amitriptyline 25mg/5ml oral solution sugar free |
| | Amitriptyline 25mg/5ml oral solution sugar free - A A H |
| 375811000001108 | Pharmaceuticals Ltd |
| 28379211000001103 | Amitriptyline 25mg/5ml oral solution sugar free - Accord Healthcare Ltd |
| 111111000001101 | Amitriptyline 25mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 22589511000001102 | Amitriptyline 25mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 13109111000001106 | Amitriptyline 25mg/5ml oral solution sugar free - Dowelhurst Ltd |
| 323711000001100 | Amitriptyline 25mg/5ml oral solution sugar free - Kent Pharmaceuticals Ltd |
| 38783111000001102 | Amitriptyline 25mg/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 75911000001101 | Amitriptyline 25mg/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd |
| 29763411000001109 | Amitriptyline 25mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc |
| 29500111000001108 | Amitriptyline 25mg/5ml oral solution sugar free - Thame Laboratories Ltd |
| 21762111000001104 | Amitriptyline 25mg/5ml oral solution sugar free - Waymade Healthcare Plc |
| 18148011000001106 | Amitriptyline 25mg/5ml oral solution sugar free - Wockhardt UK Ltd |
| 1021411000001108 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml |
| 2208711000001105 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 28379311000001106 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd |
| 2209611000001105 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 22589611000001103 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals |
| 13109311000001108 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Dowelhurst Ltd |
| 2209011000001103 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Kent Pharmaceuticals Ltd |
| 38783211000001108 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Medihealth (Northern) Ltd |
| 2209311000001100 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Rosemont Pharmaceuticals Ltd |
| 29763511000001108 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Sigma Pharmaceuticals Plc |
| 29500411000001103 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Thame Laboratories Ltd |
| 21762311000001102 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Waymade Healthcare Plc |
| 18148311000001109 | Amitriptyline 25mg/5ml oral solution sugar free 150 ml - Wockhardt UK Ltd |
| 33678311000001108 | Amitriptyline 25mg/5ml oral suspension |
| 33670911000001107 | Amitriptyline 25mg/5ml oral suspension - Special Order |
| 33670811000001102 | Amitriptyline 25mg/5ml oral suspension 1 ml |
| 33671011000001104 | Amitriptyline 25mg/5ml oral suspension 1 ml - Special Order |
| 35901511000001106 | Amitriptyline 50mg modified-release capsules |
| 321765000 | Amitriptyline 50mg modified-release capsules |
| 4533111000001107 | Amitriptyline 50mg modified-release capsules 56 capsule |
| 321747004 | Amitriptyline 50mg tablets |

| 771511000001106 | Amitriptyline 50mg tablets - A A H Pharmaceuticals Ltd |
|---|---|
| 743811000001109 | Amitriptyline 50mg tablets - Accord Healthcare Ltd |
| 698011000001106 | Amitriptyline 50mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9784911000001103 | Amitriptyline 50mg tablets - Almus Pharmaceuticals Ltd |
| 20439111000001101 | Amitriptyline 50mg tablets - Arrow Generics Ltd |
| 36613711000001102 | Amitriptyline 50mg tablets - Bristol Laboratories Ltd |
| 22590111000001100 | Amitriptyline 50mg tablets - DE Pharmaceuticals |
| 13110411000001108 | Amitriptyline 50mg tablets - Dowelhurst Ltd |
| 778911000001108 | Amitriptyline 50mg tablets - IVAX Pharmaceuticals UK Ltd |
| 55411000001107 | Amitriptyline 50mg tablets - Kent Pharmaceuticals Ltd |
| 29991911000001106 | Amitriptyline 50mg tablets - Mawdsley-Brooks & Company Ltd |
| 38784211000001106 | Amitriptyline 50mg tablets - Medihealth (Northern) Ltd |
| 34966611000001105 | Amitriptyline 50mg tablets - NorthStar Healthcare Unlimited Company |
| 17778911000001105 | Amitriptyline 50mg tablets - Phoenix Healthcare Distribution Ltd |
| 29764011000001103 | Amitriptyline 50mg tablets - Sigma Pharmaceuticals Plc |
| 540811000001101 | Amitriptyline 50mg tablets - Teva UK Ltd |
| 21763411000001100 | Amitriptyline 50mg tablets - Waymade Healthcare Plc |
| 11176811000001108 | Amitriptyline 50mg tablets - Wockhardt UK Ltd |
| 1262111000001109 | Amitriptyline 50mg tablets 28 tablet |
| 1426711000001103 | Amitriptyline 50mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1426811000001106 | Amitriptyline 50mg tablets 28 tablet - Accord Healthcare Ltd |
| 1427111000001101 | Amitriptyline 50mg tablets 28 tablet - Alliance Healthcare |
| 1427111000001101 | (Distribution) Ltd |
| 9785011000001103 | Amitriptyline 50mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 20439211000001107 | Amitriptyline 50mg tablets 28 tablet - Arrow Generics Ltd |
| 36613811000001105 | Amitriptyline 50mg tablets 28 tablet - Bristol Laboratories Ltd |
| 22590211000001106 | Amitriptyline 50mg tablets 28 tablet - DE Pharmaceuticals |
| 13110611000001106 | Amitriptyline 50mg tablets 28 tablet - Dowelhurst Ltd |
| 1427211000001107 | Amitriptyline 50mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1427011000001102 | Amitriptyline 50mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 29992011000001104 | Amitriptyline 50mg tablets 28 tablet - Mawdsley-Brooks & Company<br>Ltd |
| 38784311000001103 | Amitriptyline 50mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 34966711000001101 | Amitriptyline 50mg tablets 28 tablet - NorthStar Healthcare Unlimited Company |
| 17779011000001101 | Amitriptyline 50mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 29764111000001102 | Amitriptyline 50mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1426911000001101 | Amitriptyline 50mg tablets 28 tablet - Teva UK Ltd |
| 21763611000001102 | Amitriptyline 50mg tablets 28 tablet - Waymade Healthcare Plc |
| 11176911000001103 | Amitriptyline 50mg tablets 28 tablet - Wockhardt UK Ltd |
| 35901611000001105 | Amitriptyline 50mg/5ml oral solution sugar free |
| 321762002 | Amitriptyline 50mg/5ml oral solution sugar free |
| 686711000001108 | Amitriptyline 50mg/5ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 28379411000001104 | Amitriptyline 50mg/5ml oral solution sugar free - Accord Healthcare<br>Ltd |
| 895511000001104 | Amitriptyline 50mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 22589311000001108 | Amitriptyline 50mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 13109611000001103 | Amitriptyline 50mg/5ml oral solution sugar free - Dowelhurst Ltd |

| Amitriptyline 50mg/5ml oral solution sugar free - Medihealth (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free - Phoenix Healthon Distribution Ltd 563711000001107 Amitriptyline 50mg/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd 29763611000001107 Amitriptyline 50mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc Amitriptyline 50mg/5ml oral solution sugar free - Thame Laborator Ltd 21762411000001109 Amitriptyline 50mg/5ml oral solution sugar free - Waymade Healthcare Plc 18146311000001105 Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Ltd 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | ies<br>d |
|---|---|
| Distribution Ltd Amitriptyline 50mg/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc 29501411000001107 Amitriptyline 50mg/5ml oral solution sugar free - Thame Laborator Ltd 21762411000001109 Amitriptyline 50mg/5ml oral solution sugar free - Waymade Healthcare Plc 18146311000001105 Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Ltd 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml 2211211000001105 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd 28379511000001100 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A Ccord Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd 22589411000001101 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals 13109711000001107 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | ies<br>d |
| Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc Amitriptyline 50mg/5ml oral solution sugar free - Thame Laborator Ltd Amitriptyline 50mg/5ml oral solution sugar free - Thame Laborator Ltd Amitriptyline 50mg/5ml oral solution sugar free - Waymade Healthcare Plc Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Lt 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A Ccord Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | d |
| Pharmaceuticals Pic Amitriptyline 50mg/5ml oral solution sugar free - Thame Laborator Ltd Amitriptyline 50mg/5ml oral solution sugar free - Waymade Healthcare Pic Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Lt 1221411000001105 Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Lt 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd 28379511000001100 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhus Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | d |
| 21762411000001107 Ltd Amitriptyline 50mg/5ml oral solution sugar free - Waymade Healthcare Plc 18146311000001105 Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Lt 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd 28379511000001100 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd 2212011000001108 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals 13109711000001107 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | d |
| Healthcare Plc Amitriptyline 50mg/5ml oral solution sugar free - Wockhardt UK Lt 1221411000001104 | st |
| 1221411000001104 Amitriptyline 50mg/5ml oral solution sugar free 150 ml 2211211000001105 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd 28379511000001100 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd 2212011000001108 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd 22589411000001101 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals 13109711000001107 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhus Ltd 38784511000001109 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | st |
| Amitriptyline 50mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhultd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| Pharmaceuticals Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd 2212011000001108 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - De Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhus Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| 2212011000001100 Healthcare Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| 22589411000001101 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhu Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| 22589411000001101 Pharmaceuticals 13109711000001107 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Dowelhul Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| 13109711000001107 Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Mediheal (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| (Northern) Ltd Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | th |
| Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Phoenix | |
| Healthcare Distribution Ltd | |
| 2211511000001108 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Rosemon Pharmaceuticals Ltd | |
| 29763711000001103 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Sigma Pharmaceuticals Plc | |
| 29502511000001103 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Thame Laboratories Ltd | |
| 21762611000001107 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Waymada Healthcare Plc | |
| 18146411000001103 Amitriptyline 50mg/5ml oral solution sugar free 150 ml - Wockhard UK Ltd | it |
| 8277911000001107 Amitriptyline 5mg/5ml oral solution | |
| 8241611000001106 Amitriptyline 5mg/5ml oral solution - Special Order | |
| 8241511000001107 Amitriptyline 5mg/5ml oral solution 1 ml | |
| 8241911000001100 Amitriptyline 5mg/5ml oral solution 1 ml - Special Order | |
| 8278011000001109 Amitriptyline 5mg/5ml oral suspension | |
| 8242711000001109 Amitriptyline 5mg/5ml oral suspension - Special Order | |
| 8242511000001104 Amitriptyline 5mg/5ml oral suspension 1 ml | |
| 8242911000001106 Amitriptyline 5mg/5ml oral suspension 1 ml - Special Order | |
| 11711711000001107 Amitriptyline 75mg/5ml oral solution | |
| 11683811000001108 Amitriptyline 75mg/5ml oral solution - Special Order | |
| 11683711000001100 Amitriptyline 75mg/5ml oral solution 1 ml | |
| 11684011000001100 Amitriptyline 75mg/5ml oral solution 1 ml - Special Order | |
| 11711811000001104 Amitriptyline 80mg/5ml oral solution | |
| 11684511000001108 Amitriptyline 80mg/5ml oral solution - Special Order | |
| 11684311000001102 Amitriptyline 80mg/5ml oral solution 1 ml | |
| 11684611000001107 Amitriptyline 80mg/5ml oral solution 1 ml - Special Order | |
| 39731711000001107 Amitriptyline 10mg / Perphenazine 2mg tablets | |
| 991011000001104 Amitriptyline 10mg / Perphenazine 2mg tablets 100 tablet | |

| 39731811000001104 | Amitriptyline 25mg / Perphenazine 2mg tablets |
|---|---|
| 1000111000001101 | Amitriptyline 25mg / Perphenazine 2mg tablets 100 tablet |
| 321894004 | Amoxapine 100mg tablets |
| 32248411000001107 | Amoxapine 100mg tablets - Special Order |
| 32248311000001100 | Amoxapine 100mg tablets 1 tablet |
| 32248511000001106 | Amoxapine 100mg tablets 1 tablet - Special Order |
| 28785311000001100 | Amoxapine 100mg tablets 30 tablet |
| 3934111000001101 | Amoxapine 100mg tablets 56 tablet |
| 321893005 | Amoxapine 50mg tablets |
| 3798511000001102 | Amoxapine 50mg tablets 84 tablet |
| 701211000001104 | Anafranil 10mg capsules - Novartis Pharmaceuticals UK Ltd |
| 1555511000001106 | Anafranil 10mg capsules 84 capsule - Novartis Pharmaceuticals UK Ltd |
| 647111000001102 | Anafranil 25mg capsules - Novartis Pharmaceuticals UK Ltd |
| 1557811000001104 | Anafranil 25mg capsules 84 capsule - Novartis Pharmaceuticals UK Ltd |
| 4551211000001104 | Anafranil 25mg/2ml solution for injection ampoules - Novartis<br>Pharmaceuticals UK Ltd |
| 4551311000001107 | Anafranil 25mg/2ml solution for injection ampoules 10 ampoule - Novartis Pharmaceuticals UK Ltd |
| 4534911000001107 | Anafranil 25mg/5ml syrup - Novartis Pharmaceuticals UK Ltd |
| 4535011000001107 | Anafranil 25mg/5ml syrup 150 ml - Novartis Pharmaceuticals UK Ltd |
| 5511000001101 | Anafranil 50mg capsules - Novartis Pharmaceuticals UK Ltd |
| 1560711000001103 | Anafranil 50mg capsules 56 capsule - Novartis Pharmaceuticals UK Ltd |
| 13828111000001103 | Anafranil SR 75mg tablets - DE Pharmaceuticals |
| 5615711000001101 | Anafranil SR 75mg tablets - Dowelhurst Ltd |
| 16138211000001108 | Anafranil SR 75mg tablets - Lexon (UK) Ltd |
| 16262311000001107 | Anafranil SR 75mg tablets - Mawdsley-Brooks & Company Ltd |
| 17584911000001106 | Anafranil SR 75mg tablets - Necessity Supplies Ltd |
| 119411000001107 | Anafranil SR 75mg tablets - Novartis Pharmaceuticals UK Ltd |
| 14193311000001106 | Anafranil SR 75mg tablets - Sigma Pharmaceuticals Plc |
| 16540611000001101 | Anafranil SR 75mg tablets - Stephar (U.K.) Ltd |
| 5333911000001100 | Anafranil SR 75mg tablets - Waymade Healthcare Plc |
| 5615911000001104 | Anafranil SR 75mg tablets 20 tablet - Dowelhurst Ltd |
| 16138311000001100 | Anafranil SR 75mg tablets 20 tablet - Lexon (UK) Ltd |
| 18522411000001109 | Anafranil SR 75mg tablets 20 tablet - Mawdsley-Brooks & Company Ltd |
| 17585011000001106 | Anafranil SR 75mg tablets 20 tablet - Necessity Supplies Ltd |
| 14193411000001104 | Anafranil SR 75mg tablets 20 tablet - Sigma Pharmaceuticals Plc |
| 16540811000001102 | Anafranil SR 75mg tablets 20 tablet - Stephar (U.K.) Ltd |
| 13618511000001106 | Anafranil SR 75mg tablets 20 tablet - Waymade Healthcare Plc |
| 13828211000001109 | Anafranil SR 75mg tablets 28 tablet - DE Pharmaceuticals |
| 5616011000001107 | Anafranil SR 75mg tablets 28 tablet - Dowelhurst Ltd |
| 16138411000001107 | Anafranil SR 75mg tablets 28 tablet - Lexon (UK) Ltd |
| 16262511000001101 | Anafranil SR 75mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 17585411000001102 | Anafranil SR 75mg tablets 28 tablet - Necessity Supplies Ltd |
| 2228711000001101 | Anafranil SR 75mg tablets 28 tablet - Novartis Pharmaceuticals UK Ltd |
| 19691811000001101 | Anafranil SR 75mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 5334011000001102 | Anafranil SR 75mg tablets 28 tablet - Waymade Healthcare Plc |
| 5616211000001102 | Anafranil SR 75mg tablets 30 tablet - Dowelhurst Ltd |
| 3934511000001105 | Asendis 100mg tablets - Mercury Pharma Group Ltd |
| 3934711000001100 | Asendis 100mg tablets 56 tablet - Mercury Pharma Group Ltd |
| 3798611000001103 | Asendis 50mg tablets - Mercury Pharma Group Ltd |

| 3798711000001107 | Asendis 50mg tablets 84 tablet - Mercury Pharma Group Ltd |
|---|---|
| 321785001 | Clomipramine 10mg capsules |
| 730311000001107 | Clomipramine 10mg capsules - A A H Pharmaceuticals Ltd |
| 244311000001107 | Clomipramine 10mg capsules - Actavis UK Ltd |
| 543911000001103 | Clomipramine 10mg capsules - Alliance Healthcare (Distribution) Ltd |
| 17965811000001107 | Clomipramine 10mg capsules - Almus Pharmaceuticals Ltd |
| 23821811000001103 | Clomipramine 10mg capsules - DE Pharmaceuticals |
| 13227611000001100 | Clomipramine 10mg capsules - Dowelhurst Ltd |
| 312211000001109 | Clomipramine 10mg capsules - IVAX Pharmaceuticals UK Ltd |
| 643411000001100 | Clomipramine 10mg capsules - Kent Pharmaceuticals Ltd |
| 30014711000001101 | Clomipramine 10mg capsules - Mawdsley-Brooks & Company Ltd |
| 38844211000001103 | Clomipramine 10mg capsules - Medihealth (Northern) Ltd |
| 286811000001103 | Clomipramine 10mg capsules - Mylan |
| 17860411000001105 | Clomipramine 10mg capsules - Phoenix Healthcare Distribution Ltd |
| 29789911000001100 | Clomipramine 10mg capsules - Sigma Pharmaceuticals Plc |
| 16411000001107 | Clomipramine 10mg capsules - Teva UK Ltd |
| 21859211000001108 | Clomipramine 10mg capsules - Waymade Healthcare Plc |
| 1020511000001100 | Clomipramine 10mg capsules 100 capsule |
| 1554211000001107 | Clomipramine 10mg capsules 100 capsule - A A H Pharmaceuticals Ltd |
| 1554811000001108 | Clomipramine 10mg capsules 100 capsule - Mylan |
| 964111000001102 | Clomipramine 10mg capsules 28 capsule |
| 1554111000001101 | Clomipramine 10mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 1554411000001106 | Clomipramine 10mg capsules 28 capsule - Actavis UK Ltd |
| 1555611000001105 | Clomipramine 10mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 17965911000001102 | Clomipramine 10mg capsules 28 capsule - Almus Pharmaceuticals Ltd |
| 23822011000001101 | Clomipramine 10mg capsules 28 capsule - DE Pharmaceuticals |
| 13227811000001101 | Clomipramine 10mg capsules 28 capsule - Dowelhurst Ltd |
| 1555011000001103 | Clomipramine 10mg capsules 28 capsule - IVAX Pharmaceuticals UK Ltd |
| 1555211000001108 | Clomipramine 10mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 30014811000001109 | Clomipramine 10mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 38844311000001106 | Clomipramine 10mg capsules 28 capsule - Medihealth (Northern) Ltd |
| 1554711000001100 | Clomipramine 10mg capsules 28 capsule - Mylan |
| 17860511000001109 | Clomipramine 10mg capsules 28 capsule - Phoenix Healthcare Distribution Ltd |
| 29790011000001108 | Clomipramine 10mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 1554611000001109 | Clomipramine 10mg capsules 28 capsule - Teva UK Ltd |
| 21859311000001100 | Clomipramine 10mg capsules 28 capsule - Waymade Healthcare Plc |
| 983311000001104 | Clomipramine 10mg capsules 84 capsule |
| 12025411000001106 | Clomipramine 10mg/5ml oral solution |
| 11958511000001106 | Clomipramine 10mg/5ml oral solution - Special Order |
| 11958411000001107 | Clomipramine 10mg/5ml oral solution 1 ml |
| 11958611000001105 | Clomipramine 10mg/5ml oral solution 1 ml - Special Order |
| 12025611000001109 | Clomipramine 10mg/5ml oral suspension |
| 11958211000001108 | Clomipramine 10mg/5ml oral suspension - Special Order |
| 11958111000001102 | Clomipramine 10mg/5ml oral suspension 1 ml |
| 11958311000001100 | Clomipramine 10mg/5ml oral suspension 1 ml - Special Order |
| 36977811000001108 | Clomipramine 250mg/5ml oral suspension |
| 36959611000001101 | Clomipramine 250mg/5ml oral suspension - Special Order |

| 36959511000001100 | Clomipramine 250mg/5ml oral suspension 1 ml |
|---|---|
| 36961711000001103 | Clomipramine 250mg/5ml oral suspension 1 ml - Special Order |
| 321786000 | Clomipramine 25mg capsules |
| 235711000001109 | Clomipramine 25mg capsules - A A H Pharmaceuticals Ltd |
| 890811000001107 | Clomipramine 25mg capsules - Actavis UK Ltd |
| 537611000001102 | Clomipramine 25mg capsules - Alliance Healthcare (Distribution) Ltd |
| 17966011000001105 | Clomipramine 25mg capsules - Almus Pharmaceuticals Ltd |
| 23823111000001106 | Clomipramine 25mg capsules - DE Pharmaceuticals |
| 13228111000001109 | Clomipramine 25mg capsules - Dowelhurst Ltd |
| 299811000001105 | Clomipramine 25mg capsules - IVAX Pharmaceuticals UK Ltd |
| 364511000001101 | Clomipramine 25mg capsules - Kent Pharmaceuticals Ltd |
| 30014911000001104 | Clomipramine 25mg capsules - Mawdsley-Brooks & Company Ltd |
| 38844411000001104 | Clomipramine 25mg capsules - Medihealth (Northern) Ltd |
| 68511000001106 | Clomipramine 25mg capsules - Mylan |
| 17860611000001108 | Clomipramine 25mg capsules - Phoenix Healthcare Distribution Ltd |
| 29790111000001109 | Clomipramine 25mg capsules - Sigma Pharmaceuticals Plc |
| 149111000001109 | Clomipramine 25mg capsules - Teva UK Ltd |
| 21859411000001107 | Clomipramine 25mg capsules - Teva OK Etu Clomipramine 25mg capsules - Waymade Healthcare Plc |
| 1289611000001105 | Clomipramine 25mg capsules 100 capsule |
| 1556711000001109 | Clomipramine 25mg capsules 100 capsule - A A H Pharmaceuticals Ltd Clomipramine 25mg capsules 100 capsule - Alliance Healthcare |
| 1558411000001102 | (Distribution) Ltd |
| 13228611000001101 | Clomipramine 25mg capsules 100 capsule - Dowelhurst Ltd |
| 1598011000001100 | Clomipramine 25mg capsules 100 capsule - Kent Pharmaceuticals Ltd |
| 1557211000001100 | Clomipramine 25mg capsules 100 capsule - Mylan |
| 1030211000001101 | Clomipramine 25mg capsules 28 capsule |
| 1556611000001100 | Clomipramine 25mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 1556811000001101 | Clomipramine 25mg capsules 28 capsule - Actavis UK Ltd |
| 1558211000001101 | Clomipramine 25mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 17966111000001106 | Clomipramine 25mg capsules 28 capsule - Almus Pharmaceuticals Ltd |
| 23824211000001102 | Clomipramine 25mg capsules 28 capsule - DE Pharmaceuticals |
| 13228211000001103 | Clomipramine 25mg capsules 28 capsule - Dowelhurst Ltd |
| 1557411000001101 | Clomipramine 25mg capsules 28 capsule - IVAX Pharmaceuticals UK Ltd |
| 1557511000001102 | Clomipramine 25mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 30015011000001104 | Clomipramine 25mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 38844511000001100 | Clomipramine 25mg capsules 28 capsule - Medihealth (Northern) Ltd |
| 1557111000001106 | Clomipramine 25mg capsules 28 capsule - Mylan |
| 17860711000001104 | Clomipramine 25mg capsules 28 capsule - Phoenix Healthcare Distribution Ltd |
| 29790211000001103 | Clomipramine 25mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 1556911000001106 | Clomipramine 25mg capsules 28 capsule - Teva UK Ltd |
| 21859511000001106 | Clomipramine 25mg capsules 28 capsule - Waymade Healthcare Plc |
| 1219711000001103 | Clomipramine 25mg capsules 84 capsule |
| 321789007 | Clomipramine 25mg/2ml solution for injection ampoules |
| 36089011000001108 | Clomipramine 25mg/2ml solution for injection ampoules |
| 4551111000001105 | Clomipramine 25mg/2ml solution for injection ampoules 10 ampoule |
| 4557811000001105 | Clomipramine 25mg/5ml oral solution |
| 8372211000001108 | Clomipramine 25mg/5ml oral solution - Special Order |
| -5000001100 | Section Sectio |

| 8371911000001105 | Clomipramine 25mg/5ml oral solution 1 ml |
|---|---|
| 8372511000001106 | Clomipramine 25mg/5ml oral solution 1 ml - Special Order |
| 4534811000001102 | Clomipramine 25mg/5ml oral solution 150 ml |
| 8377211000001106 | Clomipramine 25mg/5ml oral suspension |
| 8371411000001100 | Clomipramine 25mg/5ml oral suspension - Special Order |
| 8371111000001107 | Clomipramine 25mg/5ml oral suspension 1 ml |
| 8371511000001107 | Clomipramine 25mg/5ml oral suspension 1 ml - Special Order |
| 8368311000001108 | |
| | Clomipramine 37.5mg/5ml oral solution |
| 8369011000001100 | Clomipramine 37.5mg/5ml oral solution - Special Order |
| 8365711000001100 | Clomipramine 37.5mg/5ml oral solution 1 ml |
| 8369311000001102 | Clomipramine 37.5mg/5ml oral solution 1 ml - Special Order |
| 8370111000001101 | Clomipramine 37.5mg/5ml oral suspension |
| 8369611000001107 | Clomipramine 37.5mg/5ml oral suspension - Special Order |
| 8369511000001108 | Clomipramine 37.5mg/5ml oral suspension 1 ml |
| 8369711000001103 | Clomipramine 37.5mg/5ml oral suspension 1 ml - Special Order |
| 321787009 | Clomipramine 50mg capsules |
| 636911000001101 | Clomipramine 50mg capsules - A A H Pharmaceuticals Ltd |
| 218611000001103 | Clomipramine 50mg capsules - Actavis UK Ltd |
| 769011000001109 | Clomipramine 50mg capsules - Alliance Healthcare (Distribution) Ltd |
| 17966211000001100 | Clomipramine 50mg capsules - Almus Pharmaceuticals Ltd |
| 23824711000001109 | Clomipramine 50mg capsules - DE Pharmaceuticals |
| 13229011000001103 | Clomipramine 50mg capsules - Dowelhurst Ltd |
| 404711000001100 | Clomipramine 50mg capsules - IVAX Pharmaceuticals UK Ltd |
| 920211000001105 | Clomipramine 50mg capsules - Kent Pharmaceuticals Ltd |
| 30015111000001103 | Clomipramine 50mg capsules - Mawdsley-Brooks & Company Ltd |
| 38844811000001102 | Clomipramine 50mg capsules - Medihealth (Northern) Ltd |
| 172911000001103 | Clomipramine 50mg capsules - Mylan |
| 17860811000001107 | Clomipramine 50mg capsules - Phoenix Healthcare Distribution Ltd |
| 29790311000001106 | Clomipramine 50mg capsules - Sigma Pharmaceuticals Plc |
| 627711000001103 | Clomipramine 50mg capsules - Teva UK Ltd |
| 21859711000001101 | Clomipramine 50mg capsules - Waymade Healthcare Plc |
| 953711000001108 | Clomipramine 50mg capsules 100 capsule |
| 1559011000001101 | Clomipramine 50mg capsules 100 capsule - A A H Pharmaceuticals Ltd |
| 3703011000001101 | Clomipramine 50mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 1560511000001108 | Clomipramine 50mg capsules 100 capsule - Kent Pharmaceuticals Ltd |
| 1559711000001104 | Clomipramine 50mg capsules 100 capsule - Mylan |
| 1313011000001108 | Clomipramine 50mg capsules 28 capsule |
| 1558911000001105 | Clomipramine 50mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 1559111000001100 | Clomipramine 50mg capsules 28 capsule - Actavis UK Ltd |
| 1560911000001101 | Clomipramine 50mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 17966311000001108 | Clomipramine 50mg capsules 28 capsule - Almus Pharmaceuticals Ltd |
| 23824911000001106 | Clomipramine 50mg capsules 28 capsule - DE Pharmaceuticals |
| 13229311000001100 | Clomipramine 50mg capsules 28 capsule - Dowelhurst Ltd |
| 1560211000001105 | Clomipramine 50mg capsules 28 capsule - IVAX Pharmaceuticals UK Ltd |
| 1560311000001102 | Clomipramine 50mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 30015211000001109 | Clomipramine 50mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 38844911000001107 | Clomipramine 50mg capsules 28 capsule - Medihealth (Northern) Ltd |
| | 1 |

| 1559611000001108 | Clomipramine 50mg capsules 28 capsule - Mylan |
|---|---|
| | Clomipramine 50mg capsules 28 capsule - Phoenix Healthcare |
| 17861011000001105 | Distribution Ltd |
| 29790411000001104 | Clomipramine 50mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 1559311000001103 | Clomipramine 50mg capsules 28 capsule - Teva UK Ltd |
| 21859811000001109 | Clomipramine 50mg capsules 28 capsule - Waymade Healthcare Plc |
| 1314711000001107 | Clomipramine 50mg capsules 56 capsule |
| 8377511000001109 | Clomipramine 50mg/5ml oral solution |
| 8370611000001109 | Clomipramine 50mg/5ml oral solution - Special Order |
| 8370511000001105 | Clomipramine 50mg/5ml oral solution 1 ml |
| 8370811000001108 | Clomipramine 50mg/5ml oral solution 1 ml - Special Order |
| 8377611000001108 | Clomipramine 50mg/5ml oral suspension |
| 8371311000001109 | Clomipramine 50mg/5ml oral suspension - Drug Tariff Special Order |
| 8370911000001103 | Clomipramine 50mg/5ml oral suspension 1 ml |
| 8371611000001104 | Clomipramine 50mg/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 30836011000001104 | Clomipramine 50mg/5ml oral suspension 100 ml |
| 30836111000001103 | Clomipramine 50mg/5ml oral suspension 100 ml - Drug Tariff Special Order |
| 8370211000001107 | Clomipramine 5mg/5ml oral solution |
| 8369211000001105 | Clomipramine 5mg/5ml oral solution - Special Order |
| 8369111000001104 | Clomipramine 5mg/5ml oral solution 1 ml |
| 8369411000001109 | Clomipramine 5mg/5ml oral solution 1 ml - Special Order |
| 8370311000001104 | Clomipramine 5mg/5ml oral suspension |
| 8370011000001102 | Clomipramine 5mg/5ml oral suspension - Special Order |
| 8369811000001106 | Clomipramine 5mg/5ml oral suspension 1 ml |
| 8370411000001106 | Clomipramine 5mg/5ml oral suspension 1 ml - Special Order |
| 321790003 | Clomipramine 75mg modified-release tablets |
| 36089111000001109 | Clomipramine 75mg modified-release tablets |
| 35992611000001101 | Clomipramine 75mg modified-release tablets - Special Order |
| 35992511000001100 | Clomipramine 75mg modified-release tablets 1 tablet |
| 35992711000001105 | Clomipramine 75mg modified-release tablets 1 tablet - Special Order |
| 5615311000001100 | Clomipramine 75mg modified-release tablets 20 tablet |
| 1171211000001100 | Clomipramine 75mg modified-release tablets 28 tablet |
| 5615511000001106 | Clomipramine 75mg modified-release tablets 30 tablet |
| 28802211000001104 | Defanyl 100mg tablets - Imported (France) |
| 28802311000001107 | Defanyl 100mg tablets 30 tablet - Imported (France) |
| 321805008 | Dosulepin 25mg capsules |
| 1228711000001100 | Dosulepin 25mg capsules 100 capsule |
| 947111000001101 | Dosulepin 25mg capsules 28 capsule |
| 1326311000001108 | Dosulepin 25mg capsules 600 capsule |
| 1003111000001108 | Dosulepin 25mg capsules 84 capsule |
| 321806009 | Dosulepin 75mg tablets |
| 1305411000001103 | Dosulepin 75mg tablets 28 tablet |
| 1255211000001101 | Dosulepin 75mg tablets 500 tablet |
| 29834411000001102 | Dosulepin 25mg capsules - Sigma Pharmaceuticals Plc |
| 29834511000001103 | Dosulepin 25mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 30123011000001102 | Dosulepin 75mg tablets - Mawdsley-Brooks & Company Ltd |
| 30123011000001102 | Dosulepin 75mg tablets - Mawdsley-Brooks & Company Ltd Dosulepin 75mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 17893811000001101 | Dosulepin 75mg tablets 28 tablet - Mawusiey-Brooks & Company Ltu Dosulepin 75mg tablets - Phoenix Healthcare Distribution Ltd |
| 1,02301100001107 | Dosulepin 73mg tablets - Phoenix Healthcare Distribution Ltd |

| 17893911000001107 | Dosulepin 75mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
|---|---|
| 566611000001109 | Dosulepin 75mg tablets - Sterwin Medicines |
| 1452711000001103 | Dosulepin 75mg tablets 28 tablet - Sterwin Medicines |
| 18281711000001109 | Dosulepin 75mg tablets - Strides Pharma UK Ltd |
| 18281811000001101 | Dosulepin 75mg tablets 28 tablet - Strides Pharma UK Ltd |
| 9792111000001105 | Dosulepin 25mg capsules - Almus Pharmaceuticals Ltd |
| 9792211000001104 | Dosulepin 25mg capsules 28 capsule - Almus Pharmaceuticals Ltd |
| 17893611000001101 | Dosulepin 25mg capsules - Phoenix Healthcare Distribution Ltd |
| 17893711000001105 | Dosulepin 25mg capsules 28 capsule - Phoenix Healthcare Distribution Ltd |
| 21932811000001107 | Dosulepin 25mg capsules - Waymade Healthcare Plc |
| 21932911000001102 | Dosulepin 25mg capsules 28 capsule - Waymade Healthcare Plc |
| 32799511000001101 | Dosulepin 75mg tablets - Genesis Pharmaceuticals Ltd |
| 32799611000001102 | Dosulepin 75mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 29834711000001108 | Dosulepin 75mg tablets - Sigma Pharmaceuticals Plc |
| 29834911000001105 | Dosulepin 75mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 241511000001103 | Dosulepin 75mg tablets - Teva UK Ltd |
| 1449311000001107 | Dosulepin 75mg tablets 28 tablet - Teva UK Ltd |
| 23880011000001107 | Dosulepin 25mg capsules - DE Pharmaceuticals |
| 23880111000001108 | Dosulepin 25mg capsules 28 capsule - DE Pharmaceuticals |
| 12058211000001104 | Dosulepin 125mg/5ml oral solution - Special Order |
| 12058411000001100 | Dosulepin 125mg/5ml oral solution 1 ml - Special Order |
| 619511000001105 | Dosulepin 25mg capsules - Kent Pharma (UK) Ltd |
| 1445711000001109 | Dosulepin 25mg capsules 28 capsule - Kent Pharma (UK) Ltd |
| 1445911000001106 | Dosulepin 25mg capsules 100 capsule - Kent Pharma (UK) Ltd |
| 1446111000001102 | Dosulepin 25mg capsules 600 capsule - Kent Pharma (UK) Ltd |
| 30122811000001100 | Dosulepin 25mg capsules - Mawdsley-Brooks & Company Ltd |
| 30122911000001105 | Dosulepin 25mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 582911000001100 | Dosulepin 25mg capsules - Mylan |
| 1445111000001108 | Dosulepin 25mg capsules 28 capsule - Mylan |
| 1445211000001102 | Dosulepin 25mg capsules 100 capsule - Mylan |
| 1445311000001105 | Dosulepin 25mg capsules 600 capsule - Mylan |
| 17197611000001101 | Dosulepin 25mg capsules - Sovereign Medical Ltd |
| 17197711000001105 | Dosulepin 25mg capsules 28 capsule - Sovereign Medical Ltd |
| 408611000001104 | Dosulepin 25mg capsules - Sterwin Medicines |
| 1447511000001108 | Dosulepin 25mg capsules 100 capsule - Sterwin Medicines |
| 18281511000001104 | Dosulepin 25mg capsules - Strides Pharma UK Ltd |
| 18281611000001100 | Dosulepin 25mg capsules 28 capsule - Strides Pharma UK Ltd |
| 62611000001108 | Dosulepin 75mg tablets - A A H Pharmaceuticals Ltd |
| 1448511000001107 | Dosulepin 75mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1448611000001106 | Dosulepin 75mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 397111000001102 | Dosulepin 25mg capsules - Actavis UK Ltd |
| 1444011000001108 | Dosulepin 25mg capsules 28 capsule - Actavis UK Ltd |
| 344311000001104 | Dosulepin 75mg tablets - IVAX Pharmaceuticals UK Ltd |
| 1450611000001106 | Dosulepin 75mg tablets 1994 That MacCathean on Eta Dosulepin 75mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 161411000001107 | Dosulepin 75mg tablets - Kent Pharma (UK) Ltd |
| 1450811000001105 | Dosulepin 75mg tablets - Kent Friarma (UK) Ltd Dosulepin 75mg tablets 28 tablet - Kent Pharma (UK) Ltd |
| 1451011000001108 | Dosulepin 75mg tablets 500 tablet - Kent Pharma (UK) Ltd |
| 851011000001104 | Dosulepin 75mg tablets - Mylan Dosulepin 75mg tablets - Mylan |
| 631011000001104 | Dozniehiii 12iiik ranierz - Milaii |

| 1450011000001104 | Dosulepin 75mg tablets 28 tablet - Mylan |
|---|---|
| 1450211000001109 | Dosulepin 75mg tablets 500 tablet - Mylan |
| 12060511000001106 | Dosulepin 37.5mg/5ml oral solution - Special Order |
| 12060611000001105 | Dosulepin 37.5mg/5ml oral solution 1 ml - Special Order |
| 12061711000001109 | Dosulepin 5mg/5ml oral solution - Special Order |
| 12061811000001101 | Dosulepin 5mg/5ml oral solution 1 ml - Special Order |
| 459411000001103 | Dosulepin 25mg capsules - Alliance Healthcare (Distribution) Ltd |
| | Dosulepin 25mg capsules 28 capsule - Alliance Healthcare |
| 1447811000001106 | (Distribution) Ltd |
| 3703211000001106 | Dosulepin 25mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 1448011000001104 | Dosulepin 25mg capsules 600 capsule - Alliance Healthcare (Distribution) Ltd |
| 12057211000001103 | Dosulepin 100mg/5ml oral solution - Special Order |
| 12057311000001106 | Dosulepin 100mg/5ml oral solution 1 ml - Special Order |
| 32797711000001103 | Dosulepin 25mg capsules - Genesis Pharmaceuticals Ltd |
| 32798111000001103 | Dosulepin 25mg capsules 28 capsule - Genesis Pharmaceuticals Ltd |
| 496511000001101 | Dosulepin 25mg capsules - IVAX Pharmaceuticals UK Ltd |
| 1445511000001104 | Dosulepin 25mg capsules 28 capsule - IVAX Pharmaceuticals UK Ltd |
| 1445611000001100 | Dosulepin 25mg capsules 100 capsule - IVAX Pharmaceuticals UK Ltd |
| 39328011000001101 | Dosulepin 25mg capsules - Medihealth (Northern) Ltd |
| 39328111000001100 | Dosulepin 25mg capsules 28 capsule - Medihealth (Northern) Ltd |
| 543311000001104 | Dosulepin 25mg capsules - Sandoz Ltd |
| 1446811000001109 | Dosulepin 25mg capsules 28 capsule - Sandoz Ltd |
| 600711000001109 | Dosulepin 75mg tablets - Actavis UK Ltd |
| 1448911000001100 | Dosulepin 75mg tablets 28 tablet - Actavis UK Ltd |
| 9792411000001100 | Dosulepin 75mg tablets - Almus Pharmaceuticals Ltd |
| 9792511000001101 | Dosulepin 75mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 12058711000001106 | Dosulepin 150mg/5ml oral solution - Special Order |
| 12058911000001108 | Dosulepin 150mg/5ml oral solution 1 ml - Special Order |
| 21933011000001105 | Dosulepin 75mg tablets - Waymade Healthcare Plc |
| 21933111000001106 | Dosulepin 75mg tablets 28 tablet - Waymade Healthcare Plc |
| 12059311000001101 | Dosulepin 20mg/5ml oral solution - Special Order |
| 12059411000001108 | Dosulepin 20mg/5ml oral solution 1 ml - Special Order |
| 254111000001108 | Dosulepin 25mg capsules - A A H Pharmaceuticals Ltd |
| 1443611000001104 | Dosulepin 25mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 1443811000001100 | Dosulepin 25mg capsules 100 capsule - A A H Pharmaceuticals Ltd |
| 1443911000001105 | Dosulepin 25mg capsules 600 capsule - A A H Pharmaceuticals Ltd |
| 8449011000001101 | Dosulepin 25mg/5ml oral solution - Drug Tariff Special Order |
| 8449211000001106 | Dosulepin 25mg/5ml oral solution 1 ml - Drug Tariff Special Order |
| 22245311000001105 | Dosulepin 25mg/5ml oral solution 500 ml - Drug Tariff Special Order |
| 148811000001109 | Dosulepin 25mg capsules - Teva UK Ltd |
| 1444111000001109 | Dosulepin 25mg capsules 28 capsule - Teva UK Ltd |
| 918611000001104 | Dosulepin 75mg tablets - Alliance Healthcare (Distribution) Ltd |
| 1452911000001101 | Dosulepin 75mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 1453011000001109 | Dosulepin 75mg tablets 500 tablet - Alliance Healthcare (Distribution) Ltd |
| 12061011000001107 | Dosulepin 50mg/5ml oral solution - Special Order |
| 12061111000001108 | Dosulepin 50mg/5ml oral solution 1 ml - Special Order |
| 8448611000001104 | Dosulepin 75mg/5ml oral solution - Drug Tariff Special Order |

| 8448811000001100 | Dosulepin 75mg/5ml oral solution 1 ml - Drug Tariff Special Order |
|---|---|
| 23390711000001107 | Dosulepin 75mg/5ml oral solution 150 ml - Drug Tariff Special Order |
| 12057711000001105 | Dosulepin 10mg/5ml oral solution - Special Order |
| 12057811000001102 | Dosulepin 10mg/5ml oral solution 1 ml - Special Order |
| 12059911000001100 | Dosulepin 250mg/5ml oral solution - Special Order |
| 12060111000001102 | Dosulepin 250mg/5ml oral solution 1 ml - Special Order |
| 23880411000001103 | Dosulepin 75mg tablets - DE Pharmaceuticals |
| 23880511000001104 | Dosulepin 75mg tablets 28 tablet - DE Pharmaceuticals |
| 5503211000001103 | Dosulepin 75mg tablets - Dowelhurst Ltd |
| 5503311000001106 | Dosulepin 75mg tablets 28 tablet - Dowelhurst Ltd |
| 8449911000001102 | Dosulepin 25mg/5ml oral suspension - Special Order |
| 8450211000001101 | Dosulepin 25mg/5ml oral suspension 1 ml - Special Order |
| 39237511000001102 | Dosulepin 75mg tablets - Medihealth (Northern) Ltd |
| 39237611000001103 | Dosulepin 75mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 407811000001104 | Dosulepin 75mg tablets - Sandoz Ltd |
| 1451911000001107 | Dosulepin 75mg tablets - Sandoz Ltd Dosulepin 75mg tablets 28 tablet - Sandoz Ltd |
| 17197811000001107 | Dosulepin 75mg tablets - Sovereign Medical Ltd |
| 17197911000001107 | Dosulepin 75mg tablets - Sovereign Medical Ltd Dosulepin 75mg tablets 28 tablet - Sovereign Medical Ltd |
| 8449411000001107 | Dosulepin 75mg/5ml oral suspension - Special Order |
| 8449811000001107 | Dosulepin 75mg/5ml oral suspension 1 ml - Special Order |
| 23390911000001107 | |
| 12082611000001109 | Dosulepin 75mg/5ml oral suspension 150 ml - Special Order |
| | Dosulepin 125mg/5ml oral solution |
| 12058111000001100 | Dosulepin 125mg/5ml oral solution 1 ml |
| 12083011000001106 | Dosulepin 37.5mg/5ml oral solution |
| 12060311000001100 | Dosulepin 37.5mg/5ml oral solution 1 ml |
| 12083211000001101 | Dosulepin 5mg/5ml oral solution |
| 12061611000001100 | Dosulepin 5mg/5ml oral solution 1 ml |
| 12082411000001106 | Dosulepin 100mg/5ml oral solution |
| 12057111000001109<br>12082711000001100 | Dosulepin 100mg/5ml oral solution 1 ml |
| | Dosulepin 150mg/5ml oral solution |
| 12058511000001101<br>8454111000001103 | Dosulepin 150mg/5ml oral solution 1 ml Dosulepin 75mg/5ml oral solution |
| 8448511000001103 | Dosulepin 75mg/5ml oral solution Dosulepin 75mg/5ml oral solution 1 ml |
| 23390611000001103<br>12082811000001108 | Dosulepin 75mg/5ml oral solution 150 ml |
| | Dosulepin 20mg/5ml oral solution |
| 12059011000001104 | Dosulepin 20mg/5ml oral solution 1 ml |
| 8454311000001101 | Dosulepin 25mg/5ml oral solution |
| 8448711000001108 | Dosulepin 25mg/5ml oral solution 1 ml |
| 22245211000001102 | Dosulepin 25mg/5ml oral solution 500 ml |
| 12083111000001107 | Dosulepin 50mg/5ml oral solution |
| 12060811000001109 | Dosulepin 50mg/5ml oral solution 1 ml |
| 12082511000001105 | Dosulepin 10mg/5ml oral solution |
| 12057611000001101 | Dosulepin 10mg/5ml oral solution 1 ml |
| 12082911000001103 | Dosulepin 250mg/5ml oral solution |
| 12059711000001102 | Dosulepin 250mg/5ml oral solution 1 ml |
| 8454211000001109 | Dosulepin 25mg/5ml oral suspension |
| 8449711000001104 | Dosulepin 25mg/5ml oral suspension 1 ml |
| 8454011000001104 | Dosulepin 75mg/5ml oral suspension |
| 8449311000001103 | Dosulepin 75mg/5ml oral suspension 1 ml |

| 23390811000001104 | Dosulepin 75mg/5ml oral suspension 150 ml |
|---|---|
| 14911000001107 | Dothapax 25 capsules - Ashbourne Pharmaceuticals Ltd |
| 1444311000001106 | Dothapax 25 capsules 84 capsule - Ashbourne Pharmaceuticals Ltd |
| 927011000001104 | Dothapax 75 tablets - Ashbourne Pharmaceuticals Ltd |
| 1449511000001101 | Dothapax 75 tablets 28 tablet - Ashbourne Pharmaceuticals Ltd |
| 321811006 | Doxepin 10mg capsules |
| 28417811000001106 | Doxepin 10mg capsules - Special Order |
| 28417711000001103 | Doxepin 10mg capsules 1 capsule |
| 28417911000001101 | Doxepin 10mg capsules 1 capsule - Special Order |
| 1254311000001105 | Doxepin 10mg capsules 56 capsule |
| 321812004 | Doxepin 25mg capsules |
| 24619811000001104 | Doxepin 25mg capsules - A A H Pharmaceuticals Ltd |
| 24538711000001100 | Doxepin 25mg capsules - Alliance Healthcare (Distribution) Ltd |
| 38748011000001102 | Doxepin 25mg capsules - Crescent Pharma Ltd |
| 37300811000001107 | Doxepin 25mg capsules - DE Pharmaceuticals |
| 24442311000001108 | Doxepin 25mg capsules - Marlborough Pharmaceuticals Ltd |
| 38876711000001102 | Doxepin 25mg capsules - Medihealth (Northern) Ltd |
| 24669011000001109 | Doxepin 25mg capsules - Waymade Healthcare Plc |
| 39333311000001108 | Doxepin 25mg capsules - Zentiva Pharma UK Ltd |
| 1064511000001102 | Doxepin 25mg capsules 28 capsule |
| 24619911000001109 | Doxepin 25mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 24538811000001108 | Doxepin 25mg capsules 28 capsule - Alliance Healthcare (Distribution) |
| 38748211000001107 | Ltd Doxepin 25mg capsules 28 capsule - Crescent Pharma Ltd |
| 37300911000001107 | Doxepin 25mg capsules 28 capsule - Clescent Flama Ltu Doxepin 25mg capsules 28 capsule - DE Pharmaceuticals |
| 24442411000001101 | Doxepin 25mg capsules 28 capsule - Marlborough Pharmaceuticals Ltd |
| 38876811000001101 | Doxepin 25mg capsules 28 capsule - Mariborough Friatmaceuticals Ltu Doxepin 25mg capsules 28 capsule - Medihealth (Northern) Ltd |
| 24669111000001105 | Doxepin 25mg capsules 28 capsule - Waymade Healthcare Plc |
| 39333611000001103 | Doxepin 25mg capsules 28 capsule - Waymade Healthcare Fic |
| 321813009 | Doxepin 50mg capsules Doxepin 50mg capsules |
| 24620011000001106 | Doxepin 50mg capsules - A A H Pharmaceuticals Ltd |
| 24538911000001103 | Doxepin 50mg capsules - Alliance Healthcare (Distribution) Ltd |
| 38738511000001109 | Doxepin 50mg capsules - Amarice Healthcare (Distribution) Etu |
| 37301011000001105 | Doxepin 50mg capsules - Crescent Pharma Ltu Doxepin 50mg capsules - DE Pharmaceuticals |
| 24442511000001102 | Doxepin 50mg capsules - De Friarmaceuticals Doxepin 50mg capsules - Marlborough Pharmaceuticals Ltd |
| 38876911000001102 | Doxepin 50mg capsules - Medihealth (Northern) Ltd |
| 24668811000001105 | Doxepin 50mg capsules - Waymade Healthcare Plc |
| 39333711000001107 | Doxepin 50mg capsules - Waymade Healthcare Fit |
| 1322011000001107 | Doxepin 50mg capsules - Zentiva Friarma OK Ltu Doxepin 50mg capsules 28 capsule |
| 24620111000001107 | Doxepin 50mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| | Doxepin 50mg capsules 28 capsule - A A in Priarmaceuticals Ltd Doxepin 50mg capsules 28 capsule - Alliance Healthcare (Distribution) |
| 24539011000001107 | Ltd |
| 38738611000001108 | Doxepin 50mg capsules 28 capsule - Crescent Pharma Ltd |
| 37301111000001106 | Doxepin 50mg capsules 28 capsule - DE Pharmaceuticals |
| 24442611000001103 | Doxepin 50mg capsules 28 capsule - Marlborough Pharmaceuticals Ltd |
| 38877011000001101 | Doxepin 50mg capsules 28 capsule - Medihealth (Northern) Ltd |
| 24668911000001100 | Doxepin 50mg capsules 28 capsule - Waymade Healthcare Plc |
| 39333811000001104 | Doxepin 50mg capsules 28 capsule - Zentiva Pharma UK Ltd |
| 8484811000001101 | Doxepin 50mg/5ml oral solution |
| 8460711000001100 | Doxepin 50mg/5ml oral solution - Special Order |

| 846(0411000001106 Doxepin S0mg/Sml oral solution 1 ml - Special Order 846(1011000001106 Doxepin S0mg/Sml oral solution 1 ml - Special Order 846(1111000001107 Doxepin S0mg/Sml oral suspension 846(1111000001107 Doxepin S0mg/Sml oral suspension - Special Order 846(1111000001104 Doxepin S0mg/Sml oral suspension 1 ml - Special Order 946(1111000001102 Doxepin S0mg/Sml oral suspension 1 ml - Special Order 940(11000001102 Doxepin 75mg capsules 940(11000001102 Doxepin 75mg capsules 28 capsule 940(11000001102 Doxepin 75mg capsules 28 capsule 940(11000001102 Eperpapax 70mg tablets - Ashbourne Pharmaceuticals Ltd 950(11000001106 Germanil 70mg tablets - Ashbourne Pharmaceuticals Ltd 950(11000001108 Gamanil 70mg tablets - Merck Serono Ltd 950(11000001103 Gamanil 70mg tablets - Merck Serono Ltd 12538911000001104 Imipramine 100mg/Sml oral solution - Special Order 12538911000001109 Imipramine 100mg/Sml oral suspension 1 12538911000001100 Imipramine 100mg/Sml oral suspension 1 ml 12538911000001101 Imipramine 10mg tablets - March Serial Order 1253811000001104 Imipramine 10mg tablets - March Serial Order <th></th> <th></th> | | |
|---|---|---|
| 8484911000001106 Doxepin 50mg/5ml oral suspension 8461311000001107 Doxepin 50mg/5ml oral suspension - Special Order 8461111000001107 Doxepin 50mg/5ml oral suspension 1 ml 8461111000001102 Doxepin 50mg/5ml oral suspension 1 ml - Special Order 321814003 Doxepin 75mg capsules 28 capsule 694011000001102 Doxepin 75mg capsules 28 capsule 694011000001103 Feprapax 70mg tablets - Ashbourne Pharmaceuticals Ltd 93011000001106 Gamanil 70mg tablets - Merck Serono Ltd 933811000001103 Gamanil 70mg tablets 56 tablet - Merck Serono Ltd 2338211000001106 Gamanil 70mg tablets 50 tablet - Merck Serono Ltd 12598411000001106 Gamanil 70mg tablets 50 tablet - Merck Serono Ltd 12598411000001100 Imipramine 100mg/5ml oral solution - Special Order 12598411000001100 Imipramine 100mg/5ml oral suspension 12598111000001100 Imipramine 100mg/5ml oral suspension 1 ml 12598111000001101 Imipramine 10mg tablets - Ala P Pharmaceuticals Ltd 24421100001101 Imipramine 10mg tablets - Alamace Healthcare Ltd 137816001 Imipramine 10mg tablets - Almus Pharmaceuticals Ltd 1442811000001101 Imipramine 10mg tablets - Almus Pharmaceuticals | 8460411000001106 | Doxepin 50mg/5ml oral solution 1 ml |
| 8461311000001109 Doxepin 50mg/5ml oral suspension - Special Order 8461311000001104 Doxepin 50mg/5ml oral suspension 1 ml 8461611000001102 Doxepin 50mg/5ml oral suspension 1 ml - Special Order 321814003 Doxepin 75mg capsules 1061211000001102 Feprapax 70mg tablets - Ashbourne Pharmaceuticals Ltd 69011000001102 Feprapax 70mg tablets 56 tablet - Ashbourne Pharmaceuticals Ltd 95011000001103 Gamanil 70mg tablets 56 tablet - Merck Serono Ltd 2338211000001103 Gamanil 70mg tablets 55 tablet - Merck Serono Ltd 2338211000001103 Gamanil 70mg tablets 55 tablet - Merck Serono Ltd 12598311000001102 Imipramine 100mg/5ml oral solution - Special Order 12598311000001102 Imipramine 100mg/5ml oral solution 1 ml - Special Order 12598311000001109 Imipramine 100mg/5ml oral suspension - Special Order 12598111000001100 Imipramine 100mg/5ml oral suspension - Special Order 12598111000001100 Imipramine 100mg/5ml oral suspension - Special Order 12598111000001100 Imipramine 100mg/5ml oral suspension 1 ml - Special Order 12598111000001104 Imipramine 100mg/5ml oral suspension 1 ml - Special Order 12598111000001104 Imipramine 100mg/5ml oral suspension 1 ml - Special Order 12598111000001100 Imipramine 10mg tablets - A A H Pharmaceuticals Ltd 1424211000001100 Imipramine 10mg tablets - A K A H Pharmaceuticals Ltd 1424211000001101 Imipramine 10mg tablets - Aliance Healthcare (Distribution) Ltd 13411811000001101 Imipramine 10mg tablets - Aliance Healthcare (Distribution) Ltd 13411811000001101 Imipramine 10mg tablets - Crescent Pharma Ltd 143612711000001104 Imipramine 10mg tablets - Disketh Laboratories Ltd 1439347811000001105 Imipramine 10mg tablets - Special Pharmaceuticals Ltd 1439347811000001106 Imipramine 10mg tablets - Special Pharmaceuticals Ltd 1439347811000001106 Imipramine 10mg tablets - Special Pharmaceuticals Ltd 1439347811000001100 Imipramine 10mg tablets - Special Pharmaceuticals Ltd 1439347811000001100 Imipramine 10mg tablets - Special Pharmaceuticals Ltd 1439347811000001101 Imipramine 10mg tablets - Sto tablet - A H Pharmaceuticals Lt | 8461011000001106 | Doxepin 50mg/5ml oral solution 1 ml - Special Order |
| 8461111000001107 Doxepin 50mg/5ml oral suspension 1 ml 8461611000001104 Doxepin 75mg capsules 1061211000001102 Doxepin 75mg capsules 28 capsule 694011000001106 Feprapax 70mg tablets - Ashbourne Pharmaceuticals Ltd 2335811000001106 Feprapax 70mg tablets - S6 tablet - Ashbourne Pharmaceuticals Ltd 2335811000001108 Gamanil 70mg tablets 56 tablet - Merck Serono Ltd 2338211000001103 Gamanil 70mg tablets 55 tablet - Merck Serono Ltd 2338211000001103 Gamanil 70mg tablets 55 tablet - Merck Serono Ltd 2338211000001100 Imipramine 100mg/5ml oral solution - Special Order 12598411000001109 Imipramine 100mg/5ml oral suspension - Special Order 12637511000001105 Imipramine 100mg/5ml oral suspension - Special Order 12598911000001100 Imipramine 100mg/5ml oral suspension 1 ml 12598111000001104 Imipramine 100mg/5ml oral suspension 1 ml - Special Order 12598111000001105 Imipramine 10mg tablets - A A H Pharmaceuticals Ltd 424211000001101 Imipramine 10mg tablets - A H Pharmaceuticals Ltd 424211000001105 Imipramine 10mg tablets - Alliance Healthcare (Distribution) Ltd 13411811000001101 Imipramine 10mg tablets - Crescent Pharmaceuticals Ltd | 8484911000001106 | Doxepin 50mg/5ml oral suspension |
| Doxepin 50mg/5ml oral suspension 1 ml - Special Order | 8461311000001109 | Doxepin 50mg/5ml oral suspension - Special Order |
| Doxepin 75mg capsules | 8461111000001107 | Doxepin 50mg/5ml oral suspension 1 ml |
| Doxepin 75mg capsules 28 capsule | 8461611000001104 | Doxepin 50mg/5ml oral suspension 1 ml - Special Order |
| Feprapax 70mg tablets - Ashbourne Pharmaceuticals Ltd | 321814003 | Doxepin 75mg capsules |
| 2335811000001106 | 1061211000001102 | Doxepin 75mg capsules 28 capsule |
| 95011000001108 | 694011000001102 | Feprapax 70mg tablets - Ashbourne Pharmaceuticals Ltd |
| 2338211000001103 Gamanil 70mg tablets 250 tablet - Merck Serono Ltd | 2335811000001106 | Feprapax 70mg tablets 56 tablet - Ashbourne Pharmaceuticals Ltd |
| 2337911000001106 Gamanil 70mg tablets 56 tablet - Merck Serono Ltd 12598311000001102 Imipramine 100mg/Sml oral solution - Special Order 12598411000001105 Imipramine 100mg/Sml oral solution 1 ml - Special Order 12597911000001100 Imipramine 100mg/Sml oral suspension 12597911000001102 Imipramine 100mg/Sml oral suspension - Special Order 12597911000001104 Imipramine 100mg/Sml oral suspension 1 ml 12598111000001104 Imipramine 100mg/Sml oral suspension 1 ml 12598111000001105 Imipramine 10mg tablets 1254311000001105 Imipramine 10mg tablets - A A H Pharmaceuticals Ltd 124211000001100 Imipramine 10mg tablets - A A H Pharmaceuticals Ltd 13411811000001101 Imipramine 10mg tablets - Accord Healthcare (Distribution) Ltd 13411811000001101 Imipramine 10mg tablets - Almus Pharmaceuticals Ltd 134438111000001101 Imipramine 10mg tablets - Crescent Pharma Ltd 134938111000001104 Imipramine 10mg tablets - Oalkeith Laboratories Ltd 13947811000001104 Imipramine 10mg tablets - De Pharmaceuticals 138997511000001106 Imipramine 10mg tablets - Wedihealth (Northern) Ltd 17932011000001106 Imipramine 10mg tablets - Medihealth (Northern) Ltd 17932011000001106 Imipramine 10mg tablets - Sigma Pharmaceuticals Plc 1850911000001106 Imipramine 10mg tablets - Sigma Pharmaceuticals Plc 1850911000001106 Imipramine 10mg tablets - Sigma Pharmaceuticals Plc 1877911000001100 Imipramine 10mg tablets - Sigma Pharmaceuticals Plc 1878811000001101 Imipramine 10mg tablets 250 tablet 1878811000001104 Imipramine 10mg tablets 250 tablet - A H Pharmaceuticals Ltd 1877811000001109 Imipramine 10mg tablets 250 tablet - A H Pharmaceuticals Ltd 1877811000001101 Imipramine 10mg tablets 28 tablet - Daleith Laboratories Ltd 1877811000001101 Imipramine 10mg tablets 28 tablet - A H Pharmaceuticals Ltd 1878811000001101 Imipramine 10mg tablets 28 tablet - A H Pharmaceuticals Ltd 1878811000001101 Imipramine 10mg tablets 28 tablet - De Pharmaceuticals Ltd 187897611000001103 Imipramine 10mg tablets 28 tablet - De Pharmaceu | 95011000001108 | Gamanil 70mg tablets - Merck Serono Ltd |
| 1259831100001102 | 2338211000001103 | Gamanil 70mg tablets 250 tablet - Merck Serono Ltd |
| 12598411000001109 | 2337911000001106 | Gamanil 70mg tablets 56 tablet - Merck Serono Ltd |
| 12537511000001105 | 12598311000001102 | Imipramine 100mg/5ml oral solution - Special Order |
| 12598011000001100 | 12598411000001109 | Imipramine 100mg/5ml oral solution 1 ml - Special Order |
| 12597911000001102 | 12637511000001105 | Imipramine 100mg/5ml oral suspension |
| 12598111000001104 | 12598011000001100 | Imipramine 100mg/5ml oral suspension - Special Order |
| Imipramine 10mg tablets Imipramine 10mg tablets A A H Pharmaceuticals Ltd | 12597911000001102 | Imipramine 100mg/5ml oral suspension 1 ml |
| Imipramine 10mg tablets - A A H Pharmaceuticals Ltd | 12598111000001104 | Imipramine 100mg/5ml oral suspension 1 ml - Special Order |
| A2421100001100 | 321816001 | Imipramine 10mg tablets |
| Imipramine 10mg tablets - Alliance Healthcare (Distribution) Ltd | 254311000001105 | Imipramine 10mg tablets - A A H Pharmaceuticals Ltd |
| 1341181100001101 | 424211000001100 | Imipramine 10mg tablets - Accord Healthcare Ltd |
| Imipramine 10mg tablets - Crescent Pharma Ltd | 557411000001101 | Imipramine 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| Imipramine 10mg tablets - Dalkeith Laboratories Ltd | 13411811000001101 | Imipramine 10mg tablets - Almus Pharmaceuticals Ltd |
| Imipramine 10mg tablets - DE Pharmaceuticals | 34438111000001109 | Imipramine 10mg tablets - Crescent Pharma Ltd |
| Imipramine 10mg tablets - Kent Pharmaceuticals Ltd | 36512711000001104 | Imipramine 10mg tablets - Dalkeith Laboratories Ltd |
| Imipramine 10mg tablets - Medihealth (Northern) Ltd | 23947811000001101 | Imipramine 10mg tablets - DE Pharmaceuticals |
| 17932011000001100 | 907411000001103 | Imipramine 10mg tablets - Kent Pharmaceuticals Ltd |
| Imipramine 10mg tablets - Sigma Pharmaceuticals Plc | 38997511000001106 | Imipramine 10mg tablets - Medihealth (Northern) Ltd |
| Imipramine 10mg tablets - Teva UK Ltd | 17932011000001100 | Imipramine 10mg tablets - Phoenix Healthcare Distribution Ltd |
| Imipramine 10mg tablets - Waymade Healthcare Plc | 29877211000001105 | Imipramine 10mg tablets - Sigma Pharmaceuticals Plc |
| Imipramine 10mg tablets 250 tablet 2378611000001104 | 8150911000001106 | Imipramine 10mg tablets - Teva UK Ltd |
| Imipramine 10mg tablets 250 tablet - Alliance Healthcare (Distribution) | 22057711000001109 | Imipramine 10mg tablets - Waymade Healthcare Plc |
| Ltd 2378311000001109 | 1125611000001101 | Imipramine 10mg tablets 250 tablet |
| 990711000001105 | 2378611000001104 | |
| 2377411000001101 Imipramine 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd | 2378311000001109 | Imipramine 10mg tablets 250 tablet - Kent Pharmaceuticals Ltd |
| 2377611000001103 | 990711000001105 | Imipramine 10mg tablets 28 tablet |
| Imipramine 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 13411911000001106 Imipramine 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd 34438211000001103 Imipramine 10mg tablets 28 tablet - Crescent Pharma Ltd 36512811000001107 Imipramine 10mg tablets 28 tablet - Dalkeith Laboratories Ltd 23947911000001106 Imipramine 10mg tablets 28 tablet - DE Pharmaceuticals 2378211000001101 Imipramine 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd 38997611000001105 Imipramine 10mg tablets 28 tablet - Medihealth (Northern) Ltd 17932111000001104 Imipramine 10mg tablets 28 tablet - Phoenix Healthcare Distribution | 2377411000001101 | Imipramine 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 13411911000001106 | 2377611000001103 | Imipramine 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 34438211000001103 | 2378511000001103 | |
| 36512811000001107 | 13411911000001106 | Imipramine 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 23947911000001106 | 34438211000001103 | Imipramine 10mg tablets 28 tablet - Crescent Pharma Ltd |
| 2378211000001101 Imipramine 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd 38997611000001105 Imipramine 10mg tablets 28 tablet - Medihealth (Northern) Ltd 17932111000001104 Imipramine 10mg tablets 28 tablet - Phoenix Healthcare Distribution | 36512811000001107 | Imipramine 10mg tablets 28 tablet - Dalkeith Laboratories Ltd |
| 38997611000001105 Imipramine 10mg tablets 28 tablet - Medihealth (Northern) Ltd 17932111000001104 Imipramine 10mg tablets 28 tablet - Phoenix Healthcare Distribution | 23947911000001106 | Imipramine 10mg tablets 28 tablet - DE Pharmaceuticals |
| 17932111000001104 Imipramine 10mg tablets 28 tablet - Phoenix Healthcare Distribution | 2378211000001101 | Imipramine 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 1 1/932111000001104 | 38997611000001105 | <u> </u> |
| | 17932111000001104 | |
| 29877311000001102 | Imipramine 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
|---|---|
| 8151011000001103 | Imipramine 10mg tablets 28 tablet - Teva UK Ltd |
| 22057811000001101 | Imipramine 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 8561111000001100 | Imipramine 10mg/5ml oral solution |
| 8541711000001109 | Imipramine 10mg/5ml oral solution - Special Order |
| 8541611000001100 | Imipramine 10mg/5ml oral solution 1 ml |
| 8541911000001106 | Imipramine 10mg/5ml oral solution 1 ml - Special Order |
| 8561211000001106 | Imipramine 10mg/5ml oral suspension |
| 8542311000001101 | Imipramine 10mg/5ml oral suspension - Special Order |
| 8542211000001109 | Imipramine 10mg/5ml oral suspension 1 ml |
| 8542411000001108 | Imipramine 10mg/5ml oral suspension 1 ml - Special Order |
| 8561311000001103 | Imipramine 12.5mg/5ml oral solution |
| 8542911000001100 | Imipramine 12.5mg/5ml oral solution - Special Order |
| 8542811000001105 | Imipramine 12.5mg/5ml oral solution 1 ml |
| 8543011000001108 | Imipramine 12.5mg/5ml oral solution 1 ml - Special Order |
| 8561411000001105 | Imipramine 12.5mg/5ml oral suspension |
| 8543411000001104 | Imipramine 12.5mg/5ml oral suspension - Special Order |
| 8543211000001103 | Imipramine 12.5mg/5ml oral suspension 1 ml |
| 8543611000001101 | Imipramine 12.5mg/5ml oral suspension 1 ml - Special Order |
| 15356411000001103 | Imipramine 125mg/5ml oral solution |
| 15350611000001102 | Imipramine 125mg/5ml oral solution - Special Order |
| 15350511000001101 | Imipramine 125mg/5ml oral solution 1 ml |
| 15350811000001103 | Imipramine 125mg/5ml oral solution 1 ml - Special Order |
| 15356311000001105 | Imipramine 125mg/5ml oral suspension |
| 15351111000001104 | Imipramine 125mg/5ml oral suspension - Special Order |
| 15351011000001100 | Imipramine 125mg/5ml oral suspension 1 ml |
| 15351311000001102 | Imipramine 125mg/5ml oral suspension 1 ml - Special Order |
| 321817005 | Imipramine 25mg tablets |
| 569911000001107 | Imipramine 25mg tablets - A A H Pharmaceuticals Ltd |
| 572011000001105 | Imipramine 25mg tablets - Accord Healthcare Ltd |
| 709011000001108 | Imipramine 25mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9806411000001104 | Imipramine 25mg tablets - Almus Pharmaceuticals Ltd |
| 34437911000001106 | Imipramine 25mg tablets - Crescent Pharma Ltd |
| 36512911000001102 | Imipramine 25mg tablets - Dalkeith Laboratories Ltd |
| 23948011000001108 | Imipramine 25mg tablets - DE Pharmaceuticals |
| 667611000001100 | Imipramine 25mg tablets - Kent Pharmaceuticals Ltd |
| 38997711000001101 | Imipramine 25mg tablets - Medihealth (Northern) Ltd |
| 17932211000001105 | Imipramine 25mg tablets - Phoenix Healthcare Distribution Ltd |
| 39225211000001105 | Imipramine 25mg tablets - Relonchem Ltd |
| 29877411000001109 | Imipramine 25mg tablets - Sigma Pharmaceuticals Plc |
| 8151111000001102 | Imipramine 25mg tablets - Teva UK Ltd |
| 3511000001100 | Imipramine 25mg tablets - The Boots Company Plc |
| 22058011000001108 | Imipramine 25mg tablets - Waymade Healthcare Plc |
| 5424911000001108 | Imipramine 25mg tablets 100 tablet |
| 987311000001106 | Imipramine 25mg tablets 28 tablet |
| 2379411000001105 | Imipramine 25mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 2379611000001108 | Imipramine 25mg tablets 28 tablet - Accord Healthcare Ltd |
| 2381511000001102 | Imipramine 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 9806711000001105 | Imipramine 25mg tablets 28 tablet - Almus Pharmaceuticals Ltd |

| 34438011000001108 | Imipramine 25mg tablets 28 tablet - Crescent Pharma Ltd |
|---|---|
| 36513011000001105 | Imipramine 25mg tablets 28 tablet - Dalkeith Laboratories Ltd |
| 23948111000001109 | Imipramine 25mg tablets 28 tablet - DE Pharmaceuticals |
| 2380411000001105 | Imipramine 25mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 38997811000001109 | Imipramine 25mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 17934711000001108 | Imipramine 25mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 39225311000001102 | Imipramine 25mg tablets 28 tablet - Relonchem Ltd |
| 29877511000001108 | Imipramine 25mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 8151211000001108 | Imipramine 25mg tablets 28 tablet - Teva UK Ltd |
| 22058111000001109 | Imipramine 25mg tablets 28 tablet - Waymade Healthcare Plc |
| 1127611000001108 | Imipramine 25mg tablets 500 tablet |
| 2381711000001107 | Imipramine 25mg tablets 500 tablet - Alliance Healthcare (Distribution) Ltd |
| 2380511000001109 | Imipramine 25mg tablets 500 tablet - Kent Pharmaceuticals Ltd |
| 2380011000001101 | Imipramine 25mg tablets 500 tablet - The Boots Company Plc |
| 1299111000001103 | Imipramine 25mg tablets 84 tablet |
| 36046511000001104 | Imipramine 25mg/5ml oral solution |
| 321825007 | Imipramine 25mg/5ml oral solution |
| 8545711000001106 | Imipramine 25mg/5ml oral solution - Special Order |
| 8546011000001100 | Imipramine 25mg/5ml oral solution 1 ml - Special Order |
| 8545511000001101 | Imipramine 25mg/5ml oral solution 1 mllmipramine 25mg/5ml oral solution 1 ml |
| 968811000001101 | Imipramine 25mg/5ml oral solution 150 ml |
| 16423411000001100 | Imipramine 25mg/5ml oral solution sugar free |
| 16731611000001108 | Imipramine 25mg/5ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 17630311000001102 | Imipramine 25mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 22624911000001106 | Imipramine 25mg/5ml oral solution sugar free - Colorama Pharmaceuticals Ltd |
| 24026811000001107 | Imipramine 25mg/5ml oral solution sugar free - CST Pharma Ltd |
| 21834911000001104 | Imipramine 25mg/5ml oral solution sugar free - Cubic Pharmaceuticals Ltd |
| 37422211000001109 | Imipramine 25mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 26369111000001106 | Imipramine 25mg/5ml oral solution sugar free - Ennogen Healthcare Ltd |
| 27998911000001105 | Imipramine 25mg/5ml oral solution sugar free - J M McGill Ltd |
| 28917111000001102 | Imipramine 25mg/5ml oral solution sugar free - Niche Pharma Ltd |
| 16422011000001100 | Imipramine 25mg/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd |
| 18717511000001100 | Imipramine 25mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc |
| 22057411000001103 | Imipramine 25mg/5ml oral solution sugar free - Waymade Healthcare Plc |
| 16421911000001107 | Imipramine 25mg/5ml oral solution sugar free 150 ml |
| 16731711000001104 | Imipramine 25mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 17630411000001109 | Imipramine 25mg/5ml oral solution sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 22625011000001106 | Imipramine 25mg/5ml oral solution sugar free 150 ml - Colorama Pharmaceuticals Ltd |
| 24026911000001102 | Imipramine 25mg/5ml oral solution sugar free 150 ml - CST Pharma<br>Ltd |

| Pharmaceuticals Ltd Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Imipramine 25mg/5ml oral solution sugar free 15 Healthcare Ltd Pharmaceuticals Imipramine 25mg/5ml oral solution sugar free 15 Healthcare Ltd Imipramine 25mg/5ml oral solution sugar free 15 Ltd Imipramine 25mg/5ml oral solution sugar free 15 Ltd Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Ltd Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Ltd Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Plc Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Plc Imipramine 25mg/5ml oral solution sugar free 15 Healthcare Plc Imipramine 25mg/5ml oral suspension Imipramine 25mg/5ml oral suspension - Special oral suspens | 50 ml - Ennogen<br>50 ml - J M McGill Ltd<br>50 ml - Niche Pharma<br>50 ml - Rosemont<br>50 ml - Sigma |
|---|---|
| Imipramine 25mg/5ml oral solution sugar free 19 | 50 ml - J M McGill Ltd<br>50 ml - Niche Pharma<br>50 ml - Rosemont<br>50 ml - Sigma |
| Imipramine 25mg/5ml oral solution sugar free 15 | 50 ml - Niche Pharma<br>50 ml - Rosemont<br>50 ml - Sigma |
| Ltd 16422111000001104 Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Ltd 18717611000001101 Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Plc 22057511000001104 Imipramine 25mg/5ml oral solution sugar free 15 Healthcare Plc 8561511000001109 Imipramine 25mg/5ml oral suspension 8546511000001108 Imipramine 25mg/5ml oral suspension - Special 6 | 50 ml - Rosemont<br>50 ml - Sigma |
| Pharmaceuticals Ltd Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Plc Imipramine 25mg/5ml oral solution sugar free 15 Pharmaceuticals Plc Imipramine 25mg/5ml oral solution sugar free 15 Healthcare Plc Imipramine 25mg/5ml oral suspension Imipramine 25mg/5ml oral suspension - Special 6 | 50 ml - Sigma |
| Pharmaceuticals Plc 22057511000001104 | |
| ### Healthcare Plc 8561511000001104 Healthcare Plc | 50 ml - Waymade |
| 8546511000001108 Imipramine 25mg/5ml oral suspension - Special 0 | |
| 05.46244.0000044.05 | Order |
| 8546211000001105 Imipramine 25mg/5ml oral suspension 1 ml | |
| 8546611000001107 Imipramine 25mg/5ml oral suspension 1 ml - Spe | ecial Order |
| 12637611000001109 Imipramine 40mg/5ml oral solution | |
| 12598911000001101 Imipramine 40mg/5ml oral solution - Special Ord | der |
| 12598811000001106 Imipramine 40mg/5ml oral solution 1 ml | |
| 12599011000001105 Imipramine 40mg/5ml oral solution 1 ml - Specia | al Order |
| 12637711000001100 Imipramine 40mg/5ml oral suspension | |
| 12598611000001107 Imipramine 40mg/5ml oral suspension - Special 0 | Order |
| 12598511000001108 Imipramine 40mg/5ml oral suspension 1 ml | |
| 12598711000001103 Imipramine 40mg/5ml oral suspension 1 ml - Spe | ecial Order |
| 4534311000001106 Lentizol 25mg modified-release capsules - Pfizer | Ltd |
| 4534411000001104 Lentizol 25mg modified-release capsules 56 caps | sule - Pfizer Ltd |
| 4533611000001104 Lentizol 50mg modified-release capsules - Pfizer | Ltd |
| 4534111000001109 Lentizol 50mg modified-release capsules 56 caps | sule - Pfizer Ltd |
| 12760311000001103 Lofepramine 140mg/5ml oral solution | |
| 12739311000001103 Lofepramine 140mg/5ml oral solution - Special C | Order |
| 12739011000001101 Lofepramine 140mg/5ml oral solution 1 ml | |
| 12739511000001109 Lofepramine 140mg/5ml oral solution 1 ml - Spe | cial Order |
| 12760411000001105 Lofepramine 140mg/5ml oral suspension | |
| 12746511000001103 Lofepramine 140mg/5ml oral suspension - Specia | al Order |
| 12737911000001109 Lofepramine 140mg/5ml oral suspension 1 ml | |
| 12746611000001104 Lofepramine 140mg/5ml oral suspension 1 ml - S | Special Order |
| 12760511000001109 Lofepramine 23mg/5ml oral solution | |
| 12740811000001102 Lofepramine 23mg/5ml oral solution - Special Or | rder |
| 12740611000001101 Lofepramine 23mg/5ml oral solution 1 ml | |
| Lofepramine 23mg/5ml oral solution 1 ml - Speci | ial Order |
| 12760611000001108 Lofepramine 23mg/5ml oral suspension | |
| 12740211000001103 Lofepramine 23mg/5ml oral suspension - Special | l Order |
| 12740011000001108 Lofepramine 23mg/5ml oral suspension 1 ml | |
| 12740311000001106 Lofepramine 23mg/5ml oral suspension 1 ml - Sp | pecial Order |
| 12760711000001104 Lofepramine 35mg/5ml oral solution | |
| 12742211000001102 Lofepramine 35mg/5ml oral solution - Special Or | rder |
| 12742011000001107 Lofepramine 35mg/5ml oral solution 1 ml | - |
| 12742311000001105 Lofepramine 35mg/5ml oral solution 1 ml - Speci | ial Order |
| 12760811000001107 Lofepramine 35mg/5ml oral suspension | |

| 12741611000001106 | Lofepramine 35mg/5ml oral suspension - Special Order |
|---|---|
| 12741511000001107 | Lofepramine 35mg/5ml oral suspension 1 ml |
| 12741811000001105 | Lofepramine 35mg/5ml oral suspension 1 ml - Special Order |
| 12812511000001109 | Lofepramine 5mg/5ml oral solution |
| 12799111000001107 | Lofepramine 5mg/5ml oral solution - Special Order |
| 12799011000001106 | Lofepramine 5mg/5ml oral solution 1 ml |
| 12799211000001101 | Lofepramine 5mg/5ml oral solution 1 ml - Special Order |
| 12812611000001108 | Lofepramine 5mg/5ml oral suspension |
| 12798811000001107 | Lofepramine 5mg/5ml oral suspension - Special Order |
| 12798411000001105 | Lofepramine 5mg/5ml oral suspension 1 ml |
| 12798911000001102 | Lofepramine 5mg/5ml oral suspension 1 ml - Special Order |
| 321835001 | Lofepramine 70mg tablets |
| 39699211000001104 | Lofepramine 70mg tablets |
| 493911000001102 | Lofepramine 70mg tablets - A A H Pharmaceuticals Ltd |
| 555511000001106 | Lofepramine 70mg tablets - Accord Healthcare Ltd |
| 668611000001101 | Lofepramine 70mg tablets - Alliance Healthcare (Distribution) Ltd |
| 17971511000001102 | Lofepramine 70mg tablets - Almus Pharmaceuticals Ltd |
| 13404411000001104 | Lofepramine 70mg tablets - Arrow Generics Ltd |
| 24369211000001107 | Lofepramine 70mg tablets - DE Pharmaceuticals |
| 686911000001105 | Lofepramine 70mg tablets - IVAX Pharmaceuticals UK Ltd |
| 798411000001105 | Lofepramine 70mg tablets - Kent Pharmaceuticals Ltd |
| 30222211000001104 | Lofepramine 70mg tablets - Mawdsley-Brooks & Company Ltd |
| 39028711000001103 | Lofepramine 70mg tablets - Medihealth (Northern) Ltd |
| 13804311000001102 | Lofepramine 70mg tablets - Merck Serono Ltd |
| 720011000001106 | Lofepramine 70mg tablets - Mylan |
| 38090011000001107 | Lofepramine 70mg tablets - NorthStar Healthcare Unlimited Company |
| 17937811000001109 | Lofepramine 70mg tablets - Phoenix Healthcare Distribution Ltd |
| 7488611000001103 | Lofepramine 70mg tablets - Sandoz Ltd |
| 29892311000001107 | Lofepramine 70mg tablets - Sigma Pharmaceuticals Plc |
| 373011000001103 | Lofepramine 70mg tablets - Sterwin Medicines |
| 113011000001101 | Lofepramine 70mg tablets - Teva UK Ltd |
| 22073011000001103 | Lofepramine 70mg tablets - Waymade Healthcare Plc |
| 30276711000001106 | Lofepramine 70mg tablets - Zentiva Pharma UK Ltd |
| 1111711000001100 | Lofepramine 70mg tablets 250 tablet |
| 2335111000001104 | Lofepramine 70mg tablets 250 tablet - A A H Pharmaceuticals Ltd |
| 13404611000001101 | Lofepramine 70mg tablets 250 tablet - Arrow Generics Ltd |
| 2336611000001102 | Lofepramine 70mg tablets 250 tablet - Mylan |
| 1279011000001106 | Lofepramine 70mg tablets 56 tablet |
| 2334911000001100 | Lofepramine 70mg tablets 56 tablet - A A H Pharmaceuticals Ltd |
| 2335311000001102 | Lofepramine 70mg tablets 56 tablet - Accord Healthcare Ltd |
| 2338911000001107 | Lofepramine 70mg tablets 56 tablet - Alliance Healthcare (Distribution) Ltd |
| 17971711000001107 | Lofepramine 70mg tablets 56 tablet - Almus Pharmaceuticals Ltd |
| 13404511000001100 | Lofepramine 70mg tablets 56 tablet - Arrow Generics Ltd |
| 24369311000001104 | Lofepramine 70mg tablets 56 tablet - DE Pharmaceuticals |
| 2337011000001107 | Lofepramine 70mg tablets 56 tablet - IVAX Pharmaceuticals UK Ltd |
| 2337311000001105 | Lofepramine 70mg tablets 56 tablet - Kent Pharmaceuticals Ltd |
| 30222311000001107 | Lofepramine 70mg tablets 56 tablet - Mawdsley-Brooks & Company<br>Ltd |
| 39028811000001106 | Lofepramine 70mg tablets 56 tablet - Medihealth (Northern) Ltd |

| 13804411000001109 | Lofepramine 70mg tablets 56 tablet - Merck Serono Ltd |
|---|---|
| 2336311000001107 | Lofepramine 70mg tablets 56 tablet - Mylan |
| 38090211000001102 | Lofepramine 70mg tablets 56 tablet - NorthStar Healthcare Unlimited Company |
| 17937911000001104 | Lofepramine 70mg tablets 56 tablet - Phoenix Healthcare Distribution Ltd |
| 29892411000001100 | Lofepramine 70mg tablets 56 tablet - Sigma Pharmaceuticals Plc |
| 2338611000001101 | Lofepramine 70mg tablets 56 tablet - Sterwin Medicines |
| 2335611000001107 | Lofepramine 70mg tablets 56 tablet - Teva UK Ltd |
| 22073111000001102 | Lofepramine 70mg tablets 56 tablet - Waymade Healthcare Plc |
| 30276811000001103 | Lofepramine 70mg tablets 56 tablet - Zentiva Pharma UK Ltd |
| 12812711000001104 | Lofepramine 70mg/5ml oral solution |
| 12800211000001108 | Lofepramine 70mg/5ml oral solution - Special Order |
| 12800011000001103 | Lofepramine 70mg/5ml oral solution 1 ml |
| 12800411000001107 | Lofepramine 70mg/5ml oral solution 1 ml - Special Order |
| 12812811000001107 | Lofepramine 70mg/5ml oral suspension |
| 12799411000001102 | Lofepramine 70mg/5ml oral suspension - Special Order |
| 12799311000001109 | Lofepramine 70mg/5ml oral suspension 1 ml |
| 12799611000001104 | Lofepramine 70mg/5ml oral suspension 1 ml - Special Order |
| 36040411000001100 | Lofepramine 70mg/5ml oral suspension sugar free |
| 321834002 | Lofepramine 70mg/5ml oral suspension sugar free |
| 33557811000001109 | Lofepramine 70mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd |
| 4071511000001101 | Lofepramine 70mg/5ml oral suspension sugar free - Alliance<br>Healthcare (Distribution) Ltd |
| 28776911000001104 | Lofepramine 70mg/5ml oral suspension sugar free - Colorama Pharmaceuticals Ltd |
| 24369011000001102 | Lofepramine 70mg/5ml oral suspension sugar free - DE Pharmaceuticals |
| 26853211000001108 | Lofepramine 70mg/5ml oral suspension sugar free - Ennogen<br>Healthcare Ltd |
| 28377211000001109 | Lofepramine 70mg/5ml oral suspension sugar free - J M McGill Ltd |
| 29854911000001109 | Lofepramine 70mg/5ml oral suspension sugar free - Niche Pharma Ltd |
| 32758711000001107 | Lofepramine 70mg/5ml oral suspension sugar free - Rosemont Pharmaceuticals Ltd |
| 4071211000001104 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml |
| 33557911000001104 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - A A H<br>Pharmaceuticals Ltd |
| 4071611000001102 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 28777011000001100 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - Colorama Pharmaceuticals Ltd |
| 24369111000001101 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - DE Pharmaceuticals |
| 26853311000001100 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - Ennogen Healthcare Ltd |
| 28377311000001101 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - J M McGill Ltd |
| 29855011000001109 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - Niche<br>Pharma Ltd |
| 32758811000001104 | Lofepramine 70mg/5ml oral suspension sugar free 150 ml - Rosemont Pharmaceuticals Ltd |
| 4071311000001107 | Lomont 70mg/5ml oral suspension - Rosemont Pharmaceuticals Ltd |
| 4071411000001100 | Lomont 70mg/5ml oral suspension 150 ml - Rosemont Pharmaceuticals Ltd |
| 491811000001108 | Motipress tablets - Sanofi-Synthelabo Ltd |

| 2729511000001107 | Motipress tablets 28 tablet - Sanofi-Synthelabo Ltd |
|---|---|
| 39692711000001100 | Nortriptyline 30mg / Fluphenazine 1.5mg tablets |
| 125111000001109 | Motival 10mg/500microgram tablets - Sanofi |
| 2365311000001107 | Motival 10mg/500microgram tablets 100 tablet - Sanofi |
| 39692911000001103 | Nortriptyline 10mg / Fluphenazine 500microgram tablets |
| 1290111000001108 | Nortriptyline 10mg / Fluphenazine 500microgram tablets 100 tablet |
| 1313711000001105 | Nortriptyline 30mg / Fluphenazine 1.5mg tablets 28 tablet |
| 38285811000001101 | Nortriptyline 10mg capsules |
| 39081211000001105 | Nortriptyline 10mg capsules - Alliance Healthcare (Distribution) Ltd |
| 38236211000001104 | Nortriptyline 10mg capsules - Kent Pharmaceuticals Ltd |
| 38236011000001109 | Nortriptyline 10mg capsules 100 capsule |
| 39081311000001102 | Nortriptyline 10mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 38236311000001107 | Nortriptyline 10mg capsules 100 capsule - Kent Pharmaceuticals Ltd |
| 321861002 | Nortriptyline 10mg tablets |
| 39701411000001105 | Nortriptyline 10mg tablets |
| 18310811000001100 | Nortriptyline 10mg tablets - A A H Pharmaceuticals Ltd |
| 24647911000001108 | Nortriptyline 10mg tablets - Accord Healthcare Ltd |
| 34033011000001105 | Nortriptyline 10mg tablets - Advanz Pharma |
| 34694411000001100 | Nortriptyline 10mg tablets - Alissa Healthcare Research Ltd |
| 18865411000001108 | Nortriptyline 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37462011000001107 | Nortriptyline 10mg tablets - DE Pharmaceuticals |
| 36721211000001106 | Nortriptyline 10mg tablets - Flamingo Pharma (UK) Ltd |
| 18670211000001104 | Nortriptyline 10mg tablets - King Pharmaceuticals Ltd |
| 37502911000001101 | Nortriptyline 10mg tablets - Macleods Pharma UK Ltd |
| 39061311000001100 | Nortriptyline 10mg tablets - Medihealth (Northern) Ltd |
| 36044611000001109 | Nortriptyline 10mg tablets - Medreich Plc |
| 37423711000001105 | Nortriptyline 10mg tablets - Mylan |
| 36617511000001102 | Nortriptyline 10mg tablets - Ria Generics Ltd |
| 29951911000001102 | Nortriptyline 10mg tablets - Teva UK Ltd |
| 23931311000001100 | Nortriptyline 10mg tablets - Waymade Healthcare Plc |
| 34105711000001106 | Nortriptyline 10mg tablets - Zentiva Pharma UK Ltd |
| 1088711000001102 | Nortriptyline 10mg tablets 100 tablet |
| 18310911000001105 | Nortriptyline 10mg tablets 100 tablet - A A H Pharmaceuticals Ltd |
| 24648011000001105 | Nortriptyline 10mg tablets 100 tablet - Accord Healthcare Ltd |
| 34033711000001107 | Nortriptyline 10mg tablets 100 tablet - Advanz Pharma |
| 34694511000001101 | Nortriptyline 10mg tablets 100 tablet - Alissa Healthcare Research Ltd |
| 18865511000001107 | Nortriptyline 10mg tablets 100 tablet - Alliance Healthcare (Distribution) Ltd |
| 37462111000001108 | Nortriptyline 10mg tablets 100 tablet - DE Pharmaceuticals |
| 36721311000001103 | Nortriptyline 10mg tablets 100 tablet - Flamingo Pharma (UK) Ltd |
| 18670411000001100 | Nortriptyline 10mg tablets 100 tablet - King Pharmaceuticals Ltd |
| 37503011000001109 | Nortriptyline 10mg tablets 100 tablet - Macleods Pharma UK Ltd |
| 39061411000001107 | Nortriptyline 10mg tablets 100 tablet - Medihealth (Northern) Ltd |
| 36044911000001103 | Nortriptyline 10mg tablets 100 tablet - Medreich Plc |
| 37423911000001107 | Nortriptyline 10mg tablets 100 tablet - Mylan |
| 37100211000001103 | Nortriptyline 10mg tablets 100 tablet - Ria Generics Ltd |
| 29952011000001109 | Nortriptyline 10mg tablets 100 tablet - Teva UK Ltd |
| 23931411000001107 | Nortriptyline 10mg tablets 100 tablet - Waymade Healthcare Plc |
| 34105811000001103 | Nortriptyline 10mg tablets 100 tablet - Zentiva Pharma UK Ltd |

| 36617611000001103 | Nortriptyline 10mg tablets 28 tablet |
|---|---|
| 37873911000001101 | Nortriptyline 10mg tablets 28 tablet - Alliance Healthcare |
| 3/8/3911000001101 | (Distribution) Ltd |
| 36617911000001109 | Nortriptyline 10mg tablets 28 tablet - Ria Generics Ltd |
| 34033311000001108 | Nortriptyline 10mg tablets 30 tablet |
| 34468211000001106 | Nortriptyline 10mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 34033511000001102 | Nortriptyline 10mg tablets 30 tablet - Advanz Pharma |
| 34196111000001102 | Nortriptyline 10mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 39413311000001106 | Nortriptyline 10mg tablets 30 tablet - Flamingo Pharma (UK) Ltd |
| 37423811000001102 | Nortriptyline 10mg tablets 30 tablet - Mylan |
| 36617811000001104 | Nortriptyline 10mg tablets 84 tablet |
| 37874011000001103 | Nortriptyline 10mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd |
| 37760111000001100 | Nortriptyline 10mg tablets 84 tablet - DE Pharmaceuticals |
| 36618211000001101 | Nortriptyline 10mg tablets 84 tablet - Ria Generics Ltd |
| 15000611000001107 | Nortriptyline 10mg/5ml oral solution |
| 14986211000001108 | Nortriptyline 10mg/5ml oral solution - Special Order |
| 14986111000001102 | Nortriptyline 10mg/5ml oral solution 1 ml |
| 14986311000001100 | Nortriptyline 10mg/5ml oral solution 1 ml - Special Order |
| 37868911000001103 | Nortriptyline 10mg/5ml oral solution sugar free |
| 37875011000001104 | Nortriptyline 10mg/5ml oral solution sugar free - Alliance Healthcare |
| | (Distribution) Ltd |
| 37857311000001107 | Nortriptyline 10mg/5ml oral solution sugar free - Colonis Pharma Ltd |
| 37857211000001104 | Nortriptyline 10mg/5ml oral solution sugar free 250 ml |
| 37875111000001103 | Nortriptyline 10mg/5ml oral solution sugar free 250 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 37857411000001100 | Nortriptyline 10mg/5ml oral solution sugar free 250 ml - Colonis<br>Pharma Ltd |
| 15000711000001103 | Nortriptyline 10mg/5ml oral suspension |
| 14986511000001106 | Nortriptyline 10mg/5ml oral suspension - Special Order |
| 14986411000001107 | Nortriptyline 10mg/5ml oral suspension 1 ml |
| 14986611000001105 | Nortriptyline 10mg/5ml oral suspension 1 ml - Special Order |
| 34349511000001102 | Nortriptyline 10mg/5ml oral suspension 100 ml |
| 34349611000001103 | Nortriptyline 10mg/5ml oral suspension 100 ml - Special Order |
| 38285911000001106 | Nortriptyline 25mg capsules |
| 39081411000001109 | Nortriptyline 25mg capsules - Alliance Healthcare (Distribution) Ltd |
| 38235811000001106 | Nortriptyline 25mg capsules - Kent Pharmaceuticals Ltd |
| 38235711000001103 | Nortriptyline 25mg capsules 100 capsule |
| 39081511000001108 | Nortriptyline 25mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 38235911000001101 | Nortriptyline 25mg capsules 100 capsule - Kent Pharmaceuticals Ltd |
| 321864005 | Nortriptyline 25mg tablets |
| 39701511000001109 | Nortriptyline 25mg tablets |
| 18311011000001102 | Nortriptyline 25mg tablets - A A H Pharmaceuticals Ltd |
| 24648311000001108 | Nortriptyline 25mg tablets - Accord Healthcare Ltd |
| 34033211000001100 | Nortriptyline 25mg tablets - Advanz Pharma |
| 34694211000001104 | Nortriptyline 25mg tablets - Alissa Healthcare Research Ltd |
| 19359611000001102 | Nortriptyline 25mg tablets - Alliance Healthcare (Distribution) Ltd |
| 19618311000001102 | Nortriptyline 25mg tablets - DE Pharmaceuticals |
| 37760211000001106 | Nortriptyline 25mg tablets - DE Pharmaceuticals |
| 36721411000001105 | Nortriptyline 25mg tablets - Flamingo Pharma (UK) Ltd |
| L | 1 7 3 5 5 1 N 7 1 2 |

| 16214311000001104 Nortriptyline 25mg tablets - Macleods Pharma UK Ltd | 18876511000001109 | Nortriptyline 25mg tablets - King Pharmaceuticals Ltd |
|---|---|---|
| 37503311000001107 Nortriptyline 25mg tablets - Medilenath (Northern) Ltd | | |
| 30061511000001106 Nortriptyline 25mg tablets - Medinealth (Northern) Ltd 3004511000001105 Nortriptyline 25mg tablets - Medireich Pic 37424011000001105 Nortriptyline 25mg tablets - Medireich Pic 37424011000001101 Nortriptyline 25mg tablets - Ria Generics Ltds 4327311000001101 Nortriptyline 25mg tablets - Sigma Pharmaceuticals Pic 39952111000001105 Nortriptyline 25mg tablets - Sigma Pharmaceuticals Pic 34105911000001108 Nortriptyline 25mg tablets - Valymade Healthcare Pic 34105911000001100 Nortriptyline 25mg tablets - Valymade Healthcare Pic 34105911000001100 Nortriptyline 25mg tablets 100 tablet 34105911000001101 Nortriptyline 25mg tablets 100 tablet - A A H Pharmaceuticals Ltd 34033611000001101 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 346934311000001102 Nortriptyline 25mg tablets 100 tablet - Alisas Healthcare Ltd 34033611000001103 Nortriptyline 25mg tablets 100 tablet - Alisas Healthcare Research Ltd 34033611000001107 Nortriptyline 25mg tablets 100 tablet - Alisas Healthcare Research Ltd 34033611000001109 Nortriptyline 25mg tablets 100 tablet - Alisance Healthcare 34693411000001109 Nortriptyline 25mg tablets 100 tablet - De Pharmaceuticals 34760511000001109 Nortriptyline 25mg tablets 100 tablet - De Pharmaceuticals 347760511000001104 Nortriptyline 25mg tablets 100 tablet - De Pharmaceuticals 3472711000001104 Nortriptyline 25mg tablets 100 tablet - De Pharmaceuticals 3472711000001106 Nortriptyline 25mg tablets 100 tablet - Nortriptyline 25mg tablets | | |
| Nortriptyline 25mg tablets - Medreich Plc | | |
| 37424011000001105 Nortriptyline 25mg tablets - Mylan 36618711000001105 Nortriptyline 25mg tablets - Sigma Pharmaceuticals Ptc 37411000001101 Nortriptyline 25mg tablets - Sigma Pharmaceuticals Ptc 37411000001100 Nortriptyline 25mg tablets - Teva UK Ltd 37411000001100 Nortriptyline 25mg tablets - Teva UK Ltd 37411000001100 Nortriptyline 25mg tablets - Waymade Healthcare Ptc 374011100001101 Nortriptyline 25mg tablets 100 tablet 374011100001101 Nortriptyline 25mg tablets 100 tablet 37401100001101 Nortriptyline 25mg tablets 100 tablet - AA H Pharmaceuticals Ltd 37401100001101 Nortriptyline 25mg tablets 100 tablet - ACord Healthcare Ltd 374033611000001103 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 374033611000001107 Nortriptyline 25mg tablets 100 tablet - Aliance Healthcare Ltd 3740311000001100 Nortriptyline 25mg tablets 100 tablet - Aliance Healthcare (Distribution) Ltd 3740311000001100 Nortriptyline 25mg tablets 100 tablet - Aliance Healthcare (Distribution) Ltd 374011000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 374011000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 374011000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 3740111000001109 Nortriptyline 25mg tablets 100 tablet - Leon (UK) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Leon (UK) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Leon (UK) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Wedihealth (Northern) Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 374011000001100 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 374011000001100 Nortriptyline 25mg tablets 25 tablet 374011000001100 Nortriptyline 25mg | | |
| Nortriptyline 25mg tablets - Ria Generics Ltds | | |
| 14377311000001101 Nortriptyline 25mg tablets - Sigma Pharmaceuticals Pic 29952111000001105 Nortriptyline 25mg tablets - Teva UK Ltd 21204111000001100 Nortriptyline 25mg tablets - Waymade Healthcare Pic 34105911000001100 Nortriptyline 25mg tablets - Waymade Healthcare Pic 34105911000001100 Nortriptyline 25mg tablets 100 tablet - A A H Pharmaceuticals Ltd 34033611000001101 Nortriptyline 25mg tablets 100 tablet - A A H Pharmaceuticals Ltd 34033611000001101 Nortriptyline 25mg tablets 100 tablet - Accord Healthcare Ltd 34033611000001107 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34694311000001107 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34694311000001107 Nortriptyline 25mg tablets 100 tablet - Alissa Healthcare Research Ltd 19360211000001100 Nortriptyline 25mg tablets 100 tablet - Alissa Healthcare (Distribution) Ltd 19360211000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001109 Nortriptyline 25mg tablets 100 tablet - Fiamingo Pharma (UK) Ltd 18876611000001108 Nortriptyline 25mg tablets 100 tablet - Hamingo Pharma (UK) Ltd 18703411000001106 Nortriptyline 25mg tablets 100 tablet - Handedos Pharmaceuticals Ltd 1871411000001106 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18703411000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18703411000001107 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18703711000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18704711000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18704711000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 18704711000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Pic 18704711000001100 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Pic 18704711000001100 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Pic 18704711000001100 Nortriptyline 25mg tablets 25 tablet - Sigma | | |
| 29952111000001105 Nortriptyline 25mg tablets - Teva UK Ltd 34105911000001108 Nortriptyline 25mg tablets - Waynmade Healthcare Plc 34105911000001100 Nortriptyline 25mg tablets - Waynmade Healthcare Plc 34105911000001101 Nortriptyline 25mg tablets 100 tablet - AA H Pharmaceuticals Ltd 34033611000001101 Nortriptyline 25mg tablets 100 tablet - AA H Pharmaceuticals Ltd 34033611000001103 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34033611000001107 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34093811000001107 Nortriptyline 25mg tablets 100 tablet - Alisas Healthcare Research Ltd 19360211000001100 Nortriptyline 25mg tablets 100 tablet - Alisas Healthcare Research Ltd 19360211000001100 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001108 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Ltd 18876611000001106 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Ltd 187503411000001100 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Ltd 18703111000001105 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 187424211000001107 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 187424211000001100 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Plc 18952211000001104 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Plc 19697011000001105 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Plc 1807011000001106 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Plc 1807011000001100 Nortriptyline 25mg tablets 100 tablet - Nariage Pharmaceuticals Plc 1807011000001100 Nortriptyline 25mg tablets 25 tablet 1807011000001100 Nortriptyline 25mg tablets 25 tablet 1807011000001100 Nortriptyline 25mg tablets 25 tablet 1807011000001100 Nortriptyline 25mg tablets 28 tab | | |
| 21204111000001100 Nortriptyline 25mg tablets - Waymade Healthcare Plc 34105911000001100 Nortriptyline 25mg tablets - Zentiva Pharma UK Ltd 969711000001101 Nortriptyline 25mg tablets 100 tablet 18311111000001101 Nortriptyline 25mg tablets 100 tablet - A A H Pharmaceuticals Ltd 24648411000001101 Nortriptyline 25mg tablets 100 tablet - Accord Healthcare Ltd 34033611000001103 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34694311000001107 Nortriptyline 25mg tablets 100 tablet - Aliance Healthcare (Obstribution) Ltd 19360211000001100 Nortriptyline 25mg tablets 100 tablet - Aliance Healthcare (Obstribution) Ltd 19618411000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001108 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001108 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 18876611000001100 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 19061611000001100 Nortriptyline 25mg tablets 100 tablet - Macledos Pharma UK Ltd 19061611000001107 Nortriptyline 25mg tablets 100 tablet - Medrich Plc 1970424211000001107 Nortriptyline 25mg tablets 100 tablet - Medrich Plc 1970424211000001107 Nortriptyline 25mg tablets 100 tablet - Medrich Plc 1970424211000001100 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001104 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 19704211000001104 Nortriptyline 25mg tablets 100 tablet - Vaymade Healthcare Plc 1970411000001106 Nortriptyline 25mg tablets 25 tablet 1970411000001106 Nortriptyline 25mg tablets 25 tablet 1970411000001106 Nortriptyline 25mg tablets 25 tablet 1970411000001106 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals Ltd 19704111000001100 Nortriptyline 25mg tablets 28 tablet - Aliance Healthcare (Di | | |
| 34105911000001108 Nortriptyline 25mg tablets - Zentiva Pharma UK Ltd | | |
| Nortriptyline 25mg tablets 100 tablet | | |
| 18311111000001101 Nortriptyline 25mg tablets 100 tablet - A A H Pharmaceuticals Ltd 24648411000001101 Nortriptyline 25mg tablets 100 tablet - Accord Healthcare Ltd 34033611000001103 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma 34694311000001100 Nortriptyline 25mg tablets 100 tablet - Alissa Healthcare Research Ltd 19360211000001100 Nortriptyline 25mg tablets 100 tablet - Alissa Healthcare Research Ltd 19360411000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001104 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 18214411000001106 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 16214411000001106 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 36045411000001100 Nortriptyline 25mg tablets 100 tablet - Medinealth (Northern) Ltd 37100711000001100 Nortriptyline 25mg tablets 100 tablet - Midenalth (Northern) Ltd 37100711000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 39952211000001104 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 34106011000001106 Nortriptyline 25mg tablets 100 tablet - Tentiva Pharma UK Ltd 4053611000001100 Nortriptyline 25mg tablets 100 tablet - Vaymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 25 tablet 3437611000001101 Nortriptyline 25mg tablets 25 tablet 3437611000001101 Nortriptyline 25mg tablets 25 tablet 3437611000001101 Nortriptyline 25mg tablets 25 tablet - Alliance Healthcare (Distribution) Ltd 3403311000001100 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033111000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmac | | |
| 24648411000001101 Nortriptyline 25mg tablets 100 tablet - Actord Healthcare Ltd | | |
| 3403361100001103 Nortriptyline 25mg tablets 100 tablet - Advanz Pharma | | |
| Nortriptyline 25mg tablets 100 tablet - Alissa Healthcare Research Ltd | | |
| Nortriptyline 25mg tablets 100 tablet - Alliance Healthcare (Distribution) Ltd 19618411000001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001104 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001108 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 16214411000001106 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 37503411000001100 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 39061611000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 390645411000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 390711000001105 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 41063611000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 410453611000001100 Nortriptyline 25mg tablets 25 tablet 4377611000001101 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 25 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 30433411000001100 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 3742411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000 | | |
| Clistribution) Ltd Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 37760511000001104 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001108 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001106 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 16214411000001106 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 37503411000001100 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001107 Nortriptyline 25mg tablets 100 tablet - Medriech Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Medriech Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 34106011000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 25 tablet 31000001100 Nortriptyline 25mg tablets 25 tablet 31000001100 Nortriptyline 25mg tablets 25 tablet 31000001101 Nortriptyline 25mg tablets 25 tablet 31000001101 Nortriptyline 25mg tablets 28 tablet 31000001101 Nortriptyline 25mg tablets 28 tablet 31000001102 Nortriptyline 25mg tablets 28 tablet 31000001103 Nortriptyline 25mg tablets 28 tablet 31000001103 Nortriptyline 25mg tablets 28 tablet 31000001104 Nortriptyline 25mg tablets 28 tablet 310000001106 Nortriptyline 25mg tablets 30 tablet A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet A A H Pharmaceuticals Ltd 34033411000001103 Nortriptyline 25 | | · · · - |
| 3776051100001109 Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals 36721711000001104 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd 18876611000001106 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 1621441100001106 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 37503411000001100 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Medriealth (Northern) Ltd 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001102 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 3410601100001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001100 Nortriptyline 25mg tablets 25 tablet 1437761100001101 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001101 Nortriptyline 25mg tablets 28 tablet - Sigma Pharmaceuticals Plc 37760411000001101 Nortriptyline 25mg tablets 28 tablet - Maymade Healthcare (Distribution) Ltd 37760411000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 3784811000001100 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 378403411000001100 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 34033411000001100 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 34033411000001100 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 34033411000001100 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 376618611000001104 No | 19360211000001100 | (Distribution) Ltd |
| 36721711000001104 Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd | 19618411000001109 | Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals |
| 18876611000001108 Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd 16214411000001106 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 37503411000001100 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001104 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 34053611000001104 Nortriptyline 25mg tablets 25 tablet 3407611000001106 Nortriptyline 25mg tablets 25 tablet 3618511000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 3618511000001103 Nortriptyline 25mg tablets 28 tablet - Waymade Healthcare Plc 37760411000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 34033111000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 3618811000001105 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34033411000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 84 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37760511000001109 | Nortriptyline 25mg tablets 100 tablet - DE Pharmaceuticals |
| 16214411000001106 Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd 37503411000001100 Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 1969701100001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14377611000001106 Nortriptyline 25mg tablets 25 tablet 14377611000001101 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Ibitribution) Ltd 37760411000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Ibitribution) Ltd 34033111000001105 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 84 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 36721711000001104 | Nortriptyline 25mg tablets 100 tablet - Flamingo Pharma (UK) Ltd |
| Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd | 18876611000001108 | Nortriptyline 25mg tablets 100 tablet - King Pharmaceuticals Ltd |
| 39061611000001105 Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 25 tablet 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001102 Nortriptyline 25mg tablets 28 tablet - Waymade Healthcare Plc 37760411000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - A H Pharmaceuticals Ltd 3403411000001104 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Hamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Hamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd | 16214411000001106 | Nortriptyline 25mg tablets 100 tablet - Lexon (UK) Ltd |
| 36045411000001107 Nortriptyline 25mg tablets 100 tablet - Medreich Plc 37424211000001100 Nortriptyline 25mg tablets 100 tablet - Mylan 37100711000001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 19697011000001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 25 tablet 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet - Waymade Healthcare Plc 37760411000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37875711000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001104 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37503411000001100 | Nortriptyline 25mg tablets 100 tablet - Macleods Pharma UK Ltd |
| 3742421100001100 Nortriptyline 25mg tablets 100 tablet - Mylan 3710071100001105 Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd 1969701100001102 Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 2995221100001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 2120421100001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 3410601100001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 1405361100001104 Nortriptyline 25mg tablets 25 tablet 1437761100001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 3027241100001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 3661851100001103 Nortriptyline 25mg tablets 28 tablet 3787411100001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 3776041100001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 3661881100001100 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 3403311100001106 Nortriptyline 25mg tablets 30 tablet 3446831100001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 3403341100001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 3419621100001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 39061611000001105 | Nortriptyline 25mg tablets 100 tablet - Medihealth (Northern) Ltd |
| Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd | 36045411000001107 | Nortriptyline 25mg tablets 100 tablet - Medreich Plc |
| Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc 19952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 12104211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 14106011000001100 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 14053611000001104 Nortriptyline 25mg tablets 25 tablet 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 14377611000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 14377611000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 14377611000001102 Nortriptyline 25mg tablets 28 tablet - Waymade Healthcare Plc 1437761100001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 1457641100001102 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 14618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 14033111000001106 Nortriptyline 25mg tablets 30 tablet 14468311000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 14033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 14196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 14037424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 14037424111000001104 Nortriptyline 25mg tablets 84 tablet 150376711000001104 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37424211000001100 | Nortriptyline 25mg tablets 100 tablet - Mylan |
| 29952211000001104 Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd 21204211000001106 Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 25 tablet 1437761100001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 3776041100001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001101 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37100711000001105 | Nortriptyline 25mg tablets 100 tablet - Ria Generics Ltd |
| Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc 34106011000001100 Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 25 tablet 1437761100001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 3027241100001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 3661851100001103 Nortriptyline 25mg tablets 28 tablet Nortriptyline 25mg tablets 28 tablet Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 3661881100001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 3403311100001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 19697011000001102 | Nortriptyline 25mg tablets 100 tablet - Sigma Pharmaceuticals Plc |
| Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd 14053611000001104 Nortriptyline 25mg tablets 25 tablet 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 29952211000001104 | Nortriptyline 25mg tablets 100 tablet - Teva UK Ltd |
| 14053611000001104 Nortriptyline 25mg tablets 25 tablet 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37875711000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 21204211000001106 | Nortriptyline 25mg tablets 100 tablet - Waymade Healthcare Plc |
| 14377611000001106 Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 34106011000001100 | Nortriptyline 25mg tablets 100 tablet - Zentiva Pharma UK Ltd |
| 30272411000001101 Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 14053611000001104 | Nortriptyline 25mg tablets 25 tablet |
| 36618511000001103 Nortriptyline 25mg tablets 28 tablet 37874111000001102 Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 14377611000001106 | Nortriptyline 25mg tablets 25 tablet - Sigma Pharmaceuticals Plc |
| Nortriptyline 25mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd Nortriptyline 25mg tablets 30 tablet Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd Nortriptyline 25mg tablets 30 tablet - Advanz Pharma Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd Nortriptyline 25mg tablets 30 tablet - Mylan Nortriptyline 25mg tablets 30 tablet - Mylan Nortriptyline 25mg tablets 30 tablet - Mylan Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 30272411000001101 | Nortriptyline 25mg tablets 25 tablet - Waymade Healthcare Plc |
| 37874111000001102 (Distribution) Ltd 37760411000001105 Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 36618511000001103 | · · · - |
| 36618811000001100 Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001104 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37874111000001102 | · · · · |
| 34033111000001106 Nortriptyline 25mg tablets 30 tablet 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37760411000001105 | Nortriptyline 25mg tablets 28 tablet - DE Pharmaceuticals |
| 34468311000001103 Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 36618811000001100 | Nortriptyline 25mg tablets 28 tablet - Ria Generics Ltd |
| 34033411000001101 Nortriptyline 25mg tablets 30 tablet - Advanz Pharma 34196211000001108 Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 34033111000001106 | Nortriptyline 25mg tablets 30 tablet |
| Nortriptyline 25mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd Nortriptyline 25mg tablets 30 tablet - Mylan Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 34468311000001103 | Nortriptyline 25mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 34196211000001108 (Distribution) Ltd 39413411000001104 Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 34033411000001101 | · · · |
| 37424111000001106 Nortriptyline 25mg tablets 30 tablet - Mylan 36618611000001104 Nortriptyline 25mg tablets 84 tablet 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 34196211000001108 | · · · · |
| 36618611000001104 Nortriptyline 25mg tablets 84 tablet Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 39413411000001104 | Nortriptyline 25mg tablets 30 tablet - Flamingo Pharma (UK) Ltd |
| 37875711000001102 Nortriptyline 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd | 37424111000001106 | Nortriptyline 25mg tablets 30 tablet - Mylan |
| 3/8/5/11000001102 (Distribution) Ltd | 36618611000001104 | Nortriptyline 25mg tablets 84 tablet |
| 277C0211000001102 | 37875711000001102 | ' ' ' |
| 3770U311UUUUU11U3 NOrtriptyiine 25mg tablets 84 tablet - DE Pharmaceuticals | 37760311000001103 | Nortriptyline 25mg tablets 84 tablet - DE Pharmaceuticals |

| 36618911000001105 | Nortriptyline 25mg tablets 84 tablet - Ria Generics Ltd |
|---|---|
| 14057111000001104 | Nortriptyline 25mg/5ml oral solution |
| 14019611000001108 | Nortriptyline 25mg/5ml oral solution - Special Order |
| 14019511000001109 | Nortriptyline 25mg/5ml oral solution 1 ml |
| 14019311000001103 | Nortriptyline 25mg/5ml oral solution 1 ml - Special Order |
| 37869011000001107 | Nortriptyline 25mg/5ml oral solution sugar free |
| | Nortriptyline 25mg/5ml oral solution sugar free - Alliance Healthcare |
| 37875211000001109 | (Distribution) Ltd |
| 37857611000001102 | Nortriptyline 25mg/5ml oral solution sugar free - Colonis Pharma Ltd |
| 37857511000001101 | Nortriptyline 25mg/5ml oral solution sugar free 250 ml |
| 37875311000001101 | Nortriptyline 25mg/5ml oral solution sugar free 250 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 37857711000001106 | Nortriptyline 25mg/5ml oral solution sugar free 250 ml - Colonis<br>Pharma Ltd |
| 14057211000001105 | Nortriptyline 25mg/5ml oral suspension |
| 14019911000001102 | Nortriptyline 25mg/5ml oral suspension - Special Order |
| 14019811000001107 | Nortriptyline 25mg/5ml oral suspension 1 ml |
| 14020011000001100 | Nortriptyline 25mg/5ml oral suspension 1 ml - Special Order |
| 34034111000001108 | Nortriptyline 50mg tablets |
| 34468511000001109 | Nortriptyline 50mg tablets - A A H Pharmaceuticals Ltd |
| 34033911000001109 | Nortriptyline 50mg tablets - Advanz Pharma |
| 34196311000001100 | Nortriptyline 50mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37462411000001103 | Nortriptyline 50mg tablets - DE Pharmaceuticals |
| 39061111000001102 | Nortriptyline 50mg tablets - Medihealth (Northern) Ltd |
| 37424311000001108 | Nortriptyline 50mg tablets - Mylan |
| 34033811000001104 | Nortriptyline 50mg tablets 30 tablet |
| 34468611000001108 | Nortriptyline 50mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 34034011000001107 | Nortriptyline 50mg tablets 30 tablet - Advanz Pharma |
| 34196411000001107 | Nortriptyline 50mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 37462511000001104 | Nortriptyline 50mg tablets 30 tablet - DE Pharmaceuticals |
| 39061211000001108 | Nortriptyline 50mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 37424411000001101 | Nortriptyline 50mg tablets 30 tablet - Mylan |
| 35611511000001105 | Nortriptyline 50mg/5ml oral solution |
| 35605011000001102 | Nortriptyline 50mg/5ml oral solution - Special Order |
| 35604911000001102 | Nortriptyline 50mg/5ml oral solution 1 ml |
| 35605111000001101 | Nortriptyline 50mg/5ml oral solution 1 ml - Special Order |
| 34841011000001109 | Nortriptyline 50mg/5ml oral suspension |
| 34824911000001108 | Nortriptyline 50mg/5ml oral suspension - Special Order |
| 34824811000001103 | Nortriptyline 50mg/5ml oral suspension 1 ml |
| 34825011000001108 | Nortriptyline 50mg/5ml oral suspension 1 ml - Special Order |
| 329511000001107 | Prepadine 75mg tablets - Teva UK Ltd |
| 1449911000001108 | Prepadine 75mg tablets 28 tablet - Teva UK Ltd |
| 397711000001101 | Prepadine 25mg capsules - Teva UK Ltd |
| 1444611000001101 | Prepadine 25mg capsules 28 capsule - Teva UK Ltd |
| 16228611000001105 | Prothiaden 25mg capsules - Lexon (UK) Ltd |
| 14344411000001102 | Prothiaden 25mg capsules - Sigma Pharmaceuticals Plc |
| 16586411000001105 | Prothiaden 25mg capsules - Stephar (U.K.) Ltd |
| 208811000001101 | Prothiaden 25mg capsules - Teofarma S.r.l. |
| 10528711000001102 | Prothiaden 25mg capsules - Waymade Healthcare Plc |
| 16228711000001101 | Prothiaden 25mg capsules 100 capsule - Lexon (UK) Ltd |
| | The state of the s |

| 4424454400004402 | D 11: 1 25 1 400 1 6: D1 1: 1 D1 |
|---|---|
| 14344511000001103 | Prothiaden 25mg capsules 100 capsule - Sigma Pharmaceuticals Plc |
| 16586511000001109 | Prothiaden 25mg capsules 100 capsule - Stephar (U.K.) Ltd |
| 1446311000001100 | Prothiaden 25mg capsules 100 capsule - Teofarma S.r.l. |
| 10528911000001100 | Prothiaden 25mg capsules 100 capsule - Waymade Healthcare Plc |
| 17589611000001101 | Prothiaden 25mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 12660011000001106 | Prothiaden 25mg capsules 28 capsule - Teofarma S.r.l. |
| 1446511000001106 | Prothiaden 25mg capsules 600 capsule - Teofarma S.r.l. |
| 5575311000001101 | Prothiaden 75mg tablets - Dowelhurst Ltd |
| 733111000001103 | Prothiaden 75mg tablets - Teofarma S.r.l. |
| 5403111000001102 | Prothiaden 75mg tablets - Waymade Healthcare Plc |
| 5575411000001108 | Prothiaden 75mg tablets 28 tablet - Dowelhurst Ltd |
| 1451511000001100 | Prothiaden 75mg tablets 28 tablet - Teofarma S.r.l. |
| 5403311000001100 | Prothiaden 75mg tablets 28 tablet - Waymade Healthcare Plc |
| 1451711000001105 | Prothiaden 75mg tablets 500 tablet - Teofarma S.r.l. |
| 376651008 | Protriptyline 10mg tablets |
| 11498111000001108 | Protriptyline 10mg tablets 100 tablet |
| 376650009 | Protriptyline 5mg tablets |
| 11498411000001103 | Protriptyline 5mg tablets 100 tablet |
| 11044311000001104 | Sinepin 25mg capsules - Marlborough Pharmaceuticals Ltd |
| 11044411000001106 | Sinepin 25mg capsules 28 capsule - Marlborough Pharmaceuticals Ltd |
| 11044611000001109 | Sinepin 50mg capsules - Marlborough Pharmaceuticals Ltd |
| 11044811000001108 | Sinepin 50mg capsules 28 capsule - Marlborough Pharmaceuticals Ltd |
| 259211000001103 | Sinequan 10mg capsules - Pfizer Ltd |
| 2690011000001105 | Sinequan 10mg capsules 56 capsule - Pfizer Ltd |
| 400611000001102 | Sinequan 25mg capsules - Pfizer Ltd |
| 2691511000001109 | Sinequan 25mg capsules 28 capsule - Pfizer Ltd |
| 621711000001107 | Sinequan 50mg capsules - Pfizer Ltd |
| 2692011000001109 | Sinequan 50mg capsules 28 capsule - Pfizer Ltd |
| 276511000001108 | Sinequan 75mg capsules - Pfizer Ltd |
| 2692911000001108 | Sinequan 75mg capsules 28 capsule - Pfizer Ltd |
| 908011000001108 | Surmontil 10mg tablets - Sanofi |
| 2399811000001102 | Surmontil 10mg tablets 28 tablet - Sanofi |
| 2399611000001101 | Surmontil 10mg tablets 84 tablet - Sanofi |
| 498211000001103 | Surmontil 25mg tablets - Sanofi |
| 2398811000001109 | Surmontil 25mg tablets 28 tablet - Sanofi |
| 2398611000001105 | Surmontil 25mg tablets 84 tablet - Sanofi |
| 101711000001102 | Surmontil 50mg capsules - Sanofi |
| 14622311000001109 | Surmontil 50mg capsules - Sigma Pharmaceuticals Plc |
| 2400111000001106 | Surmontil 50mg capsules 28 capsule - Sanofi |
| 14622411000001102 | Surmontil 50mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 709611000001101 | Thaden 75mg tablets - Opus Pharmaceuticals Ltd |
| 1452211000001105 | Thaden 75mg tablets 28 tablet - Opus Pharmaceuticals Ltd |
| 398211000001107 | Thaden 25mg capsules - Opus Pharmaceuticals Ltd |
| 1447011000001100 | Thaden 25mg capsules 84 capsule - Opus Pharmaceuticals Ltd |
| 16276511000001109 | Tofranil 25mg tablets - Lexon (UK) Ltd |
| 53511000001107 | Tofranil 25mg tablets - Novartis Pharmaceuticals UK Ltd |
| 5425111000001109 | Tofranil 25mg tablets - Novartis Pharmaceuticals OK Etd Tofranil 25mg tablets - Waymade Healthcare Plc |
| 16276611000001108 | Tofranii 25mg tablets 100 tablet - Lexon (UK) Ltd |
| 5425311000001106 | Tofranil 25mg tablets 100 tablet - Waymade Healthcare Plc |

| 2381011000001105 | Tofranil 25mg tablets 84 tablet - Novartis Pharmaceuticals UK Ltd |
|---|---|
| 214311000001103 | Tofranil 25mg/5ml syrup - Novartis Pharmaceuticals UK Ltd |
| 2357211000001103 | Tofranil 25mg/5ml syrup 150 ml - Novartis Pharmaceuticals UK Ltd |
| 321887002 | Trimipramine 10mg tablets |
| 9710311000001109 | Trimipramine 10mg tablets - A A H Pharmaceuticals Ltd |
| 29924711000001102 | Trimipramine 10mg tablets - Advanz Pharma |
| 10350011000001100 | Trimipramine 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37742111000001108 | Trimipramine 10mg tablets - CST Pharma Ltd |
| 37829711000001104 | Trimipramine 10mg tablets - DE Pharmaceuticals |
| 4819911000001102 | Trimipramine 10mg tablets - Kent Pharmaceuticals Ltd |
| 17866611000001105 | Trimipramine 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 37735311000001100 | Trimipramine 10mg tablets - Pilsco Ltd |
| 15200511000001100 | Trimipramine 10mg tablets - Sigma Pharmaceuticals Plc |
| 21906811000001101 | Trimipramine 10mg tablets - Waymade Healthcare Plc |
| 21374111000001103 | Trimipramine 10mg tablets - Zentiva Pharma UK Ltd |
| 37735411000001107 | Trimipramine 10mg tablets 25 tablet |
| 37735511000001106 | Trimipramine 10mg tablets 25 tablet - Pilsco Ltd |
| 1202511000001101 | Trimipramine 10mg tablets 28 tablet |
| 9710411000001102 | Trimipramine 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 29925011000001100 | Trimipramine 10mg tablets 28 tablet - Advanz Pharma |
| 10350111000001104 | Trimipramine 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 37829811000001107 | Trimipramine 10mg tablets 28 tablet - DE Pharmaceuticals |
| 4820211000001105 | Trimipramine 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 17866711000001101 | Trimipramine 10mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 15200611000001101 | Trimipramine 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 21906911000001106 | Trimipramine 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 21374211000001109 | Trimipramine 10mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 37735611000001105 | Trimipramine 10mg tablets 50 tablet |
| 37742211000001102 | Trimipramine 10mg tablets 50 tablet - CST Pharma Ltd |
| 37735911000001104 | Trimipramine 10mg tablets 50 tablet - Pilsco Ltd |
| 1027311000001107 | Trimipramine 10mg tablets 84 tablet |
| 11529711000001104 | Trimipramine 10mg tablets 84 tablet - A A H Pharmaceuticals Ltd |
| 11142711000001103 | Trimipramine 10mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd |
| 4820611000001107 | Trimipramine 10mg tablets 84 tablet - Kent Pharmaceuticals Ltd |
| 17866811000001109 | Trimipramine 10mg tablets 84 tablet - Phoenix Healthcare Distribution<br>Ltd |
| 15200711000001105 | Trimipramine 10mg tablets 84 tablet - Sigma Pharmaceuticals Plc |
| 21907011000001105 | Trimipramine 10mg tablets 84 tablet - Waymade Healthcare Plc |
| 13455011000001100 | Trimipramine 10mg/5ml oral solution |
| 13446011000001107 | Trimipramine 10mg/5ml oral solution - Special Order |
| 13445911000001104 | Trimipramine 10mg/5ml oral solution 1 ml |
| 13446111000001108 | Trimipramine 10mg/5ml oral solution 1 ml - Special Order |
| 13455111000001104 | Trimipramine 10mg/5ml oral suspension |
| 13446611000001100 | Trimipramine 10mg/5ml oral suspension - Special Order |
| 13446511000001104 | Trimipramine 10mg/5ml oral suspension 1 ml |
| 13446711000001109 | Trimipramine 10mg/5ml oral suspension 1 ml - Special Order |
| 13455211000001105 | Trimipramine 125mg/5ml oral solution |
| 13446911000001106 | Trimipramine 125mg/5ml oral solution - Special Order |

| 13446811000001101 | Trimipramine 125mg/5ml oral solution 1 ml |
|---|---|
| 13447011000001105 | Trimipramine 125mg/5ml oral solution 1 ml - Special Order |
| 13455311000001102 | Trimipramine 125mg/5ml oral suspension |
| 13447211000001100 | Trimipramine 125mg/5ml oral suspension - Special Order |
| 13447111000001106 | Trimipramine 125mg/5ml oral suspension 1 ml |
| 13447311000001108 | Trimipramine 125mg/5ml oral suspension 1 ml - Special Order |
| 321888007 | Trimipramine 25mg tablets |
| 9710511000001103 | Trimipramine 25mg tablets - A A H Pharmaceuticals Ltd |
| 29925111000001104 | Trimipramine 25mg tablets - Advanz Pharma |
| 10350211000001105 | Trimipramine 25mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37708211000001108 | Trimipramine 25mg tablets - CST Pharma Ltd |
| 38171811000001108 | Trimipramine 25mg tablets - DE Pharmaceuticals |
| 37829911000001102 | Trimipramine 25mg tablets - DE Pharmaceuticals |
| 4819311000001103 | Trimipramine 25mg tablets - Kent Pharmaceuticals Ltd |
| 17866911000001104 | Trimipramine 25mg tablets - Phoenix Healthcare Distribution Ltd |
| 37736111000001104 | Trimipramine 25mg tablets - Pilsco Ltd |
| 15200811000001102 | Trimipramine 25mg tablets - Pilsco Ltu Trimipramine 25mg tablets - Sigma Pharmaceuticals Plc |
| 21907111000001106 | Trimipramine 25mg tablets - Sigma Pharmaceuticals Pic Trimipramine 25mg tablets - Waymade Healthcare Pic |
| 21373911000001100 | |
| 37711911000001105 | Trimipramine 25mg tablets - Zentiva Pharma UK Ltd |
| | Trimipramine 25mg tablets 100 tablet Trimipramine 25mg tablets 100 tablet. CST Pharma Ltd. |
| 37712011000001103 | Trimipramine 25mg tablets 100 tablet - CST Pharma Ltd |
| 37736211000001102 | Trimipramine 25mg tablets 100 tablet - Pilsco Ltd |
| 984311000001102 | Trimipramine 25mg tablets 28 tablet |
| 9710711000001108 | Trimipramine 25mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 29925211000001105 | Trimipramine 25mg tablets 28 tablet - Advanz Pharma Trimipramine 25mg tablets 28 tablet - Alliance Healthcare |
| 10350311000001102 | (Distribution) Ltd |
| 37830011000001107 | Trimipramine 25mg tablets 28 tablet - DE Pharmaceuticals |
| 4819511000001109 | Trimipramine 25mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 17867111000001104 | Trimipramine 25mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 15200911000001107 | Trimipramine 25mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 21907211000001100 | Trimipramine 25mg tablets 28 tablet - Waymade Healthcare Plc |
| 21374011000001104 | Trimipramine 25mg tablets 28 tablet - Zentiva Pharma UK Ltd |
| 37708011000001103 | Trimipramine 25mg tablets 50 tablet |
| 37708411000001107 | Trimipramine 25mg tablets 50 tablet - CST Pharma Ltd |
| 38171911000001103 | Trimipramine 25mg tablets 50 tablet - DE Pharmaceuticals |
| 1298211000001104 | Trimipramine 25mg tablets 84 tablet |
| 9710811000001100 | Trimipramine 25mg tablets 84 tablet - A A H Pharmaceuticals Ltd |
| 10350411000001109 | Trimipramine 25mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd |
| 4819611000001108 | Trimipramine 25mg tablets 84 tablet - Kent Pharmaceuticals Ltd |
| 17867011000001100 | Trimipramine 25mg tablets 84 tablet - Phoenix Healthcare Distribution Ltd |
| 15201011000001104 | Trimipramine 25mg tablets 84 tablet - Sigma Pharmaceuticals Plc |
| 21907311000001108 | Trimipramine 25mg tablets 84 tablet - Waymade Healthcare Plc |
| 13455411000001109 | Trimipramine 25mg/5ml oral solution |
| 13447811000001104 | Trimipramine 25mg/5ml oral solution - Special Order |
| 13447611000001103 | Trimipramine 25mg/5ml oral solution 1 ml |
| 13448011000001106 | Trimipramine 25mg/5ml oral solution 1 ml - Special Order |
| 13455511000001108 | Trimipramine 25mg/5ml oral suspension |

| 13448211000001101 | Trimipramine 25mg/5ml oral suspension - Special Order |
|---|---|
| 13448111000001107 | Trimipramine 25mg/5ml oral suspension 1 ml |
| 13448311000001109 | Trimipramine 25mg/5ml oral suspension 1 ml - Special Order |
| 321886006 | Trimipramine 50mg capsules |
| 9709811000001106 | Trimipramine 50mg capsules - A A H Pharmaceuticals Ltd |
| 29924311000001101 | Trimipramine 50mg capsules - Advanz Pharma |
| 10349811000001104 | Trimipramine 50mg capsules - Alliance Healthcare (Distribution) Ltd |
| 37659511000001102 | Trimipramine 50mg capsules - CST Pharma Ltd |
| 38171611000001109 | Trimipramine 50mg capsules - DE Pharmaceuticals |
| 4819011000001101 | Trimipramine 50mg capsules - Kent Pharmaceuticals Ltd |
| 30942511000001102 | Trimipramine 50mg capsules - Mawdsley-Brooks & Company Ltd |
| 39076511000001106 | Trimipramine 50mg capsules - Pharmaram Ltd |
| 17866411000001107 | Trimipramine 50mg capsules - Phoenix Healthcare Distribution Ltd |
| 37736311000001105 | Trimipramine 50mg capsules - Pilsco Ltd |
| 15201211000001109 | Trimipramine 50mg capsules - Sigma Pharmaceuticals Plc |
| 21906611000001100 | Trimipramine 50mg capsules - Waymade Healthcare Plc |
| 21373711000001104 | Trimipramine 50mg capsules - Zentiva Pharma UK Ltd |
| 1063111000001109 | Trimipramine 50mg capsules 28 capsule |
| 9710211000001101 | Trimipramine 50mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 29924511000001107 | Trimipramine 50mg capsules 28 capsule - Advanz Pharma |
| 10349911000001109 | Trimipramine 50mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 37659611000001103 | Trimipramine 50mg capsules 28 capsule - CST Pharma Ltd |
| 38171711000001100 | Trimipramine 50mg capsules 28 capsule - DE Pharmaceuticals |
| 4819211000001106 | Trimipramine 50mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 30942611000001103 | Trimipramine 50mg capsules 28 capsule - Mawdsley-Brooks & Company Ltd |
| 39076611000001105 | Trimipramine 50mg capsules 28 capsule - Pharmaram Ltd |
| 17866511000001106 | Trimipramine 50mg capsules 28 capsule - Phoenix Healthcare Distribution Ltd |
| 37736711000001109 | Trimipramine 50mg capsules 28 capsule - Pilsco Ltd |
| 15201411000001108 | Trimipramine 50mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 21906711000001109 | Trimipramine 50mg capsules 28 capsule - Waymade Healthcare Plc |
| 21373811000001107 | Trimipramine 50mg capsules 28 capsule - Zentiva Pharma UK Ltd |
| 13455611000001107 | Trimipramine 50mg/5ml oral solution |
| 13448911000001105 | Trimipramine 50mg/5ml oral solution - Special Order |
| 13448711000001108 | Trimipramine 50mg/5ml oral solution 1 ml |
| 13449011000001101 | Trimipramine 50mg/5ml oral solution 1 ml - Special Order |
| 13455711000001103 | Trimipramine 50mg/5ml oral suspension |
| 13449411000001105 | Trimipramine 50mg/5ml oral suspension - Special Order |
| 13449311000001103 | Trimipramine 50mg/5ml oral suspension 1 ml |
| 13449511000001109 | Trimipramine 50mg/5ml oral suspension 1 ml - Special Order |
| 479411000001101 | Triptafen-M tablets - Mercury Pharma Group Ltd |
| 2195411000001109 | Triptafen-M tablets 100 tablet - Mercury Pharma Group Ltd |
| 514611000001101 | Triptafen tablets - Advanz Pharma |
| 2196511000001101 | Triptafen tablets 100 tablet - Advanz Pharma |
| 11498211000001102 | Vivactil 10mg tablets - Imported (United States) |
| 11498311000001105 | Vivactil 10mg tablets 100 tablet - Imported (United States) |
| 11498511000001104 | Vivactil 5mg tablets - Imported (United States) |
| 11498611000001100 | Vivactil 5mg tablets 100 tablet - Imported (United States) |

| MAOIs | | |
|---|---|---|
| Read V2 Code | Term ID | Description |
| d81 | All | PHENELZINE |
| d811. | All | NARDIL 15mg tablets |
| d81z. | All | PHENELZINE 15mg tablets |
| d83 | All | ISOCARBOXAZID |
| d831. | All | *MARPLAN 10mg tablets |
| d83z. | All | ISOCARBOXAZID 10mg tablets |
| d84 | All | TRANYLCYPROMINE |
| d841. | All | *PARNATE 10mg tablets |
| d84z. | All | TRANYLCYPROMINE 10mg tablets |
| d85 | All | MOCLOBEMIDE |
| d851. | All | MANERIX 150mg tablets |
| d852. | All | MOCLOBEMIDE 150mg tablets |
| d853. | All | MANERIX 300mg tablets |
| d854. | All | MOCLOBEMIDE 300mg tablets |
| Read CTV3 Code | Term ID | Description |
| d83 | All | Isocarboxazid |
| d83z. | All | Isocarboxazid 10mg tablet |
| d831. | All | Marplan 10mg tablet |
| d81 | All | Phenelzine |
| d81z. | All | Phenelzine 15mg tablet |
| d811. | All | Nardil 15mg tablet |
| d84 | All | Tranylcypromine |
| d84z. | All | Tranylcypromine 10mg tablet |
| d841. | All | Parnate 10mg tablet |
| d85 | All | Moclobemide |
| d852. | All | Moclobemide 150mg tablet |
| d851. | All | Manerix 150mg tablet |
| d854. | All | Moclobemide 300mg tablet |
| d853. | All | Manerix 300mg tablet |
| SNOMED Code | Term ID | Description |
| 321908006 | | Isocarboxazid 10mg tablets |
| 3752311000001104 | | Isocarboxazid 10mg tablets - A A H Pharmaceuticals Ltd |
| 3752911000001103 | | Isocarboxazid 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 3752711000001100 | | Isocarboxazid 10mg tablets - Alliance Pharmaceuticals Ltd |
| 26376511000001103 | | Isocarboxazid 10mg tablets - Ennogen Healthcare Ltd |
| 3752111000001101 | | Isocarboxazid 10mg tablets 56 tablet |
| 3752411000001106 | | Isocarboxazid 10mg tablets 56 tablet - A A H Pharmaceuticals Ltd |
| 3753011000001106 | | Isocarboxazid 10mg tablets 56 tablet - Alliance Healthcare (Distribution) Ltd |
| 3752811000001108 | | Isocarboxazid 10mg tablets 56 tablet - Alliance Pharmaceuticals Ltd |
| 26376611000001104 | | Isocarboxazid 10mg tablets 56 tablet - Ennogen Healthcare Ltd |
| 12639611000001104 | | Isocarboxazid 20mg/5ml oral suspension |
| 12610111000001106 | | Isocarboxazid 20mg/5ml oral suspension - Special Order |
| 12610011000001105 | | Isocarboxazid 20mg/5ml oral suspension 1 ml |
| 12610211000001100 | | Isocarboxazid 20mg/5ml oral suspension 1 ml - Special Order |
| 37383611000001103 | | Manerix 150mg tablets - CST Pharma Ltd |
| 5556211000001101 | | Manerix 150mg tablets - Dowelhurst Ltd |

| 538111000001106 | Manerix 150mg tablets - Mylan |
|---|---|
| 17607311000001108 | Manerix 150mg tablets - Necessity Supplies Ltd |
| 14479911000001104 | Manerix 150mg tablets - Sigma Pharmaceuticals Plc |
| 5386611000001108 | Manerix 150mg tablets - Waymade Healthcare Plc |
| 5556711000001108 | Manerix 150mg tablets 100 tablet - Dowelhurst Ltd |
| 37383711000001107 | Manerix 150mg tablets 30 tablet - CST Pharma Ltd |
| 5556311000001109 | Manerix 150mg tablets 30 tablet - Dowelhurst Ltd |
| 2633811000001103 | Manerix 150mg tablets 30 tablet - Mylan |
| 17607411000001101 | Manerix 150mg tablets 30 tablet - Necessity Supplies Ltd |
| 14481111000001108 | Manerix 150mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 5386711000001104 | Manerix 150mg tablets 30 tablet - Waymade Healthcare Plc |
| 37395711000001107 | Manerix 300mg tablets - CST Pharma Ltd |
| 5558211000001100 | Manerix 300mg tablets - Dowelhurst Ltd |
| 48311000001107 | Manerix 300mg tablets - Mylan |
| 17607511000001102 | Manerix 300mg tablets - Necessity Supplies Ltd |
| 5386911000001102 | Manerix 300mg tablets - Waymade Healthcare Plc |
| 37395811000001104 | Manerix 300mg tablets 30 tablet - CST Pharma Ltd |
| 5558411000001101 | Manerix 300mg tablets 30 tablet - Dowelhurst Ltd |
| 2635811000001104 | Manerix 300mg tablets 30 tablet - Mylan |
| 17607611000001103 | Manerix 300mg tablets 30 tablet - Necessity Supplies Ltd |
| 5387011000001103 | Manerix 300mg tablets 30 tablet - Waymade Healthcare Plc |
| 5558811000001104 | Manerix 300mg tablets 60 tablet - Dowelhurst Ltd |
| 321913005 | Moclobemide 150mg tablets |
| 409811000001107 | Moclobemide 150mg tablets - A A H Pharmaceuticals Ltd |
| 906511000001101 | Moclobemide 150mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37687911000001108 | Moclobemide 150mg tablets - CST Pharma Ltd |
| 24401111000001108 | Moclobemide 150mg tablets - DE Pharmaceuticals |
| 5495411000001108 | Moclobemide 150mg tablets - Dowelhurst Ltd |
| 735511000001106 | Moclobemide 150mg tablets - Kent Pharmaceuticals Ltd |
| 30832211000001108 | Moclobemide 150mg tablets - Mawdsley-Brooks & Company Ltd |
| 4621911000001100 | Moclobemide 150mg tablets - Mylan |
| 129211000001100 | Moclobemide 150mg tablets - Sandoz Ltd |
| 15232911000001101 | Moclobemide 150mg tablets - Sigma Pharmaceuticals Plc |
| 823011000001104 | Moclobemide 150mg tablets - Teva UK Ltd |
| 13758911000001104 | Moclobemide 150mg tablets - Tillomed Laboratories Ltd |
| 10541811000001102 | Moclobemide 150mg tablets - Waymade Healthcare Plc |
| 21805611000001100 | Moclobemide 150mg tablets - Waymade Healthcare Plc |
| 5495311000001101 | Moclobemide 150mg tablets 100 tablet |
| 5495711000001102 | Moclobemide 150mg tablets 100 tablet - Dowelhurst Ltd |
| 1132611000001107 | Moclobemide 150mg tablets 30 tablet |
| 2631911000001107 | Moclobemide 150mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 2634411000001102 | Moclobemide 150mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 37688111000001106 | Moclobemide 150mg tablets 30 tablet - CST Pharma Ltd |
| 24401211000001102 | Moclobemide 150mg tablets 30 tablet - DE Pharmaceuticals |
| 5495611000001106 | Moclobemide 150mg tablets 30 tablet - Dowelhurst Ltd |
| 2633211000001104 | Moclobemide 150mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 30832311000001100 | Moclobemide 150mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 4622211000001102 | Moclobemide 150mg tablets 30 tablet - Mylan |

| 2633411000001100 | Moclobemide 150mg tablets 30 tablet - Sandoz Ltd |
|---|---|
| 15233011000001109 | Moclobemide 150mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 2632511000001108 | Moclobemide 150mg tablets 30 tablet - Teva UK Ltd |
| 13759111000001109 | Moclobemide 150mg tablets 30 tablet - Tillomed Laboratories Ltd |
| 10541911000001107 | Moclobemide 150mg tablets 30 tablet - Waymade Healthcare Plc |
| 21806011000001103 | Moclobemide 150mg tablets 30 tablet - Waymade Healthcare Plc |
| 13000111000001109 | Moclobemide 150mg/5ml oral suspension |
| 12981511000001106 | Moclobemide 150mg/5ml oral suspension - Special Order |
| 12981611000001105 | Moclobemide 150mg/5ml oral suspension 1 ml - Special Order |
| 321915003 | Moclobemide 300mg tablets |
| 898011000001104 | Moclobemide 300mg tablets - A A H Pharmaceuticals Ltd |
| 668311000001106 | Moclobemide 300mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37707611000001106 | Moclobemide 300mg tablets - CST Pharma Ltd |
| 24401311000001105 | Moclobemide 300mg tablets - DE Pharmaceuticals |
| 5495911000001100 | Moclobemide 300mg tablets - Dowelhurst Ltd |
| 38961911000001105 | Moclobemide 300mg tablets - Imported |
| 502511000001108 | Moclobemide 300mg tablets - Kent Pharmaceuticals Ltd |
| 4936811000001104 | Moclobemide 300mg tablets - Mylan |
| 934511000001101 | Moclobemide 300mg tablets - Sandoz Ltd |
| 15233111000001105 | Moclobemide 300mg tablets - Sigma Pharmaceuticals Plc |
| 554811000001108 | Moclobemide 300mg tablets - Teva UK Ltd |
| 13759311000001106 | Moclobemide 300mg tablets - Tillomed Laboratories Ltd |
| 1012511000001108 | Moclobemide 300mg tablets 30 tablet |
| 2634811000001100 | Moclobemide 300mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 2636011000001101 | Moclobemide 300mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 37707711000001102 | Moclobemide 300mg tablets 30 tablet - CST Pharma Ltd |
| 24401411000001103 | Moclobemide 300mg tablets 30 tablet - DE Pharmaceuticals |
| 5496011000001108 | Moclobemide 300mg tablets 30 tablet - Dowelhurst Ltd |
| 38962011000001103 | Moclobemide 300mg tablets 30 tablet - Imported |
| 2635211000001100 | Moclobemide 300mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 4936911000001109 | Moclobemide 300mg tablets 30 tablet - Mylan |
| 2635511000001102 | Moclobemide 300mg tablets 30 tablet - Sandoz Ltd |
| 15233211000001104 | Moclobemide 300mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 2635111000001106 | Moclobemide 300mg tablets 30 tablet - Teva UK Ltd |
| 13759411000001104 | Moclobemide 300mg tablets 30 tablet - Tillomed Laboratories Ltd |
| 5495811000001105 | Moclobemide 300mg tablets 60 tablet |
| 5496111000001109 | Moclobemide 300mg tablets 60 tablet - Dowelhurst Ltd |
| 13000211000001103 | Moclobemide 50mg/5ml oral suspension |
| 12982211000001101 | Moclobemide 50mg/5ml oral suspension - Special Order |
| 12981911000001104 | Moclobemide 50mg/5ml oral suspension 1 ml |
| 12982511000001103 | Moclobemide 50mg/5ml oral suspension 1 ml - Special Order |
| 32511000001104 | Nardil 15mg tablets - Neon Healthcare Ltd |
| 2308511000001108 | Nardil 15mg tablets 100 tablet - Neon Healthcare Ltd |
| 38976911000001105 | Phenelzine 15mg capsules |
| 39000111000001109 | Phenelzine 15mg capsules - Imported |
| 38947211000001100 | Phenelzine 15mg capsules - Special Order |
| 38947111000001106 | |
| | Phenelzine 15mg capsules 1 capsule |
| 38947411000001101 | Phenelzine 15mg capsules 1 capsule Phenelzine 15mg capsules 1 capsule - Special Order |

| 39000211000001103 | Phenelzine 15mg capsules 60 capsule - Imported |
|---|---|
| 321902007 | Phenelzine 15mg tablets |
| 37614011000001103 | Phenelzine 15mg tablets - Special Order |
| 37614111000001102 | Phenelzine 15mg tablets 1 tablet |
| 37614211000001108 | Phenelzine 15mg tablets 1 tablet - Special Order |
| 1040811000001104 | Phenelzine 15mg tablets 100 tablet |
| 39708811000001101 | Tranylcypromine 10mg tablets |
| 321910008 | Tranylcypromine 10mg tablets |
| 300511000001109 | Tranylcypromine 10mg tablets - A A H Pharmaceuticals Ltd |
| 845511000001108 | Tranylcypromine 10mg tablets - Advanz Pharma |
| 477311000001103 | Tranylcypromine 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 37686011000001106 | Tranylcypromine 10mg tablets - CST Pharma Ltd |
| 30105311000001105 | Tranylcypromine 10mg tablets - DE Pharmaceuticals |
| 37707211000001109 | Tranylcypromine 10mg tablets - Pilsco Ltd |
| 30991711000001107 | Tranylcypromine 10mg tablets - Teva UK Ltd |
| 28277611000001104 | Tranylcypromine 10mg tablets - Waymade Healthcare Plc |
| 1258911000001104 | Tranylcypromine 10mg tablets 28 tablet |
| 2452811000001107 | Tranylcypromine 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 2453111000001106 | Tranylcypromine 10mg tablets 28 tablet - Advanz Pharma |
| 2453211000001100 | Tranylcypromine 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 37686211000001101 | Tranylcypromine 10mg tablets 28 tablet - CST Pharma Ltd |
| 30105411000001103 | Tranylcypromine 10mg tablets 28 tablet - DE Pharmaceuticals |
| 37707311000001101 | Tranylcypromine 10mg tablets 28 tablet - Pilsco Ltd |
| 30991811000001104 | Tranylcypromine 10mg tablets 28 tablet - Teva UK Ltd |
| 28277711000001108 | Tranylcypromine 10mg tablets 28 tablet - Waymade Healthcare Plc |

| Anxiolytics | | |
|--------------|---------|------------------------------------|
| Read V2 Code | Term ID | Description |
| d21 | All | DIAZEPAM [ANXIOLYTIC] |
| d211. | All | *DIAZEPAM 2mg capsules |
| d212. | All | *DIAZEPAM 5mg capsules |
| d213. | All | DIAZEPAM 2mg tablets |
| d214. | All | DIAZEPAM 5mg tablets |
| d215. | All | DIAZEPAM 10mg tablets |
| d216. | All | DIAZEPAM 2mg/5mL elixir |
| d217. | All | *ALUPRAM 2mg tablets |
| d218. | All | *ALUPRAM 5mg tablets |
| d219. | All | *ALUPRAM 10mg tablets |
| d21A. | All | DIAZEPAM 5mg/5mL oral solution |
| d21B. | All | *RIMAPAM 2mg tablets |
| d21C. | All | *RIMAPAM 5mg tablets |
| d21D. | All | *RIMAPAM 10mg tablets |
| d21E. | All | DIALAR 2mg/5mL syrup |
| d21F. | All | DIALAR 5mg/5mL syrup |
| d21G. | All | *VALCLAIR 10mg suppositories |
| d21J. | All | DIAZEPAM 10mg/5mL suspension |
| d21a. | All | *ATENSINE 2mg tablets |
| d21b. | All | *ATENSINE 5mg tablets |
| d21c. | All | *ATENSINE 10mg tablets |
| d21d. | All | DIAZEMULS 10mg/2mL ampoules |
| d21e. | All | *EVACALM 2mg tablets |
| d21f. | All | *EVACALM 5mg tablets |
| d21g. | All | *SOLIS 2mg capsules |
| d21h. | All | *SOLIS 5mg capsules |
| d21i. | All | *STESOLID 10mg/2mL injection |
| d21j. | All | *STESOLID 20mg/4mL injection |
| d21k. | All | STESOLID 5mg rectal solution |
| d21l. | All | STESOLID 10mg rectal solution |
| d21m. | All | TENSIUM 2mg tablets |
| d21n. | All | TENSIUM 5mg tablets |
| d21o. | All | TENSIUM 10mg tablets |
| d21p. | All | *VALIUM 2mg capsules |
| d21q. | All | *VALIUM 5mg capsules |
| d21r. | All | *VALIUM 2mg tablets |
| d21s. | All | *VALIUM 5mg tablets |
| d21t. | All | *VALIUM 10mg tablets |
| d21u. | All | *VALIUM 2mg/5mL syrup |
| d21v. | All | VALIUM [ANXIOL] 10mg/2mL injection |
| d21w. | All | *VALIUM DUP DEL injection |
| d21x. | All | *VALIUM 5mg suppositories |
| d21y. | All | *VALIUM 10mg suppositories |
| d21z. | All | *DIAZEPAM 10mg suppositories |
| d22 | All | ALPRAZOLAM |
| d221. | All | XANAX 250micrograms tablets |
| d222. | All | XANAX 500micrograms tablets |
| | / 111 | |

| d22y. | All | ALPRAZOLAM 250microgram tablets |
|---|---|---|
| d22z. | All | ALPRAZOLAM 500microgram tablets |
| d24 | All | CHLORDIAZEPOXIDE |
| d241. | All | CHLORDIAZEPOXIDE 5mg capsules |
| d242. | All | CHLORDIAZEPOXIDE 10mg capsules |
| d243. | All | CHLORDIAZER OXIDE TOTAL CAPSULES CHLORDIAZEROXIDE HYDROCHLORIDE 5mg tablets |
| d244. | All | CHLORDIAZEPOXIDE HYDROCHLORIDE 10mg tablets |
| d245. | All | CHLORDIAZEPOXIDE HYDROCHLORIDE 25mg tablets |
| d246. | All | *CHLORDIAZEPOXIDE 5mg tablets |
| d247. | All | *CHLORDIAZEFOXIDE 10mg tablets |
| d248. | All | *CHLORDIAZET OXIDE 10mg tablets *CHLORDIAZEPOXIDE 25mg tablets |
| d249. | All | LIBRIUM 5mg capsules |
| d24a. | All | LIBRIUM 10mg capsules |
| | All | *LIBRIUM 5mg tablets |
| d24b.<br>d24c. | All | *LIBRIUM 10mg tablets |
| | _ | |
| d24c. | All | *LIBRIUM 10mg tablets |
| d24e. | All | *LIBRIUM 100mg injection |
| d24f. | All | TROPIUM 5mg capsules |
| d24g. | All | *TROPIUM 10mg capsules |
| d24h. | All | TROPIUM 5mg tablets |
| d24i. | All | TROPIUM 10mg tablets |
| d24j. | All | *TROPIUM 25mg tablets |
| d26 | All | CLOBAZAM |
| d261. | All | *CLOBAZAM 10mg capsules |
| d262. | All | *FRISIUM 10mg capsules |
| d263. | All | CLOBAZAM 10mg tablets |
| d264. | All | FRISIUM 10mg tablets |
| d265. | All | TAPCLOB 5mg/5mL oral suspension |
| d266. | All | CLOBAZAM 5mg/5mL oral suspension |
| d267. | All | TAPCLOB 10mg/5mL oral suspension |
| d268. | All | CLOBAZAM 10mg/5mL oral suspension |
| d2a | All | LORAZEPAM [ANXIOLYTIC] |
| d2a1. | All | LORAZEPAM 1mg tablets |
| d2a2. | All | LORAZEPAM 2.5mg tablets |
| d2a3. | All | *ALMAZINE 1mg tablets |
| d2a4. | All | *ALMAZINE 2.5mg tablets |
| d2a5. | All | *ATIVAN 1mg tablets |
| d2a6. | All | *ATIVAN 2.5mg tablets |
| d2a7. | All | ATIVAN 4mg/1mL injection |
| d2ax. | All | *ATIVAN 4mg/mL injection |
| d2az. | All | LORAZEPAM 4mg/1mL injection |
| d2d | All | OXAZEPAM |
| d2d1. | All | *OXAZEPAM 30mg capsules |
| d2d2. | All | OXAZEPAM 10mg tablets |
| d2d3. | All | OXAZEPAM 15mg tablets |
| d2d4. | All | OXAZEPAM 30mg tablets |
| d2d5. | All | *OXANID 10mg tablets |
| | All | OVAINID TOTING tablets |
| d2d6. | All | *OXANID 10Hig tablets *OXANID 15mg tablets |

| dn4 | All | CLONAZEPAM [EPILEPSY CONTROL] |
|----------------|---------|-----------------------------------------------|
| dn41. | All | *RIVOTRIL 500mcg tablets |
| dn42. | All | *RIVOTRIL 2mg tablets |
| dn4w. | All | CLONAZEPAM 0.5mg/5mL sugar free oral solution |
| dn4x. | All | CLONAZEPAM 2mg/5mL sugar free oral solution |
| dn4y. | All | CLONAZEPAM 500microgram tablets |
| dn4z. | All | CLONAZEPAM 2mg tablets |
| Read CTV3 Code | Term ID | Description |
| d24 | All | Chlordiazepoxide |
| d246. | All | Chlordiazepoxide 5mg tablet |
| d24b. | All | Librium 5mg tablet |
| d247. | All | Chlordiazepoxide 10mg tablet |
| d24c. | All | Librium 10mg tablet |
| d248. | All | Chlordiazepoxide 25mg tablet |
| d24d. | All | Librium 25mg tablet |
| d241. | All | Chlordiazepoxide hydrochloride 5mg capsule |
| d249. | All | Librium 5mg capsule |
| d24f. | All | Tropium 5mg capsule |
| d242. | All | Chlordiazepoxide hydrochloride 10mg capsule |
| d24a. | All | Librium 10mg capsule |
| d24g. | All | Tropium 10mg capsule |
| d243. | All | Chlordiazepoxide hydrochloride 5mg tablet |
| d24h. | All | Tropium 5mg tablet |
| d244. | All | Chlordiazepoxide hydrochloride 10mg tablet |
| d24i. | All | Tropium 10mg tablet |
| d245. | All | Chlordiazepoxide hydrochloride 25mg tablet |
| d24j. | All | Tropium 25mg tablet |
| d24e. | All | Librium 100mg injection |
| d22 | All | Alprazolam |
| d22y. | All | Alprazolam 250micrograms tablet |
| d221. | All | Xanax 250mcg tablet |
| d22z. | All | Alprazolam 500micrograms tablet |
| d222. | All | Xanax 500mcg tablet |
| x02Lk | All | Clonazepam |
| dn4y. | All | Clonazepam 500micrograms tablet |
| dn41. | All | Rivotril 500mcg tablet |
| dn4z. | All | Clonazepam 2mg tablet |
| dn42. | All | Rivotril 2mg tablet |
| do2z. | All | Clonazepam 1mg/1mL injection |
| do21. | All | Rivotril 1mg/1mL injection |
| dn4w. | All | Clonazepam 0.5mg/5mL s/f oral solution |
| dn4x. | All | Clonazepam 2mg/5mL s/f oral solution |
| dn4 | All | Clonazepam [epilepsy control] |
| do2 | All | Clonazepam [status epilepsy] |
| x02LM | All | Diazepam |
| x01BA | All | Oral diazepam |
| d213. | All | Diazepam 2mg tablet |
| d217. | All | Alupram 2mg tablet |
| d21a. | All | Atensine 2mg tablet |

| d21e. | All | Evacalm 2mg tablet |
|-------|-----|---------------------------------------|
| d21B. | All | Rimapam 2mg tablet |
| d21m. | All | Tensium 2mg tablet |
| d21r. | All | Valium 2mg tablet |
| d214. | All | Diazepam 5mg tablet |
| d218. | All | Alupram 5mg tablet |
| d21n. | All | Tensium 5mg tablet |
| d21s. | All | Valium 5mg tablet |
| d215. | All | Diazepam 10mg tablet |
| d219. | All | Alupram 10mg tablet |
| d21c. | All | Atensine 10mg tablet |
| d21D. | All | Rimapam 10mg tablet |
| d21o. | All | Tensium 10mg tablet |
| d21t. | All | Valium 10mg tablet |
| d211. | All | Diazepam 2mg capsule |
| d21g. | All | Solis 2mg capsule |
| d21p. | All | Valium 2mg capsule |
| d212. | All | Diazepam 5mg capsule |
| d21q. | All | Valium 5mg capsule |
| d21H. | All | Diazepam 1mg/5mL suspension |
| d216. | All | Diazepam 2mg/5mL oral solution |
| d21u. | All | Valium 2mg/5mL syrup |
| d21F. | All | Dialar 5mg/5mL syrup |
| d21J. | All | Diazepam 10mg/5mL suspension |
| x01BB | All | Parenteral diazepam |
| do1w. | All | Diazepam 10mg/2mL injection |
| d21i. | All | Stesolid 10mg/2mL injection |
| do12. | All | Stesolid [ep] 10mg/2mL injection |
| o534. | All | Valium 10mg/2mL injection |
| d21v. | All | Valium [anxiol] 10mg/2ml injection |
| do16. | All | Valium [ep] 10mg/2mL injection |
| d21w. | All | Valium dup del injection |
| do1v. | All | Diazepam 10mg/2mL injection emulsion |
| do11. | All | Diazemuls [ep] 10mg/2mL injection |
| do1z. | All | Diazepam 20mg/4mL injection |
| do17. | All | Valium [ep] 20mg/4mL injection |
| x01BC | All | Rectal diazepam |
| d21x. | All | Valium 5mg suppository |
| d21z. | All | Diazepam 10mg suppository |
| d21y. | All | Valium 10mg suppository |
| do1t. | All | Diazepam 2.5mg/1.25mL rectal solution |
| do1A. | All | Diazepam 2.5mg/1.25mL RecTube |
| do1x. | All | Diazepam 5mg/2.5mL rectal solution |
| do18. | All | Diazepam 5mg/2.5mL RecTube |
| d21k. | All | Stesolid 5mg rectal solution |
| do1y. | All | Diazepam 10mg/2.5mL rectal solution |
| do19. | All | Diazepam 10mg/2.5mL RecTube |
| d21l. | All | Stesolid 10mg rectal solution |
| do1u. | All | Diazepam 20mg/5mL rectal solution |
| | / | - alepan Long, one rectal solution |

| do1B. | All | Diazepam 20mg/5mL RecTube |
|--------------|-----|-------------------------------------|
| d21 | All | Diazepam [anxiolytic] |
| do1 | All | Diazepam [epilepsy use] |
| j81 | All | Diazepam [skeletal muscle relaxant] |
| o53 | All | Diazepam [anaesthesia] |
| x02LN | All | Lorazepam |
| x01BD | All | Oral lorazepam |
| d2a1. | All | Lorazepam 1mg tablet |
| d2a3. | All | Almazine 1mg tablet |
| d2a5. | All | Ativan 1mg tablet |
| d2a2. | All | Lorazepam 2.5mg tablet |
| d2a4. | All | Almazine 2.5mg tablet |
| d2a6. | All | Ativan 2.5mg tablet |
| x01BE | All | Parenteral lorazepam |
| d2az. | All | Lorazepam 4mg/1mL injection |
| d2a7. | All | Ativan 4mg/1mL injection |
| do41. | All | Ativan [ep] 4mg/mL injection |
| d2a | All | Lorazepam [anxiolytic] |
| do4 | All | Lorazepam [epilepsy] |
| o56 | All | Lorazepam [anaesthesia] |
| d2d | All | Oxazepam |
| d2d2. | All | Oxazepam 10mg tablet |
| d2d5. | All | Oxanid 10mg tablet |
| d2d3. | All | Oxazepam 15mg tablet |
| d2d6. | All | Oxanid 15mg tablet |
| d2d4. | All | Oxazepam 30mg tablet |
| d2d7. | All | Oxanid 30mg tablet |
| d2d1. | All | Oxazepam 30mg capsule |
| d1a2. | All | Temazepam 15mg capsule |
| d1a3. | All | Temazepam 20mg capsule |
| d1a7. | All | Normison 20mg capsule |
| d1b | All | Triazolam |
| d1b1. | All | Triazolam 125micrograms tablet |
| d1b3. | All | Halcion 125micrograms tablet |
| d1b2. | All | Triazolam 250micrograms tablet |
| d1b4. | All | Halcion 250micrograms tablet |
| x02Ml | All | Temazepam |
| d1a1. | All | Temazepam 10mg capsule |
| d1a6. | All | Normison 10mg capsule |
| x01BH | All | Buspirone |
| d2f1. | All | Buspirone hydrochloride 5mg tablet |
| d2f2. | All | Buspar 5mg tablet |
| d2f3. | All | Buspar 5mg tablets x126 |
| d2f5. | All | Buspirone hydrochloride 10mg tablet |
| d2f4. | All | Buspar 10mg tablet |
| d2f | All | Buspirone hydrochloride |
| | 1 | <u> </u> |
| d26 | All | Clobazam |
| d26<br>d261. | All | Clobazam Clobazam 10mg capsule |

| dnc1. | All | Clobazam SLS 10mg capsules |
|---|---|---|
| d263. | All | Clobazam 10mg tablet |
| d264. | All | Frisium 10mg tablet |
| d265. | All | TAPCLOB 5mg/5mL oral suspension |
| d266. | All | CLOBAZAM 5mg/5mL oral suspension |
| d267. | All | TAPCLOB 10mg/5mL oral suspension |
| d268. | All | CLOBAZAM 10mg/5mL oral suspension |
| d269. | All | PERIZAM 1mg/mL oral suspension |
| d26A. | All | PERIZAM 2mg/mL oral suspension |
| dnc | All | Clobazam [epilepsy only] |
| d2c | All | Meprobamate |
| d2c1. | All | Meprobamate 200mg tablet |
| d2c3. | All | Equanil 200mg tablet |
| d2c2. | All | Meprobamate 400mg tablet |
| d2c4. | All | Equanil 400mg tablet |
| d2c5. | All | Meprate 400mg tablet |
| d2c6. | All | Tenavoid tablet |
| SNOMED Code | Term ID | Description |
| 321241004 | | Alprazolam 250microgram tablets |
| 4658311000001107 | | Alprazolam 250microgram tablets 60 tablet |
| 4659211000001109 | | Alprazolam 500microgram tablets |
| 3925811000001106 | | Ativan 4mg/1ml solution for injection ampoules - Pfizer Ltd |
| 2026011000001100 | | Ativan 4mg/1ml solution for injection ampoules 10 ampoule - Pfizer |
| 3926011000001109 | | Ltd |
| 39320611000001105 | | Ativan 4mg/1ml solution for injection vials - Imported (Canada) |
| 39320711000001101 | | Ativan 4mg/1ml solution for injection vials 25 vial - Imported (Canada) |
| 737311000001108 | | Buspirone 10mg tablets |
| 10838511000001105 | | Buspirone 10mg tablets 20 tablet |
| 972911000001101 | | Buspirone 10mg tablets 30 tablet |
| 1040411000001101 | | Buspirone 10mg tablets 90 tablet |
| 5107411000001104 | | Buspirone 10mg tablets 100 tablet |
| 19817311000001106 | | Buspirone 5mg tablets - Almus Pharmaceuticals Ltd |
| 17896011000001100 | | Buspirone 5mg tablets - Sigma Pharmaceuticals Plc |
| 1102211000001102 | | Buspirone 5mg tablets 30 tablet |
| 5339211000001106 | | Buspirone 5mg tablets 60 tablet |
| 1195011000001104 | | Buspirone 5mg tablets 90 tablet |
| 16627711000001104 | | Buspirone 10mg tablets - Mylan |
| 15062011000001102 | | Buspirone 10mg tablets - Sigma Pharmaceuticals Plc |
| 22624511000001104 | | Buspirone 5mg tablets - DE Pharmaceuticals |
| 34564611000001106 | | Buspirone 5mg tablets - Teva UK Ltd |
| 292211000001101 | | Buspirone 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 13188711000001102 | | Buspirone 10mg tablets - Dowelhurst Ltd |
| 741511000001107 | | Buspirone 5mg tablets - Accord Healthcare Ltd |
| 32707711000001100 | | Buspirone 5mg tablets - Alissa Healthcare Research Ltd |
| 8299111000001107 | | Buspirone 5mg/5ml oral solution - Special Order |
| 15062211000001107 | | Buspirone 5mg tablets - Sigma Pharmaceuticals Plc |
| 8304411000001106 | | Buspirone 5mg/5ml oral solution |
| 37227511000001106 | | Buspirone 7.5mg tablets - Strides Pharma UK Ltd |

| | Buspirone 10mg tablets - Alissa Healthcare Research Ltd |
|---|---|
| | Buspirone 10mg tablets - DE Pharmaceuticals |
| | Buspirone 10mg tablets - Mawdsley-Brooks & Company Ltd |
| | Buspirone 10mg tablets - Teva UK Ltd |
| | Buspirone 5mg tablets - Dowelhurst Ltd |
| | Buspirone 5mg tablets - Medihealth (Northern) Ltd |
| | Buspirone 10mg tablets - A A H Pharmaceuticals Ltd |
| | Buspirone 10mg tablets - Accord Healthcare Ltd |
| | Buspirone 10mg tablets - Almus Pharmaceuticals Ltd |
| | Buspirone 10mg tablets - Medihealth (Northern) Ltd |
| | Buspirone 10mg tablets - Phoenix Healthcare Distribution Ltd |
| | Buspirone 10mg tablets - Waymade Healthcare Plc |
| | Buspirone 5mg tablets - A A H Pharmaceuticals Ltd |
| | Buspirone 5mg tablets - Alliance Healthcare (Distribution) Ltd |
| | Buspirone 5mg tablets - Kent Pharma (UK) Ltd |
| | Buspirone 5mg tablets - Mawdsley-Brooks & Company Ltd |
| | Buspirone 5mg tablets - Mylan |
| | Buspirone 5mg tablets - Phoenix Healthcare Distribution Ltd |
| | Buspirone 5mg tablets 30 tablet - Waymade Healthcare Plc |
| | Buspirone 5mg tablets - Waymade Healthcare Plc |
| | Buspirone 5mg/5ml oral suspension - Special Order |
| | Buspirone 5mg/5ml oral suspension 1 ml - Special Order |
| | Buspirone 5mg tablets 30 tablet - Mylan |
| | Buspirone 5mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| | Buspirone 5mg tablets 30 tablet - Kent Pharma (UK) Ltd |
| P | Buspirone 5mg tablets 30 tablet - Alliance Healthcare (Distribution) |
| 1 1933011000001107 | Ltd |
| 1932011000001103 | Buspirone 5mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 21807511000001108 | Buspirone 10mg tablets 30 tablet - Waymade Healthcare Plc |
| 22204511000001105 | Buspirone 10mg tablets 30 tablet - Phoenix Healthcare Distribution<br>Ltd |
| 38813211000001107 E | Buspirone 10mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 19817211000001103 | Buspirone 10mg tablets 30 tablet - Almus Pharmaceuticals Ltd |
| 1933311000001105 | Buspirone 10mg tablets 30 tablet - Accord Healthcare Ltd |
| 1933211000001102 | Buspirone 10mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 38813411000001106 | Buspirone 5mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 13189211000001104 E | Buspirone 5mg tablets 30 tablet - Dowelhurst Ltd |
| 34819311000001100 | Buspirone 10mg tablets 30 tablet - Teva UK Ltd |
| 30006011000001105 | Buspirone 10mg tablets 30 tablet - Mawdsley-Brooks & Company Ltd |
| 22624411000001103 E | Buspirone 10mg tablets 30 tablet - DE Pharmaceuticals |
| 32709811000001100 E | Buspirone 10mg tablets 30 tablet - Alissa Healthcare Research Ltd |
| 8299411000001102 E | Buspirone 5mg/5ml oral solution 1 ml - Special Order |
| 37227611000001105 | Buspirone 7.5mg tablets 30 tablet - Strides Pharma UK Ltd |
| 15062311000001104 E | Buspirone 5mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 32709611000001104 E | Buspirone 5mg tablets 30 tablet - Alissa Healthcare Research Ltd |
| 1932211000001108 E | Buspirone 5mg tablets 30 tablet - Accord Healthcare Ltd |
| 13188811000001105 | Buspirone 10mg tablets 30 tablet - Dowelhurst Ltd |
| 1 19338 1 1000001 101 | Buspirone 10mg tablets 30 tablet - Alliance Healthcare (Distribution)<br>Ltd |
| | Buspirone 5mg tablets 30 tablet - Teva UK Ltd |

| 22624611000001100 Buspirone 5mg tablets 30 tablet - DE Pharmaceuticals 15062111000001101 Buspirone 10mg tablets 30 tablet - Sigma Pharmaceuticals Plc 16627911000001102 Buspirone 10mg tablets 30 tablet - Mylan 17896111000001104 Buspirone 5mg tablets 60 tablet - Sigma Pharmaceuticals Plc 19817411000001104 Buspirone 5mg tablets 30 tablet - Almus Pharmaceuticals Ltd 8299811000001100 Buspirone 5mg/5ml oral suspension 1 ml 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001101 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd 16350511000001104 Buspar 10mg tablets - Mawdsley-Brooks & Company Ltd |
|---|
| 16627911000001102 Buspirone 10mg tablets 30 tablet - Mylan 17896111000001104 Buspirone 5mg tablets 60 tablet - Sigma Pharmaceuticals Plc 19817411000001104 Buspirone 5mg tablets 30 tablet - Almus Pharmaceuticals Ltd 8299811000001100 Buspirone 5mg/5ml oral suspension 1 ml 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets - Lexon (UK) Ltd |
| 17896111000001104 Buspirone 5mg tablets 60 tablet - Sigma Pharmaceuticals Plc 19817411000001104 Buspirone 5mg tablets 30 tablet - Almus Pharmaceuticals Ltd 8299811000001100 Buspirone 5mg/5ml oral suspension 1 ml 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001100 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 1933411000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 19817411000001104 Buspirone 5mg tablets 30 tablet - Almus Pharmaceuticals Ltd 8299811000001100 Buspirone 5mg/5ml oral suspension 1 ml 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 8299811000001100 Buspirone 5mg/5ml oral suspension 1 ml 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets - Lexon (UK) Ltd |
| 8304311000001104 Buspirone 5mg/5ml oral suspension 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 37227411000001107 Buspirone 7.5mg tablets 30 tablet 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 5526911000001106 Buspar 5mg tablets - Dowelhurst Ltd 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 5527011000001105 Buspar 5mg tablets 60 tablet - Dowelhurst Ltd 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 737211000001100 Buspar 10mg tablets - IXL Pharma Ltd 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 1933411000001103 Buspar 10mg tablets 90 tablet - IXL Pharma Ltd 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 5107911000001107 Buspar 10mg tablets 100 tablet - IXL Pharma Ltd 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 13838811000001107 Buspar 10mg tablets - DE Pharmaceuticals 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 18548011000001100 Buspar 10mg tablets 20 tablet - DE Pharmaceuticals 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 13839311000001109 Buspar 10mg tablets 30 tablet - DE Pharmaceuticals 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 16143211000001101 Buspar 10mg tablets - Lexon (UK) Ltd |
| 16350711000001109 Buspar 10mg tablets 20 tablet - Mawdsley-Brooks & Company Ltd |
| 16350911000001106 Buspar 10mg tablets 90 tablet - Mawdsley-Brooks & Company Ltd |
| 14300511000001104 Buspar 10mg tablets - Sigma Pharmaceuticals Plc |
| 14301111000001102 Buspar 10mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 5339011000001101 Buspar 10mg tablets - Waymade Healthcare Plc |
| 10838611000001109 Buspar 10mg tablets 20 tablet - Waymade Healthcare Plc |
| 5339111000001100 Buspar 10mg tablets 30 tablet - Waymade Healthcare Plc |
| 14753711000001105 Buspar 10mg tablets 90 tablet - Waymade Healthcare Plc |
| 16143011000001106 Buspar 5mg tablets - Lexon (UK) Ltd |
| 16143111000001107 Buspar 5mg tablets 60 tablet - Lexon (UK) Ltd |
| 5339411000001105 Buspar 5mg tablets - Waymade Healthcare Plc |
| 5339511000001109 Buspar 5mg tablets 60 tablet - Waymade Healthcare Plc |
| 14754011000001105 Buspar 5mg tablets 90 tablet - Waymade Healthcare Plc |
| 5526311000001105 Buspar 10mg tablets - Dowelhurst Ltd |
| 5526511000001104 Buspar 10mg tablets 30 tablet - Dowelhurst Ltd |
| 5526811000001101 Buspar 10mg tablets 90 tablet - Dowelhurst Ltd |
| 365311000001106 Buspar 5mg tablets - IXL Pharma Ltd |
| 1932411000001107 Buspar 5mg tablets 90 tablet - IXL Pharma Ltd |
| 14301511000001106 Buspar 5mg tablets - Sigma Pharmaceuticals Plc |
| 14301811000001109 Buspar 5mg tablets 60 tablet - Sigma Pharmaceuticals Plc |
| 16349311000001104 Buspar 5mg tablets - Mawdsley-Brooks & Company Ltd |
| 16349711000001100 Buspar 5mg tablets 60 tablet - Mawdsley-Brooks & Company Ltd |
| 16349511000001105 Buspar 5mg tablets 90 tablet - Mawdsley-Brooks & Company Ltd |
| 610411000001101 Chlordiazepoxide 10mg capsules - A A H Pharmaceuticals Ltd |
| 805211000001104 Chlordiazepoxide 10mg capsules - Actavis UK Ltd |
| 679411000001104 Chlordiazepoxide 10mg capsules - Alliance Healthcare (Distribution Ltd |
| 28923211000001108 Chlordiazepoxide 10mg capsules - Crescent Pharma Ltd |
| 23815311000001100 Chlordiazepoxide 10mg capsules - DE Pharmaceuticals |
| 13214911000001108 Chlordiazepoxide 10mg capsules - Dowelhurst Ltd |
| 11013611000001101 Chlordiazepoxide 10mg capsules - Dr Reddys Laboratories (UK) Ltd |
| 688011000001105 Chlordiazepoxide 10mg capsules - Kent Pharmaceuticals Ltd |

| 30013111000001104 | Chlordiazepoxide 10mg capsules - Mawdsley-Brooks & Company Ltd |
|---|---|
| 38829611000001104 | Chlordiazepoxide 10mg capsules - Medihealth (Northern) Ltd |
| 17855311000001101 | Chlordiazepoxide 10mg capsules - Phoenix Healthcare Distribution Ltd |
| 3696311000001101 | Chlordiazepoxide 10mg capsules - Ranbaxy (UK) Ltd |
| 7487911000001108 | Chlordiazepoxide 10mg capsules - Sandoz Ltd |
| 15075111000001100 | Chlordiazepoxide 10mg capsules - Sigma Pharmaceuticals Plc |
| 21836311000001106 | Chlordiazepoxide 10mg capsules - Waymade Healthcare Plc |
| 8425211000001106 | Chlordiazepoxide 10mg capsules 100 capsule - A A H Pharmaceuticals Ltd |
| 2305111000001109 | Chlordiazepoxide 10mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 28923311000001100 | Chlordiazepoxide 10mg capsules 100 capsule - Crescent Pharma Ltd |
| 23815511000001106 | Chlordiazepoxide 10mg capsules 100 capsule - DE Pharmaceuticals |
| 11014111000001106 | Chlordiazepoxide 10mg capsules 100 capsule - Dr Reddys Laboratories (UK) Ltd |
| 4324411000001100 | Chlordiazepoxide 10mg capsules 100 capsule - Kent Pharmaceuticals Ltd |
| 30013311000001102 | Chlordiazepoxide 10mg capsules 100 capsule - Mawdsley-Brooks & Company Ltd |
| 38829811000001100 | Chlordiazepoxide 10mg capsules 100 capsule - Medihealth (Northern) Ltd |
| 17855411000001108 | Chlordiazepoxide 10mg capsules 100 capsule - Phoenix Healthcare Distribution Ltd |
| 3696411000001108 | Chlordiazepoxide 10mg capsules 100 capsule - Ranbaxy (UK) Ltd |
| 15075211000001106 | Chlordiazepoxide 10mg capsules 100 capsule - Sigma Pharmaceuticals Plc |
| 21836411000001104 | Chlordiazepoxide 10mg capsules 100 capsule - Waymade Healthcare Plc |
| 28962611000001106 | Chlordiazepoxide 10mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 28878211000001106 | Chlordiazepoxide 10mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 30029711000001106 | Chlordiazepoxide 10mg capsules 28 capsule - DE Pharmaceuticals |
| 28992511000001109 | Chlordiazepoxide 10mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 29785511000001109 | Chlordiazepoxide 10mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 2303311000001105 | Chlordiazepoxide 10mg capsules 500 capsule - A A H Pharmaceuticals Ltd |
| 2303811000001101 | Chlordiazepoxide 10mg capsules 500 capsule - Actavis UK Ltd |
| 2305311000001106 | Chlordiazepoxide 10mg capsules 500 capsule - Alliance Healthcare (Distribution) Ltd |
| 13215011000001108 | Chlordiazepoxide 10mg capsules 500 capsule - Dowelhurst Ltd |
| 11014311000001108 | Chlordiazepoxide 10mg capsules 500 capsule - Dr Reddys Laboratories (UK) Ltd |
| 2304511000001101 | Chlordiazepoxide 10mg capsules 500 capsule - Kent Pharmaceuticals Ltd |
| 17855511000001107 | Chlordiazepoxide 10mg capsules 500 capsule - Phoenix Healthcare Distribution Ltd |
| 3696511000001107 | Chlordiazepoxide 10mg capsules 500 capsule - Ranbaxy (UK) Ltd |
| 7488011000001105 | Chlordiazepoxide 10mg capsules 500 capsule - Sandoz Ltd |
| 8425711000001104 | Chlordiazepoxide 10mg tablets - A A H Pharmaceuticals Ltd |
| 33311000001100 | Chlordiazepoxide 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 23817311000001108 | Chlordiazepoxide 10mg tablets - DE Pharmaceuticals |
| 11014911000001109 | Chlordiazepoxide 10mg tablets - Dr Reddys Laboratories (UK) Ltd |

| 17855811000001105 | Chlordiazepoxide 10mg tablets - Phoenix Healthcare Distribution Ltd |
|---|---|
| 21837211000001101 | Chlordiazepoxide 10mg tablets - Waymade Healthcare Plc |
| 8425811000001107 | Chlordiazepoxide 10mg tablets 100 tablet - A A H Pharmaceuticals Ltd |
| 2455011000001106 | Chlordiazepoxide 10mg tablets 100 tablet - Alliance Healthcare (Distribution) Ltd |
| 23817511000001102 | Chlordiazepoxide 10mg tablets 100 tablet - DE Pharmaceuticals |
| 11015111000001105 | Chlordiazepoxide 10mg tablets 100 tablet - Dr Reddys Laboratories (UK) Ltd |
| 17855911000001100 | Chlordiazepoxide 10mg tablets 100 tablet - Phoenix Healthcare Distribution Ltd |
| 21837411000001102 | Chlordiazepoxide 10mg tablets 100 tablet - Waymade Healthcare Plc |
| 8425911000001102 | Chlordiazepoxide 10mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 2455111000001107 | Chlordiazepoxide 10mg tablets 500 tablet - Alliance Healthcare (Distribution) Ltd |
| 21837511000001103 | Chlordiazepoxide 10mg tablets 500 tablet - Waymade Healthcare Plc |
| 12404111000001101 | Chlordiazepoxide 10mg/5ml oral solution - Special Order |
| 12404411000001106 | Chlordiazepoxide 10mg/5ml oral solution 1 ml - Special Order |
| 12402811000001102 | Chlordiazepoxide 10mg/5ml oral suspension - Special Order |
| 12402911000001107 | Chlordiazepoxide 10mg/5ml oral suspension 1 ml - Special Order |
| 16133911000001109 | Chlordiazepoxide 2.5mg/5ml oral solution - Special Order |
| 16134011000001107 | Chlordiazepoxide 2.5mg/5ml oral solution 1 ml - Special Order |
| 16134611000001100 | Chlordiazepoxide 2.5mg/5ml oral suspension - Special Order |
| 16134711000001109 | Chlordiazepoxide 2.5mg/5ml oral suspension 1 ml - Special Order |
| 20159211000001109 | Chlordiazepoxide 2.5mg/5ml oral suspension 50 ml - Special Order |
| 12406911000001106 | Chlordiazepoxide 4mg/5ml oral solution - Special Order |
| 12407111000001106 | Chlordiazepoxide 4mg/5ml oral solution 1 ml - Special Order |
| 12405811000001109 | Chlordiazepoxide 4mg/5ml oral suspension - Special Order |
| 12406111000001108 | Chlordiazepoxide 4mg/5ml oral suspension 1 ml - Special Order |
| 299111000001103 | Chlordiazepoxide 5mg capsules - A A H Pharmaceuticals Ltd |
| 620311000001103 | Chlordiazepoxide 5mg capsules - Actavis UK Ltd |
| 202211000001104 | Chlordiazepoxide 5mg capsules - Alliance Healthcare (Distribution) Ltd |
| 28923011000001103 | Chlordiazepoxide 5mg capsules - Crescent Pharma Ltd |
| 23816311000001105 | Chlordiazepoxide 5mg capsules - DE Pharmaceuticals |
| 13215111000001109 | Chlordiazepoxide 5mg capsules - Dowelhurst Ltd |
| 11012911000001100 | Chlordiazepoxide 5mg capsules - Dr Reddys Laboratories (UK) Ltd |
| 47111000001109 | Chlordiazepoxide 5mg capsules - Kent Pharmaceuticals Ltd |
| 38829911000001105 | Chlordiazepoxide 5mg capsules - Medihealth (Northern) Ltd |
| 17855011000001104 | Chlordiazepoxide 5mg capsules - Phoenix Healthcare Distribution Ltd |
| 3696011000001104 | Chlordiazepoxide 5mg capsules - Ranbaxy (UK) Ltd |
| 7487311000001107 | Chlordiazepoxide 5mg capsules - Sandoz Ltd |
| 15075311000001103 | Chlordiazepoxide 5mg capsules - Sigma Pharmaceuticals Plc |
| 21834311000001100 | Chlordiazepoxide 5mg capsules - Waymade Healthcare Plc |
| 8425111000001100 | Chlordiazepoxide 5mg capsules 100 capsule - A A H Pharmaceuticals Ltd |
| 2307211000001106 | Chlordiazepoxide 5mg capsules 100 capsule - Alliance Healthcare (Distribution) Ltd |
| 28923111000001102 | Chlordiazepoxide 5mg capsules 100 capsule - Crescent Pharma Ltd |
| 23816711000001109 | Chlordiazepoxide 5mg capsules 100 capsule - DE Pharmaceuticals |
| 11013111000001109 | Chlordiazepoxide 5mg capsules 100 capsule - Dr Reddys Laboratories (UK) Ltd |

| 4224241000001107 | Chlordiazepoxide 5mg capsules 100 capsule - Kent Pharmaceuticals |
|---|---|
| 4324311000001107 | Ltd |
| 38830011000001100 | Chlordiazepoxide 5mg capsules 100 capsule - Medihealth (Northern) Ltd |
| 17855111000001103 | Chlordiazepoxide 5mg capsules 100 capsule - Phoenix Healthcare Distribution Ltd |
| 3696111000001103 | Chlordiazepoxide 5mg capsules 100 capsule - Ranbaxy (UK) Ltd |
| 15075411000001105 | Chlordiazepoxide 5mg capsules 100 capsule - Sigma Pharmaceuticals Plc |
| 21834411000001107 | Chlordiazepoxide 5mg capsules 100 capsule - Waymade Healthcare Plc |
| 28962511000001107 | Chlordiazepoxide 5mg capsules 28 capsule - A A H Pharmaceuticals Ltd |
| 28878011000001101 | Chlordiazepoxide 5mg capsules 28 capsule - Alliance Healthcare (Distribution) Ltd |
| 30029511000001101 | Chlordiazepoxide 5mg capsules 28 capsule - DE Pharmaceuticals |
| 28992411000001105 | Chlordiazepoxide 5mg capsules 28 capsule - Kent Pharmaceuticals Ltd |
| 29785611000001108 | Chlordiazepoxide 5mg capsules 28 capsule - Sigma Pharmaceuticals Plc |
| 2306111000001103 | Chlordiazepoxide 5mg capsules 500 capsule - A A H Pharmaceuticals Ltd |
| 2306411000001108 | Chlordiazepoxide 5mg capsules 500 capsule - Actavis UK Ltd |
| 2307411000001105 | Chlordiazepoxide 5mg capsules 500 capsule - Alliance Healthcare (Distribution) Ltd |
| 13215211000001103 | Chlordiazepoxide 5mg capsules 500 capsule - Dowelhurst Ltd |
| 11013311000001106 | Chlordiazepoxide 5mg capsules 500 capsule - Dr Reddys Laboratories (UK) Ltd |
| 2307111000001100 | Chlordiazepoxide 5mg capsules 500 capsule - Kent Pharmaceuticals Ltd |
| 17855211000001109 | Chlordiazepoxide 5mg capsules 500 capsule - Phoenix Healthcare Distribution Ltd |
| 3696211000001109 | Chlordiazepoxide 5mg capsules 500 capsule - Ranbaxy (UK) Ltd |
| 7487611000001102 | Chlordiazepoxide 5mg capsules 500 capsule - Sandoz Ltd |
| 8425311000001103 | Chlordiazepoxide 5mg tablets - A A H Pharmaceuticals Ltd |
| 257511000001107 | Chlordiazepoxide 5mg tablets - Alliance Healthcare (Distribution) Ltd |
| 11014511000001102 | Chlordiazepoxide 5mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 28879611000001104 | Chlordiazepoxide 5mg tablets - Ennogen Healthcare Ltd |
| 17855611000001106 | Chlordiazepoxide 5mg tablets - Phoenix Healthcare Distribution Ltd |
| 21836511000001100 | Chlordiazepoxide 5mg tablets - Waymade Healthcare Plc |
| 8425511000001109 | Chlordiazepoxide 5mg tablets 100 tablet - A A H Pharmaceuticals Ltd |
| 2455811000001100 | Chlordiazepoxide 5mg tablets 100 tablet - Alliance Healthcare (Distribution) Ltd |
| 11014611000001103 | Chlordiazepoxide 5mg tablets 100 tablet - Dr Reddys Laboratories (UK) Ltd |
| 28879711000001108 | Chlordiazepoxide 5mg tablets 100 tablet - Ennogen Healthcare Ltd |
| 17855711000001102 | Chlordiazepoxide 5mg tablets 100 tablet - Phoenix Healthcare Distribution Ltd |
| 21836711000001105 | Chlordiazepoxide 5mg tablets 100 tablet - Waymade Healthcare Plc |
| 8425611000001108 | Chlordiazepoxide 5mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 2456011000001102 | Chlordiazepoxide 5mg tablets 500 tablet - Alliance Healthcare (Distribution) Ltd |
| 8337411000001108 | Chlordiazepoxide 5mg/5ml oral suspension - Special Order |
| 8337711000001102 | Chlordiazepoxide 5mg/5ml oral suspension 1 ml - Special Order |
| 23318011000001108 | Chlordiazepoxide 7.5mg/5ml oral suspension - Special Order |
| 23318111000001109 | Chlordiazepoxide 7.5mg/5ml oral suspension 1 ml - Special Order |
| | . 3, 1, |

| 23318211000001103 | Chlordiazepoxide 7.5mg/5ml oral suspension 100 ml - Special Order |
|---|---|
| 14410111000001100 | Clobazam 1.25mg/5ml oral solution |
| 14349311000001105 | Clobazam 1.25mg/5ml oral solution - Special Order |
| 14349111000001108 | Clobazam 1.25mg/5ml oral solution 1 ml |
| 14349511000001104 | Clobazam 1.25mg/5ml oral solution 1 ml - Special Order |
| 14410211000001106 | Clobazam 1.25mg/5ml oral suspension |
| 14350111000001101 | Clobazam 1.25mg/5ml oral suspension - Special Order |
| 14349811000001101 | Clobazam 1.25mg/5ml oral suspension 1 ml |
| 14350311000001104 | Clobazam 1.25mg/5ml oral suspension 1 ml - Special Order |
| 12021911000001100 | Clobazam 1.5mg/5ml oral solution |
| 11959111000001109 | Clobazam 1.5mg/5ml oral solution - Special Order |
| 11959011000001108 | Clobazam 1.5mg/5ml oral solution 1 ml |
| 11959211000001103 | Clobazam 1.5mg/5ml oral solution 1 ml - Special Order |
| 12022011000001107 | Clobazam 1.5mg/5ml oral suspension |
| 11958811000001109 | Clobazam 1.5mg/5ml oral suspension - Special Order |
| 11958711000001103 | Clobazam 1.5mg/5ml oral suspension 1 ml |
| 11958911000001101 | Clobazam 1.5mg/5ml oral suspension 1 ml - Special Order |
| 12022111000001108 | Clobazam 100mg/5ml oral solution |
| 11959611000001101 | Clobazam 100mg/5ml oral solution - Special Order |
| 11959711000001101 | |
| 11959811000001103 | Clobazam 100mg/5ml oral solution 1 ml |
| 12022211000001102 | Clobazam 100mg/5ml oral solution 1 ml - Special Order |
| | Clobazam 100mg/5ml oral suspension |
| 11959411000001104 | Clobazam 100mg/5ml oral suspension - Special Order |
| 11959311000001106 | Clobazam 100mg/5ml oral suspension 1 ml |
| 11959511000001100 | Clobazam 100mg/5ml oral suspension 1 ml - Special Order |
| 321272000<br>10356611000001109 | Clobazam 10mg tablets Clobazam 10mg tablets - A A H Pharmaceuticals Ltd |
| 15628011000001102 | Clobazam 10mg tablets - Accord Healthcare Ltd |
| 16641011000001109 | Clobazam 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 30042411000001109 | Clobazam 10mg tablets - Alliance Healthcare (Distribution) Eta Clobazam 10mg tablets - DE Pharmaceuticals |
| 32397611000001108 | Clobazam 10mg tablets - Kent Pharmaceuticals Ltd |
| 38843311000001109 | Clobazam 10mg tablets - Medihealth (Northern) Ltd |
| 17860211000001109 | Clobazam 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 29789511000001107 | Clobazam 10mg tablets - Frioemx Healthcare Distribution Eta Clobazam 10mg tablets - Sigma Pharmaceuticals Plc |
| 18389711000001107 | Clobazam 10mg tablets - Signia Pharmaceuticals Pic Clobazam 10mg tablets - Teva UK Ltd |
| 21858711000001104 | |
| | Clobazam 10mg tablets - Waymade Healthcare Plc |
| 30280311000001100 | Clobazam 10mg tablets - Waymade Healthcare Plc |
| 13164511000001102 | Clobazam 10mg tablets 20 tablet Clobazam 10mg tablets 20 tablet. Waymado Healtheare Blo |
| 30280411000001107 | Clobazam 10mg tablets 20 tablet - Waymade Healthcare Plc |
| 1034311000001101 | Clobazam 10mg tablets 30 tablet |
| 10356711000001100 | Clobazam 10mg tablets 30 tablet - A A H Pharmaceuticals Ltd |
| 15628111000001101 | Clobazam 10mg tablets 30 tablet - Accord Healthcare Ltd |
| 16641111000001105 | Clobazam 10mg tablets 30 tablet - Alliance Healthcare (Distribution) Ltd |
| 30042511000001108 | Clobazam 10mg tablets 30 tablet - DE Pharmaceuticals |
| 32397811000001107 | Clobazam 10mg tablets 30 tablet - Kent Pharmaceuticals Ltd |
| 38843411000001102 | Clobazam 10mg tablets 30 tablet - Medihealth (Northern) Ltd |
| 17860311000001103 | Clobazam 10mg tablets 30 tablet - Phoenix Healthcare Distribution Ltd |
| 29789611000001106 | Clobazam 10mg tablets 30 tablet - Sigma Pharmaceuticals Plc |

| 10200011000001107 | Claharana 10ma tahlata 20 tahlat. Tana 117 Ital |
|---|---|
| 18389811000001107 | Clobazam 10mg tablets 30 tablet - Teva UK Ltd |
| 21858811000001102 | Clobazam 10mg tablets 30 tablet - Waymade Healthcare Plc |
| 14243711000001104 | Clobazam 10mg tablets 50 tablet |
| 12560411000001109 | Clobazam 10mg tablets 60 tablet |
| 8360711000001105 | Clobazam 10mg/5ml oral solution |
| 8352311000001102 | Clobazam 10mg/5ml oral solution - Special Order |
| 8351411000001104 | Clobazam 10mg/5ml oral solution 1 ml |
| 8352911000001101 | Clobazam 10mg/5ml oral solution 1 ml - Special Order |
| 19595911000001100 | Clobazam 10mg/5ml oral solution 50 ml |
| 19596111000001109 | Clobazam 10mg/5ml oral solution 50 ml - Special Order |
| 8360811000001102 | Clobazam 10mg/5ml oral suspension |
| 8354811000001100 | Clobazam 10mg/5ml oral suspension - Special Order |
| 8354211000001101 | Clobazam 10mg/5ml oral suspension 1 ml |
| 8356011000001101 | Clobazam 10mg/5ml oral suspension 1 ml - Special Order |
| 19933411000001109 | Clobazam 10mg/5ml oral suspension 100 ml |
| 19933511000001108 | Clobazam 10mg/5ml oral suspension 100 ml - Special Order |
| 19596211000001103 | Clobazam 10mg/5ml oral suspension 50 ml |
| 19596411000001104 | Clobazam 10mg/5ml oral suspension 50 ml - Special Order |
| 21856411000001100 | Clobazam 10mg/5ml oral suspension sugar free |
| 29933611000001106 | Clobazam 10mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd |
| 38336811000001105 | Clobazam 10mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd |
| 37471111000001107 | Clobazam 10mg/5ml oral suspension sugar free - Atnahs Pharma UK |
| 37225911000001109 | Clobazam 10mg/5ml oral suspension sugar free - DE Pharmaceuticals |
| 38843511000001103 | Clobazam 10mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd |
| 31954311000001108 | Clobazam 10mg/5ml oral suspension sugar free - Thame Laboratories Ltd |
| 37921711000001106 | Clobazam 10mg/5ml oral suspension sugar free - Wockhardt UK Ltd |
| 21803311000001109 | Clobazam 10mg/5ml oral suspension sugar free 150 ml |
| 29933711000001102 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 38336911000001100 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 37471611000001104 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - Atnahs<br>Pharma UK Ltd |
| 37226011000001101 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - DE Pharmaceuticals |
| 38843611000001104 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - Medihealth (Northern) Ltd |
| 31954511000001102 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - Thame Laboratories Ltd |
| 37921811000001103 | Clobazam 10mg/5ml oral suspension sugar free 150 ml - Wockhardt UK Ltd |
| 30926011000001107 | Clobazam 10mg/5ml oral suspension sugar free 250 ml |
| 31064311000001105 | Clobazam 10mg/5ml oral suspension sugar free 250 ml - A A H Pharmaceuticals Ltd |
| 8360011000001108 | Clobazam 12.5mg/5ml oral solution |
| 8344911000001107 | Clobazam 12.5mg/5ml oral solution - Special Order |
| 8344711000001105 | Clobazam 12.5mg/5ml oral solution 1 ml |
| 8345011000001107 | Clobazam 12.5mg/5ml oral solution 1 ml - Special Order |
| 8360111000001109 | Clobazam 12.5mg/5ml oral suspension |
| | - 0, |

| 8345411000001103 | Clobazam 12.5mg/5ml oral suspension - Special Order |
|-------------------|----------------------------------------------------------|
| 8345211000001102 | Clobazam 12.5mg/5ml oral suspension 1 ml |
| 8345511000001104 | Clobazam 12.5mg/5ml oral suspension 1 ml - Special Order |
| 12022311000001105 | Clobazam 120mg/5ml oral solution |
| 11960311000001107 | Clobazam 120mg/5ml oral solution - Special Order |
| 11960211000001104 | Clobazam 120mg/5ml oral solution 1 ml |
| 11960411000001100 | Clobazam 120mg/5ml oral solution 1 ml - Special Order |
| 12022411000001103 | Clobazam 120mg/5ml oral suspension |
| 11960011000001109 | Clobazam 120mg/5ml oral suspension - Special Order |
| 11959911000001107 | Clobazam 120mg/5ml oral suspension 1 ml |
| 11960111000001105 | Clobazam 120mg/5ml oral suspension 1 ml - Special Order |
| 8360911000001107 | Clobazam 15mg/5ml oral solution |
| 8352711000001103 | Clobazam 15mg/5ml oral solution - Special Order |
| 8352511000001108 | Clobazam 15mg/5ml oral solution 1 ml |
| 8353111000001105 | Clobazam 15mg/5ml oral solution 1 ml - Special Order |
| 8361011000001104 | Clobazam 15mg/5ml oral suspension |
| 8355011000001105 | Clobazam 15mg/5ml oral suspension - Special Order |
| 8354311000001109 | Clobazam 15mg/5ml oral suspension 1 ml |
| 8355811000001104 | Clobazam 15mg/5ml oral suspension 1 ml - Special Order |
| 8360211000001103 | Clobazam 1mg/5ml oral solution |
| 8348911000001100 | Clobazam 1mg/5ml oral solution - Special Order |
| 8348411000001108 | Clobazam 1mg/5ml oral solution 1 ml |
| 8349811000001103 | Clobazam 1mg/5ml oral solution 1 ml - Special Order |
| 8361111000001103 | Clobazam 1mg/5ml oral suspension |
| 8352611000001107 | Clobazam 1mg/5ml oral suspension - Special Order |
| 8352411000001109 | Clobazam 1mg/5ml oral suspension 1 ml |
| 8352811000001106 | Clobazam 1mg/5ml oral suspension 1 ml - Special Order |
| 8792211000001101 | Clobazam 2.5mg capsules |
| 8747011000001101 | Clobazam 2.5mg capsules - Special Order |
| 8746911000001100 | Clobazam 2.5mg capsules 1 capsule |
| 8748211000001105 | Clobazam 2.5mg capsules 1 capsule - Special Order |
| 8361211000001109 | Clobazam 2.5mg/5ml oral solution |
| 8356711000001104 | Clobazam 2.5mg/5ml oral solution - Special Order |
| 8356411000001105 | Clobazam 2.5mg/5ml oral solution 1 ml |
| 8356911000001102 | Clobazam 2.5mg/5ml oral solution 1 ml - Special Order |
| 8361311000001101 | Clobazam 2.5mg/5ml oral suspension |
| 8357211000001108 | Clobazam 2.5mg/5ml oral suspension - Special Order |
| 8357011000001103 | Clobazam 2.5mg/5ml oral suspension 1 ml |
| 8357811000001109 | Clobazam 2.5mg/5ml oral suspension 1 ml - Special Order |
| 8366211000001101 | Clobazam 20mg/5ml oral solution |
| 8362811000001101 | Clobazam 20mg/5ml oral solution - Special Order |
| 8362311000001105 | Clobazam 20mg/5ml oral solution 1 ml |
| 8363111000001102 | Clobazam 20mg/5ml oral solution 1 ml - Special Order |
| 8366311000001109 | Clobazam 20mg/5ml oral suspension |
| 8366111000001107 | Clobazam 20mg/5ml oral suspension - Special Order |
| 8365911000001103 | Clobazam 20mg/5ml oral suspension 1 ml |
| 8368211000001100 | Clobazam 20mg/5ml oral suspension 1 ml - Special Order |
| 12022511000001104 | Clobazam 250micrograms/5ml oral solution |
| 11961411000001109 | Clobazam 250micrograms/5ml oral solution - Special Order |
| <u> </u> | |

| 11961311000001102 | Clobazam 250micrograms/5ml oral solution 1 ml |
|---|---|
| 11961511000001108 | Clobazam 250micrograms/5ml oral solution 1 ml - Special Order |
| 12022611000001100 | Clobazam 250micrograms/5ml oral suspension |
| 11961111000001104 | Clobazam 250micrograms/5ml oral suspension - Special Order |
| 11960511000001101 | Clobazam 250micrograms/5ml oral suspension 1 ml |
| 11961211000001105 | Clobazam 250micrograms/5ml oral suspension 1 ml - Special Order |
| 8366411000001102 | Clobazam 25mg/5ml oral solution |
| 8362011000001107 | Clobazam 25mg/5ml oral solution - Special Order |
| 8361811000001105 | Clobazam 25mg/5ml oral solution 1 ml |
| 8362211000001102 | Clobazam 25mg/5ml oral solution 1 ml - Special Order |
| 8366611000001104 | Clobazam 25mg/5ml oral suspension |
| 8363211000001108 | Clobazam 25mg/5ml oral suspension - Special Order |
| 8362911000001106 | Clobazam 25mg/5ml oral suspension 1 ml |
| 8363411000001107 | Clobazam 25mg/5ml oral suspension 1 ml - Special Order |
| 8366711000001108 | Clobazam 2mg/5ml oral solution |
| 8363011000001103 | Clobazam 2mg/5ml oral solution - Special Order |
| 8362711000001109 | Clobazam 2mg/5ml oral solution 1 ml |
| 8363311000001100 | Clobazam 2mg/5ml oral solution 1 ml - Special Order |
| 8366811000001100 | Clobazam 2mg/5ml oral suspension |
| 8363911000001104 | Clobazam 2mg/5ml oral suspension - Special Order |
| 8363711000001101 | Clobazam 2mg/5ml oral suspension 1 ml |
| 8364211000001106 | Clobazam 2mg/5ml oral suspension 1 ml - Special Order |
| 8366911000001105 | Clobazam 3.5mg/5ml oral solution |
| 8361911000001100 | Clobazam 3.5mg/5ml oral solution - Special Order |
| 8361711000001102 | Clobazam 3.5mg/5ml oral solution 1 ml |
| 8362111000001108 | Clobazam 3.5mg/5ml oral solution 1 ml - Special Order |
| 8367111000001105 | Clobazam 3.5mg/5ml oral suspension |
| 8362511000001104 | Clobazam 3.5mg/5ml oral suspension - Special Order |
| 8362411000001103 | Clobazam 3.5mg/5ml oral suspension 1 ml |
| 8362611000001100 | Clobazam 3.5mg/5ml oral suspension 1 ml - Special Order |
| 12022811000001101 | Clobazam 3.75mg/5ml oral solution |
| 11962311000001106 | Clobazam 3.75mg/5ml oral solution - Special Order |
| 11962211000001103 | Clobazam 3.75mg/5ml oral solution 1 ml |
| 11962411000001104 | Clobazam 3.75mg/5ml oral solution 1 ml - Special Order |
| 12022911000001106 | Clobazam 3.75mg/5ml oral suspension |
| 11962011000001108 | Clobazam 3.75mg/5ml oral suspension - Special Order |
| 11961911000001101 | Clobazam 3.75mg/5ml oral suspension 1 ml |
| 11962111000001109 | Clobazam 3.75mg/5ml oral suspension 1 ml - Special Order |
| 12023011000001103 | Clobazam 32.5mg/5ml oral solution |
| 11962911000001107 | Clobazam 32.5mg/5ml oral solution - Special Order |
| 11962811000001102 | Clobazam 32.5mg/5ml oral solution 1 ml |
| 11963011000001104 | Clobazam 32.5mg/5ml oral solution 1 ml - Special Order |
| 12023111000001102 | Clobazam 32.5mg/5ml oral suspension |
| 11962611000001101 | Clobazam 32.5mg/5ml oral suspension - Special Order |
| 11962511000001100 | Clobazam 32.5mg/5ml oral suspension 1 ml |
| 11962711000001105 | Clobazam 32.5mg/5ml oral suspension 1 ml - Special Order |
| 8367211000001104 | Clobazam 4mg/5ml oral solution |
| 8363611000001105 | Clobazam 4mg/5ml oral solution - Special Order |
| 8363511000001106 | Clobazam 4mg/5ml oral solution 1 ml |

| Sa64411000001105 | | |
|---|---|---|
| | 8367411000001100 | Clobazam 4mg/5ml oral suspension |
| Clobazam 500m//sml oral suspension 1 ml - Special Order | 8364411000001105 | Clobazam 4mg/5ml oral suspension - Special Order |
| 12023311000001100 | 8364011000001101 | Clobazam 4mg/5ml oral suspension 1 ml |
| 11963511000001107 | 8364911000001102 | Clobazam 4mg/5ml oral suspension 1 ml - Special Order |
| 11963411000001108 | 12023311000001100 | Clobazam 500micrograms/5ml oral solution |
| 1963611000001106 | 11963511000001107 | Clobazam 500micrograms/5ml oral solution - Special Order |
| 12023511000001106 | 11963411000001108 | Clobazam 500micrograms/5ml oral solution 1 ml |
| 11963211000001109 | 11963611000001106 | Clobazam 500micrograms/5ml oral solution 1 ml - Special Order |
| 11963111000001101 | 12023511000001106 | Clobazam 500micrograms/5ml oral suspension |
| 11963311000001101 | 11963211000001109 | Clobazam 500micrograms/5ml oral suspension - Special Order |
| Sa67511000001101 | 11963111000001103 | Clobazam 500micrograms/5ml oral suspension 1 ml |
| Sa64311000001103 | 11963311000001101 | Clobazam 500micrograms/5ml oral suspension 1 ml - Special Order |
| Sa6411100001100 | 8367511000001101 | Clobazam 50mg/5ml oral solution |
| 3364111000001100 | 8364311000001103 | Clobazam 50mg/5ml oral solution - Special Order |
| 384511000001109 | | |
| Sa67611000001102 | 8364511000001109 | |
| S36471100001104 | | |
| Sa6481100001108 | | |
| Sa6841100001107 | | |
| Sa68611000001103 | | - ' |
| Sa67711000001106 | | |
| Sa67011000001109 Clobazam Smg/5ml oral solution 1 ml | | |
| Sa68111000001106 | | |
| 19596611000001101 | | |
| 19605611000001104 Clobazam 5mg/5ml oral solution 100 ml - Special Order | | |
| Sa6881100001104 Clobazam Smg/5ml oral suspension | | |
| Sa6871100001107 Clobazam 5mg/5ml oral suspension - Special Order | | |
| Sa6841100001101 Clobazam 5mg/5ml oral suspension 1 ml | | |
| Clobazam 5mg/5ml oral suspension 1 ml - Special Order | | |
| 19596811000001102 Clobazam 5mg/5ml oral suspension 100 ml 19597011000001101 Clobazam 5mg/5ml oral suspension 100 ml - Special Order 21856511000001101 Clobazam 5mg/5ml oral suspension sugar free 29933411000001108 Clobazam 5mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd 38337011000001101 Clobazam 5mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd 37471711000001108 Clobazam 5mg/5ml oral suspension sugar free - Atnahs Pharma UK Ltd 37225711000001107 Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals 2010 Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd 21953611000001101 Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd 21802611000001104 Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd 21802611000001109 Clobazam 5mg/5ml oral suspension sugar free 150 ml 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd 38337111000001100 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | | |
| 19597011000001106 Clobazam 5mg/5ml oral suspension 100 ml - Special Order 21856511000001101 Clobazam 5mg/5ml oral suspension sugar free 29933411000001108 Clobazam 5mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd 38337011000001101 Clobazam 5mg/5ml oral suspension sugar free - Aliance Healthcare (Distribution) Ltd 37471711000001108 Clobazam 5mg/5ml oral suspension sugar free - Atnahs Pharma UK Ltd 37225711000001107 Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd 37921211000001104 Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd 21802611000001109 Clobazam 5mg/5ml oral suspension sugar free 150 ml 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd | | i i |
| 21856511000001101 Clobazam 5mg/5ml oral suspension sugar free 29933411000001108 Clobazam 5mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd 38337011000001101 Clobazam 5mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd 37471711000001108 Clobazam 5mg/5ml oral suspension sugar free - Atnahs Pharma UK Ltd 37225711000001107 Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd 31953611000001101 Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd 37921211000001104 Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd 21802611000001109 Clobazam 5mg/5ml oral suspension sugar free 150 ml 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd 38337111000001100 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | | |
| Clobazam 5mg/5ml oral suspension sugar free - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free - Atnahs Pharma UK Ltd Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | | |
| Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free - Atnahs Pharma UK Ltd Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals Smg/5ml oral suspension sugar free - DE Pharmaceuticals Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 21856511000001101 | |
| (Distribution) Ltd | 29933411000001108 | Pharmaceuticals Ltd |
| 37471711000001108 Ltd Clobazam 5mg/5ml oral suspension sugar free - DE Pharmaceuticals Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Clobazam 5mg/5ml oral suspension sugar free 150 ml - A H Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 38337011000001101 | |
| Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 37471711000001108 | |
| Clobazam 5mg/5ml oral suspension sugar free - Medihealth (Northern) Ltd 31953611000001101 Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 37225711000001107 | |
| Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 38843711000001108 | |
| 37921211000001104 Clobazam 5mg/5ml oral suspension sugar free - Wockhardt UK Ltd 21802611000001109 Clobazam 5mg/5ml oral suspension sugar free 150 ml 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd 38337111000001100 Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 31953611000001101 | Clobazam 5mg/5ml oral suspension sugar free - Thame Laboratories |
| 21802611000001109 Clobazam 5mg/5ml oral suspension sugar free 150 ml 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 37921211000001104 | |
| 29933511000001107 Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H Pharmaceuticals Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | | |
| 38337111000001100 Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance Healthcare (Distribution) Ltd Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | | Clobazam 5mg/5ml oral suspension sugar free 150 ml - A A H |
| Clobazam 5mg/5ml oral suspension sugar free 150 ml - Atnahs | 38337111000001100 | Clobazam 5mg/5ml oral suspension sugar free 150 ml - Alliance |
| I Harring OK Etg | 37471811000001100 | |

| 27225044000004404 | Clobazam 5mg/5ml oral suspension sugar free 150 ml - DE |
|---|---|
| 37225811000001104 | Pharmaceuticals |
| 38843811000001100 | Clobazam 5mg/5ml oral suspension sugar free 150 ml - Medihealth (Northern) Ltd |
| 31954011000001105 | Clobazam 5mg/5ml oral suspension sugar free 150 ml - Thame<br>Laboratories Ltd |
| 37921311000001107 | Clobazam 5mg/5ml oral suspension sugar free 150 ml - Wockhardt UK Ltd |
| 30926211000001102 | Clobazam 5mg/5ml oral suspension sugar free 250 ml |
| 31064211000001102 | Clobazam 5mg/5ml oral suspension sugar free 250 ml - A A H Pharmaceuticals Ltd |
| 12023611000001105 | Clobazam 600micrograms/5ml oral solution |
| 11964111000001101 | Clobazam 600micrograms/5ml oral solution - Special Order |
| 11964011000001102 | Clobazam 600micrograms/5ml oral solution 1 ml |
| 11964211000001107 | Clobazam 600micrograms/5ml oral solution 1 ml - Special Order |
| 12023811000001109 | Clobazam 600micrograms/5ml oral suspension |
| 11963811000001105 | Clobazam 600micrograms/5ml oral suspension - Special Order |
| 11963711000001102 | Clobazam 600micrograms/5ml oral suspension 1 ml |
| 11963911000001100 | Clobazam 600micrograms/5ml oral suspension 1 ml - Special Order |
| 8367811000001103 | Clobazam 6mg/5ml oral solution |
| 8365111000001101 | Clobazam 6mg/5ml oral solution - Special Order |
| 8365011000001102 | Clobazam 6mg/5ml oral solution 1 ml |
| 8365211000001107 | Clobazam 6mg/5ml oral solution 1 ml - Special Order |
| 8368011000001105 | Clobazam 6mg/5ml oral suspension |
| 8365411000001106 | Clobazam 6mg/5ml oral suspension - Special Order |
| 8365311000001104 | Clobazam 6mg/5ml oral suspension 1 ml |
| 8365511000001105 | Clobazam 6mg/5ml oral suspension 1 ml - Special Order |
| 12024011000001101 | Clobazam 7.5mg/5ml oral solution |
| 11964711000001100 | Clobazam 7.5mg/5ml oral solution - Special Order |
| 11964611000001109 | Clobazam 7.5mg/5ml oral solution 1 ml |
| 11964811000001108 | Clobazam 7.5mg/5ml oral solution 1 ml - Special Order |
| 12024111000001100 | Clobazam 7.5mg/5ml oral suspension |
| 11964411000001106 | Clobazam 7.5mg/5ml oral suspension - Special Order |
| 11964311000001104 | Clobazam 7.5mg/5ml oral suspension 1 ml |
| 11964511000001105 | Clobazam 7.5mg/5ml oral suspension 1 ml - Special Order |
| 12024311000001103 | Clobazam 750micrograms/5ml oral solution |
| 11965311000001100 | Clobazam 750micrograms/5ml oral solution - Special Order |
| 11965211000001108 | Clobazam 750micrograms/5ml oral solution 1 ml |
| 11965411000001107 | Clobazam 750micrograms/5ml oral solution 1 ml - Special Order |
| 12024411000001105 | Clobazam 750micrograms/5ml oral suspension |
| 11965011000001103 | Clobazam 750micrograms/5ml oral suspension - Special Order |
| 11964911000001103 | Clobazam 750micrograms/5ml oral suspension 1 ml |
| 11965111000001102 | Clobazam 750micrograms/5ml oral suspension 1 ml - Special Order |
| 12024511000001109 | Clobazam 7mg/5ml oral solution |
| 11965911000001104 | Clobazam 7mg/5ml oral solution - Special Order |
| 11965811000001109 | Clobazam 7mg/5ml oral solution 1 ml |
| 11966011000001107 | Clobazam 7mg/5ml oral solution 1 ml - Special Order |
| 12024611000001108 | Clobazam 7mg/5ml oral suspension |
| 11965611000001105 | Clobazam 7mg/5ml oral suspension - Special Order |
| 11965511000001106 | Clobazam 7mg/5ml oral suspension 1 ml |
| 11965711000001101 | Clobazam 7mg/5ml oral suspension 1 ml - Special Order |
| 11707/11000001101 | Cionazam 7mg/2mii orai saspension 1 mii - speciai oraei |

| 12024811000001107 | Clobazam 8mg/5ml oral solution |
|---|---|
| 11966511000001104 | Clobazam 8mg/5ml oral solution - Special Order |
| 11966411000001103 | Clobazam 8mg/5ml oral solution 1 ml |
| 11966611000001100 | Clobazam 8mg/5ml oral solution 1 ml - Special Order |
| 12024911000001102 | Clobazam 8mg/5ml oral suspension |
| 11966211000001102 | Clobazam 8mg/5ml oral suspension - Special Order |
| 11966111000001108 | Clobazam 8mg/5ml oral suspension 1 ml |
| 11966311000001105 | Clobazam 8mg/5ml oral suspension 1 ml - Special Order |
| 12025011000001102 | Clobazam 9mg/5ml oral solution |
| 11967111000001106 | Clobazam 9mg/5ml oral solution - Special Order |
| 11967011000001105 | Clobazam 9mg/5ml oral solution 1 ml |
| 11967211000001100 | Clobazam 9mg/5ml oral solution 1 ml - Special Order |
| 12025111000001101 | Clobazam 9mg/5ml oral suspension |
| 11966811000001101 | Clobazam 9mg/5ml oral suspension - Special Order |
| 11966711000001109 | Clobazam 9mg/5ml oral suspension 1 ml |
| 11966911000001106 | Clobazam 9mg/5ml oral suspension 1 ml - Special Order |
| 8382211000001104 | Clonazepam 1.25mg/5ml oral solution |
| 8372811000001109 | Clonazepam 1.25mg/5ml oral solution - Special Order |
| 8372611000001105 | Clonazepam 1.25mg/5ml oral solution 1 ml |
| 8373211000001103 | Clonazepam 1.25mg/5ml oral solution 1 ml - Special Order |
| 8382311000001107<br>8374311000001107 | Clonazepam 1.25mg/5ml oral suspension Clonazepam 1.25mg/5ml oral suspension - Special Order |
| 8373711000001107 | Clonazepam 1.25mg/5ml oral suspension 1 ml |
| 8374511000001109 | Clonazepam 1.25mg/5ml oral suspension 1 ml - Special Order |
| 11943811000001101 | Clonazepam 1.2mg/5ml oral solution |
| 11938711000001101 | Clonazepam 1.2mg/5ml oral solution - Special Order |
| 11938711000001102 | Clonazepam 1.2mg/5ml oral solution 1 ml |
| 11938811000001105 | Clonazepam 1.2mg/5ml oral solution 1 ml - Special Order |
| 11943911000001106 | Clonazepam 1.2mg/5ml oral suspension |
| 11938411000001108 | Clonazepam 1.2mg/5ml oral suspension - Special Order |
| 11938311000001101 | Clonazepam 1.2mg/5ml oral suspension 1 ml |
| 11938511000001101 | Clonazepam 1.2mg/5ml oral suspension 1 ml - Special Order |
| 8382411000001100 | Clonazepam 1.5mg/5ml oral solution |
| 8371211000001101 | Clonazepam 1.5mg/5ml oral solution - Special Order |
| 8371211000001101 | Clonazepam 1.5mg/5ml oral solution 1 ml |
| 8371711000001108 | Clonazepam 1.5mg/5ml oral solution 1 ml - Special Order |
| 8382511000001101 | Clonazepam 1.5mg/5ml oral suspension |
| 837211100001101 | Clonazepam 1.5mg/5ml oral suspension - Special Order |
| 837211100001102 | Clonazepam 1.5mg/5ml oral suspension 1 ml |
| 8372411000001107 | Clonazepam 1.5mg/5ml oral suspension 1 ml - Special Order |
| 11939311000001107 | Clonazepam 100micrograms/5ml oral solution - Special Order |
| 11939311000001107 | Clonazepam 100micrograms/5ml oral solution - Special Order Clonazepam 100micrograms/5ml oral solution 1 ml - Special Order |
| 11939411000001100 | Clonazepam 100micrograms/5ml oral suspension |
| 11939011000001109 | Clonazepam 100micrograms/5ml oral suspension - Special Order |
| 11938911000001109 | Clonazepam 100micrograms/5ml oral suspension 1 ml |
| | Clonazepam 100micrograms/5ml oral suspension 1 ml - Special |
| 11939111000001105 | Order |
| 20459211000001108 | Clonazepam 100micrograms/5ml oral suspension 100 ml |
| 20459311000001100 | Clonazepam 100micrograms/5ml oral suspension 100 ml - Special Order |

| 8382911000001108 | Clonazepam 10mg/5ml oral solution |
|---|---|
| 8373411000001103 | Clonazepam 10mg/5ml oral solution - Special Order |
| 8373311000001105 | Clonazepam 10mg/5ml oral solution 1 ml |
| 8373511000001104 | Clonazepam 10mg/5ml oral solution 1 ml - Special Order |
| 8383011000001100 | Clonazepam 10mg/5ml oral suspension |
| 8374111000001105 | Clonazepam 10mg/5ml oral suspension - Special Order |
| 8374011000001109 | Clonazepam 10mg/5ml oral suspension 1 ml |
| 8374211000001104 | Clonazepam 10mg/5ml oral suspension 1 ml - Special Order |
| 11944211000001104 | Clonazepam 12.5mg/5ml oral solution |
| 11939911000001108 | Clonazepam 12.5mg/5ml oral solution - Special Order |
| 11939811000001103 | Clonazepam 12.5mg/5ml oral solution 1 ml |
| 11940011000001102 | Clonazepam 12.5mg/5ml oral solution 1 ml - Special Order |
| 11944311000001107 | Clonazepam 12.5mg/5ml oral suspension |
| 11939611000001102 | Clonazepam 12.5mg/5ml oral suspension - Special Order |
| 11939511000001101 | Clonazepam 12.5mg/5ml oral suspension 1 ml |
| 11939711000001106 | Clonazepam 12.5mg/5ml oral suspension 1 ml - Special Order |
| 11944411000001100 | Clonazepam 120micrograms/5ml oral solution |
| 11940511000001105 | Clonazepam 120micrograms/5ml oral solution - Special Order |
| 11940411000001106 | Clonazepam 120micrograms/5ml oral solution 1 ml |
| 11940611000001109 | Clonazepam 120micrograms/5ml oral solution 1 ml - Special Order |
| 11944511000001101 | Clonazepam 120micrograms/5ml oral suspension |
| 11940211000001107 | Clonazepam 120micrograms/5ml oral suspension - Special Order |
| 11940111000001101 | Clonazepam 120micrograms/5ml oral suspension 1 ml |
| | Clonazepam 120micrograms/5ml oral suspension 1 ml - Special |
| 11940311000001104 | Order |
| 11944611000001102 | Clonazepam 125micrograms/5ml oral solution |
| 11941111000001107 | Clonazepam 125micrograms/5ml oral solution - Special Order |
| 11941011000001106 | Clonazepam 125micrograms/5ml oral solution 1 ml |
| 11941211000001101 | Clonazepam 125micrograms/5ml oral solution 1 ml - Special Order |
| 11944711000001106 | Clonazepam 125micrograms/5ml oral suspension |
| 11940811000001108 | Clonazepam 125micrograms/5ml oral suspension - Special Order |
| 11940711000001100 | Clonazepam 125micrograms/5ml oral suspension 1 ml |
| 11940911000001103 | Clonazepam 125micrograms/5ml oral suspension 1 ml - Special Order |
| 11954511000001104 | Clonazepam 150micrograms/5ml oral solution |
| 11941711000001108 | Clonazepam 150micrograms/5ml oral solution - Special Order |
| 11941611000001104 | Clonazepam 150micrograms/5ml oral solution 1 ml |
| 11941811000001100 | Clonazepam 150micrograms/5ml oral solution 1 ml - Special Order |
| 11954611000001100 | Clonazepam 150micrograms/5ml oral suspension |
| 11941411000001102 | Clonazepam 150micrograms/5ml oral suspension - Special Order |
| 11941311000001109 | Clonazepam 150micrograms/5ml oral suspension 1 ml |
| 11941511000001103 | Clonazepam 150micrograms/5ml oral suspension 1 ml - Special Order |
| 11954711000001109 | Clonazepam 160micrograms/5ml oral solution |
| 11942311000001100 | Clonazepam 160micrograms/5ml oral solution - Special Order |
| 11942211000001108 | Clonazepam 160micrograms/5ml oral solution 1 ml |
| | Cl 460 : /5 |
| 11942411000001107 | Clonazepam 160micrograms/5ml oral solution 1 ml - Special Order |
| 11942411000001107<br>11954811000001101 | Clonazepam 160micrograms/5ml oral suspension Clonazepam 160micrograms/5ml oral suspension |
| 11942111000001102 | Clonazepam 160micrograms/5ml oral suspension 1 ml - Special Order |
|---|---|
| 8394911000001100 | Clonazepam 180micrograms/5ml oral solution |
| 8377711000001104 | Clonazepam 180micrograms/5ml oral solution - Special Order |
| 8376911000001100 | Clonazepam 180micrograms/5ml oral solution 1 ml |
| 8378211000001105 | Clonazepam 180micrograms/5ml oral solution 1 ml - Special Order |
| 8395011000001100 | Clonazepam 180micrograms/5ml oral suspension |
| 8378911000001101 | Clonazepam 180micrograms/5ml oral suspension - Special Order |
| 8378811000001106 | Clonazepam 180micrograms/5ml oral suspension 1 ml |
| 8379211000001100 | Clonazepam 180micrograms/5ml oral suspension 1 ml - Special Order |
| 8395111000001104 | Clonazepam 1mg/5ml oral solution |
| 8378711000001103 | Clonazepam 1mg/5ml oral solution - Special Order |
| 8378511000001108 | Clonazepam 1mg/5ml oral solution 1 ml |
| 8379011000001105 | Clonazepam 1mg/5ml oral solution 1 ml - Special Order |
| 8395211000001105 | Clonazepam 1mg/5ml oral suspension |
| 8379711000001107 | Clonazepam 1mg/5ml oral suspension - Special Order |
| 8379511000001102 | Clonazepam 1mg/5ml oral suspension 1 ml |
| 8379811000001104 | Clonazepam 1mg/5ml oral suspension 1 ml - Special Order |
| 8395311000001102 | Clonazepam 2.5mg/5ml oral solution |
| 8376711000001102 | Clonazepam 2.5mg/5ml oral solution - Special Order |
| 8376411000001108 | Clonazepam 2.5mg/5ml oral solution 1 ml |
| 8377311000001103 | Clonazepam 2.5mg/5ml oral solution 1 ml - Special Order |
| 8395411000001109 | Clonazepam 2.5mg/5ml oral suspension |
| 8378411000001109 | Clonazepam 2.5mg/5ml oral suspension - Special Order |
| 8378011000001100 | Clonazepam 2.5mg/5ml oral suspension 1 ml |
| 8378611000001107 | Clonazepam 2.5mg/5ml oral suspension 1 ml - Special Order |
| 23466511000001106 | Clonazepam 2.5mg/ml drops |
| 23403411000001101 | Clonazepam 2.5mg/ml drops - Drug Tariff Special Order |
| 23403211000001100 | Clonazepam 2.5mg/ml drops 1 ml |
| 23403711000001107 | Clonazepam 2.5mg/ml drops 1 ml - Drug Tariff Special Order |
| 23403311000001108 | Clonazepam 2.5mg/ml drops 10 ml |
| 23403511000001102 | Clonazepam 2.5mg/ml drops 10 ml - Drug Tariff Special Order |
| 7662511000001100 | Clonazepam 2.5mg/ml drops sugar free |
| 15865811000001102 | Clonazepam 2.5mg/ml drops sugar free - Special Order |
| 15865711000001105 | Clonazepam 2.5mg/ml drops sugar free 1 ml |
| 15865911000001107 | Clonazepam 2.5mg/ml drops sugar free 1 ml - Special Order |
| 7654911000001106 | Clonazepam 2.5mg/ml drops sugar free 10 ml |
| 8395511000001108 | Clonazepam 200micrograms/5ml oral solution |
| 8377011000001101 | Clonazepam 200micrograms/5ml oral solution - Special Order |
| 8376611000001106 | Clonazepam 200micrograms/5ml oral solution 1 ml |
| 8377411000001105 | Clonazepam 200micrograms/5ml oral solution 1 ml - Special Order |
| 8395611000001107 | Clonazepam 200micrograms/5ml oral suspension |
| 8378111000001104 | Clonazepam 200micrograms/5ml oral suspension - Special Order |
| 8377911000001102 | Clonazepam 200micrograms/5ml oral suspension 1 ml |
| 8378311000001102 | Clonazepam 200micrograms/5ml oral suspension 1 ml - Special Order |
| 8395711000001103 | Clonazepam 250micrograms/5ml oral solution |
| 8380311000001108 | Clonazepam 250micrograms/5ml oral solution - Special Order |
| 8379911000001109 | Clonazepam 250micrograms/5ml oral solution 1 ml |

| 8380611000001103 | Clonazepam 250micrograms/5ml oral solution 1 ml - Special Order |
|---|---|
| 8395811000001106 | Clonazepam 250micrograms/5ml oral suspension |
| 8381111000001100 | Clonazepam 250micrograms/5ml oral suspension - Special Order |
| 8381011000001101 | Clonazepam 250micrograms/5ml oral suspension 1 ml |
| 8381311000001103 | Clonazepam 250micrograms/5ml oral suspension 1 ml - Special Order |
| 20459411000001107 | Clonazepam 250micrograms/5ml oral suspension 100 ml |
| | Clonazepam 250micrograms/5ml oral suspension 100 ml - Special |
| 20459511000001106 | Order |
| 11954911000001106 | Clonazepam 25mg/5ml oral solution |
| 11943511000001104 | Clonazepam 25mg/5ml oral solution - Special Order |
| 11943411000001103 | Clonazepam 25mg/5ml oral solution 1 ml |
| 11943611000001100 | Clonazepam 25mg/5ml oral solution 1 ml - Special Order |
| 11955011000001106 | Clonazepam 25mg/5ml oral suspension |
| 11943211000001102 | Clonazepam 25mg/5ml oral suspension - Special Order |
| 11943111000001108 | Clonazepam 25mg/5ml oral suspension 1 ml |
| 11943311000001105 | Clonazepam 25mg/5ml oral suspension 1 ml - Special Order |
| 11955111000001107 | Clonazepam 25micrograms/5ml oral solution |
| 11942911000001104 | Clonazepam 25micrograms/5ml oral solution - Special Order |
| 11942811000001100 | Clonazepam 25micrograms/5ml oral solution 1 ml |
| 11943011000001107 | Clonazepam 25micrograms/5ml oral solution 1 ml - Special Order |
| 11955211000001101 | Clonazepam 25micrograms/5ml oral suspension |
| 11942611000001105 | Clonazepam 25micrograms/5ml oral suspension - Special Order |
| 11942511000001106 | Clonazepam 25micrograms/5ml oral suspension 1 ml |
| 11942711000001101 | Clonazepam 25micrograms/5ml oral suspension 1 ml - Special Order |
| 322898003 | Clonazepam 2mg tablets |
| 13655811000001108 | Clonazepam 2mg tablets - A A H Pharmaceuticals Ltd |
| 13932511000001104 | Clonazepam 2mg tablets - Alliance Healthcare (Distribution) Ltd |
| 17966811000001104 | Clonazepam 2mg tablets - Almus Pharmaceuticals Ltd |
| 37227011000001103 | Clonazepam 2mg tablets - DE Pharmaceuticals |
| 32398211000001105 | Clonazepam 2mg tablets - Kent Pharmaceuticals Ltd |
| 37054011000001100 | Clonazepam 2mg tablets - Mawdsley-Brooks & Company Ltd |
| 38845211000001102 | Clonazepam 2mg tablets - Medihealth (Northern) Ltd |
| 17861411000001101 | Clonazepam 2mg tablets - Phoenix Healthcare Distribution Ltd |
| 15077211000001103 | Clonazepam 2mg tablets - Sigma Pharmaceuticals Plc |
| 37450611000001106 | Clonazepam 2mg tablets - Star Pharmaceuticals Ltd |
| 15627511000001106 | Clonazepam 2mg tablets - Teva UK Ltd |
| 21922411000001108 | Clonazepam 2mg tablets - Waymade Healthcare Plc |
| 958011000001104 | Clonazepam 2mg tablets 100 tablet |
| 13655911000001103 | Clonazepam 2mg tablets 100 tablet - A A H Pharmaceuticals Ltd |
| 13932611000001100 | Clonazepam 2mg tablets 100 tablet - Alliance Healthcare (Distribution) Ltd |
| 17966911000001109 | Clonazepam 2mg tablets 100 tablet - Almus Pharmaceuticals Ltd |
| 32398311000001102 | Clonazepam 2mg tablets 100 tablet - Kent Pharmaceuticals Ltd |
| 37054111000001104 | Clonazepam 2mg tablets 100 tablet - Mawdsley-Brooks & Company Ltd |
| 38845411000001103 | Clonazepam 2mg tablets 100 tablet - Medihealth (Northern) Ltd |
| 17861511000001102 | Clonazepam 2mg tablets 100 tablet - Phoenix Healthcare Distribution Ltd |
| 15077411000001104 | Clonazepam 2mg tablets 100 tablet - Sigma Pharmaceuticals Plc |
| 15627611000001105 | Clonazepam 2mg tablets 100 tablet - Teva UK Ltd |

| 37226911000001102 | Clonazepam 2mg tablets 105 tablet |
|---|---|
| 37227111000001102 | Clonazepam 2mg tablets 105 tablet - DE Pharmaceuticals |
| 37451411000001104 | Clonazepam 2mg tablets 105 tablet - Star Pharmaceuticals Ltd |
| 14664011000001109 | Clonazepam 2mg tablets 60 tablet Clonazepam 2mg tablets 60 tablet |
| 8395911000001101 | Clonazepam 2mg/5ml oral solution |
| 8379411000001101 | Clonazepam 2mg/5ml oral solution - Special Order |
| 8379311000001101 | Clonazepam 2mg/5ml oral solution 1 ml |
| 8379611000001103 | Clonazepam 2mg/5ml oral solution 1 ml - Special Order |
| 20065611000001108 | Clonazepam 2mg/5ml oral solution sugar free |
| | Clonazepam 2mg/5ml oral solution sugar free - A A H |
| 20637711000001105 | Pharmaceuticals Ltd |
| 35827011000001106 | Clonazepam 2mg/5ml oral solution sugar free - Accord Healthcare Ltd |
| 20359511000001104 | Clonazepam 2mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 37226311000001103 | Clonazepam 2mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 38845811000001101 | Clonazepam 2mg/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 20019211000001108 | Clonazepam 2mg/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd |
| 29790711000001105 | Clonazepam 2mg/5ml oral solution sugar free - Sigma Pharmaceuticals Plc |
| 34886811000001101 | Clonazepam 2mg/5ml oral solution sugar free - Thame Laboratories Ltd |
| 22082011000001101 | Clonazepam 2mg/5ml oral solution sugar free - Waymade Healthcare Plc |
| 20019111000001102 | Clonazepam 2mg/5ml oral solution sugar free 150 ml |
| 20637811000001102 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 35827111000001107 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd |
| 20359611000001100 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 37226411000001105 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - DE Pharmaceuticals |
| 38845911000001106 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Medihealth (Northern) Ltd |
| 20019311000001100 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Rosemont Pharmaceuticals Ltd |
| 29790811000001102 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Sigma<br>Pharmaceuticals Plc |
| 34886911000001106 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Thame Laboratories Ltd |
| 22082111000001100 | Clonazepam 2mg/5ml oral solution sugar free 150 ml - Waymade Healthcare Plc |
| 8396011000001109 | Clonazepam 2mg/5ml oral suspension |
| 8380111000001106 | Clonazepam 2mg/5ml oral suspension - Special Order |
| 8380011000001105 | Clonazepam 2mg/5ml oral suspension 1 ml |
| 8380411000001101 | Clonazepam 2mg/5ml oral suspension 1 ml - Special Order |
| 8396111000001105 | Clonazepam 3.75mg/5ml oral solution |
| 8383311000001102 | Clonazepam 3.75mg/5ml oral solution - Special Order |
| 8382611000001102 | Clonazepam 3.75mg/5ml oral solution 1 ml |
| 8383411000001109 | Clonazepam 3.75mg/5ml oral solution 1 ml - Special Order |
| 8396211000001104 | Clonazepam 3.75mg/5ml oral suspension |
| 8383711000001103 | Clonazepam 3.75mg/5ml oral suspension - Special Order |
| 8383511000001108 | Clonazepam 3.75mg/5ml oral suspension 1 ml |

| 8383911000001101 | Clonazepam 3.75mg/5ml oral suspension 1 ml - Special Order |
|---|---|
| 11955311000001109 | Clonazepam 300micrograms/5ml oral solution |
| 11946111000001103 | Clonazepam 300micrograms/5ml oral solution - Special Order |
| 11946011000001104 | Clonazepam 300micrograms/5ml oral solution 1 ml |
| 11946211000001109 | Clonazepam 300micrograms/5ml oral solution 1 ml - Special Order |
| 11955411000001102 | Clonazepam 300micrograms/5ml oral suspension |
| 11945811000001102 | Clonazepam 300micrograms/5ml oral suspension - Special Order |
| 11945711000001105 | Clonazepam 300micrograms/5ml oral suspension 1 ml |
| 11945911000001107 | Clonazepam 300micrograms/5ml oral suspension 1 ml - Special Order |
| 11955511000001103 | Clonazepam 312.5micrograms/5ml oral solution |
| 11946711000001102 | Clonazepam 312.5micrograms/5ml oral solution - Special Order |
| 11946611000001106 | Clonazepam 312.5micrograms/5ml oral solution 1 ml |
| 11946811000001105 | Clonazepam 312.5micrograms/5ml oral solution 1 ml - Special Order |
| 11955611000001104 | Clonazepam 312.5micrograms/5ml oral suspension |
| 11946411000001108 | Clonazepam 312.5micrograms/5ml oral suspension - Special Order |
| 11946311000001101 | Clonazepam 312.5micrograms/5ml oral suspension 1 ml |
| 11946511000001107 | Clonazepam 312.5micrograms/5ml oral suspension 1 ml - Special Order |
| 11955711000001108 | Clonazepam 330micrograms/5ml oral solution |
| 11947311000001103 | Clonazepam 330micrograms/5ml oral solution - Special Order |
| 11947211000001106 | Clonazepam 330micrograms/5ml oral solution 1 ml |
| 11947411000001105 | Clonazepam 330micrograms/5ml oral solution 1 ml - Special Order |
| 11955811000001100 | Clonazepam 330micrograms/5ml oral suspension |
| 11947011000001101 | Clonazepam 330micrograms/5ml oral suspension - Special Order |
| 11946911000001100 | Clonazepam 330micrograms/5ml oral suspension 1 ml |
| 11947111000001100 | Clonazepam 330micrograms/5ml oral suspension 1 ml - Special Order |
| 11955911000001105 | Clonazepam 340micrograms/5ml oral solution |
| 11947911000001102 | Clonazepam 340micrograms/5ml oral solution - Special Order |
| 11947811000001107 | Clonazepam 340micrograms/5ml oral solution 1 ml |
| 11948011000001100 | Clonazepam 340micrograms/5ml oral solution 1 ml - Special Order |
| 11956011000001102 | Clonazepam 340micrograms/5ml oral suspension |
| 11947611000001108 | Clonazepam 340micrograms/5ml oral suspension - Special Order |
| 11947511000001109 | Clonazepam 340micrograms/5ml oral suspension 1 ml |
| 11947711000001104 | Clonazepam 340micrograms/5ml oral suspension 1 ml - Special Order |
| 8396311000001107 | Clonazepam 350micrograms/5ml oral solution |
| 8381411000001105 | Clonazepam 350micrograms/5ml oral solution - Special Order |
| 8381211000001106 | Clonazepam 350micrograms/5ml oral solution 1 ml |
| 8381511000001109 | Clonazepam 350micrograms/5ml oral solution 1 ml - Special Order |
| 8396411000001100 | Clonazepam 350micrograms/5ml oral suspension |
| 8380811000001104 | Clonazepam 350micrograms/5ml oral suspension - Special Order |
| 8380711000001107 | Clonazepam 350micrograms/5ml oral suspension 1 ml |
| 8380911000001109 | Clonazepam 350micrograms/5ml oral suspension 1 ml - Special<br>Order |
| 11956111000001101 | Clonazepam 37.5micrograms/5ml oral solution |
| 11948511000001108 | Clonazepam 37.5micrograms/5ml oral solution - Special Order |
| 11948411000001109 | Clonazepam 37.5micrograms/5ml oral solution 1 ml |
| 11948611000001107 | Clonazepam 37.5micrograms/5ml oral solution 1 ml - Special Order |

| 11948211000001105 | Clonazepam 37.5micrograms/5ml oral suspension - Special Order |
|---|---|
| 11948111000001104 | Clonazepam 37.5micrograms/5ml oral suspension 1 ml |
| 11948311000001102 | Clonazepam 37.5micrograms/5ml oral suspension 1 ml - Special Order |
| 8396511000001101 | Clonazepam 375micrograms/5ml oral solution |
| 8385411000001108 | Clonazepam 375micrograms/5ml oral solution - Special Order |
| 8384611000001105 | Clonazepam 375micrograms/5ml oral solution 1 ml |
| 8385811000001105 | Clonazepam 375micrograms/5ml oral solution 1 ml - Special Order |
| 8396611000001102 | Clonazepam 375micrograms/5ml oral suspension |
| 8387811000001100 | Clonazepam 375micrograms/5ml oral suspension - Special Order |
| 8387411000001102 | Clonazepam 375micrograms/5ml oral suspension 1 ml |
| 8388311000001105 | Clonazepam 375micrograms/5ml oral suspension 1 ml - Special Order |
| 8396711000001106 | Clonazepam 3mg/5ml oral solution |
| 8381711000001104 | Clonazepam 3mg/5ml oral solution - Special Order |
| 8381611000001108 | Clonazepam 3mg/5ml oral solution 1 ml |
| 8381811000001107 | Clonazepam 3mg/5ml oral solution 1 ml - Special Order |
| 8396811000001103 | Clonazepam 3mg/5ml oral suspension |
| 8382011000001109 | Clonazepam 3mg/5ml oral suspension - Special Order |
| 8381911000001102 | Clonazepam 3mg/5ml oral suspension 1 ml |
| 8382111000001105 | Clonazepam 3mg/5ml oral suspension 1 ml - Special Order |
| 11956311000001104 | Clonazepam 400micrograms/5ml oral solution |
| 11949111000001106 | Clonazepam 400micrograms/5ml oral solution - Special Order |
| 11949011000001105 | Clonazepam 400micrograms/5ml oral solution 1 ml |
| 11949211000001100 | Clonazepam 400micrograms/5ml oral solution 1 ml - Special Order |
| 11956411000001106 | Clonazepam 400micrograms/5ml oral suspension |
| 11948811000001106 | Clonazepam 400micrograms/5ml oral suspension - Special Order |
| 11948711000001103 | Clonazepam 400micrograms/5ml oral suspension 1 ml |
| 11948911000001101 | Clonazepam 400micrograms/5ml oral suspension 1 ml - Special Order |
| 8396911000001108 | Clonazepam 4mg/5ml oral solution |
| 8384911000001104 | Clonazepam 4mg/5ml oral solution - Special Order |
| 8384711000001101 | Clonazepam 4mg/5ml oral solution 1 ml |
| 8385011000001104 | Clonazepam 4mg/5ml oral solution 1 ml - Special Order |
| 8397011000001107 | Clonazepam 4mg/5ml oral suspension |
| 8386111000001109 | Clonazepam 4mg/5ml oral suspension - Special Order |
| 8385611000001106 | Clonazepam 4mg/5ml oral suspension 1 ml |
| 8386611000001101 | Clonazepam 4mg/5ml oral suspension 1 ml - Special Order |
| 8397111000001108 | Clonazepam 500micrograms/5ml oral solution |
| 8385311000001101 | Clonazepam 500micrograms/5ml oral solution - Special Order |
| 8385111000001103 | Clonazepam 500micrograms/5ml oral solution 1 ml |
| 8385511000001107 | Clonazepam 500micrograms/5ml oral solution 1 ml - Special Order |
| 19597411000001102 | Clonazepam 500micrograms/5ml oral solution 150 ml |
| 19597611000001104 | Clonazepam 500micrograms/5ml oral solution 150 ml - Special Order |
| 20128211000001100 | Clonazepam 500micrograms/5ml oral solution sugar free |
| 20612511000001109 | Clonazepam 500micrograms/5ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 35826811000001102 | Clonazepam 500micrograms/5ml oral solution sugar free - Accord Healthcare Ltd |
| 20359311000001105 | Clonazepam 500micrograms/5ml oral solution sugar free - Alliance<br>Healthcare (Distribution) Ltd |

| | Clonazepam 500micrograms/5ml oral solution sugar free - DE |
|---|---|
| 37226111000001100 | Pharmaceuticals |
| 38845611000001100 | Clonazepam 500micrograms/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 20018711000001105 | Clonazepam 500micrograms/5ml oral solution sugar free - Rosemont Pharmaceuticals Ltd |
| 29790511000001100 | Clonazepam 500micrograms/5ml oral solution sugar free - Sigma Pharmaceuticals Plc |
| 34886611000001100 | Clonazepam 500micrograms/5ml oral solution sugar free - Thame Laboratories Ltd |
| 22081811000001103 | Clonazepam 500micrograms/5ml oral solution sugar free - Waymade Healthcare Plc |
| 20018611000001101 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml |
| 20612611000001108 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 35826911000001107 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - Accord Healthcare Ltd |
| 20359411000001103 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - Alliance Healthcare (Distribution) Ltd |
| 37226211000001106 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - DE Pharmaceuticals |
| 38845711000001109 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - Medihealth (Northern) Ltd |
| 20018811000001102 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml -<br>Rosemont Pharmaceuticals Ltd |
| 29790611000001101 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - Sigma Pharmaceuticals Plc |
| 34886711000001109 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml -<br>Thame Laboratories Ltd |
| 22081911000001108 | Clonazepam 500micrograms/5ml oral solution sugar free 150 ml - Waymade Healthcare Plc |
| 8397211000001102 | Clonazepam 500micrograms/5ml oral suspension |
| 8386311000001106 | Clonazepam 500micrograms/5ml oral suspension - Special Order |
| 8386011000001108 | Clonazepam 500micrograms/5ml oral suspension 1 ml |
| 8386411000001104 | Clonazepam 500micrograms/5ml oral suspension 1 ml - Special Order |
| 19597811000001100 | Clonazepam 500micrograms/5ml oral suspension 100 ml |
| 19598011000001107 | Clonazepam 500micrograms/5ml oral suspension 100 ml - Special Order |
| 19933611000001107 | Clonazepam 500micrograms/5ml oral suspension 150 ml |
| 19933711000001103 | Clonazepam 500micrograms/5ml oral suspension 150 ml - Special Order |
| 11956511000001105 | Clonazepam 50micrograms/5ml oral solution |
| 11949911000001109 | Clonazepam 50micrograms/5ml oral solution - Special Order |
| 11949811000001104 | Clonazepam 50micrograms/5ml oral solution 1 ml |
| 11950011000001100 | Clonazepam 50micrograms/5ml oral solution 1 ml - Special Order |
| 11956611000001109 | Clonazepam 50micrograms/5ml oral suspension |
| 11949611000001103 | Clonazepam 50micrograms/5ml oral suspension - Special Order |
| 11949511000001102 | Clonazepam 50micrograms/5ml oral suspension 1 ml |
| 11949711000001107 | Clonazepam 50micrograms/5ml oral suspension 1 ml - Special Order |
| 8397311000001105 | Clonazepam 5mg/5ml oral solution |
| 8387211000001101 | Clonazepam 5mg/5ml oral solution - Special Order |
| 8387111000001107 | Clonazepam 5mg/5ml oral solution 1 ml |
| 8387511000001103 | Clonazepam 5mg/5ml oral solution 1 ml - Special Order |
| 8397411000001103 | Clonazepam 5mg/5ml oral suspension |
| 8388211000001102 | Clonazepam 5mg/5ml oral suspension - Special Order |

| 8388011000001107 | Clonazepam 5mg/5ml oral suspension 1 ml |
|---|---|
| 8388411000001103 | Clonazepam 5mg/5ml oral suspension 1 ml - Special Order |
| 11956711000001100 | Clonazepam 600micrograms/5ml oral solution |
| 11950511000001108 | Clonazepam 600micrograms/5ml oral solution - Special Order |
| 11950411000001109 | Clonazepam 600micrograms/5ml oral solution 1 ml |
| 11950611000001107 | Clonazepam 600micrograms/5ml oral solution 1 ml - Special Order |
| 11956811000001108 | Clonazepam 600micrograms/5ml oral suspension |
| 11950211000001105 | Clonazepam 600micrograms/5ml oral suspension - Special Order |
| 11950111000001104 | Clonazepam 600micrograms/5ml oral suspension 1 ml |
| 11950311000001102 | Clonazepam 600micrograms/5ml oral suspension 1 ml - Special Order |
| 8397511000001104 | Clonazepam 625micrograms/5ml oral solution |
| 8390911000001105 | Clonazepam 625micrograms/5ml oral solution - Special Order |
| 8390511000001103 | Clonazepam 625micrograms/5ml oral solution 1 ml |
| 8391011000001102 | Clonazepam 625micrograms/5ml oral solution 1 ml - Special Order |
| 8397611000001100 | Clonazepam 625micrograms/5ml oral suspension |
| 8392211000001100 | Clonazepam 625micrograms/5ml oral suspension - Special Order |
| 8391711000001100 | Clonazepam 625micrograms/5ml oral suspension 1 ml |
| 8392511000001102 | Clonazepam 625micrograms/5ml oral suspension 1 ml - Special Order |
| 8397711000001109 | Clonazepam 7.5mg/5ml oral solution |
| 8389311000001104 | Clonazepam 7.5mg/5ml oral solution - Special Order |
| 8389211000001107 | Clonazepam 7.5mg/5ml oral solution 1 ml |
| 8389411000001106 | Clonazepam 7.5mg/5ml oral solution 1 ml - Special Order |
| 8397811000001101 | Clonazepam 7.5mg/5ml oral suspension |
| 8389711000001100 | Clonazepam 7.5mg/5ml oral suspension - Special Order |
| 8389511000001105 | Clonazepam 7.5mg/5ml oral suspension 1 ml |
| 8390111000001107 | Clonazepam 7.5mg/5ml oral suspension 1 ml - Special Order |
| 11956911000001103 | Clonazepam 700micrograms/5ml oral solution |
| 11951111000001105 | Clonazepam 700micrograms/5ml oral solution - Special Order |
| 11951011000001109 | Clonazepam 700micrograms/5ml oral solution 1 ml |
| 11951211000001104 | Clonazepam 700micrograms/5ml oral solution 1 ml - Special Order |
| 11957011000001104 | Clonazepam 700micrograms/5ml oral suspension |
| 11950811000001106 | Clonazepam 700micrograms/5ml oral suspension - Special Order |
| 11950711000001103 | Clonazepam 700micrograms/5ml oral suspension 1 ml |
| 11950911000001101 | Clonazepam 700micrograms/5ml oral suspension 1 ml - Special Order |
| 11957111000001103 | Clonazepam 750micrograms/5ml oral solution |
| 11951711000001106 | Clonazepam 750micrograms/5ml oral solution - Special Order |
| 11951611000001102 | Clonazepam 750micrograms/5ml oral solution 1 ml |
| 11951811000001103 | Clonazepam 750micrograms/5ml oral solution 1 ml - Special Order |
| 11957211000001109 | Clonazepam 750micrograms/5ml oral suspension |
| 11951411000001100 | Clonazepam 750micrograms/5ml oral suspension - Special Order |
| 11951311000001107 | Clonazepam 750micrograms/5ml oral suspension 1 ml |
| 11951511000001101 | Clonazepam 750micrograms/5ml oral suspension 1 ml - Special Order |
| 11957311000001101 | Clonazepam 80micrograms/5ml oral solution |
| 11952311000001103 | Clonazepam 80micrograms/5ml oral solution - Special Order |
| 11952211000001106 | Clonazepam 80micrograms/5ml oral solution 1 ml |
| 11952411000001105 | Clonazepam 80micrograms/5ml oral solution 1 ml - Special Order |
| 11957411000001108 | Clonazepam 80micrograms/5ml oral suspension |

| 11952011000001101 | Clonazepam 80micrograms/5ml oral suspension - Special Order |
|---|---|
| 11951911000001108 | Clonazepam 80micrograms/5ml oral suspension 1 ml |
| 11952111000001100 | Clonazepam 80micrograms/5ml oral suspension 1 ml - Special Order |
| 11957511000001107 | Clonazepam 875micrograms/5ml oral solution |
| 11952911000001102 | Clonazepam 875micrograms/5ml oral solution - Special Order |
| 11952811000001107 | Clonazepam 875micrograms/5ml oral solution 1 ml |
| 11953011000001105 | Clonazepam 875micrograms/5ml oral solution 1 ml - Special Order |
| 11957611000001106 | Clonazepam 875micrograms/5ml oral suspension |
| 11952611000001108 | Clonazepam 875micrograms/5ml oral suspension - Special Order |
| 11952511000001109 | Clonazepam 875micrograms/5ml oral suspension 1 ml |
| 11952711000001104 | Clonazepam 875micrograms/5ml oral suspension 1 ml - Special Order |
| 11957711000001102 | Clonazepam 900micrograms/5ml oral solution |
| 11953511000001102 | Clonazepam 900micrograms/5ml oral solution - Special Order |
| 11953411000001101 | Clonazepam 900micrograms/5ml oral solution 1 ml |
| 11953611000001103 | Clonazepam 900micrograms/5ml oral solution 1 ml - Special Order |
| 11957811000001105 | Clonazepam 900micrograms/5ml oral suspension |
| 11953211000001100 | Clonazepam 900micrograms/5ml oral suspension - Special Order |
| 11953111000001106 | Clonazepam 900micrograms/5ml oral suspension 1 ml |
| 11953311000001108 | Clonazepam 900micrograms/5ml oral suspension 1 ml - Special Order |
| 3971111000001102 | Diazemuls 10mg/2ml emulsion for injection ampoules - Accord Healthcare Ltd |
| 3971311000001100 | Diazemuls 10mg/2ml emulsion for injection ampoules 10 ampoule - Accord Healthcare Ltd |
| 26811000001102 | Diazepam 10mg RecTubes - Wockhardt UK Ltd |
| 2638611000001109 | Diazepam 10mg RecTubes 5 tube - Wockhardt UK Ltd |
| 321238008 | Diazepam 10mg suppositories |
| 27320211000001103 | Diazepam 10mg suppositories - Special Order |
| 27320511000001100 | Diazepam 10mg suppositories 1 suppository |
| 27320711000001105 | Diazepam 10mg suppositories 1 suppository - Special Order |
| 3823911000001106 | Diazepam 10mg suppositories 6 suppository |
| 321198003 | Diazepam 10mg tablets |
| 734911000001103 | Diazepam 10mg tablets - A A H Pharmaceuticals Ltd |
| 486211000001103 | Diazepam 10mg tablets - Accord Healthcare Ltd |
| 433011000001105 | Diazepam 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9790811000001104 | Diazepam 10mg tablets - Almus Pharmaceuticals Ltd |
| 10400711000001100 | Diazepam 10mg tablets - Arrow Generics Ltd |
| 28922211000001102 | Diazepam 10mg tablets - Crescent Pharma Ltd |
| 23861111000001100 | Diazepam 10mg tablets - DE Pharmaceuticals |
| 11020311000001105 | Diazepam 10mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 230211000001106 | Diazepam 10mg tablets - IVAX Pharmaceuticals UK Ltd |
| 305211000001102 | Diazepam 10mg tablets - Kent Pharmaceuticals Ltd |
| 37057611000001101 | Diazepam 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 38867711000001106 | Diazepam 10mg tablets - Medihealth (Northern) Ltd |
| 878511000001104 | Diazepam 10mg tablets - Mylan |
| 18107511000001108 | Diazepam 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 253911000001109 | Diazepam 10mg tablets - Ranbaxy (UK) Ltd |
| 29804111000001100 | Diazepam 10mg tablets - Sigma Pharmaceuticals Plc |
| 17197311000001106 | Diazepam 10mg tablets - Sovereign Medical Ltd |
| 366511000001107 | Diazepam 10mg tablets - Teva UK Ltd |

| 21925811000001103 | Diazepam 10mg tablets - Waymade Healthcare Plc |
|---|---|
| 13938311000001108 | Diazepam 10mg tablets - Wockhardt UK Ltd |
| 9106611000001109 | Diazepam 10mg tablets 100 tablet |
| 1132211000001105 | Diazepam 10mg tablets 28 tablet |
| 1420011000001103 | Diazepam 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1420811000001109 | Diazepam 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 1443411000001102 | Diazepam 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 9790911000001109 | Diazepam 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 10400811000001108 | Diazepam 10mg tablets 28 tablet - Arrow Generics Ltd |
| 28922311000001105 | Diazepam 10mg tablets 28 tablet - Crescent Pharma Ltd |
| 23861311000001103 | Diazepam 10mg tablets 28 tablet - DE Pharmaceuticals |
| 1422111000001103 | Diazepam 10mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1422711000001102 | Diazepam 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 37057711000001105 | Diazepam 10mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38868011000001105 | Diazepam 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 1422611000001106 | Diazepam 10mg tablets 28 tablet - Mylan |
| 18107611000001107 | Diazepam 10mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 1442711000001100 | Diazepam 10mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 29804211000001106 | Diazepam 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 17197411000001104 | Diazepam 10mg tablets 28 tablet - Sovereign Medical Ltd |
| 1421811000001101 | Diazepam 10mg tablets 28 tablet - Teva UK Ltd |
| 21925911000001108 | Diazepam 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 13938411000001101 | Diazepam 10mg tablets 28 tablet - Wockhardt UK Ltd |
| 1289511000001106 | Diazepam 10mg tablets 500 tablet |
| 1420311000001100 | Diazepam 10mg tablets 500 tablet - A A H Pharmaceuticals Ltd |
| 1443511000001103 | Diazepam 10mg tablets 500 tablet - Alliance Healthcare (Distribution) Ltd |
| 10400911000001103 | Diazepam 10mg tablets 500 tablet - Arrow Generics Ltd |
| 11020411000001103 | Diazepam 10mg tablets 500 tablet - Dr Reddys Laboratories (UK) Ltd |
| 1423411000001104 | Diazepam 10mg tablets 500 tablet - Kent Pharmaceuticals Ltd |
| 1443211000001101 | Diazepam 10mg tablets 500 tablet - Ranbaxy (UK) Ltd |
| 17197511000001100 | Diazepam 10mg tablets 500 tablet - Sovereign Medical Ltd |
| 23591311000001100 | Diazepam 10mg tablets 500 tablet - Waymade Healthcare Plc |
| 16431111000001106 | Diazepam 10mg tablets 500 tablet - Wockhardt UK Ltd |
| 323074003 | Diazepam 10mg/2.5ml rectal solution tube |
| 343011000001104 | Diazepam 10mg/2.5ml rectal solution tube - A A H Pharmaceuticals Ltd |
| 885611000001101 | Diazepam 10mg/2.5ml rectal solution tube - Alliance Healthcare (Distribution) Ltd |
| 22198411000001102 | Diazepam 10mg/2.5ml rectal solution tube - Desitin Pharma Ltd |
| 75811000001106 | Diazepam 10mg/2.5ml rectal solution tube - Sandoz Ltd |
| 29804511000001109 | Diazepam 10mg/2.5ml rectal solution tube - Sigma Pharmaceuticals Plc |
| 1057611000001101 | Diazepam 10mg/2.5ml rectal solution tube 5 tube |
| 2638411000001106 | Diazepam 10mg/2.5ml rectal solution tube 5 tube - A A H Pharmaceuticals Ltd |
| 2638811000001108 | Diazepam 10mg/2.5ml rectal solution tube 5 tube - Alliance<br>Healthcare (Distribution) Ltd |
| 22198511000001103 | Diazepam 10mg/2.5ml rectal solution tube 5 tube - Desitin Pharma Ltd |
| 2638711000001100 | Diazepam 10mg/2.5ml rectal solution tube 5 tube - Sandoz Ltd |

| 29804611000001108 | Diazepam 10mg/2.5ml rectal solution tube 5 tube - Sigma |
|---|---|
| | Pharmaceuticals Plc |
| 36097511000001106 | Diazepam 10mg/2ml emulsion for injection ampoules |
| 323071006 | Diazepam 10mg/2ml emulsion for injection ampoules |
| 3971011000001103 | Diazepam 10mg/2ml emulsion for injection ampoules 10 ampoule |
| 36097611000001105 | Diazepam 10mg/2ml solution for injection ampoules |
| 323072004 | Diazepam 10mg/2ml solution for injection ampoules |
| 434211000001102 | Diazepam 10mg/2ml solution for injection ampoules - A A H Pharmaceuticals Ltd |
| 155811000001103 | Diazepam 10mg/2ml solution for injection ampoules - Alliance Healthcare (Distribution) Ltd |
| 5083111000001106 | Diazepam 10mg/2ml solution for injection ampoules - hameln pharma Ltd |
| 687511000001101 | Diazepam 10mg/2ml solution for injection ampoules - Wockhardt UK Ltd |
| 1306411000001107 | Diazepam 10mg/2ml solution for injection ampoules 10 ampoule |
| 2759311000001100 | Diazepam 10mg/2ml solution for injection ampoules 10 ampoule - A A H Pharmaceuticals Ltd |
| 2759711000001101 | Diazepam 10mg/2ml solution for injection ampoules 10 ampoule - Alliance Healthcare (Distribution) Ltd |
| 5083211000001100 | Diazepam 10mg/2ml solution for injection ampoules 10 ampoule - hameln pharma Ltd |
| 2759611000001105 | Diazepam 10mg/2ml solution for injection ampoules 10 ampoule - Wockhardt UK Ltd |
| 8792711000001108 | Diazepam 10mg/5ml oral solution |
| 22328211000001103 | Diazepam 10mg/5ml oral solution - AM Distributions (Yorkshire) Ltd |
| 8781111000001101 | Diazepam 10mg/5ml oral solution - Special Order |
| 8781011000001102 | Diazepam 10mg/5ml oral solution 1 ml |
| 8781311000001104 | Diazepam 10mg/5ml oral solution 1 ml - Special Order |
| 20443911000001100 | Diazepam 10mg/5ml oral solution 100 ml |
| 20444411000001106 | Diazepam 10mg/5ml oral solution 100 ml - Special Order |
| 22327611000001100 | Diazepam 10mg/5ml oral solution 200 ml |
| 22328311000001106 | Diazepam 10mg/5ml oral solution 200 ml - AM Distributions (Yorkshire) Ltd |
| 13893211000001109 | Diazepam 10mg/5ml oral suspension |
| 13883811000001109 | Diazepam 10mg/5ml oral suspension - Special Order |
| 13883611000001105 | Diazepam 10mg/5ml oral suspension 1 ml |
| 13884011000001101 | Diazepam 10mg/5ml oral suspension 1 ml - Special Order |
| 21310311000001103 | Diazepam 10mg/5ml oral suspension 200 ml |
| 21310411000001105 | Diazepam 10mg/5ml oral suspension 200 ml - Special Order |
| 22371411000001107 | Diazepam 15mg/5ml oral solution - Special Order |
| 22371511000001106 | Diazepam 15mg/5ml oral solution 1 ml - Special Order |
| 22371611000001105 | Diazepam 15mg/5ml oral solution 100 ml - Special Order |
| 283311000001103 | Diazepam 2.5mg RecTubes - Wockhardt UK Ltd |
| 2645111000001107 | Diazepam 2.5mg RecTubes 5 tube - Wockhardt UK Ltd |
| 323069006 | Diazepam 2.5mg/1.25ml rectal solution tube |
| 945211000001104 | Diazepam 2.5mg/1.25ml rectal solution tube 5 tube |
| 8792911000001105 | Diazepam 2.5mg/5ml oral solution |
| 8780511000001103 | Diazepam 2.5mg/5ml oral solution - Special Order |
| 8780411000001102 | Diazepam 2.5mg/5ml oral solution 1 ml |
| 8780611000001104 | Diazepam 2.5mg/5ml oral solution 1 ml - Special Order |
| 13893311000001101 | Diazepam 2.5mg/5ml oral suspension |
| 13892111000001109 | Diazepam 2.5mg/5ml oral suspension - Special Order |

| 13892011000001108 | Diazepam 2.5mg/5ml oral suspension 1 ml |
|---|---|
| 13892211000001103 | Diazepam 2.5mg/5ml oral suspension 1 ml - Special Order |
| 426016003 | Diazepam 25mg/5ml oral solution |
| 8793011000001102 | Diazepam 25mg/5ml oral solution |
| 8780811000001100 | Diazepam 25mg/5ml oral solution - Special Order |
| 8780711000001108 | Diazepam 25mg/5ml oral solution 1 ml |
| 8780911000001105 | Diazepam 25mg/5ml oral solution 1 ml - Special Order |
| 321196004 | Diazepam 2mg tablets |
| 889411000001101 | Diazepam 2mg tablets - A A H Pharmaceuticals Ltd |
| 790811000001109 | Diazepam 2mg tablets - Accord Healthcare Ltd |
| 28611000001100 | Diazepam 2mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9790311000001108 | Diazepam 2mg tablets - Almus Pharmaceuticals Ltd |
| 10400111000001101 | Diazepam 2mg tablets - Arrow Generics Ltd |
| 28922011000001107 | Diazepam 2mg tablets - Crescent Pharma Ltd |
| 13577011000001103 | Diazepam 2mg tablets - DE Pharmaceuticals |
| 11019911000001105 | Diazepam 2mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 52211000001103 | Diazepam 2mg tablets - IVAX Pharmaceuticals UK Ltd |
| 708811000001109 | Diazepam 2mg tablets - Kent Pharmaceuticals Ltd |
| 30021611000001103 | Diazepam 2mg tablets - Mawdsley-Brooks & Company Ltd |
| 38868111000001106 | Diazepam 2mg tablets - Medihealth (Northern) Ltd |
| 849711000001101 | Diazepam 2mg tablets - Mylan |
| 18107111000001104 | Diazepam 2mg tablets - Phoenix Healthcare Distribution Ltd |
| 463011000001103 | Diazepam 2mg tablets - Ranbaxy (UK) Ltd |
| 125411000001104 | Diazepam 2mg tablets - Sandoz Ltd |
| 15081411000001104 | Diazepam 2mg tablets - Sigma Pharmaceuticals Plc |
| 17196711000001107 | Diazepam 2mg tablets - Sovereign Medical Ltd |
| 223511000001101 | Diazepam 2mg tablets - Teva UK Ltd |
| 790211000001108 | Diazepam 2mg tablets - The Boots Company Plc |
| 21925411000001100 | Diazepam 2mg tablets - Waymade Healthcare Plc |
| 13937911000001108 | Diazepam 2mg tablets - Wockhardt UK Ltd |
| 9107011000001104 | Diazepam 2mg tablets 100 tablet |
| 998211000001100 | Diazepam 2mg tablets 1000 tablet |
| 1423611000001101 | Diazepam 2mg tablets 1000 tablet - A A H Pharmaceuticals Ltd |
| 1424811000001104 | Diazepam 2mg tablets 1000 tablet - Alliance Healthcare (Distribution) Ltd |
| 10400311000001104 | Diazepam 2mg tablets 1000 tablet - Arrow Generics Ltd |
| 13577111000001102 | Diazepam 2mg tablets 1000 tablet - DE Pharmaceuticals |
| 11020011000001107 | Diazepam 2mg tablets 1000 tablet - Dr Reddys Laboratories (UK) Ltd |
| 1424211000001100 | Diazepam 2mg tablets 1000 tablet - Kent Pharmaceuticals Ltd |
| 23654011000001100 | Diazepam 2mg tablets 1000 tablet - Phoenix Healthcare Distribution Ltd |
| 1424511000001102 | Diazepam 2mg tablets 1000 tablet - Ranbaxy (UK) Ltd |
| 17196911000001109 | Diazepam 2mg tablets 1000 tablet - Sovereign Medical Ltd |
| 1423911000001107 | Diazepam 2mg tablets 1000 tablet - The Boots Company Plc |
| 23591111000001102 | Diazepam 2mg tablets 1000 tablet - Waymade Healthcare Plc |
| 16430911000001102 | Diazepam 2mg tablets 1000 tablet - Wockhardt UK Ltd |
| 1257511000001107 | Diazepam 2mg tablets 28 tablet |
| 1423511000001100 | Diazepam 2mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1423711000001105 | Diazepam 2mg tablets 28 tablet - Accord Healthcare Ltd |

| 1424011000001100 | Diazepam 2mg tablets 28 tablet - Alliance Healthcare (Distribution) |
|---|---|
| 1424911000001109 | Ltd |
| 9790511000001102 | Diazepam 2mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 10400211000001107 | Diazepam 2mg tablets 28 tablet - Arrow Generics Ltd |
| 28922111000001108 | Diazepam 2mg tablets 28 tablet - Crescent Pharma Ltd |
| 23861611000001108 | Diazepam 2mg tablets 28 tablet - DE Pharmaceuticals |
| 1424111000001106 | Diazepam 2mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1424311000001108 | Diazepam 2mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 30021911000001109 | Diazepam 2mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38868211000001100 | Diazepam 2mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 1424011000001105 | Diazepam 2mg tablets 28 tablet - Mylan |
| 18107211000001105 | Diazepam 2mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 1424711000001107 | Diazepam 2mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 1424411000001101 | Diazepam 2mg tablets 28 tablet - Sandoz Ltd |
| 15081511000001100 | Diazepam 2mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 17196811000001104 | Diazepam 2mg tablets 28 tablet - Sovereign Medical Ltd |
| 1423811000001102 | Diazepam 2mg tablets 28 tablet - Teva UK Ltd |
| 21925511000001101 | Diazepam 2mg tablets 28 tablet - Waymade Healthcare Plc |
| 13938011000001105 | Diazepam 2mg tablets 28 tablet - Wockhardt UK Ltd |
| 9107111000001103 | Diazepam 2mg tablets 500 tablet |
| 321199006 | Diazepam 2mg/5ml oral solution |
| 753911000001101 | Diazepam 2mg/5ml oral solution - A A H Pharmaceuticals Ltd |
| 8892111000001109 | Diazepam 2mg/5ml oral solution - Actavis UK Ltd |
| 11248711000001102 | Diazepam 2mg/5ml oral solution - Alliance Healthcare (Distribution) Ltd |
| 182011000001108 | Diazepam 2mg/5ml oral solution - Sandoz Ltd |
| 15106611000001102 | Diazepam 2mg/5ml oral solution - Sigma Pharmaceuticals Plc |
| 1133111000001105 | Diazepam 2mg/5ml oral solution 100 ml |
| 2639211000001102 | Diazepam 2mg/5ml oral solution 100 ml - A A H Pharmaceuticals Ltd |
| 8892511000001100 | Diazepam 2mg/5ml oral solution 100 ml - Actavis UK Ltd |
| 11248811000001105 | Diazepam 2mg/5ml oral solution 100 ml - Alliance Healthcare (Distribution) Ltd |
| 2639411000001103 | Diazepam 2mg/5ml oral solution 100 ml - Sandoz Ltd |
| 1292611000001104 | Diazepam 2mg/5ml oral solution 500 ml |
| 2639311000001105 | Diazepam 2mg/5ml oral solution 500 ml - A A H Pharmaceuticals Ltd |
| 2639511000001104 | Diazepam 2mg/5ml oral solution 500 ml - Sandoz Ltd |
| 15106811000001103 | Diazepam 2mg/5ml oral solution 500 ml - Sigma Pharmaceuticals Plc |
| 38894311000001101 | Diazepam 2mg/5ml oral solution sugar free |
| 398895004 | Diazepam 2mg/5ml oral solution sugar free |
| 19571011000001105 | Diazepam 2mg/5ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 9765211000001106 | Diazepam 2mg/5ml oral solution sugar free - Accord Healthcare Ltd |
| 28972511000001100 | Diazepam 2mg/5ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 30762111000001108 | Diazepam 2mg/5ml oral solution sugar free - Almus Pharmaceuticals Ltd |
| 37297811000001102 | Diazepam 2mg/5ml oral solution sugar free - DE Pharmaceuticals |
| 30850511000001109 | Diazepam 2mg/5ml oral solution sugar free - Mawdsley-Brooks & Company Ltd |
| 38869411000001109 | Diazepam 2mg/5ml oral solution sugar free - Medihealth (Northern) Ltd |
| 9765111000001100 | Diazepam 2mg/5ml oral solution sugar free 100 ml |

| | Diazepam 2mg/5ml oral solution sugar free 100 ml - A A H |
|---|---|
| 19571111000001106 | Pharmaceuticals Ltd |
| 9765311000001103 | Diazepam 2mg/5ml oral solution sugar free 100 ml - Accord Healthcare Ltd |
| 28972711000001105 | Diazepam 2mg/5ml oral solution sugar free 100 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 30762211000001102 | Diazepam 2mg/5ml oral solution sugar free 100 ml - Almus Pharmaceuticals Ltd |
| 37297911000001107 | Diazepam 2mg/5ml oral solution sugar free 100 ml - DE Pharmaceuticals |
| 30850611000001108 | Diazepam 2mg/5ml oral solution sugar free 100 ml - Mawdsley-<br>Brooks & Company Ltd |
| 38869511000001108 | Diazepam 2mg/5ml oral solution sugar free 100 ml - Medihealth (Northern) Ltd |
| 19677811000001102 | Diazepam 2mg/5ml oral suspension |
| 32903011000001104 | Diazepam 2mg/5ml oral suspension - A A H Pharmaceuticals Ltd |
| 32782211000001108 | Diazepam 2mg/5ml oral suspension - Alliance Healthcare (Distribution) Ltd |
| 32635111000001108 | Diazepam 2mg/5ml oral suspension - Sandoz Ltd |
| 19674911000001101 | Diazepam 2mg/5ml oral suspension - Special Order |
| 19674811000001106 | Diazepam 2mg/5ml oral suspension 1 ml |
| 19675011000001101 | Diazepam 2mg/5ml oral suspension 1 ml - Special Order |
| 32635011000001107 | Diazepam 2mg/5ml oral suspension 100 ml |
| 32903111000001103 | Diazepam 2mg/5ml oral suspension 100 ml - A A H Pharmaceuticals Ltd |
| 32782311000001100 | Diazepam 2mg/5ml oral suspension 100 ml - Alliance Healthcare (Distribution) Ltd |
| 32635211000001102 | Diazepam 2mg/5ml oral suspension 100 ml - Sandoz Ltd |
| 603811000001108 | Diazepam 5mg RecTubes - Wockhardt UK Ltd |
| 2640411000001109 | Diazepam 5mg RecTubes 5 tube - Wockhardt UK Ltd |
| 224211000001101 | Diazepam 5mg tablets - A A H Pharmaceuticals Ltd |
| 61811000001103 | Diazepam 5mg tablets - Accord Healthcare Ltd |
| 521111000001100 | Diazepam 5mg tablets - Alliance Healthcare (Distribution) Ltd |
| 9790611000001103 | Diazepam 5mg tablets - Almus Pharmaceuticals Ltd |
| 10400411000001106 | Diazepam 5mg tablets - Arrow Generics Ltd |
| 28921811000001105 | Diazepam 5mg tablets - Crescent Pharma Ltd |
| 13577211000001108 | Diazepam 5mg tablets - DE Pharmaceuticals |
| 11020111000001108 | Diazepam 5mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 833711000001100 | Diazepam 5mg tablets - IVAX Pharmaceuticals UK Ltd |
| 644911000001105 | Diazepam 5mg tablets - Kent Pharmaceuticals Ltd |
| 30022111000001101 | Diazepam 5mg tablets - Mawdsley-Brooks & Company Ltd |
| 38869111000001104 | Diazepam 5mg tablets - Medihealth (Northern) Ltd |
| 606511000001102 | Diazepam 5mg tablets - Mylan |
| 18107311000001102 | Diazepam 5mg tablets - Phoenix Healthcare Distribution Ltd |
| 924411000001103 | Diazepam 5mg tablets - Ranbaxy (UK) Ltd |
| 10286311000001104 | Diazepam 5mg tablets - Relonchem Ltd |
| 213011000001103 | Diazepam 5mg tablets - Sandoz Ltd |
| 15081611000001101 | Diazepam 5mg tablets - Sigma Pharmaceuticals Plc |
| 17197011000001108 | Diazepam 5mg tablets - Sovereign Medical Ltd |
| 647011000001103 | Diazepam 5mg tablets - Teva UK Ltd |
| 21925611000001102 | Diazepam 5mg tablets - Waymade Healthcare Plc |
| 13938111000001106 | Diazepam 5mg tablets - Wockhardt UK Ltd |
| 1419611000001106 | Diazepam 5mg tablets 1000 tablet - A A H Pharmaceuticals Ltd |

| 1421411000001102 | Diazepam 5mg tablets 1000 tablet - Alliance Healthcare |
|---|---|
| 1421411000001103 | (Distribution) Ltd |
| 10400611000001109 | Diazepam 5mg tablets 1000 tablet - Arrow Generics Ltd |
| 13577311000001100 | Diazepam 5mg tablets 1000 tablet - DE Pharmaceuticals |
| 11020211000001102 | Diazepam 5mg tablets 1000 tablet - Dr Reddys Laboratories (UK) Ltd |
| 1420611000001105 | Diazepam 5mg tablets 1000 tablet - Kent Pharmaceuticals Ltd |
| 23654111000001104 | Diazepam 5mg tablets 1000 tablet - Phoenix Healthcare Distribution Ltd |
| 1421011000001107 | Diazepam 5mg tablets 1000 tablet - Ranbaxy (UK) Ltd |
| 10286611000001109 | Diazepam 5mg tablets 1000 tablet - Relonchem Ltd |
| 8826811000001109 | Diazepam 5mg tablets 1000 tablet - Sandoz Ltd |
| 17197211000001103 | Diazepam 5mg tablets 1000 tablet - Sovereign Medical Ltd |
| 23591211000001108 | Diazepam 5mg tablets 1000 tablet - Waymade Healthcare Plc |
| 16431011000001105 | Diazepam 5mg tablets 1000 tablet - Wockhardt UK Ltd |
| 1419411000001108 | Diazepam 5mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1419711000001102 | Diazepam 5mg tablets 28 tablet - Accord Healthcare Ltd |
| 1421311000001105 | Diazepam 5mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 9790711000001107 | Diazepam 5mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 10400511000001105 | Diazepam 5mg tablets 28 tablet - Arrow Generics Ltd |
| 28921911000001100 | Diazepam 5mg tablets 28 tablet - Crescent Pharma Ltd |
| 23862111000001105 | Diazepam 5mg tablets 28 tablet - DE Pharmaceuticals |
| 1420211000001108 | Diazepam 5mg tablets 28 tablet - IVAX Pharmaceuticals UK Ltd |
| 1420511000001106 | Diazepam 5mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 30022211000001107 | Diazepam 5mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 38869211000001105 | Diazepam 5mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 1419911000001100 | Diazepam 5mg tablets 28 tablet - Mylan |
| 18107411000001109 | Diazepam 5mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 1420911000001104 | Diazepam 5mg tablets 28 tablet - Ranbaxy (UK) Ltd |
| 10286511000001105 | Diazepam 5mg tablets 28 tablet - Relonchem Ltd |
| 1421711000001109 | Diazepam 5mg tablets 28 tablet - Sandoz Ltd |
| 15081711000001105 | Diazepam 5mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 17197111000001109 | Diazepam 5mg tablets 28 tablet - Sovereign Medical Ltd |
| 1419811000001105 | Diazepam 5mg tablets 28 tablet - Teva UK Ltd |
| 21925711000001106 | Diazepam 5mg tablets 28 tablet - Waymade Healthcare Plc |
| 13938211000001100 | Diazepam 5mg tablets 28 tablet - Wockhardt UK Ltd |
| 39709411000001106 | Diazepam 5mg/2.5ml rectal solution tube |
| 323073009 | Diazepam 5mg/2.5ml rectal solution tube |
| 636111000001104 | Diazepam 5mg/2.5ml rectal solution tube - A A H Pharmaceuticals Ltd |
| 463611000001105 | Diazepam 5mg/2.5ml rectal solution tube - Alliance Healthcare (Distribution) Ltd |
| 22198211000001101 | Diazepam 5mg/2.5ml rectal solution tube - Desitin Pharma Ltd |
| 707111000001103 | Diazepam 5mg/2.5ml rectal solution tube - Sandoz Ltd |
| 29804711000001104 | Diazepam 5mg/2.5ml rectal solution tube - Sigma Pharmaceuticals Plc |
| 121611000001104 | Diazepam 5mg/2.5ml rectal solution tube - The Boots Company Plc |
| 1234411000001104 | Diazepam 5mg/2.5ml rectal solution tube 5 tube |
| 2640011000001100 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - A A H Pharmaceuticals Ltd |
| 2640811000001106 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - Alliance Healthcare (Distribution) Ltd |

| 22198311000001109 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - Desitin Pharma |
|---|---|
| | Ltd |
| 2640511000001108 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - Sandoz Ltd |
| 29804811000001107 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - Sigma Pharmaceuticals Plc |
| 2640211000001105 | Diazepam 5mg/2.5ml rectal solution tube 5 tube - The Boots Company Plc |
| 109111000001104 | Diazepam 5mg/5ml oral solution - A A H Pharmaceuticals Ltd |
| 22326511000001101 | Diazepam 5mg/5ml oral solution - AM Distributions (Yorkshire) Ltd |
| 798311000001103 | Diazepam 5mg/5ml oral solution - Sandoz Ltd |
| 2645711000001108 | Diazepam 5mg/5ml oral solution 100 ml - A A H Pharmaceuticals Ltd |
| 2645911000001105 | Diazepam 5mg/5ml oral solution 100 ml - Sandoz Ltd |
| 32903211000001109 | Diazepam 5mg/5ml oral suspension - A A H Pharmaceuticals Ltd |
| 32635511000001104 | Diazepam 5mg/5ml oral suspension - Sandoz Ltd |
| 32903311000001101 | Diazepam 5mg/5ml oral suspension 100 ml - A A H Pharmaceuticals Ltd |
| 32635911000001106 | Diazepam 5mg/5ml oral suspension 100 ml - Sandoz Ltd |
| 13881411000001108 | Frisium 10mg tablets - DE Pharmaceuticals |
| 13164611000001103 | Frisium 10mg tablets - Dowelhurst Ltd |
| 16182211000001104 | Frisium 10mg tablets - Lexon (UK) Ltd |
| 16275711000001107 | Frisium 10mg tablets - Mawdsley-Brooks & Company Ltd |
| 929911000001107 | Frisium 10mg tablets - Sanofi |
| 14240711000001108 | Frisium 10mg tablets - Sigma Pharmaceuticals Plc |
| 5367711000001103 | Frisium 10mg tablets - Waymade Healthcare Plc |
| 13881611000001106 | Frisium 10mg tablets 30 tablet - DE Pharmaceuticals |
| 16182311000001107 | Frisium 10mg tablets 30 tablet - Lexon (UK) Ltd |
| 2177011000001101 | Frisium 10mg tablets 30 tablet - Sanofi |
| 14240911000001105 | Frisium 10mg tablets 30 tablet - Sigma Pharmaceuticals Plc |
| 5368011000001104 | Frisium 10mg tablets 30 tablet - Waymade Healthcare Plc |
| 14243811000001107 | Frisium 10mg tablets 50 tablet - Sigma Pharmaceuticals Plc |
| 12560511000001108 | Frisium 10mg tablets 60 tablet - Waymade Healthcare Plc |
| 17996511000001100 | Klonopin 0.5mg oral lyophilisates - Imported (United States) |
| 17996611000001101 | Klonopin 0.5mg oral lyophilisates 60 tablet - Imported (United States) |
| 218811000001104 | Librium 10mg capsules - Mylan |
| 2304311000001107 | Librium 10mg capsules 100 capsule - Mylan |
| 849211000001108 | Librium 5mg capsules - Mylan |
| 2306611000001106 | Librium 5mg capsules 100 capsule - Mylan |
| 12813311000001108 | Lorazepam 1.125mg/5ml oral solution |
| 12807211000001107 | Lorazepam 1.125mg/5ml oral solution - Special Order |
| 12807111000001101 | Lorazepam 1.125mg/5ml oral solution 1 ml |
| 12807311000001104 | Lorazepam 1.125mg/5ml oral solution 1 ml - Special Order |
| 12813411000001101 | Lorazepam 1.125mg/5ml oral suspension |
| 12806911000001101 | Lorazepam 1.125mg/5ml oral suspension - Special Order |
| 12806811000001106 | Lorazepam 1.125mg/5ml oral suspension 1 ml |
| 12807011000001102 | Lorazepam 1.125mg/5ml oral suspension 1 ml - Special Order |
| 37600511000001104 | Lorazepam 1mg orodispersible tablets |
| 37364611000001102 | Lorazepam 1mg orodispersible tablets - Aristo Pharma Ltd |
| 37363711000001109 | Lorazepam 1mg orodispersible tablets 28 tablet |
| 37365011000001108 | Lorazepam 1mg orodispersible tablets 28 tablet - Aristo Pharma Ltd |
| 321294008 | Lorazepam 1mg trablets |
| J21234000 | rotazehatit Titik ranierz |

| 295711000001104 | Lorazepam 1mg tablets - A A H Pharmaceuticals Ltd |
|---|---|
| 15434211000001100 | Lorazepam 1mg tablets - Accord Healthcare Ltd |
| 814311000001105 | Lorazepam 1mg tablets - Alliance Healthcare (Distribution) Ltd |
| 13403911000001105 | Lorazepam 1mg tablets - Almus Pharmaceuticals Ltd |
| 37899711000001106 | Lorazepam 1mg tablets - Aristo Pharma Ltd |
| 10387311000001105 | Lorazepam 1mg tablets - Arrow Generics Ltd |
| 24370411000001108 | Lorazepam 1mg tablets - DE Pharmaceuticals |
| 18589811000001109 | Lorazepam 1mg tablets - DE Pharmaceuticals |
| 20324811000001104 | Lorazepam 1mg tablets - Genesis Pharmaceuticals Ltd |
| 917211000001100 | Lorazepam 1mg tablets - Genus Pharmaceuticals Ltd |
| 701811000001103 | Lorazepam 1mg tablets - Kent Pharmaceuticals Ltd |
| 37119211000001108 | Lorazepam 1mg tablets - Mawdsley-Brooks & Company Ltd |
| 39029911000001109 | Lorazepam 1mg tablets - Medihealth (Northern) Ltd |
| 24134311000001103 | Lorazepam 1mg tablets - Morningside Healthcare Ltd |
| 9480811000001109 | Lorazepam 1mg tablets - Mylan |
| 17938411000001106 | Lorazepam 1mg tablets - Phoenix Healthcare Distribution Ltd |
| 12533011000001103 | Lorazepam 1mg tablets - Sandoz Ltd |
| 17568411000001109 | Lorazepam 1mg tablets - Sigma Pharmaceuticals Plc |
| 29896911000001107 | Lorazepam 1mg tablets - Sigma Pharmaceuticals Plc |
| 842411000001101 | Lorazepam 1mg tablets - Teva UK Ltd |
| 10545011000001105 | Lorazepam 1mg tablets - Waymade Healthcare Plc |
| 22073811000001109 | Lorazepam 1mg tablets - Waymade Healthcare Plc |
| 15171111000001109 | Lorazepam 1mg tablets 100 tablet |
| 15171311000001106 | Lorazepam 1mg tablets 100 tablet - Waymade Healthcare Plc |
| 15473311000001108 | Lorazepam 1mg tablets 1000 tablet |
| 15473411000001101 | Lorazepam 1mg tablets 1000 tablet - Alliance Healthcare (Distribution) Ltd |
| 1114711000001102 | Lorazepam 1mg tablets 28 tablet |
| 1855511000001105 | Lorazepam 1mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 15434311000001108 | Lorazepam 1mg tablets 28 tablet - Accord Healthcare Ltd |
| 1857811000001103 | Lorazepam 1mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 13404011000001108 | Lorazepam 1mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 37899811000001103 | Lorazepam 1mg tablets 28 tablet - Aristo Pharma Ltd |
| 10387611000001100 | Lorazepam 1mg tablets 28 tablet - Arrow Generics Ltd |
| 24370511000001107 | Lorazepam 1mg tablets 28 tablet - DE Pharmaceuticals |
| 20324911000001109 | Lorazepam 1mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 1856511000001103 | Lorazepam 1mg tablets 28 tablet - Genus Pharmaceuticals Ltd |
| 1857411000001100 | Lorazepam 1mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 37119311000001100 | Lorazepam 1mg tablets 28 tablet - Mawdsley-Brooks & Company Ltd |
| 39030011000001104 | Lorazepam 1mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 35957811000001107 | Lorazepam 1mg tablets 28 tablet - Morningside Healthcare Ltd |
| 9481011000001107 | Lorazepam 1mg tablets 28 tablet - Mylan |
| 17938511000001105 | Lorazepam 1mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 12533111000001102 | Lorazepam 1mg tablets 28 tablet - Sandoz Ltd |
| 29897011000001106 | Lorazepam 1mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1856911000001105 | Lorazepam 1mg tablets 28 tablet - Teva UK Ltd |
| 22073911000001104 | Lorazepam 1mg tablets 28 tablet - Waymade Healthcare Plc |
| 10545111000001106 | Lorazepam 1mg tablets 30 tablet |

| 24134411000001105 | Lorazepam 1mg tablets 30 tablet - Morningside Healthcare Ltd |
|---|---|
| 10545211000001100 | Lorazepam 1mg tablets 30 tablet - Waymade Healthcare Plc |
| 15171011000001108 | Lorazepam 1mg tablets 50 tablet |
| 18590111000001108 | Lorazepam 1mg tablets 50 tablet - DE Pharmaceuticals |
| 17568511000001108 | Lorazepam 1mg tablets 50 tablet - Sigma Pharmaceuticals Plc |
| 15171211000001103 | Lorazepam 1mg tablets 50 tablet - Sigma Pharmaceuticals Pic Lorazepam 1mg tablets 50 tablet - Waymade Healthcare Pic |
| 8624311000001104 | Lorazepam 1mg/5ml oral solution |
| 8596311000001109 | Lorazepam 1mg/5ml oral solution - Drug Tariff Special Order |
| 8596111000001107 | Lorazepam 1mg/5ml oral solution 1 ml |
| 8596411000001102 | Lorazepam 1mg/5ml oral solution 1 ml - Drug Tariff Special Order |
| 19597711000001108 | Lorazepam 1mg/5ml oral solution 150 ml |
| 19597911000001105 | Lorazepam 1mg/5ml oral solution 150 ml - Drug Tariff Special Order |
| 8624511000001105 | Lorazepam 1mg/5ml oral suspension |
| 8596811000001100 | Lorazepam 1mg/5ml oral suspension - Drug Tariff Special Order |
| 8596711000001108 | Lorazepam 1mg/5ml oral suspension 1 ml |
| 8596911000001105 | Lorazepam 1mg/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 19598411000001103 | Lorazepam 1mg/5ml oral suspension 100 ml |
| 19598611000001100 | Lorazepam 1mg/5ml oral suspension 100 ml - Drug Tariff Special Order |
| 34697811000001107 | Lorazepam 1mg/ml oral solution sugar free |
| 35108511000001103 | Lorazepam 1mg/ml oral solution sugar free - A A H Pharmaceuticals Ltd |
| 34979011000001104 | Lorazepam 1mg/ml oral solution sugar free - Alliance Healthcare (Distribution) Ltd |
| 34612211000001107 | Lorazepam 1mg/ml oral solution sugar free - Thame Laboratories Ltd |
| 34612111000001101 | Lorazepam 1mg/ml oral solution sugar free 150 ml |
| 35108611000001104 | Lorazepam 1mg/ml oral solution sugar free 150 ml - A A H Pharmaceuticals Ltd |
| 34979311000001101 | Lorazepam 1mg/ml oral solution sugar free 150 ml - Alliance<br>Healthcare (Distribution) Ltd |
| 34612311000001104 | Lorazepam 1mg/ml oral solution sugar free 150 ml - Thame Laboratories Ltd |
| 37600611000001100 | Lorazepam 2.5mg orodispersible tablets |
| 37367111000001100 | Lorazepam 2.5mg orodispersible tablets - Aristo Pharma Ltd |
| 37366811000001105 | Lorazepam 2.5mg orodispersible tablets 28 tablet |
| 37367411000001105 | Ltd Lorazepam 2.5mg orodispersible tablets 28 tablet - Aristo Pharma |
| 321295009 | Lorazepam 2.5mg tablets |
| 771611000001105 | Lorazepam 2.5mg tablets - A A H Pharmaceuticals Ltd |
| 15434411000001101 | Lorazepam 2.5mg tablets - Accord Healthcare Ltd |
| 115511000001108 | Lorazepam 2.5mg tablets - Alliance Healthcare (Distribution) Ltd |
| 13403411000001102 | Lorazepam 2.5mg tablets - Almus Pharmaceuticals Ltd |
| 37904511000001107 | Lorazepam 2.5mg tablets - Aristo Pharma Ltd |
| 10389311000001100 | Lorazepam 2.5mg tablets - Arrow Generics Ltd |
| 24370611000001106 | Lorazepam 2.5mg tablets - DE Pharmaceuticals |
| 20325111000001105 | Lorazepam 2.5mg tablets - Genesis Pharmaceuticals Ltd |
| 845311000001102 | Lorazepam 2.5mg tablets - Genus Pharmaceuticals Ltd |
| 585511000001101 | Lorazepam 2.5mg tablets - Kent Pharmaceuticals Ltd |
| 39030511000001107 | Lorazepam 2.5mg tablets - Medihealth (Northern) Ltd |
| 24134611000001108 | Lorazepam 2.5mg tablets - Morningside Healthcare Ltd |
| 9481211000001102 | Lorazepam 2.5mg tablets - Mylan |
| 17938611000001109 | Lorazepam 2.5mg tablets - Phoenix Healthcare Distribution Ltd |

| 12533211000001108 | Lorazepam 2.5mg tablets - Sandoz Ltd |
|---|---|
| 15108811000001102 | Lorazepam 2.5mg tablets - Sigma Pharmaceuticals Plc |
| 478511000001108 | Lorazepam 2.5mg tablets - Teva UK Ltd |
| 22074011000001101 | Lorazepam 2.5mg tablets - Waymade Healthcare Plc |
| 1128211000001105 | Lorazepam 2.5mg tablets 28 tablet |
| 1859111000001104 | Lorazepam 2.5mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 15434511000001102 | Lorazepam 2.5mg tablets 28 tablet - Accord Healthcare Ltd |
| 1860611000001106 | Lorazepam 2.5mg tablets 28 tablet - Alliance Healthcare |
| | (Distribution) Ltd |
| 13403611000001104 | Lorazepam 2.5mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 37904711000001102 | Lorazepam 2.5mg tablets 28 tablet - Aristo Pharma Ltd |
| 10389511000001106 | Lorazepam 2.5mg tablets 28 tablet - Arrow Generics Ltd |
| 24370711000001102 | Lorazepam 2.5mg tablets 28 tablet - DE Pharmaceuticals |
| 20325211000001104 | Lorazepam 2.5mg tablets 28 tablet - Genesis Pharmaceuticals Ltd |
| 1859311000001102 | Lorazepam 2.5mg tablets 28 tablet - Genus Pharmaceuticals Ltd |
| 4582311000001108 | Lorazepam 2.5mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 1860011000001104 | Lorazepam 2.5mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 39030611000001106 | Lorazepam 2.5mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 35959111000001106 | Lorazepam 2.5mg tablets 28 tablet - Morningside Healthcare Ltd |
| 9481311000001105 | Lorazepam 2.5mg tablets 28 tablet - Mylan |
| 17938711000001100 | Lorazepam 2.5mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 12533311000001100 | Lorazepam 2.5mg tablets 28 tablet - Sandoz Ltd |
| 15108911000001107 | Lorazepam 2.5mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 1859711000001103 | Lorazepam 2.5mg tablets 28 tablet - Teva UK Ltd |
| 22074111000001100 | Lorazepam 2.5mg tablets 28 tablet - Waymade Healthcare Plc |
| 24134811000001107 | Lorazepam 2.5mg tablets 30 tablet |
| 24135211000001107 | Lorazepam 2.5mg tablets 30 tablet - Morningside Healthcare Ltd |
| 8659111000001104 | Lorazepam 250micrograms/5ml oral solution |
| 8597211000001104 | Lorazepam 250micrograms/5ml oral solution - Special Order |
| 8597011000001109 | Lorazepam 250micrograms/5ml oral solution 1 ml |
| 8597311000001107 | Lorazepam 250micrograms/5ml oral solution 1 ml - Special Order |
| 8659211000001105 | Lorazepam 250micrograms/5ml oral suspension |
| 8597711000001106 | Lorazepam 250micrograms/5ml oral suspension - Special Order |
| 8597611000001102 | Lorazepam 250micrograms/5ml oral suspension 1 ml |
| 8597911000001108 | Lorazepam 250micrograms/5ml oral suspension 1 ml - Special Order |
| 23675911000001104 | Lorazepam 2mg/1ml solution for injection ampoules |
| 23670011000001109 | Lorazepam 2mg/1ml solution for injection ampoules - Special Order |
| 23669911000001105 | Lorazepam 2mg/1ml solution for injection ampoules 1 ampoule |
| 23670111000001105 | Lorazepam 2mg/1ml solution for injection ampoules 1 ampoule - Special Order |
| 38926811000001104 | Lorazepam 2mg/1ml solution for injection Carpuject cartridges - Imported (United States) |
| 38926911000001109 | Lorazepam 2mg/1ml solution for injection Carpuject cartridges 10 cartridge - Imported (United States) |
| 38931911000001102 | Lorazepam 2mg/1ml solution for injection cartridges |
| 38926511000001102 | Lorazepam 2mg/1ml solution for injection cartridges 10 cartridge |
| 36108111000001105 | Lorazepam 2mg/1ml solution for injection vials |
| 36011311000001105 | Lorazepam 2mg/1ml solution for injection vials - Imported (United States) |
| 36011211000001102 | Lorazepam 2mg/1ml solution for injection vials 10 vial |

| | Lorazepam 2mg/1ml solution for injection vials 10 vial - Imported |
|---|---|
| 36011411000001103 | (United States) |
| 8659411000001109 | Lorazepam 2mg/5ml oral solution |
| 8597411000001100 | Lorazepam 2mg/5ml oral solution - Special Order |
| 8597111000001105 | Lorazepam 2mg/5ml oral solution 1 ml |
| 8597511000001101 | Lorazepam 2mg/5ml oral solution 1 ml - Special Order |
| 8659511000001108 | Lorazepam 2mg/5ml oral suspension |
| 8598011000001105 | Lorazepam 2mg/5ml oral suspension - Special Order |
| 8597811000001103 | Lorazepam 2mg/5ml oral suspension 1 ml |
| 8598111000001106 | Lorazepam 2mg/5ml oral suspension 1 ml - Special Order |
| 12813511000001102 | Lorazepam 3.75mg/5ml oral solution |
| 12809611000001104 | Lorazepam 3.75mg/5ml oral solution - Special Order |
| 12808911000001102 | Lorazepam 3.75mg/5ml oral solution 1 ml |
| 12809711000001108 | Lorazepam 3.75mg/5ml oral solution 1 ml - Special Order |
| 12813611000001103 | Lorazepam 3.75mg/5ml oral suspension |
| 12808711000001104 | Lorazepam 3.75mg/5ml oral suspension - Special Order |
| 12808311000001103 | Lorazepam 3.75mg/5ml oral suspension 1 ml |
| 12808811000001107 | Lorazepam 3.75mg/5ml oral suspension 1 ml - Special Order |
| 12817711000001102 | Lorazepam 400micrograms/5ml oral solution |
| 12810811000001106 | Lorazepam 400micrograms/5ml oral solution - Special Order |
| 12810711000001103 | Lorazepam 400micrograms/5ml oral solution 1 ml |
| 12810911000001101 | Lorazepam 400micrograms/5ml oral solution 1 ml - Special Order |
| 12817811000001105 | Lorazepam 400micrograms/5ml oral suspension |
| 12810311000001102 | Lorazepam 400micrograms/5ml oral suspension - Special Order |
| 12810111000001104 | Lorazepam 400micrograms/5ml oral suspension 1 ml |
| 12810511000001108 | Lorazepam 400micrograms/5ml oral suspension 1 ml - Special Order |
| 36040511000001101 | Lorazepam 4mg/1ml solution for injection ampoules |
| 321302003 | Lorazepam 4mg/1ml solution for injection ampoules |
| 39502711000001107 | Lorazepam 4mg/1ml solution for injection ampoules - Macure Pharma UK Ltd |
| 3925311000001102 | Lorazepam 4mg/1ml solution for injection ampoules 10 ampoule |
| 39502811000001104 | Lorazepam 4mg/1ml solution for injection ampoules 10 ampoule - Macure Pharma UK Ltd |
| 39332011000001101 | Lorazepam 4mg/1ml solution for injection vials |
| 39320511000001106 | Lorazepam 4mg/1ml solution for injection vials 25 vial |
| 12817911000001100 | Lorazepam 4mg/5ml oral solution |
| 12811411000001100 | Lorazepam 4mg/5ml oral solution - Special Order |
| 12811311000001107 | Lorazepam 4mg/5ml oral solution 1 ml |
| 12811511000001101 | Lorazepam 4mg/5ml oral solution 1 ml - Special Order |
| 12818011000001103 | Lorazepam 4mg/5ml oral suspension |
| 12811111000001105 | Lorazepam 4mg/5ml oral suspension - Special Order |
| 12811011000001109 | Lorazepam 4mg/5ml oral suspension 1 ml |
| 12811211000001104 | Lorazepam 4mg/5ml oral suspension 1 ml - Special Order |
| 377147002 | Lorazepam 500microgram tablets |
| 37480811000001104 | Lorazepam 500microgram tablets - A A H Pharmaceuticals Ltd |
| 37230311000001103 | Lorazepam 500microgram tablets - Advanz Pharma |
| 37660711000001108 | Lorazepam 500microgram tablets - Alliance Healthcare (Distribution) Ltd |
| 37230211000001106 | Lorazepam 500microgram tablets 28 tablet |
| 37480911000001109 | Lorazepam 500microgram tablets 28 tablet - A A H Pharmaceuticals Ltd |

| 37230411000001105 | Lorazepam 500microgram tablets 28 tablet - Advanz Pharma |
|---|---|
| 37660811000001100 | Lorazepam 500microgram tablets 28 tablet - Alliance Healthcare |
| 37000811000001100 | (Distribution) Ltd |
| 8659611000001107 | Lorazepam 500micrograms/5ml oral solution |
| 8598611000001103 | Lorazepam 500micrograms/5ml oral solution - Drug Tariff Special Order |
| 8598511000001102 | Lorazepam 500micrograms/5ml oral solution 1 ml |
| 8598811000001104 | Lorazepam 500micrograms/5ml oral solution 1 ml - Drug Tariff Special Order |
| 19598811000001101 | Lorazepam 500micrograms/5ml oral solution 150 ml |
| 19599111000001101 | Lorazepam 500micrograms/5ml oral solution 150 ml - Drug Tariff Special Order |
| 8659811000001106 | Lorazepam 500micrograms/5ml oral suspension |
| 8599511000001108 | Lorazepam 500micrograms/5ml oral suspension - Drug Tariff Special Order |
| 8599411000001109 | Lorazepam 500micrograms/5ml oral suspension 1 ml |
| 8599611000001107 | Lorazepam 500micrograms/5ml oral suspension 1 ml - Drug Tariff Special Order |
| 19599211000001107 | Lorazepam 500micrograms/5ml oral suspension 100 ml |
| 19599411000001106 | Lorazepam 500micrograms/5ml oral suspension 100 ml - Drug Tariff Special Order |
| 8599111000001104 | Lorazepam 5mg/5ml oral solution - Special Order |
| 8599211000001105 | Lorazepam 5mg/5ml oral solution 1 ml - Special Order |
| 8660011000001104 | Lorazepam 5mg/5ml oral suspension |
| 8599811000001106 | Lorazepam 5mg/5ml oral suspension - Special Order |
| 8599711000001103 | Lorazepam 5mg/5ml oral suspension 1 ml |
| 8599911000001101 | Lorazepam 5mg/5ml oral suspension 1 ml - Special Order |
| 3642111000001107 | Meprobamate 400mg tablets - Thornton & Ross Ltd |
| 3642211000001101 | Meprobamate 400mg tablets 84 tablet - Thornton & Ross Ltd |
| 3642611000001104 | Meprobamate 400mg tablets - Kent Pharma (UK) Ltd |
| 3642911000001105 | Meprobamate 400mg tablets 84 tablet - Kent Pharma (UK) Ltd |
| 3641811000001109 | Meprobamate 400mg tablets - A A H Pharmaceuticals Ltd |
| 3642011000001106 | Meprobamate 400mg tablets 84 tablet - A A H Pharmaceuticals Ltd |
| 12694111000001101 | Meprobamate 5mg/5ml oral suspension - Special Order |
| 12694311000001104 | Meprobamate 5mg/5ml oral suspension 1 ml - Special Order |
| 3643011000001102 | Meprobamate 400mg tablets - Alliance Healthcare (Distribution) Ltd |
| 3643311000001104 | Meprobamate 400mg tablets 84 tablet - Alliance Healthcare (Distribution) Ltd |
| 12694711000001100 | Meprobamate 5mg/5ml oral solution - Special Order |
| 12694811000001108 | Meprobamate 5mg/5ml oral solution 1 ml - Special Order |
| 29905711000001108 | Meprobamate 400mg tablets - Sigma Pharmaceuticals Plc |
| 29905811000001100 | Meprobamate 400mg tablets 84 tablet - Sigma Pharmaceuticals Plc |
| 321308004 | Meprobamate 400mg tablets |
| 3640711000001109 | Meprobamate 400mg tablets 84 tablet |
| 12701311000001107 | Meprobamate 5mg/5ml oral solution |
| 12694611000001109 | Meprobamate 5mg/5ml oral solution 1 ml |
| 12701411000001100 | Meprobamate 5mg/5ml oral suspension |
| 321314006 | Oxazepam 10mg tablets |
| 498511000001100 | Oxazepam 10mg tablets - A A H Pharmaceuticals Ltd |
| 214711000001104 | Oxazepam 10mg tablets - Accord Healthcare Ltd |
| 682511000001104 | Oxazepam 10mg tablets - Alliance Healthcare (Distribution) Ltd |
| 19819411000001108 | Oxazepam 10mg tablets - Almus Pharmaceuticals Ltd |

| 30069511000001106 | Oxazepam 10mg tablets - DE Pharmaceuticals |
|---|---|
| 616111000001109 | Oxazepam 10mg tablets - Genus Pharmaceuticals Ltd |
| 384111000001108 | Oxazepam 10mg tablets - Kent Pharmaceuticals Ltd |
| 39068111000001105 | Oxazepam 10mg tablets - Medihealth (Northern) Ltd |
| 17950111000001102 | Oxazepam 10mg tablets - Phoenix Healthcare Distribution Ltd |
| 29974111000001104 | Oxazepam 10mg tablets - Sigma Pharmaceuticals Plc |
| 39490011000001104 | Oxazepam 10mg tablets - Tillomed Laboratories Ltd |
| 21828411000001100 | Oxazepam 10mg tablets - Waymade Healthcare Plc |
| 1217911000001108 | Oxazepam 10mg tablets 28 tablet |
| 1928811000001109 | Oxazepam 10mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1928911000001104 | Oxazepam 10mg tablets 28 tablet - Accord Healthcare Ltd |
| 1929211000001103 | Oxazepam 10mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 19819511000001107 | Oxazepam 10mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| 30069611000001105 | Oxazepam 10mg tablets 28 tablet - DE Pharmaceuticals |
| 1929011000001108 | Oxazepam 10mg tablets 28 tablet - Genus Pharmaceuticals Ltd |
| 1929111000001109 | Oxazepam 10mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 39068211000001104 | Oxazepam 10mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 17950211000001108 | Oxazepam 10mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 29974211000001105 | Oxazepam 10mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 39490111000001103 | Oxazepam 10mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 21828511000001101 | Oxazepam 10mg tablets 28 tablet - Waymade Healthcare Plc |
| 12141711000001106 | Oxazepam 10mg/5ml oral suspension |
| 12133911000001108 | Oxazepam 10mg/5ml oral suspension - Special Order |
| 12133811000001103 | Oxazepam 10mg/5ml oral suspension 1 ml |
| 12134011000001106 | Oxazepam 10mg/5ml oral suspension 1 ml - Special Order |
| 12141811000001103 | Oxazepam 12.5mg/5ml oral suspension |
| 12133211000001104 | Oxazepam 12.5mg/5ml oral suspension - Special Order |
| 12133111000001105 | Oxazepam 12.5mg/5ml oral suspension 1 ml |
| 12133311000001107 | Oxazepam 12.5mg/5ml oral suspension 1 ml - Special Order |
| 321315007 | Oxazepam 15mg tablets |
| 647511000001106 | Oxazepam 15mg tablets - A A H Pharmaceuticals Ltd |
| 191811000001107 | Oxazepam 15mg tablets - Accord Healthcare Ltd |
| 37611000001102 | Oxazepam 15mg tablets - Alliance Healthcare (Distribution) Ltd |
| 19819611000001106 | Oxazepam 15mg tablets - Almus Pharmaceuticals Ltd |
| 30069711000001101 | Oxazepam 15mg tablets - DE Pharmaceuticals |
| 500711000001102 | Oxazepam 15mg tablets - Genus Pharmaceuticals Ltd |
| 762211000001107 | Oxazepam 15mg tablets - Kent Pharmaceuticals Ltd |
| 39068311000001107 | Oxazepam 15mg tablets - Medihealth (Northern) Ltd |
| 17950311000001100 | Oxazepam 15mg tablets - Phoenix Healthcare Distribution Ltd |
| 29974311000001102 | Oxazepam 15mg tablets - Sigma Pharmaceuticals Plc |
| 39490511000001107 | Oxazepam 15mg tablets - Tillomed Laboratories Ltd |
| 21828611000001102 | Oxazepam 15mg tablets - Waymade Healthcare Plc |
| 1202211000001104 | Oxazepam 15mg tablets 28 tablet |
| 1929311000001106 | Oxazepam 15mg tablets 28 tablet - A A H Pharmaceuticals Ltd |
| 1929411000001104 | Oxazepam 15mg tablets 28 tablet - Accord Healthcare Ltd |
| 1929711000001105 | Oxazepam 15mg tablets 28 tablet - Alliance Healthcare (Distribution) Ltd |
| 19819711000001102 | Oxazepam 15mg tablets 28 tablet - Almus Pharmaceuticals Ltd |
| | · |

| 30069811000001109 | Oxazepam 15mg tablets 28 tablet - DE Pharmaceuticals |
|---|---|
| 1929511000001100 | Oxazepam 15mg tablets 28 tablet - Genus Pharmaceuticals Ltd |
| 1929611000001101 | Oxazepam 15mg tablets 28 tablet - Kent Pharmaceuticals Ltd |
| 39068511000001101 | Oxazepam 15mg tablets 28 tablet - Medihealth (Northern) Ltd |
| 17950411000001107 | Oxazepam 15mg tablets 28 tablet - Phoenix Healthcare Distribution Ltd |
| 29974411000001109 | Oxazepam 15mg tablets 28 tablet - Sigma Pharmaceuticals Plc |
| 39490611000001106 | Oxazepam 15mg tablets 28 tablet - Tillomed Laboratories Ltd |
| 21828711000001106 | Oxazepam 15mg tablets 28 tablet - Waymade Healthcare Plc |
| 12141911000001108 | Oxazepam 2.5mg/5ml oral suspension |
| 12132911000001101 | Oxazepam 2.5mg/5ml oral suspension - Special Order |
| 12132811000001106 | Oxazepam 2.5mg/5ml oral suspension 1 ml |
| 12133011000001109 | Oxazepam 2.5mg/5ml oral suspension 1 ml - Special Order |
| 12142011000001101 | Oxazepam 2mg/5ml oral suspension |
| 12132611000001107 | Oxazepam 2mg/5ml oral suspension - Special Order |
| 12131911000001107 | Oxazepam 2mg/5ml oral suspension 1 ml |
| 12132711000001103 | Oxazepam 2mg/5ml oral suspension 1 ml - Special Order |
| 29794011000001101 | Perizam 1mg/ml oral suspension - Rosemont Pharmaceuticals Ltd |
| 29794111000001100 | Perizam 1mg/ml oral suspension 150 ml - Rosemont Pharmaceuticals Ltd |
| 29794211000001106 | Perizam 2mg/ml oral suspension - Rosemont Pharmaceuticals Ltd |
| 29794311000001103 | Perizam 2mg/ml oral suspension 150 ml - Rosemont Pharmaceuticals Ltd |
| 7655011000001106 | Rivotril 2.5mg/1ml drops - Imported (Switzerland) |
| 7655111000001107 | Rivotril 2.5mg/1ml drops 10 ml - Imported (Switzerland) |
| 291011000001103 | Rivotril 2mg tablets - Roche Products Ltd |
| 14664211000001104 | Rivotril 2mg tablets - Sigma Pharmaceuticals Plc |
| 5406711000001108 | Rivotril 2mg tablets - Waymade Healthcare Plc |
| 2168411000001101 | Rivotril 2mg tablets 100 tablet - Roche Products Ltd |
| 5406811000001100 | Rivotril 2mg tablets 100 tablet - Waymade Healthcare Plc |
| 14664411000001100 | Rivotril 2mg tablets 60 tablet - Sigma Pharmaceuticals Plc |
| 142611000001108 | Stesolid 10mg rectal tube - Accord Healthcare Ltd |
| 2638511000001105 | Stesolid 10mg rectal tube 5 tube - Accord Healthcare Ltd |
| 82011000001104 | Stesolid 5mg rectal tube - Accord Healthcare Ltd |
| 2640111000001104 | Stesolid 5mg rectal tube 5 tube - Accord Healthcare Ltd |
| 21803611000001104 | Tapclob 10mg/5ml oral suspension - Martindale Pharmaceuticals Ltd |
| 21803911000001105 | Tapclob 10mg/5ml oral suspension 150 ml - Martindale Pharmaceuticals Ltd |
| 30926111000001108 | Tapclob 10mg/5ml oral suspension 250 ml - Martindale Pharmaceuticals Ltd |
| 21802811000001108 | Tapclob 5mg/5ml oral suspension - Martindale Pharmaceuticals Ltd |
| 21803011000001106 | Tapclob 5mg/5ml oral suspension 150 ml - Martindale Pharmaceuticals Ltd |
| 30926311000001105 | Tapclob 5mg/5ml oral suspension 250 ml - Martindale Pharmaceuticals Ltd |
| 9106811000001108 | Tensium 10mg tablets - DDSA Pharmaceuticals Ltd |
| 9106911000001103 | Tensium 10mg tablets 100 tablet - DDSA Pharmaceuticals Ltd |
| 9107211000001109 | Tensium 2mg tablets - DDSA Pharmaceuticals Ltd |
| 9107411000001108 | Tensium 2mg tablets 100 tablet - DDSA Pharmaceuticals Ltd |
| 9107511000001107 | Tensium 2mg tablets 500 tablet - DDSA Pharmaceuticals Ltd |
| 511311000001108 | Tropium 10mg capsules - Dr Reddys Laboratories (UK) Ltd |

| 2304711000001106 | Tropium 10mg capsules 100 capsule - Dr Reddys Laboratories (UK)<br>Ltd |
|---|---|
| 2304811000001103 | Tropium 10mg capsules 500 capsule - Dr Reddys Laboratories (UK)<br>Ltd |
| 153811000001102 | Tropium 10mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 2455311000001109 | Tropium 10mg tablets 100 tablet - Dr Reddys Laboratories (UK) Ltd |
| 2455411000001102 | Tropium 10mg tablets 500 tablet - Dr Reddys Laboratories (UK) Ltd |
| 307711000001103 | Tropium 5mg capsules - Dr Reddys Laboratories (UK) Ltd |
| 2306811000001105 | Tropium 5mg capsules 100 capsule - Dr Reddys Laboratories (UK) Ltd |
| 2306911000001100 | Tropium 5mg capsules 500 capsule - Dr Reddys Laboratories (UK) Ltd |
| 204011000001103 | Tropium 5mg tablets - Dr Reddys Laboratories (UK) Ltd |
| 2455511000001103 | Tropium 5mg tablets 100 tablet - Dr Reddys Laboratories (UK) Ltd |
| 2455611000001104 | Tropium 5mg tablets 500 tablet - Dr Reddys Laboratories (UK) Ltd |
| 3824311000001107 | Valclair 10mg suppositories - Durbin Plc |
| 3824411000001100 | Valclair 10mg suppositories 6 suppository - Durbin Plc |
| 4658511000001101 | Xanax 250microgram tablets - Upjohn UK Ltd |
| 4658611000001102 | Xanax 250microgram tablets 60 tablet - Upjohn UK Ltd |
| 4659411000001108 | Xanax 500microgram tablets - Upjohn UK Ltd |
| 4659511000001107 | Xanax 500microgram tablets 60 tablet - Upjohn UK Ltd |
| 34247011000001105 | Zacco 10mg/5ml oral suspension - Thame Laboratories Ltd |
| 34247211000001100 | Zacco 10mg/5ml oral suspension 150 ml - Thame Laboratories Ltd |
| 34246711000001109 | Zacco 5mg/5ml oral suspension - Thame Laboratories Ltd |
| 34246811000001101 | Zacco 5mg/5ml oral suspension 150 ml - Thame Laboratories Ltd |

## Appendix 4

Below is a list of the variables to be extracted and utilised for the study

| Variable | Role Data s | | Operational |
|---|---|---|---|
| | | | definition |
| Vitiligo | Case definition | OPCRD | As defined using the |
| | | | codes listed in |
| | | | Appendix 1 |
| Vitiligo exclusion | Case definition | OPCRD | As defined using the |
| conditions | | | codes listed in |
| | | | Appendix 1 and |
| | | | summarised in |
| | | | Appendix 2 |
| Depressive episode | Primary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Recurrent depressive | Primary outcome | OPCRD | Identified from coding |
| disorder | variable | | in the clinical record |
| Non-phobia related | Primary outcome | OPCRD | Identified from coding |
| anxiety disorder | variable | | in the clinical record |
| Social phobia | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Adjustment disorder | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Substance abuse | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Self-harm | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Suicide attempt | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Parasuicide | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Primary care visit | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Secondary care | Secondary outcome | OPCRD | Identified from coding |
| dermatology referral | variable | | in the clinical record |
| Med 3 certificates | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Unemployment | Secondary outcome | OPCRD | Identified from coding |
| | variable | | in the clinical record |
| Age | Baseline characteristic, | OPCRD | Defined as age at the |
| | predictor variable | | start of follow up |
| Gender | Baseline characteristic, | OPCRD | Primary care recorded |
| | predictor variable | | patient gender |
| dermatology referral Med 3 certificates Unemployment Age | Secondary outcome variable Secondary outcome variable Secondary outcome variable Baseline characteristic, predictor variable Baseline characteristic, | OPCRD OPCRD | Identified from cool in the clinical record in the clinical record in the clinical record Identified from cool in the clinical record in the clinical record Defined as age at the start of follow up |

| Variable | Role | Data source(s) | Operational |
|---|---|---|---|
| | | | definition |
| Socioeconomic status | Baseline characteristic, | OPCRD | Defined using patient |
| (SES) | predictor variable | | index of multiple |
| | | | deprivation quintile |
| Ethnicity | Baseline characteristic, | OPCRD | Defined using office of |
| | predictor variable | | national statistics |
| | | | census categories using |
| | | | clinically coded |
| | | | ethnicity data |
| Smoking status | Baseline characteristic, | OPCRD | Using most recent |
| | predictor variable | | clinically recorded |
| | | | smoking status |
| | | | information |
| Alcohol use | Baseline characteristic, | OPCRD | Using most recent |
| | predictor variable | | clinically recorded |
| | | | alcohol use status |
| | | | information |
| Body mass index (BMI) | Baseline characteristic, | OPCRD | Defined using most |
| | predictor variable | | recent clinically |
| | | | recorded BMI |
| | | | information |
| Death | Censoring event | OPCRD | Identified from coding |
| | | | in the clinical record |
| Deregistration from GP | Censoring event | OPCRD | Identified from coding |
| | | | in the clinical record |
| Atrial fibrillation | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Angina | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Myocardial infarction | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Congestive heart failure | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Stroke | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Diabetes type | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| Hyperlipidaemia | Baseline characteristic, | OPCRD | Identified using clinical |
| | predictor variable | | codes for the condition |
| II | Baseline characteristic, | OPCRD | Identified using clinical |
| Hypertension | predictor variable | | codes for the condition |
| | r · | | The state of the condition |

| Variable | Role | Data source(s) | Operational |
|---|---|---|---|
| | | | definition |
| Chronic kidney disease stages 3-5 | Baseline characteristic, predictor variable | OPCRD | Identified using clinical codes for the condition and lab test results |
| Chronic obstructive pulmonary disease | Baseline characteristic, predictor variable | OPCRD | Identified using clinical codes for the condition |
| Asthma | Baseline characteristic, predictor variable | OPCRD | Identified using clinical codes for the condition |
| Chronic liver disease | Baseline characteristic, predictor variable | OPCRD | Identified using clinical codes for the condition |
| Dementia | Baseline characteristic, predictor variable | OPCRD | Identified using clinical codes for the condition |